

#### Statistical Analysis Plan

A RANDOMIZED, OPEN-LABEL, 2-SEQUENCE, 3-TREATMENT, CROSSOVER STUDY TO EVALUATE THE PHARMACOKINETICS OF SINGLE DOSES OF DIAZEPAM BUCCAL FILM (DBF) (AQUESTIVE THERAPEUTICS) COMPARED WITH DIASTAT® RECTAL GEL (VALEANT PHARMACEUTICALS NORTH AMERICA) IN ADULT MALE AND FEMALE SUBJECTS ON A CONCOMITANT REGIMEN OF ANTIEPILEPTIC DRUGS (AED) FOR THE TREATMENT OF EPILEPSY

Sponsor Protocol No. 180323 inVentiv Health Clinique inc. Project No. 180323

Final Version: 1.0 Date: 28-JUN-2019

Contract Research Organization: inVentiv Health Clinique Inc. ("inVentiv"), a Syneos Health company 2500, rue Einstein Québec (Québec) Canada, G1P 0A2 Sponsor: Aquestive Therapeutics 30 Technology Drive Warren, NJ 07059 USA

CONFIDENTIAL

#### **SIGNATURES**

Sponsor Protocol No. 180323

inVentiv Project No.: 180323

Study Title: A Randomized, Open-Label, 2-Sequence, 3-Treatment, Crossover Study to

Evaluate the Pharmacokinetics of Single Doses of Diazepam Buccal Film (DBF) (Aquestive Therapeutics) Compared with Diastat® Rectal Gel (Valeant Pharmaceuticals North America) in Adult Male and Female Subjects on a Concomitant Regimen of Antiepileptic Drugs (AED) for the Treatment of

**Epilepsy** 

Author:

Claude Lapointe, M. Sc.

Principal Statistician

in Ventiv

Signature: Claude Japante

Date: 02-Jul- 2019

Sponsor's

Representative: Allen H Heller, MD, MPH

Founder and CEO, Pharma Study

Design LLC (Consultant to Aquestive

Therapeutics)

Signature: Oll N. N. Date: 28 June 2019



## TABLE OF CONTENTS

| SIGN. | ATURES | 2 |
|---|---|---|
| LIST | OF ABBREVIATIONS | 5 |
| 1. | Introduction | 7 |
| 2. | Study Objectives | 8 |
| 2.1 | Primary Objective | 8 |
| 2.2 | Secondary Objectives | 8 |
| 3. | Study Design | 9 |
| 3.1 | General Design | 9 |
| 3.2 | Study Procedures | 9 |
| 3.3 | Treatment Description | 9 |
| 3.4 | Sample Size | 10 |
| 3.5 | Subject Withdrawal and Replacement | 11 |
| 4. | Change From the Protocol | 12 |
| 5. | Primary and Secondary Parameters | 13 |
| 6. | Analysis Populations | 14 |
| 6.1 | Safety Population | 14 |
| 6.2 | Pharmacokinetic Population and Pharmacokinetic Analysis Data Set | 14 |
| 7. | Interim Analyses | 15 |
| 8. | Study Population and Exposure | 16 |
| 8.1 | Subject Disposition | 16 |
| 8.2 | Protocol Deviations | 16 |
| 8.3 | Demographics and Baseline Characteristics | 16 |
| 8.4 | Medical History | 16 |
| 8.5 | Prior and Concomitant Medications | 16 |
| 8.6 | Study Drug Administration | 16 |
| 9. | Safety Analyses | 17 |
| 9.1 | Physical Examination Findings | 17 |
| 9.2 | Adverse Events | 17 |
| 9.3 | Laboratory Parameters | 19 |
| 9.4 | Vital Signs | 20 |
| 9.5 | Electrocardiogram | |
| 9.6 | DBF Application Site Inspection | 21 |
| 10. | Pharmacokinetic Analyses. | 22 |
| 10.1 | Handling of the Below the Lower Limit of Quantitation (BLQ) and the No | |
| | Reportable Concentration Values | 22 |



| Statistical A | Malysis | Plan |
|---------------|---------|------|
| Project No. | 180323 | |

Aquestive Therapeutics

| 10.2 Handling of the Difference Between the Schedule | ed and the Actual Sampling |
|---|---|
| Times | 22 |
| 10.3 Pharmacokinetic Parameters | 22 |
| 10.4 Statistical Analyses | 23 |
| 10.4.1 Treatment Comparison DBF (Test) versus D | |
| Moderate-Fat Meal | 24 |
| 10.4.2 Treatment Comparison DBF (Test) versus D | ORG (Reference) Following |
| Different Meal Conditions | 24 |
| 11. Percentages and Decimal Places | 25 |
| 12. Data Handling | 26 |
| 13. Handling of Missing Data | 27 |
| 14. Software to be Used | 28 |
| 15. Reference List | 29 |

Statistical Analysis Plan Aquestive Therapeutics Project No. 180323

#### LIST OF ABBREVIATIONS

**A** Abnormal

**AE** Adverse event

**AED** Antiepileptic drug

**ALP** Alkaline phosphatase

**ALT** Alanine aminotransferase

**ANOVA** Analysis of variance

**AST** Aspartate aminotransferase

**AUC** Area under the concentration-time curve

**AUC**<sub>0-inf</sub> Area under the concentration-time curve from time 0 to infinity (extrapolated)

 $AUC_{0-t}$  Area under the concentration-time curve from time 0 to the last non-zero

concentration

**BLQ** Below the lower limit of quantitation

BMI Body mass index
BP Blood Pressure
CK Creatine Kinase

CI/F Apparent total clearance

Cl/F/kg Apparent total clearance normalized for the subject body weight in kg

C<sub>last</sub> The last observed non-zero concentration
C<sub>max</sub> Maximal observed plasma concentration

**CSR** Clinical study report

CV Coefficient of variation (equivalent to C.V.)

DBF Diazepam Buccal Film
 DRG Diastat® Rectal Gel
 ECG Electrocardiogram

**FDA** Food and Drug Administration

H Above normal range

**HBsAg** Surface Antigen of the Hepatitis B Virus

**HCV** Human Hepatitis C Virus

**HEENT** Head, eyes, ears, nose and throat **HIV** Human immunodeficiency virus

**HR** Heart rate

**K**<sub>el</sub> Terminal elimination rate constant

 $K_{el \ Lower}$  The actual sampling time where  $K_{el}$  calculation begins

 $\mathbf{K}_{\text{el Upper}}$  The actual sampling time of the last measurable concentration used to estimate  $\mathbf{K}_{\text{el}}$ 

kg Kilogram



Aquestive Therapeutics

L Below normal range (conflicting with Liter)

Max Maximum (equivalent to max.)

MDMA 3,4-methylenedioxy-N-methylamphetamine MedDRA® Medical Dictionary for Regulatory Activities

mg Milligram

Min Minimum (equivalent to min.)

mL Milliliter

N Number of observations

PCP Phencyclidine
PK Pharmacokinetic

PT MedDRA® Preferred Term

**QUALIFIED INVESTIGATOR** 

**QRS** The QRS complex is a structure on the ECG that corresponds to the depolarization

of the ventricles

**QT** Time from electrocardiogram Q wave to the end of the T wave corresponding to

electrical systole

**QTcB** QT Corrected with Bazett formula

**QTcF** QT Corrected with Fridericia's formula

**RR** Respiratory Rate

SAE Serious Adverse Event
SAP Statistical Analysis Plan
SAS® Statistical Analysis System

**SD** Standard Deviation

SOC MedDRA® System Organ ClassSOP Standard Operating Procedure

**TEAE** Treatment-Emergent Adverse Event

T<sub>½ el</sub> Elimination half-life
THC Tetrahydrocannabinol

T<sub>max</sub> Time of maximal observed plasma concentration

vs Versus

 $V_d/F$  Apparent volume of distribution

 $V_d/F/kg$  Apparent volume of distribution normalized for the subject body weight in kg

**WHO DD** World Health Organization Drug Dictionary



Aquestive Therapeutics

#### 1. Introduction

This statistical analysis plan (SAP) is intended to give a detailed description of the summaries and the analyses that will be generated for the present study by inVentiv. Analyses specified in this plan are based on Aquestive Therapeutics study Protocol No. 180323 Amendment III, dated 24 May 2019 (inVentiv Project No. 180323). Safety, tolerability and pharmacokinetic (PK) analyses will all be described.

The plan may change due to unforeseen circumstances and any changes made after the plan has been finalized will be documented. If additional analyses are required to supplement the planned analyses described in the SAP, the changes and justification for the changes will be outlined in the clinical study report (CSR). No change will be made without prior approval of the study sponsor. No revision to the SAP is required for changes which do not affect the statistical analysis methods, definitions, or rules defined in this document.

When applicable, all methodology and related processes will be conducted according to inVentiv's Standard Operating Procedures (SOPs). Protocol deviations occurring during the study will be listed.

Shells for all statistical tables, figures and listings referred to in this SAP will be displayed in a separate document.

Aquestive Therapeutics

#### 2. Study Objectives

#### 2.1 Primary Objective

• Evaluate the pharmacokinetics (PK) of single doses of Diazepam Buccal Film (DBF) at the recommended dose regimen (range 10 mg to 17.5 mg according to body weight) compared with Diastat<sup>®</sup> Rectal Gel (DRG) at the labeled dose regimen (range 10 mg to 20 mg according to body weight) in adult male and female subjects on a stable concomitant regimen of antiepileptic drugs (AED) for the treatment of epilepsy, following a moderate-fat meal.

#### 2.2 Secondary Objectives

- Evaluate the PK of single doses of DBF following a high-fat meal compared with DRG following a moderate-fat meal at the recommended dose regimen in adult male and female subjects on a stable concomitant regimen of AED for the treatment of epilepsy.
- Assess the safety-tolerability of single doses of DBF and DRG administered to adult male and female subjects on a stable concomitant regimen of AEDs under fed conditions.

Aquestive Therapeutics

#### 3. Study Design

#### 3.1 General Design

This will be a randomized, multiple centers, single-dose, open-label, three-period, three treatment, two-sequence crossover study under fed conditions.

The study will evaluate single doses of DBF compared with DRG administered according to weight category in adult male and female subjects on a stable concomitant regimen of AED for the treatment of epilepsy. A stable regimen of AED is defined as no change in the prescribed AED regimen during the 30 day period prior to the first study drug administration and no change anticipated in the prescribed AED regimen over the course of study participation until the last PK blood sample collection.

Subjects will receive Treatment A and Treatment B (DBF and DRG following a moderate-fat meal) in Period 1 and Period 2 in a randomized sequence, and at a dosage specific to body weight. DBF will be administered according to the currently recommended dose regimen (derived by Aquestive from population PK modeling in healthy volunteers). DRG will be administered depending on weight category according to the current product labeling for Diastat<sup>®</sup>. Subjects may be asked to participate in a third period, on a voluntary basis. Subjects who volunteer to participate in a third period will receive a second dose of DBF administered in exactly the same manner as the earlier dose of DBF with the exception that DBF in Period 3 will be administered following a high-fat meal. There will be a washout of 28 days between doses.

A maximum of 32 eligible subjects will be enrolled in an effort to complete Period 2 with at least 16 subjects with representation of both genders, representation across the five weight categories of subjects taking one or more AEDs known to induce diazepam metabolism, and representation of subjects taking sodium divalproex/valproic acid. Subjects who are eligible may be enrolled without regard to weight category. Since only exploratory PK data will be gathered from treatment period 3, no more than 50% of the subjects who complete Period 1 and Period 2 will participate in Period 3.

This study is intended for filing under FDA regulations.

#### 3.2 Study Procedures

The overall schedule of procedures and assessments is provided in the protocol.

#### 3.3 Treatment Description

Subjects will be administered each treatment according to the 3-period, 2-sequence, block randomization scheme produced by inVentiv. At admission to the clinic, subjects who meet the inclusion/exclusion criteria will be assigned between the 2-sequence arms (ABC or BAC) according to the randomization schedule. inVentiv will inform the site about the medication to be dispensed to each particular subject at the time of subject's randomization and at the prospective

Aquestive Therapeutics

protocol visits. The clinic will administer the study treatment as described in Table 3-1, according to the subject's weight obtained at screening visit.

The randomization code will not be available to the Bioanalytical Division until the clinical and analytical phases of the study have been completed.

Table 3-1 Study Treatment Administration According to Weight Category

| Product | Meal<br>Condition | Weight<br>Category | Weight (kg) | Dose |
|---|---|---|---|---|
| Test (Treatment A): | Moderate-Fat | A1 | 38-50 | 1 x 10 mg |
| Diazepam Buccal Film | Meal | A2 | 51-62 | 1 x 12.5 mg |
| (Aquestive Therapeutics, USA) | | A3 | 63-75 | 1 x 15 mg |
| | | A4 | 76-87 | 1 x 15 mg |
| | | A5 | 88-111* | 1 x 17.5 mg |
| Reference (Treatment B): | Moderate-Fat | B1 | 38-50 | 2 mL (10 mg) |
| Diastat® AcuDial <sup>TM</sup> rectal gel | Meal | B2 | 51-62 | 2.5 mL (12.5 mg) |
| (Valeant Pharmaceuticals, USA) | | В3 | 63-75 | 3 mL (15 mg) |
| | | B4 | 76-87 | 3.5 mL (17.5 mg) |
| | | B5 | 88-111* | 4 mL (20 mg) |
| Test (Treatment C): | High-Fat | A1 | 38-50 | 1 x 10 mg |
| Diazepam Buccal Film | Meal | A2 | 51-62 | 1 x 12.5 mg |
| (Aquestive Therapeutics, USA) | | A3 | 63-75 | 1 x 15 mg |
| | | A4 | 76-87 | 1 x 15 mg |
| | | A5 | 88-111* | 1 x 17.5 mg |

<sup>\*</sup>Subjects eligible for study with weights in the range of 112 to 134 kg will be dosed at the 88-111 kg weight range as shown above.

#### 3.4 Sample Size

Subjects will be enrolled to attain a sample size of no more than 32 subjects (and a minimum of 16 completed subjects in Period 2). Because this is not a formal hypothesis testing study, the sample size is proposed based on the desired level of precision for estimating pharmacokinetic parameters and the relationship between pharmacokinetic parameters. In principle, the expected precision of the estimates of the ratios of geometric means of interest can be estimated from the intra-subject variability observed in Aquestive Study 162021 (pharmacokinetic crossover of DBF 15 mg with DRG 5, 12.5, and 20 mg in healthy volunteers). Aquestive has not undertaken a formal analysis to predict the expected precision.



Aquestive Therapeutics

#### 3.5 Subject Withdrawal and Replacement

Subjects will be advised that they are free to withdraw from the study at any time. Over the course of the study, the Sponsor and the Investigator or a delegate may withdraw any subject from the study for one of the reasons described below:

- safety reason;
- non-compliance with protocol requirements;
- significant protocol deviation;
- positive alcohol breath test;
- positive drug screen (except for subjects using prescribed marijuana and THC containing products as AED treatment);
- positive pregnancy test.

Positive result to the urine benzodiazepine screen (urine drug screen) in Period 2 and Period 3 may derive from residual concentrations from study drug administered in the previous period(s). Therefore, it is not required that subjects with a positive result to that test in Period 2 and Period 3 be withdrawn from the study. Continued subject participation in the study will be evaluated by the Principal Investigator.

Subjects experiencing emesis within 4 hours following DBF administration will be evaluated on a case-by-case basis by the Principal Investigator/Sub-Investigator, the CRO PK Scientist, and the Sponsor, and a decision on their continued participation will be made. Subjects experiencing a bowel movement within 4 hours following DRG administration or clinically significant leakage of the rectal gel within 4 hours post-dose will be evaluated on a case-by-case basis by the Principal Investigator/Sub-Investigator, the CRO PK Scientist, and the Sponsor, and a decision on their continued participation will be made. All decisions will be made prior to the bioanalytical laboratory commencing bioanalysis.

Subjects who withdraw or are withdrawn from the study after dosing will not be replaced. However, in the event that the number of drop-outs exceeds initial expectations, subjects who withdraw or are withdrawn might be replaced at the discretion of the Sponsor. Such replacement resulting in dosing of more subjects than planned in this protocol would be documented in a protocol amendment.

Subjects who withdraw or are withdrawn will be asked to remain at the clinic until the Investigator or a delegate agrees that the subject is fine and can be discharged. As soon as subject withdrawal is confirmed, blood sampling will be stopped. Study exit procedures will be performed at the time of withdrawal from the study or as soon as possible thereafter.



Aquestive Therapeutics

### 4. Change From the Protocol

No changes in planned analyses were done compared to the protocol. However, for B vs C comparison, the period will not be included in the ANOVA since Treatment C is confounded with Period 3.



Aquestive Therapeutics

#### 5. Primary and Secondary Parameters

For PK analyses (A vs B comparison),  $AUC_{0-t}$ ,  $AUC_{0-inf}$ , and  $C_{max}$  calculated using diazepam plasma concentrations will be regarded as the primary endpoints. All other PK parameters (including those calculated using nordiazepam) will be regarded as secondary endpoints (refer to Section 10.3).

The safety and tolerability parameters will be regarded as secondary endpoints (refer to Section 9).



Aquestive Therapeutics

#### 6. Analysis Populations

The analysis of safety and tolerability parameters will be based on the safety population detailed in Section 6.1 below. The analysis of PK parameters will be based on the PK population detailed in Section 6.2 below. Treatment assignment will be according to the actual treatment received.

#### 6.1 Safety Population

The safety population is defined as all subjects who received at least one dose of the study medication.

#### 6.2 Pharmacokinetic Population and Pharmacokinetic Analysis Data Set

The pharmacokinetic population will include all subjects completing at least Period 1 and Period 2 with no significant violation of study restrictions, and for whom the pharmacokinetic profile can be adequately characterized. Any subject who completes only one period will be presented in the concentrations and pharmacokinetic tables but excluded from descriptive statistics and ANOVA.

A violation of the requirement to maintain a stable regimen of AEDs or a stable regimen of other concomitant drugs with the potential to influence diazepam pharmacokinetics will be considered a significant violation of study restrictions. A change of drug in the prescribed AED regimen and/or change in the dose of a prescribed AED will be considered a departure from a stable regimen. Any subject who does not maintain a stable AED regimen in the course of the study will be presented in the concentrations and pharmacokinetic tables but excluded from descriptive statistics and ANOVA. For cases in which a departure from a stable AED regimen is a matter of judgment, the decision will be made by the Principal Investigator/Sub-Investigator and/or by the CRO PK Scientist in consultation with the Sponsor prior to bioanalysis.

Any subject with diazepam or nordiazepam pre-dose concentrations will be presented in the concentrations and pharmacokinetic tables but excluded from descriptive statistics and ANOVA if the pre-dose concentration is greater than 5% of the  $C_{max}$  value for that analyte of that period for that subject.

Subjects withdrawn due to vomiting episodes as per criterion established under section 3.5 or due to adverse events will be presented but excluded from the statistical analyses (i.e., descriptive statistics and ANOVA).

Data from subjects who experienced emesis during the sampling interval and who were not withdrawn as per criterion established under section 3.5 may be evaluated after completion of the pharmacokinetic analysis. Any subject who experienced emesis within 2 times median  $T_{max}$  of the current study (based on the reference product) will be excluded from the statistical analysis (i.e., descriptive statistics and ANOVA).

Aquestive Therapeutics

## 7. Interim Analyses

No interim analysis will be performed.



Aquestive Therapeutics

#### 8. Study Population and Exposure

No inferential analysis will be done. Only observed data will be used.

#### 8.1 Subject Disposition

Subject disposition will be summarized for the number of subjects who were screened, enrolled, randomized and dosed, completed the study, and who were withdrawn from the study and the reason. The data will be presented by treatment and overall (frequency and the percentage of subjects) and listed.

#### 8.2 Protocol Deviations

The protocol deviations will be categorized and listed by subject.

#### 8.3 Demographics and Baseline Characteristics

The descriptive statistics (mean, median, standard deviation [SD], minimum [Min], maximum [Max], and sample size) will be calculated for continuous variables (age, body mass index [BMI], height, and weight) considering last results (scheduled or unscheduled) obtained at screening. Frequency counts and percentages will be tabulated for categorical variables (age group, gender, ethnicity, and race). Results will be presented overall and by treatment group for each study population (only if populations are different). All demographic characteristics will be listed by subject.

#### **8.4** Medical History

Medical history at screening will be listed by subject. The Medical Dictionary for Regulatory Activities (MedDRA®) Version 21.1 will be used to classify all medical history findings by System Organ Class (SOC) and Preferred Term (PT).

#### 8.5 Prior and Concomitant Medications

The use of prior and/or concomitant medications will be monitored throughout the study and listed by subject. The World Health Organization Drug Dictionary (WHO DD) Version Sep2018, format B3 will be used to classify all medication reported during the study.

#### 8.6 Study Drug Administration

The study drug administration details (including treatment received, start and end date and time of administration) will be listed by subject. The time of dosing will be set as the time the film is placed against the buccal mucosa.



Aquestive Therapeutics

#### 9. Safety Analyses

Safety and tolerability data will be evaluated through the assessment of AEs, clinical laboratory parameters (biochemistry, hematology, and urinalysis), 12-lead electrocardiogram (ECG), vital sign (blood pressure, heart rate, respiratory rate, pulse oximetry, and oral temperature), continuous cardiac ECG monitoring, physical examination, and visual oral inspection. Laboratory parameters, vital signs, and ECG parameters will be listed and summarized using descriptive statistics. All AEs will be listed and summarized using descriptive methodology. The incidence of AEs for each treatment will be presented by severity and association with the study drug.

Safety data will be summarized but will not be subjected to inferential analysis. The analysis of the safety variables will be based on safety population.

#### 9.1 Physical Examination Findings

A physical examination will be performed at screening and study exit. The physical examination includes at least the following components: HEENT (head, eyes, ears, nose, and throat), neck, chest and lungs, cardiovascular, abdomen, skin, and musculoskeletal evaluation.

A brief neurologic examination will be performed at screening and study exit. The neurologic assessment involves at least the following evaluation: mental status, cranial nerves, motor system, sensory system, cerebellar disorder, gait, and reflexes.

Any abnormal findings judged to be clinically significant will be documented as medical history or as an AE, depending upon whether noted at screening, prior to dosing or after dosing, as appropriate. Any physical examination findings documented as AEs will be included in the AE summaries.

#### 9.2 Adverse Events

Treatment-emergent AEs (TEAEs) and non-TEAEs (those occurring prior to administration of study medication or that first occurred prior to study drug administration and did not worsen in frequency or severity) will be listed. TEAEs will be defined as AEs that occur on or after the date and time of study drug administration, or those that first occur pre-dose but worsen in frequency or severity after study drug administration. AEs will be collected and documented from the signing of the ICF until at least 10 days following the last study drug administration, and as observed or reported spontaneously by study participants. TEAEs will be attributed to the most recent study drug taken. A TEAE with a start date and time during the wash-out period (ending at the time of study drug administration) will be attributed to the study drug taken during the previous treatment period. Any AEs, whether serious or non-serious, will be monitored throughout the study and followed to resolution or for up to 2 weeks after the last PK blood draw, after which the Investigator will decide the course of action.



Aquestive Therapeutics

The incidence of TEAEs will be summarized using the safety population. The MedDRA® dictionary Version 21.1 will be used to classify all AEs reported during the study by SOC and PT.

Incidence of subjects who experienced TEAEs (as well as number of events) will be presented by treatment and overall, by SOC, and PT, investigator-assessed relationship and also by severity. Each subject may only contribute once to each of the incidence rates, for a TEAE following a given treatment, regardless of the number of occurrences; the highest severity or highest relationship will be presented, as appropriate. In each table, SOC will be presented in descending order of overall incidence rate in terms of frequency of subjects and then in frequency of events (alphabetical order will be used in case of equal rates). For each SOC, PT will be presented the same way.

The relationship of an AE to the study drug will be assessed according to the study protocol as:

Probable: A clinical event, including laboratory test abnormality, with a reasonable

time sequence to drug administration, unlikely to be attributed to concurrent disease or other drugs or chemicals, and which follows a

clinically reasonable response on withdrawal.

Possible: A clinical event, including laboratory test abnormality, with a reasonable

time sequence to drug administration, but which could also be explained by

concurrent disease or other drugs or chemicals. Information on drug

withdrawal may be lacking or unclear.

Unlikely: A clinical event, including laboratory test abnormality, with a temporal

relationship to drug administration which makes a causal relationship improbable, and which other drugs, chemicals or underlying disease

provide plausible explanation.

Unrelated: This category is applicable to AEs which are judged to be clearly and

incontrovertibly due to extraneous causes (diseases, environment, etc.) and do not meet the criteria for drug relationship listed for the above-mentioned

conditions.

The Severity of AEs will be rated as according to the study protocol as:

Mild: AE resulting in discomfort, but not sufficient to cause interference in

normal daily activities.

Moderate: AE resulting in discomfort that is sufficient to cause interference in daily

activities.

Severe: AE resulting in discomfort causing an inability to carry out normal daily

activities.



Aquestive Therapeutics

A significant AE will be defined as any event (other than those reported as serious) that led to an intervention, including withdrawal of treatment, or significant additional concomitant therapy. Serious and significant AEs will be listed separately.

#### 9.3 Laboratory Parameters

Clinical laboratory (biochemistry, hematology, and urinalysis) results will be obtained at screening, and at study exit or early termination.

Biochemistry parameters include the following: albumin, alkaline phosphatase (ALP), aspartate aminotransferase (AST), alanine aminotransferase (ALT), urea, calcium, chloride, glucose, phosphorus, potassium, creatinine, sodium, total bilirubin, CK, lactate dehydrogenase, uric acid, total protein, magnesium, bicarbonates, and ammonia.

Hematology parameters include the following: complete blood count with differential, hemoglobin, hematocrit and platelet count.

Urinalysis parameters include the following: macroscopic examination, pH, specific gravity, protein, glucose, ketones, bilirubin, occult blood, nitrite, and leukocytes. Unless otherwise specified, microscopic examination will be performed on abnormal findings and results will be listed.

Hepatitis B (HBs Ag), Hepatitis C (HCV) antibody, and HIV antigen and antibody detection will be performed at screening.

A urine drug screen (amphetamines, methamphetamines, barbiturates, benzodiazepines, tetrahydrocannabinol, cocaine, opiates, Phencyclidine (PCP), 3, 4-methylenedioxy-N-methylamphetamine (MDMA), methadone), and an alcohol breath test will be performed at screening and before dosing of each period.

A urine pregnancy test will be performed at screening and at study exit, and a serum pregnancy test will be performed at check-in of each period.

Listings of all clinical laboratory (biochemistry, hematology, and urinalysis) results will be provided with the abnormal values flagged with "L" (low) and "H" (high) for continuous parameters, and "A" (abnormal) for categorical parameters.

Descriptive statistics (mean, median, SD, Min, Max, and sample size) for each clinical laboratory test (continuous variables) will be presented overall for screening and study exit visit. Descriptive statistics for change from screening will also be presented for study exit. Screening includes the last screening results (scheduled or unscheduled). For categorical variable (urinalysis test), the number of subjects (frequency and percentage) will be tabulated by results (e.g. negative, positive, trace...). A summary table of shifts from screening to study exit visit will be provided. Results from repeat or unscheduled tests will not be included in the summary statistics unless the repeat was required (and documented as such) due to technical reasons or an



Aquestive Therapeutics

invalid initial result, or for screening determination, if applicable. Early termination results (if any) will be included with the study exit visit for the summary statistics.

If more than one clinical laboratory is used for the study, a formula that takes into consideration the relative normal ranges of each test of laboratories used will be applied in order to normalize these data. The conversion formula used will depend on the typical distribution of the normal range for each laboratory test; the two formulae used are presented below:

Hemoglobin, hematocrit, and platelet count test results are considered to have a normal distribution (Chuang-Stein, 1992) and the following formula will be used (Karvanen J., 2003):

$$s = L_s + (x-L_x) \frac{U_s-L_s}{U_x-L_x}$$

Where U= Upper limit; L= Lower limit; s= Primary facility result; and x= Secondary facility results.

The remaining hematology, serum chemistry, and urinalysis test results are considered to have a non-normal distribution (Chuang-Stein, 1992) and the following formula will be used (Karvanen J., 2003):

$$s = \frac{x U_s}{U_x}$$

Prior to applying these formulae, if required, units will be adjusted.

#### 9.4 Vital Signs

Vital signs measurements (blood pressure (BP), heart rate (HR), respiratory rate (RR)) and digital oxygen monitoring will be measured in a sitting position (except for safety reasons) at screening, and at study exit or early termination. Oral temperature will be measured at screening, and at study exit or early termination.

Vital signs and digital oxygen monitoring will be measured before dosing and approximately 0.5, 1, 1.5, 2, 4, and 8 hours post-dose (and beyond if clinically indicated). Vital signs will also be measured approximately 12 and 24 hours post-dose.

Descriptive statistics (mean, median, SD, Min, Max, and sample size) will be presented overall for screening and study exit, and by associated current treatment for on-study measurements for each parameter where applicable. Descriptive statistics for change from screening to study exit, and for change from baseline for on-study measurements will also be presented. Screening includes the last screening results (scheduled or unscheduled). Baseline will be defined as the last results (scheduled or unscheduled) obtained prior to drug administration in each period. Results from repeat or unscheduled tests will not be included in the summary statistics unless the repeat was required (and documented as such) due to technical reasons or an invalid initial result,



Aquestive Therapeutics

or for screening or baseline determination, if applicable. Early termination results (if any) will be included with the study exit visit for the summary statistics.

A listing of all vital signs results will be provided.

#### 9.5 Electrocardiogram

Supine ECG will be performed at screening and study exit. Continuous ECG monitoring will be performed from approximately 1 hour prior to dosing until 8 hours post-dose (and extended if clinically indicated).

For supine ECG, descriptive statistics (mean, median, SD, Min, Max, and sample size), for each ECG parameter (heart rate, PR interval, QRS interval, QT interval, and QTcF interval) will be presented overall for screening and study exit visit. Descriptive statistics for change from screening will also be presented for study exit. Screening includes the last screening results (scheduled or unscheduled). Results from repeat or unscheduled tests will not be included in the summary statistics unless the repeat was required (and documented as such) due to technical reasons or an invalid initial result, or for screening determination, if applicable. Early termination results (if any) will be included with the study exit visit for the summary statistics. A listing of all supine ECG results will be provided.

#### 9.6 DBF Application Site Inspection

The Investigator or designee will make a visual inspection of the oral mucosa at screening. The application site will also be inspected prior to DBF administration and approximately 6 and 24 hours after administration. Assessments of the oral mucosa (normal/abnormal) will be conducted by the Principal Investigator/Sub-Investigator or a trained nurse. A listing will be provided.

Abnormalities observed before dosing will be recorded and evaluated regarding exclusion criteria but will not be considered AEs. Any post-dose abnormalities will be reported as AEs and followed until resolution.

Aquestive Therapeutics

#### 10. Pharmacokinetic Analyses

## 10.1 Handling of the Below the Lower Limit of Quantitation (BLQ) and the No Reportable Concentration Values

All concentration values BLQ will be set to zero, except when they occur between two non-BLQ concentrations where they will be considered as missing for pharmacokinetic calculations. Samples with no reportable value occurring prior to dosing for a given period will be replaced by "0.00", otherwise they will be set to missing for tabulation, graphical representation and calculation purposes. All samples with no reportable value observed after dosing will be set to missing.

#### 10.2 Handling of the Difference Between the Scheduled and the Actual Sampling Times

The actual clock time for dosing and the actual clock time for each collection time for the PK samples will be recorded using the electronic data capture. For all sampling times, the actual sampling times will be calculated as the difference between the sample collection actual clock time and the actual clock time of dosing. The actual post-dose sampling times expressed in hours and rounded off to three decimal digits will be used to calculate the PK parameters, except for pre-dose samples occurring prior to dosing, which will always be reported as zero (0.000), regardless of the time difference. In the PK section of the report, scheduled sampling times will be presented in concentration tables and mean graphs while actual times are presented for the individual graphs. A listing of the actual times for PKs will be provided for PK samples.

#### 10.3 Pharmacokinetic Parameters

In each period, a total of 19 blood samples will be drawn from each subject for pharmacokinetic analyses. Blood samples will be collected prior to study drug administration (0.00 hour) and 0.500, 0.750, 1.00, 1.50, 2.00, 3.00, 4.00, 6.00, 9.00, 12.0, 24.0, 48.0, 72.0, 96.0, 120, 144, 192, and 240 hours post-dose (3 mL for each sampling time). The time tolerance window for blood samples collected during the confinement period will be  $\pm 1$  minute for all samples collected before 8 hours post-dose and  $\pm 3$  minutes for subsequent samples. The time tolerance window for return visit samples will be  $\pm 60$  minutes. Blood samples will be collected as close as possible to nominal times; exact sample collection times will be recorded on the appropriate source documents and reported for each subject. The actual time of blood sample collection will be used for PK and statistical analysis.

Plasma concentrations from diazepam and nordiazepam will be used to calculate the following PK parameters by standard non-compartmental methods:

 $AUC_{0-t}$  Area under the concentration-time curve from time zero to the last non-zero

concentration and it is calculated using the linear trapezoidal method.

AUC<sub>0-inf</sub> Area under the concentration-time curve from time zero to infinity

(extrapolated), calculated as  $AUC_{0-t} + C_{last} / K_{el}$ , where  $C_{last}$  is the last

observed non-zero concentration.



Statistical Analysis Plan Aquestive Therapeutics
Project No. 180323

C<sub>max</sub> Maximal observed plasma concentration.

Residual Area Residual area, calculated as 100\*(1- AUC<sub>0-inf</sub>).

 $T_{\text{max}}$  Time when the maximal plasma concentration is observed.

K<sub>el</sub> Elimination rate constant. This parameter will be the negative of the

estimated slope of the linear regression of the ln-transformed concentration versus time profile in the elimination phase. Four non-zero observations during the elimination phase (excluding the  $C_{max}$ ) will be used to calculate  $K_{el}$ , or a minimum of 3 concentration points will be used if fewer than four observations are available. The time point where ln-linear  $K_{el}$  calculation begins ( $K_{el \ Lower}$ ), and the actual sampling time of the last quantifiable concentration used to estimate the  $K_{el}$  ( $K_{el \ Upper}$ ) will be reported with the

correlation coefficient from the linear regression to calculate K<sub>el</sub>

(Correlation).

 $T_{\frac{1}{2} \text{ el}}$  Elimination half-life, calculated as  $\ln(2) / K_{\text{el}}$ .

Cl/F Apparent total clearance, calculated as Dose / AUC<sub>0-inf</sub>.

Cl/F/kg Apparent total clearance normalized for the subject body weight in kg,

calculated as (Cl/F) / weight.

V<sub>d</sub>/F Apparent volume of distribution, calculated as Dose/(K<sub>el</sub> x AUC<sub>0-inf</sub>)

V<sub>d</sub>/F/kg Apparent volume of distribution normalized for the subject body weight in

kg, calculated as  $(V_d/F)$  / weight.

For subjects with missing or non-reportable concentrations for three or more of the last samples (e.g. timepoints pass  $T_{max}$ ), the data will be reviewed on a case-by-case basis by inVentiv pharmacokinetic scientist and/or sponsor to determine if the data are reliable for  $C_{max}$  and  $T_{max}$ . If so, only the  $C_{max}$  and  $T_{max}$  will be presented and included in the statistical analysis. Other PK parameters will not be reported. Explanations for PK parameters that could not be estimated will be provided in the CSR.

Additional PK analysis may be performed.

#### 10.4 Statistical Analyses

Individual and mean plasma concentration versus time curves will be presented for both linear and semi-log scales for diazepam and nordiazepam. Descriptive statistics (arithmetic and geometric means, SD, coefficient of variation [CV (%)], Min, Max, and median) of the plasma concentrations versus time will be presented as well for the PK parameters for diazepam and nordiazepam.



Aquestive Therapeutics

## 10.4.1 Treatment Comparison DBF (Test) versus DRG (Reference) Following a Moderate-Fat Meal

The statistical analyses below will include only data from subjects completing both Treatments A and B.

For diazepam and nordiazepam, using GLM procedures in SAS, ANOVA will be performed on untransformed  $T_{max}$ ,  $K_{el}$ , and  $T_{\frac{1}{2}el}$  and on ln-transformed  $AUC_{0-t}$ ,  $AUC_{0-inf}$ ,  $C_{max}$ , Cl/F, Cl/F/kg,  $V_d/F$ , and  $V_d/F/kg$  at the alpha level of 0.05. Factors incorporated in the model will include: Sequence, Subject(Sequence), Period, and Treatment.  $T_{max}$  will be analyzed using an additional non-parametric test (Wilcoxon signed-rank test).

The ratio of geometric means will be calculated for  $AUC_{0-t}$ ,  $AUC_{0-inf}$ , and  $C_{max}$  for the Test product versus the Reference product (Treatment A/Treatment B) irrespective of weight category. The 90% confidence interval for the ratio of geometric means, based on least-squares means from the ANOVA of the ln-transformed data will also be calculated. Intra and intersubject coefficient of variation will be estimated.

## 10.4.2 Treatment Comparison DBF (Test) versus DRG (Reference) Following Different Meal Conditions

An exploratory pair-wise analysis comparing DBF following a high-fat meal (Treatment C) with DRG following a moderate-fat meal (Treatment B) will be conducted and reported. The statistical analyses below will include only data from subjects completing both Treatments B and C.

For diazepam and nordiazepam, using GLM procedures in SAS, ANOVA will be performed on untransformed  $T_{max}$ ,  $K_{el}$ , and  $T_{\frac{1}{2}el}$  and on In-transformed AUC<sub>0-t</sub>, AUC<sub>0-inf</sub>,  $C_{max}$ , Cl/F, Cl/F/kg,  $V_d$ /F, and  $V_d$ /F/kg at the alpha level of 0.05. Factors incorporated in the model will include: Sequence, Subject(Sequence), and Treatment.  $T_{max}$  will be analyzed using an additional non-parametric test (Wilcoxon signed-rank test).

The ratio of geometric means will be calculated for  $AUC_{0-t}$ ,  $AUC_{0-inf}$ , and  $C_{max}$  for Treatment C versus Treatment B, irrespective of weight category. The 90% confidence interval for the ratio of geometric means, based on least-squares means from the ANOVA of the ln-transformed data will also be calculated. Intra and inter-subject coefficient of variation will be estimated.

Additional analyses may be performed.



Aquestive Therapeutics

#### 11. Percentages and Decimal Places

If not otherwise specified, the following rules will be applied, with the exception of PK tables and listings described below:

- Percentages will be presented to one decimal point.
- Percentages equal to 0 or 100 will be presented as such without a decimal point.
- Minimum and maximum will be presented with the same precision as the original values and, mean, standard deviation, and median will be presented with one more decimal place than the original values.

All digits will be used for pharmacokinetic and statistical PK calculations. For PK tables and listings, the final reportable results or data will be presented by rounding off to two decimal digits, except for the following situations (this applies to individual data and descriptive statistics):

- K<sub>el</sub> data: rounded off to four decimal digits.
- Pharmacokinetic parameters related to time such as T<sub>max</sub> must be reported with the same precision as the actual sampling time: rounded off to 3 decimal digits.
- Concentration versus time data, as well as C<sub>max</sub>: reported as they appear in corresponding dataset.
- Ratios and 90% confidence intervals, CV (%), Inter-CV%, Intra-CV% will be presented to two decimal places.

Aquestive Therapeutics

### 12. Data Handling

The PK plasma concentrations, safety and tolerability data will be received as SAS® datasets from the inVentiv data management facility. Screening failures and ineligible volunteer's data (subject disposition) will be received from the clinical site as source data.



Aquestive Therapeutics

#### 13. Handling of Missing Data

For PK, only observed data will be used in the data analysis except for concentration values BLQ and samples with no reportable value occurring prior to dosing as described in Section 10.1. No attempt will be made to extrapolate or interpolate estimates for missing data.

For safety,

- If an AE is recorded with an onset date corresponding to a dosing day, but the time is missing, then the AE will be assigned to the treatment.
- If an AE is recorded with an onset date that does not correspond to the dosing day, but the time is missing, then the AE will be assigned to the treatment if AE onset date is after dosing date.
- If an AE is recorded with an onset date where day and time are both missing, then the AE allocation to the treatment will be done on a case by case basis considering available information (e.g., AE onset date, AE end date, AE comments, subject disposition).



Aquestive Therapeutics

#### 14. Software to be Used

PK analysis will be performed using Phoenix WinNonlin® version 8.0 or higher, which is validated for bioequivalence/bioavailability studies by inVentiv. Inferential statistical analyses will be performed using SAS® according to FDA guidelines. The safety data tables and listings, as well as PK tables and listings will be created using SAS®, release 9.2 or a higher version. PK figures will be created using R version 3.5. The report text will be created using Microsoft® Office Word 2010, or a higher version.

Aquestive Therapeutics

#### 15. Reference List

- Chuang-Stein C. Summarizing laboratory data with different reference ranges in multi-center clinical trials. Drug Information Journal. 1992; 26:77-84.
- Karvanen J. The statistical basis of laboratory data normalization. Drug Information Journal. 2003; 37:101-107.

## **Table/Figure/Listing Shells**

#### Table/Figure/Listing Shells

A RANDOMIZED, OPEN-LABEL, 2-SEQUENCE, 3-TREATMENT, CROSSOVER STUDY TO EVALUATE THE PHARMACOKINETICS OF SINGLE DOSES OF DIAZEPAM BUCCAL FILM (DBF) (AQUESTIVE THERAPEUTICS) COMPARED WITH DIASTAT® RECTAL GEL (VALEANT PHARMACEUTICALS NORTH AMERICA) IN ADULT MALE AND FEMALE SUBJECTS ON A CONCOMITANT REGIMEN OF ANTIEPILEPTIC DRUGS (AED) FOR THE TREATMENT OF EPILEPSY

Sponsor Protocol No. 180323 inVentiv Health Clinical Inc. Project No. 180323

Final Version: 1.0 Date: 28-JUN-2019

Contract Research Organization: inVentiv Health Clinique Inc. ("inVentiv"), a Syneos Health company 2500, rue Einstein Québec (Québec) Canada, G1P 0A2

Sponsor: Aquestive Therapeutics 30 Technology Drive Warren, NJ 07059 USA

#### CONFIDENTIAL

**Aquestive Therapeutics** 

#### **SIGNATURES**

Sponsor Protocol No. 180323

inVentiv Project No.: 180323

Study Title: A Randomized, Open-Label, 2-Sequence, 3-Treatment, Crossover Study to
Evaluate the Pharmacokinetics of Single Doses of Diazepam Buccal Film
(DBF) (Aquestive Therapeutics) Compared With Diastat® Rectal Gel (Valeant
Pharmaceuticals North America) in Adult Male and Female Subjects on a
Concomitant Regimen of Antiepileptic Drugs (AED) for the Treatment of
Epilepsy

Author:

Siva Durga Prasad Sattu, M.Sc.

Statistician inVentiv

Signature:

Date: 01 Tul 9019

Sponsor's

Representative: Allen H Heller, MD, MPH

Founder and CEO, Pharma Study Design LLC (Consultant to Aquestive

Therapeutics)



Aquestive Therapeutics

### TABLE OF CONTENTS

| SIG | SNATURES | 2 |
|-----|----------------------------------------------|----|
| TAI | BLE OF CONTENTS | 3 |
| 1. | Tables, Figures and Data Listings Formatting | 4 |
| | Table 1-1 Layout Specifications | 4 |
| 2. | Summary TFLs | 5 |
| | Table 2-1 List of Table Shells | |
| | Table 2-2 List of Figures Shells | 7 |
| | Table 2-3 List of Data Listings Shells | 8 |
| 3. | CSR In-text Tables | 9 |
| 4. | Summary Tables | 14 |
| 5. | Figures | 36 |
| 6. | Listings | 43 |

Aquestive Therapeutics

#### 1. Tables, Figures and Data Listings Formatting

The table, figure, and data listing (TFL) shells are presented in order to provide a framework for displaying the study data. The shells may change due to unforeseen circumstances. The shells may not be truly representative of every aspect of the study (e.g., sampling time points, assessed laboratory parameters, calculated parameters, units), but are intended to illustrate the general layout of the tables, figures, and data listings that will be included in the final report.

The default tables, listings, and figures layout will be as presented in Table 1-1:

**Table 1-1 Layout Specifications** 

| Orientation | Portrait | Landscape |
|---|---|---|
| Paper Size | Letter | Letter |
| Margins | Top: 3.05 cm | Top: 3.05 cm |
| | Bottom: 2.54 cm | Bottom: 2.2 cm |
| | Left: 2.54 cm | Left: 1.9 cm |
| | Right: 2.54 cm | Right: 1.9 cm |
| Font | Table text: Times new Ro | Table text: Times new Roman 9 or 10 pts |
| | Table title: Times new Ro | Table title: Times new Roman 12 pts |
| | Table legend: Times new | Table legend: Times new Roman 10 pts |

The font size may be reduced as necessary to allow additional columns to be presented, but not at the expense of clarity. Also the orientation may be changed to portrait if appropriate.

Except for pharmacokinetic (PK) tables, descriptive statistics for minimum and maximum will be presented with the same decimal digits as the original values, and with one more decimal place than the original data for mean, standard Deviation, and median. For PK tables, the data presentation will be as per the appropriate inVentiv SOP.



## 2. Summary TFLs

## **Table 2-1 List of Table Shells**

| Table<br>Number | Title |
|---|---|
| | In-Text Table |
| 10.1-1 | Subject Disposition |
| 11.4.2.3-1 | Summary of Pharmacokinetic Parameters of Diazepam- PK Population |
| 11.4.2.3-2 | Ratios (A/B), 90% Geometric Confidence Intervals, Intra-Subjects CV (%), Inter-Subjects CV (%) and P-values for Plasma Pharmacokinetic Parameters of Diazepam – PK Population |
| 11.4.2.3-3 | Ratios (C/B), 90% Geometric Confidence Intervals, Intra-Subjects CV (%), Inter-Subjects CV (%) and P-values for Plasma Pharmacokinetic Parameters of Diazepam – PK Population |
| 11.4.2.3-4 | Summary of Pharmacokinetic Parameters Nordiazepam – PK Population |
| 11.4.2.3-5 | Ratios (A/B), 90% Geometric Confidence Intervals, Intra-Subjects CV (%), Inter-Subjects CV (%) and P-values for Plasma Pharmacokinetic Parameters of Nordiazepam – PK Population |
| 11.4.2.3-6 | Ratios (C/B), 90% Geometric Confidence Intervals, Intra-Subjects CV (%), Inter-Subjects CV (%) and P-values for Plasma Pharmacokinetic Parameters of Nordiazepam – PK Population |
| | Demographic Data Summary Tables |
| 14.1-1 | Summary of Demographic Characteristics of Subjects Included in the Safety Population |
| 14.1-2 | Summary of Demographic Characteristics of Subjects Included in the Pharmacokinetic Population |
| | Pharmacokinetic Tables |
| 14.2.1-1 | Descriptive Statistics for Plasma Concentration over Nominal Time by Treatment– PK Population |
| 14.2.1-2 | Descriptive Statistics of Plasma Pharmacokinetic Parameters by Treatment - PK Population |
| 14.2.1-3 | Descriptive Statistics of Individual Ratios or Individual Differences between Treatments for Pharmacokinetic Parameters - PK Population |
| 14.2.1-4 | Ratios (A/B), 90% Geometric Confidence Intervals, Intra-Subjects CV (%) and P-values for Diazepam – PK Population |
| 14.2.1-5 | Ratios (C/B), 90% Geometric Confidence Intervals, Intra-Subjects CV (%) and P-values for Diazepam – PK Population |
| 14.2.1-6 | Ratios (A/B), 90% Geometric Confidence Intervals, Intra-Subjects CV (%) and P-values for Nordiazepam – PK Population |
| 14.2.1-7 | Ratios (C/B), 90% Geometric Confidence Intervals, Intra-Subjects CV (%) and P-values for Nordiazepam – PK Population |
| | Safety Data Summary Tables |
| 14.3.1-1 | Frequency of Subjects Experiencing Treatment-Emergent Adverse Events and Number of Events Summarized per Treatment – Safety Population |
| 14.3.1-2 | Frequency of Subjects Experiencing Treatment-Emergent Adverse Events Summarized per Treatment and Severity – Safety Population |
| 14.3.1-3 | Number of Treatment-Emergent Adverse Events Summarized per Treatment and Severity – Safety Population |



Aquestive Therapeutics

| 14.3.1-4 | Frequency of Subjects Experiencing Treatment-Emergent Adverse Events Summarized per Treatment and Relationship – Safety Population |
|---|---|
| 14.3.1-5 | Number of Treatment-Emergent Adverse Events Summarized per Treatment and Relationship – Safety Population |
| 14.3.4-1 | Biochemistry Summary Descriptive Statistics and Change from Screening to Study Exit – Safety Population |
| 14.3.4-2 | Frequency of Subjects – Biochemistry Shifts from Screening to Study Exit – Safety Population |
| 14.3.4-3 | Hematology Summary Descriptive Statistics and Change from Screening to Study Exit – Safety Population |
| 14.3.4-4 | Frequency of Subjects - Hematology Shifts from Screening to Study Exit - Safety Population |
| 14.3.4-5 | Urinalysis Summary Descriptive Statistics and Change from Screening to Study Exit – Safety Population |
| 14.3.4-6 | Frequency of Subjects - Urinalysis Shifts from Screening to Study Exit, pH and Specific Gravity – Safety Population |
| 14.3.4-7 | Urinalysis Frequency Summary: Categorical Results – Safety Population |
| 14.3.4-8 | Frequency of Subjects - Urinalysis Shifts from Screening to Study Exit : Categorical Results – Safety Population |
| 14.3.4-9 | Vital Signs Summary Descriptive Statistics – Safety Population |
| 14.3.4-10 | Electrocardiogram Summary Descriptive Statistics – Safety Population |


Aquestive Therapeutics

### **Table 2-2 List of Figures Shells**

| Figure<br>Number* | Title |
|---|---|
| 14.2.2-1a to<br>14.2.2-32a** | Plasma Concentrations of Diazepam for Subject XX - Linear Scale |
| 14.2.2-1b to 14.2.2-32b** | Plasma Concentrations of Diazepam for Subject XX - Semi-Log Scale |
| 14.2.2-33a | Mean (± SD) Plasma Concentrations of Diazepam - Linear Scale |
| 14.2.2-33b | Mean (± SD) Plasma Concentrations of Diazepam - Semi-Log Scale |
| 14.2.2-34a | Overlay of Individual and Mean Plasma Concentrations of Diazepam by Treatment - Linear Scale |
| 14.2.2-34b | Overlay of Individual and Mean Plasma Concentrations of Diazepam by Treatment - Semi-Log<br>Scale |
| 14.2.2-35a to 14.2.2-66a** | Plasma Concentrations of Nordiazepam for Subject XX - Linear Scale |
| 14.2.2-35b to 14.2.2-66b** | Plasma Concentrations of Nordiazepam for Subject XX - Semi-Log Scale |
| 14.2.2-67a | Mean (± SD) Plasma Concentrations of Nordiazepam - Linear Scale |
| 14.2.2-67b | Mean (± SD) Plasma Concentrations of Nordiazepam - Semi-Log Scale |
| 14.2.2-68a | Overlay of Individual and Mean Plasma Concentrations of Nordiazepam by Treatment - Linear Scale |
| 14.2.2-68b | Overlay of Individual and Mean Plasma Concentrations of Nordiazepam by Treatment - Semi-<br>Log Scale |

<sup>\*</sup> Depending on the number of subjects included in the PK population, the figure numbering presented here may change in the report.

<sup>\*\*</sup> Similar figures will be presented for each subject who received study medication

Aquestive Therapeutics

# **Table 2-3 List of Data Listings Shells**

| Listing<br>Number | Title |
|---|---|
| | Documentation of Statistical Methods |
| 16.1.9-1 | ANOVA for Treatment Comparison of Diazepam – PK Population |
| 16.1.9-2 | ANOVA for Treatment Comparison of Nordiazepam – PK Population |
| 16.1.9-3 | Wilcoxon Signed-Rank Test for T <sub>max</sub> for Treatment Comparison of Diazepam – PK |
| | Population |
| 16.1.9-4 | Wilcoxon Signed-Rank Test for T <sub>max</sub> for Treatment Comparison of Nordiazepam – PK |
| | Population |
| | Subject Characteristics Listings |
| 16.2.1-1 | Subjects Completion and Discontinuation Information |
| 16.2.2-1 | Protocol Deviations |
| 16.2.4-1 | Demographics |
| 16.2.4-2 | Medical History Findings at Screening |
| 16.2.4-3 | Prior and Concomitant Medications |
| 16.2.4-4 | Study Drug Administration |
| 16.2.4-5 | Assignment to Analysis Populations |
| | PK Data Listings |
| 16.2.6-1 | Listing of Individual Actual Sampling Times and Pharmacokinetic Concentrations |
| 16.2.6-2 | Listing of Individual Pharmacokinetic Parameters |
| 16.2.6-3 | Listing of Individual Ratios or Differences between Treatment for Pharmacokinetic |
| | Parameters |
| | Safety Data Listings |
| 16.2.7-1 | Non-Treatment-Emergent Adverse Events |
| 16.2.7-2 | Treatment-Emergent Adverse Events |
| 16.2.7-3 | Serious Adverse Events |
| 16.2.7-4 | Significant Adverse Events |
| 16.2.8-1 | Clinical Laboratory – Biochemistry |
| 16.2.8-2 | Clinical Laboratory – Hematology |
| 16.2.8-3 | Clinical Laboratory – Urinalysis |
| 16.2.8-4 | Vital Signs Result |
| 16.2.8-5 | Electrocardiogram Result |
| 16.2.8-6 | DBF Application Site Visual Inspection |

Aquestive Therapeutics

# 3. CSR In-text Tables



Aquestive Therapeutics

**Table 10.1-1 Subject Disposition** 

| Category | Treatment A | Treatment B | Treatment C | Overall |
|---|---|---|---|---|
| Screened | - | - | - | XX |
| Screening Failures <sup>1,2</sup> | - | - | - | x(xx.x) |
| Not Enrolled <sup>1,3</sup> | - | - | - | x ( xx.x) |
| Enrolled <sup>1,4</sup> | - | - | - | x ( xx.x) |
| Dosed | xx | xx | xx | XX |
| Not Dosed | xx | XX | XX | XX |
| Completed <sup>5</sup> | x ( xx.x) | x ( xx.x) | x ( xx.x) | - |
| Completed All Treatment Periods <sup>6</sup> | - | - | - | x ( xx.x) |
| Number of Subjects Discontinued <sup>7, 8</sup> Primary Reason for Discontinuation <sup>7, 8, 9</sup> | xx | XX | XX | xx |
| Adverse Event | x ( xx.x) | x ( xx.x) | x ( xx.x) | x(xx.x) |
| Lost to Follow-up | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) |
| Non-Compliance with Protocol | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) |
| Requirements | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) |
| Positive Alcohol Breath Test | x ( xx.x) | x ( xx.x) | x ( xx.x) | x(xx.x) |
| Positive Drug Screen | x ( xx.x) | x ( xx.x) | x ( xx.x) | x(xx.x) |
| Positive Pregnancy Test | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) |
| Safety Reason | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) |
| Significant Protocol Deviation | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) |
| Study Terminated by Sponsor | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) |
| Other | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) |
| Informed Consent Withdrawn | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) |
| Investigator's decision | x ( xx.x) | x ( xx.x) | x ( xx.x) | x(xx.x) |

#### Programming Note:

28-Jun-2019 (Final 1.0)

if a subject was withdrawn from one period or more but he is included in next period(s) please add a footnote 10 to clarify, e.g.

<sup>&</sup>quot;10 Subject No. XX completed Period 1 (Treatment A) but was discontinued before dosing in Period 2 (Treatment B) and was dosed in Periods 3 (Treatment C)."

<sup>&</sup>lt;sup>1</sup> Percentage based on the number of screened subjects.



Aquestive Therapeutics

Treatment A: Diazepam Buccal Film under fed conditions (breakfast with moderate fat content);

Treatment B: Diastat® AcuDial<sup>TM</sup> rectal gel under fed conditions (breakfast with moderate fat content),

Treatment C: Diazepam Buccal Film under fed conditions (breakfast with high fat content).

Data source: Listings 16.2.1-1 and 16.2.4-4.

28-Jun-2019 (Final 1.0) 

<sup>&</sup>lt;sup>2</sup> Screening failures include volunteers who did not meet project criteria.

<sup>&</sup>lt;sup>3</sup> Not enrolled include volunteers who were judged eligible but decided not to participate on study or who were not selected to participate in the study since there was already a sufficient number of subjects.

<sup>&</sup>lt;sup>4</sup> Enrolled include volunteers who were judged eligible and accepted to participate in the trial after having signed the approved final version of the study informed consent form and also those identified as standby who may replace subjects who withdraw from the study before dosing.

<sup>&</sup>lt;sup>5</sup> Percentage based on the number of dosed subjects for a given treatment.

<sup>&</sup>lt;sup>6</sup> Percentage based on the overall number of subjects dosed (safety population).

<sup>&</sup>lt;sup>7</sup> Includes subjects who discontinued during the washout period or during the baseline assessment; these subjects are included under the last treatment received prior to discontinuation.

<sup>&</sup>lt;sup>8</sup> Overall, each subject could only contribute once to each reason for discontinuation, regardless of the number of occurrences.

<sup>&</sup>lt;sup>9</sup> Percentage based on the number of discontinued subjects per treatment group or overall, as appropriate.



Aquestive Therapeutics

Table 11.4.2.3-1 Summary of Plasma Pharmacokinetic Parameters of Diazepam – PK Population

| D | | Treat | ment A | | | Treat | ment B | | | Treat | ment C | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Parameter(unit) | N | Mean | SD | CV% | N | Mean | SD | CV% | N | Mean | SD | CV% |
| $\begin{array}{c} AUC_{0\text{-t}}\left(h^*ng/mL\right)\\ AUC_{0\text{-inf}}\left(h^*ng/mL\right)\\ Residual area (\%)\\ C_{max}\left(ng/mL\right)\\ T_{\frac{1}{2}\text{ el}}\left(h\right)\\ K_{\text{el}}\left(/h\right)\\ Cl/F\\ V_{\text{d}}/F\\ Cl/F/kg\\ V_{\text{d}}/F/kg \end{array}$ | | | | | | | | | | | | |
| Parameter (unit) | | Treat | ment A | | | Treat | ment B | | | Treat | ment C | |
| | N | Median | Min | Max | N | Median | Min | Max | N | Median | Min | Max |
| T <sub>max</sub> (h) | | | | | | | | | | | | |

N: Number of observations; SD: Standard Deviation; CV = Coefficient of Variation; Min = Minimum, Max = Maximum; '.' : Not calculated. Residual area (%) = 100\*(1- AUC<sub>0-t</sub> / AUC<sub>0-inf</sub>).

Treatment A: Diazepam Buccal Film under fed conditions (breakfast with moderate fat content);

Treatment B: Diastat® AcuDial<sup>TM</sup> rectal gel under fed conditions (breakfast with moderate fat content);

Treatment C: Diazepam Buccal Film under fed conditions (breakfast with high fat content).

Note: Similar layout will be used for Tables 11.4.2.3-4. Please adapt title and footnotes accordingly.

28-Jun-2019 (Final 1.0) 



Aquestive Therapeutics

Table 11.4.2.3-2 Ratios (A/B), 90% Geometric Confidence Intervals, Intra-Subjects CV (%), Inter-Subjects CV (%) and p-values for Plasma Pharmacokinetic Parameters of Diazepam – PK Population

| Parameter (unit) | Geometric LSM | | 90% Geometric<br>C.I. <sup>2</sup> | | | | p-values | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | Treatment A | Treatment B | Ratio <sup>1</sup> (%) | Lower (%) | Upper (%) | Intra-Subject CV (%) <sup>3</sup> | Inter-Subject CV (%) <sup>4</sup> | Sequence | Period | Treatment |
| AUC <sub>0-t</sub> (h*ng/mL) | | | | | , , | , , , | , , | | | |
| $AUC_{0\text{-}inf}\left(h*ng/mL\right)$ | | | | | | | | | | |
| $C_{max}$ (ng/mL) | | | | | | | | | | |

LSM: Least Square Mean.

Probability (p) values are derived from Type III sums of squares. p-value for the Sequence effect is tested using the Subject(Sequence) effect as the error term.

Treatment A: Diazepam Buccal Film under fed conditions (breakfast with moderate fat content);

Treatment B: Diastat® AcuDial<sup>TM</sup> rectal gel under fed conditions (breakfast with moderate fat content).

Note: Similar layout will be used for Tables 11.4.2.3-3, 11.4.2.3-5 and 11.4.2.3-6. Please adapt title and footnotes accordingly.

28-Jun-2019 (Final 1.0) 

<sup>&</sup>lt;sup>1</sup>Calculated using least-squares means according to the formula: exp (DIFFERENCE) \* 100. <sup>2</sup> 90% Geometric Confidence Interval calculated according to the formula: exp (DIFFERENCE  $\pm$  t<sub>(dfResidual)</sub>\* SE<sub>DIFFERENCE</sub>)

<sup>&</sup>lt;sup>3</sup> Calculated according to formula: SQRT (exp (MSE) – 1) \* 100

<sup>&</sup>lt;sup>4</sup> Calculated according to formula: SQRT (exp ((MS<sub>SUBJECT(SEO)</sub> - MSE)/2) – 1) \* 100

Aquestive Therapeutics

# 4. Summary Tables



Aquestive Therapeutics

Table 14.1-1 Summary of Demographic Characteristics of Subjects Included in the Safety Population

| Category | Statistic | Treatment A | Treatment B | Treatment C | Overall |
|---|---|---|---|---|---|
| Age (years) | N | XX | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X | xx.x |
| | SD. | XX.X | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X | xx.x |
| | Min, Max | XX-XX | xx-xx | xx-xx | XX-XX |
| Age Groups | | | | | |
| <18 | n (%) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) |
| 18-40 | n (%) | x ( xx.x) | x ( xx.x) | x(xx.x) | x (xx.x) |
| > 40 | n (%) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x (xx.x) |
| Sex | (0.0) | | | | |
| Female | n (%) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) |
| Male | n (%) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) |
| Ethnicity | (0./) | | | | |
| Hispanic or Latino | n (%) | x ( xx.x) | x ( xx.x) | x(xx.x) | x(xx.x) |
| Not Hispanic or Latino | n (%) | x ( xx.x) | x ( xx.x) | x(xx.x) | x(xx.x) |
| Not Reported | n (%) | x ( xx.x) | x ( xx.x) | x(xx.x) | x(xx.x) |
| Unknown | n (%) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) |
| Race | | | | | |
| Am Indian | n (%) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) |
| Asian | n (%) | x ( xx.x) | x ( xx.x) | x (xx.x) | x (xx.x) |
| Black | n (%) | x ( xx.x) | x ( xx.x) | x (xx.x) | x ( xx.x) |
| Hawaiian | n (%) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x (xx.x) |
| Islander | n (%) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x (xx.x) |
| White | n (%) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x (xx.x) |
| Other | n (%) | x ( xx.x) | x ( xx.x) | x (xx.x) | x ( xx.x) |
| Height (cm) | N | XX | XX | XX | XX |
| | Mean | XX.XX | xx.xx | XX.XX | XX.XX |
| | SD | XX.XX | xx.xx | xx.xx | XX.XX |
| | Median | XX.XX | XX.XX | xx.xx | XX.XX |
| | Min, Max | xx.x-xx.x | XX.X-XX.X | xx.x-xx.x | XX.X-XX.X |
| Weight (kg) | N | XX | XX | XX | XX |
| | Mean | XX.XX | XX.XX | XX.XX | XX.XX |
| | SD | XX.XX | XX.XX | XX.XX | XX.XX |

28-Jun-2019 (Final 1.0)



Aquestive Therapeutics

| | Median<br>Min, Max | xx.xx<br>xx.x-xx.x | xx.xx<br>xx.x-xx.x | xx.xx<br>xx.x-xx.x | xx.xx<br>xx.x-xx.x |
|---|---|---|---|---|---|
| BMI (kg/m <sup>2</sup> ) | N | XX | XX | xx | XX |
| | Mean | XX.XXX | xx.xxx | xx.xxx | xx.xxx |
| | SD | xx.xxx | XX.XXX | xx.xxx | XX.XXX |
| | Median | XX.XXX | XX.XXX | xx.xxx | XX.XXX |
| | Min, Max | XX.XX-XX.XX | XX.XX-XX.XX | XX.XX-XX.XX | xx.xx-xx.xx |

Programming Note:

1) Refer to the note below for additional instructions

N: Number of subjects dosed; n (%): Number and percent of subjects; SD: Standard Deviation.

Am Indian: American Indian or Alaskan Native; Black: Black or African American; Hawaiian: Native Hawaiian or Pacific Islander;

BMI: body mass index.

Last results (scheduled or unscheduled) obtained at screening were used to generate this table.

Treatment A: Diazepam Buccal Film under fed conditions (breakfast with moderate fat content);

Treatment B: Diastat® AcuDial<sup>TM</sup> rectal gel under fed conditions (breakfast with moderate fat content);

Treatment C: Diazepam Buccal Film under fed conditions (breakfast with high fat content).

Data source: Listing 16.2.4-1

Note: This table will be repeated for Table 14.1-2 only if PK Population is not the same as Safety Population. Otherwise, the title will be updated accordingly.

28-Jun-2019 (Final 1.0) 



Aquestive Therapeutics

Table 14.2.1-1 Descriptive Statistics for Plasma Concentration over Nominal Time by Treatment- PK Population

| Analyte | Treatment | Nominal Time | Time Unit | N | Mean | SD | CV% | Min | Median | Max | Geometric Mean Concentration Unit |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Diazepam | A | 0.000 | h | | | | | | | | |
| • | | 0.500 | h | | | | | | | | |
| | | 0.750 | h | | | | | | | | |
| | | 1 00 | h | | | | | | | | |
| | | 1.50 | h | | | | | | | | |
| | | 2.00 | h | | | | | | | | |
| | | 3.00 | h | | | | | | | | |
| | | 4.00 | h | | | | | | | | |
| | | 6.00 | h | | | | | | | | |
| | | 9.00 | h | | | | | | | | |
| | | 12.0 | h | | | | | | | | |
| | | 24.0 | h | | | | | | | | |
| | | 48.0 | h | | | | | | | | |
| | | 72.0 | h | | | | | | | | |
| | | 96.0 | h | | | | | | | | |
| | | 120 | h | | | | | | | | |
| | | 144 | h | | | | | | | | |
| | | 192 | h | | | | | | | | |
| | | 240 | h | | | | | | | | |

N: Number of observations; SD: Standard Deviation; CV: Coefficient of Variation; Min: Minimum, Max: Maximum.

Treatment A: Diazepam Buccal Film under fed conditions (breakfast with moderate fat content);

 $Treatment \ B: \ Diastat^{\circledR} \ AcuDial^{TM} \ rectal \ gel \ under \ fed \ conditions \ (breakfast \ with \ moderate \ fat \ content);$ 

Treatment C: Diazepam Buccal Film under fed conditions (breakfast with high fat content).

Data source: Listing 16.2.6-1

28-Jun-2019 (Final 1.0) 



Aquestive Therapeutics

Table 14.2.1-2 Descriptive Statistics of Plasma Pharmacokinetic Parameters by Treatment - PK Population

| Analyte | Treatment | Parameter(unit) | N | Mean | SD | CV% | Min | Median | Max | Geometric Mean |
|---|---|---|---|---|---|---|---|---|---|---|
| Diazepam | A | AUC <sub>0-t</sub> (ng*h/mL) | | | | | | | | |
| - | | $AUC_{0-inf} (ng*h/mL)$ | | | | | | | | |
| | | Residual Area (%) | | | | | | | | |
| | | C <sub>max</sub> (ng/mL) | | | | | | | | |
| | | $T_{\text{max}}$ (h) | | | | | | | | |
| | | $T_{1/2 \text{ el}}$ (h) | | | | | | | | |
| | | $K_{el}(/h)$ | | | | | | | | |
| | | Cl/F(h) | | | | | | | | |
| | | Vd/F(h) | | | | | | | | |
| | | Cl/F/kg | | | | | | | | |
| | | Vd/F/kg | | | | | | | | |
| | | ••• | | | | | | | | |

N: Number of observations; SD: Standard Deviation; CV = Coefficient of Variation; Min = Minimum, Max = Maximum; '.': Not calculated.

Treatment A: Diazepam Buccal Film under fed conditions (breakfast with moderate fat content);

Treatment B: Diastat® AcuDial<sup>TM</sup> rectal gel under fed conditions (breakfast with moderate fat content);

Treatment C: Diazepam Buccal Film under fed conditions (breakfast with high fat content).

Data source: Listing 16.2.6-2

28-Jun-2019 (Final 1.0) 

Aquestive Therapeutics

# Table 14.2.1-3 Descriptive Statistics of Individual Ratios or Individual Differences between Treatments for Pharmacokinetic Parameters - PK Population

| Analyte | Comparison | Parameter | Ratio/Difference (unit) | N | Mean | SD CV% Min Median Max Geometric Mean |
|---|---|---|---|---|---|---|
| Diazepam | A vs B | $\mathrm{AUC}_{0\text{-t}}$ | A/B (%) | | | |
| | | $\mathrm{AUC}_{0	ext{-inf}}$ | A/B (%) | | | |
| | | Residual Area | A - B (%) | | | |
| | | $C_{max}$ | A/B (%) | | | |
| | | $T_{max}$ | A - B (h) | | | |
| | | T <sub>½ el</sub> | A/B (%) | | | |
| | | $K_{el}$ | A/B (%) | | | |
| | ••• | | | | | |

N: Number of observations; SD: Standard Deviation; CV = Coefficient of Variation; Min = Minimum, Max = Maximum; '.': Not calculated.

Treatment A: Diazepam Buccal Film under fed conditions (breakfast with moderate fat content);

Treatment B: Diastat® AcuDial<sup>TM</sup> rectal gel under fed conditions (breakfast with moderate fat content);

Treatment C: Diazepam Buccal Film under fed conditions (breakfast with high fat content).

Data source: Listing 16.2.6-3

28-Jun-2019 (Final 1.0) 



Aquestive Therapeutics

### Table 14.2.1-4 Ratios (A/B), 90% Geometric Confidence Intervals, Intra-Subjects CV (%) and P-values for Diazepam – PK **Population**

| Comparison | Parameter(unit) | Geometric LSM | | | 90% Geometric C.I. <sup>2</sup> | | | | | | p-values |
|---|---|---|---|---|---|---|---|---|---|---|---|
| (Test vs. Ref.) | Parameter(unit) | Test | Ref. | Ratio <sup>1</sup> (%) | Lower (%) | Upper (%) | Intra-Subject CV (%) <sup>3</sup> | Inter-Subject<br>CV (%) <sup>4</sup> | Sequence | Period | Treatment |
| A vs B | AUC <sub>0-t</sub> (h*ng/mL) | | | | | | | | | | |
| | $AUC_{0\text{-}inf}\left(h*ng/mL\right)$ | | | | | | | | | | |
| | $C_{max} (ng/mL)$ | | | | | | | | | | |

<sup>&</sup>lt;sup>1</sup>Calculated using least-squares means according to the formula: exp (DIFFERENCE) \* 100.

LSM: Least Square Mean; Ref.: Reference.

Treatment A: Diazepam Buccal Film under fed conditions (breakfast with moderate fat content);

Treatment B: Diastat® AcuDial<sup>TM</sup> rectal gel under fed conditions (breakfast with moderate fat content).

Data Source: Listing 16.1.9-1

Note: Similar layout will be used for Table 14.2.1-5, 14.2.1-6 and 14.2.1-7. Please adapt title and footnotes accordingly.

28-Jun-2019 (Final 1.0) 

 $<sup>^2</sup>$  90% Geometric Confidence Interval calculated according to the formula: exp (DIFFERENCE  $\pm$  t<sub>(dfResidual)</sub>\* SE<sub>DIFFERENCE</sub>)  $^3$  Calculated according to formula: SQRT (exp (MSE) - 1) \* 100

<sup>&</sup>lt;sup>4</sup> Calculated according to formula: SQRT (exp ((MS<sub>SUBJECT (SEO)</sub> - MSE)/2) – 1) \* 100

Aquestive Therapeutics

Table 14.3.1-1 Frequency of Subjects Experiencing Treatment-Emergent Adverse Events and Number of Events Summarized per Treatment – Safety Population

| MedDRA® System Organ Class<br>MedDRA® Preferred Term | Statistic | Treatment A (N=XX) | Treatment B (N=XX) | Treatment C<br>(N=XX) | Overall (N=XX) |
|---|---|---|---|---|---|
| Number of TEAEs | E | XX | XX | XX | XX |
| Number of Subjects with TEAEs | n (%) | x ( xx.x) | x (xx.x) | x (xx.x) | x (xx.x) |
| MedDRA® System Organ Class 1 | n(%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| MedDRA® Preferred Term 1 | n(%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| MedDRA® Preferred Term 2 | n(%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| MedDRA® System Organ Class 2 | n(%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| MedDRA® Preferred Term 1 | n(%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| MedDRA® Preferred Term 2 | n(%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| MedDRA® System Organ Class 3 | n(%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| MedDRA® Preferred Term 1 | n(%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |
| MedDRA® Preferred Term 2 | n(%) E | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x | x ( xx.x) x |

#### Programming Notes:

1) SOC will be presented in descending order of overall incidence rate in terms of frequency of subjects and then in frequency of events (alphabetical order will be used in case of equal rates). For each SOC, PT will be presented the same way.

2) Refer to footnotes for additional instructions.

E: Number of TEAEs; N: Number of subjects dosed; n (%): Number and percent of subjects with TEAE; MedDRA®: Medical Dictionary for Regulatory Activities, version 21.1; TEAEs: Treatment-Emergent Adverse Events.

Each subject could only contribute once to each of the incidence rates, regardless of the number of occurrences.

Overall: Included results from all treatment groups.

Treatment A: Diazepam Buccal Film under fed conditions (breakfast with moderate fat content);

Treatment B: Diastat® AcuDial<sup>TM</sup> rectal gel under fed conditions (breakfast with moderate fat content);

Treatment C: Diazepam Buccal Film under fed conditions (breakfast with high fat content).

Data source: Listing 16.2.7-2

28-Jun-2019 (Final 1.0) 



**Aquestive Therapeutics** 

Table 14.3.1-2 Frequency of Subjects Experiencing Treatment-Emergent Adverse Events Summarized per Treatment and Severity – Safety Population

| MedDRA® System Organ Class<br>MedDRA® Preferred Term | | Treatment A (N=XX) | | | Treatment B (N=XX) | | |
|---|---|---|---|---|---|---|---|
| | n (%) | Mild | Moderate | Severe | Mild | Moderate | Severe |
| MedDRA® System Organ Class 1 | | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) |
| MedDRA® Preferred Term 1 | | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) |
| MedDRA® Preferred Term 2 | | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) |
| MedDRA® System Organ Class 2 | | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) |
| MedDRA® Preferred Term 1 | | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) |
| MedDRA® Preferred Term 2 | | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) |

#### Programming Notes:

- 1) SOC will be presented in descending order of overall incidence rate in terms of frequency of subjects and then in frequency of events (alphabetical order will be used in case of equal rates). For each SOC, PT will be presented the same way.
- 2) If the distribution of treatments is presented on more than one page, preserve the order of the SOC and PT as defined in the generation of the global table without severity.
- 3) Refer to footnotes for additional instructions.

N: Number of subjects dosed; n (%): Number and percent of subjects with treatment-emergent adverse events; MedDRA®: Medical Dictionary for Regulatory Activities, version 21.1.

Each subject could only contribute once to each of the incidence rates, regardless of the number of occurrence; the highest severity is presented.

Overall: Included results from all treatment groups.

Treatment A: Diazepam Buccal Film under fed conditions (breakfast with moderate fat content);

Treatment B: Diastat® AcuDial<sup>TM</sup> rectal gel under fed conditions (breakfast with moderate fat content);

Treatment C: Diazepam Buccal Film under fed conditions (breakfast with high fat content).

Data source: Listing 16.2.7-2

28-Jun-2019 (Final 1.0) 



Aquestive Therapeutics

Table 14.3.1-2 Frequency of Subjects Experiencing Treatment-Emergent Adverse Events Summarized per Treatment and Severity – Safety Population

| MedDRA® System Organ Class<br>MedDRA® Preferred Term | | Treatment C (N=XX) | | | Overall (N=XX) | | |
|---|---|---|---|---|---|---|---|
| | n (%) | Mild | Moderate | Severe | Mild | Moderate | Severe |
| MedDRA® System Organ Class 1 | | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) |
| MedDRA® Preferred Term 1 | | x (xx.x) | x(xx.x) | x (xx.x) | x (xx.x) | x(xx.x) | x (xx.x) |
| MedDRA® Preferred Term 2 | | x (xx.x) | x ( xx.x) | x ( xx.x) | x (xx.x) | x ( xx.x) | x ( xx.x) |
| MedDRA® System Organ Class 2 | | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) |
| MedDRA® Preferred Term 1 | | x (xx.x) | x(xx.x) | x(xx.x) | x (xx.x) | x ( xx.x) | x (xx.x) |
| MedDRA® Preferred Term 2 | | x(xx.x) | x(xx.x) | x(xx.x) | x (xx.x) | x(xx.x) | x (xx.x) |

#### Programming Notes:

- 1) SOC will be presented in descending order of overall incidence rate in terms of frequency of subjects and then in frequency of events (alphabetical order will be used in case of equal rates). For each SOC, PT will be presented the same way.
- 2) If the distribution of treatments is presented on more than one page, preserve the order of the SOC and PT as defined in the generation of the global table without severity.
- *Refer to footnotes for additional instructions.*

N: Number of subjects dosed; n (%): Number and percent of subjects with treatment-emergent adverse events; MedDRA®: Medical Dictionary for Regulatory Activities, version 21.1.

Each subject could only contribute once to each of the incidence rates, regardless of the number of occurrence; the highest severity is presented.

Overall: Included results from all treatment groups.

Treatment A: Diazepam Buccal Film under fed conditions (breakfast with moderate fat content);

Treatment B: Diastat® AcuDial<sup>TM</sup> rectal gel under fed conditions (breakfast with moderate fat content);

Treatment C: Diazepam Buccal Film under fed conditions (breakfast with high fat content).

Data source: Listing 16.2.7-2

28-Jun-2019 (Final 1.0) 



Aquestive Therapeutics

Table 14.3.1-3 Number of Treatment-Emergent Adverse Events Summarized per Treatment and Severity – Safety Population

| MedDRA® System Organ Class MedDRA® Preferred Term | | Treatment A (N=XX) | | Treatment B (N=XX) | | |
|---|---|---|---|---|---|---|
| I | E Mild | Moderate | Severe | Mild | Moderate | Severe |
| MedDRA® System Organ Class 1 | X | X | x | x | x | x |
| MedDRA® Preferred Term 1 | X | X | x | x | x | x |
| MedDRA® Preferred Term 2 | X | X | x | x | x | x |
| MedDRA <sup>®</sup> System Organ Class 2 | x | x | x | X | x | x |
| MedDRA <sup>®</sup> Preferred Term 1 | x | x | x | X | x | x |
| MedDRA <sup>®</sup> Preferred Term 2 | x | x | x | X | x | x |

#### Programming Notes:

E: Number of treatment-emergent adverse event; N: Number of subjects dosed; MedDRA®: Medical Dictionary for Regulatory Activities, version 21.1. Overall: Included results from all treatment groups.

Treatment A: Diazepam Buccal Film under fed conditions (breakfast with moderate fat content);

Treatment B: Diastat® AcuDial<sup>TM</sup> rectal gel under fed conditions (breakfast with moderate fat content);

Treatment C: Diazepam Buccal Film under fed conditions (breakfast with high fat content).

Data source: Listing 16.2.7-2

28-Jun-2019 (Final 1.0) 

<sup>1)</sup> SOC will be presented in descending order of overall incidence rate in terms of frequency of subjects and then in frequency of events (alphabetical order will be used in case of equal rates). For each SOC, PT will be presented the same way.

<sup>2)</sup> If the distribution of treatments is presented on more than one page, preserve the order of the SOC and PT as defined in the generation of the global table without severity.



Aquestive Therapeutics

Table 14.3.1-3 Number of Treatment-Emergent Adverse Events Summarized per Treatment and Severity – Safety Population

| MedDRA® System Organ Class<br>MedDRA® Preferred Term | | Treatment C Overall $(N=XX)$ | | | | |
|---|---|---|---|---|---|---|
| E | Mild | Moderate | Severe | Mild | Moderate | Severe |
| MedDRA® System Organ Class 1 MedDRA® Preferred Term 1 MedDRA® Preferred Term 2 | X | x | x | x | x | X |
| | X | x | x | x | x | X |
| | X | x | x | x | x | X |
| MedDRA <sup>®</sup> System Organ Class 2 | x | x | x | x | x | x |
| MedDRA <sup>®</sup> Preferred Term 1 | x | x | x | x | x | x |
| MedDRA <sup>®</sup> Preferred Term 2 | x | x | x | x | x | x |

#### Programming Notes:

1) SOC will be presented in descending order of overall incidence rate in terms of frequency of subjects and then in frequency of events (alphabetical order will be used in case of equal rates). For each SOC, PT will be presented the same way.

2) If the distribution of treatments is presented on more than one page, preserve the order of the SOC and PT as defined in the generation of the global table without severity.

E: Number of treatment-emergent adverse event; N: Number of subjects dosed; MedDRA®: Medical Dictionary for Regulatory Activities, version 21.1. Overall: Included results from all treatment groups.

Treatment A: Diazepam Buccal Film under fed conditions (breakfast with moderate fat content);

Treatment B: Diastat® AcuDial<sup>TM</sup> rectal gel under fed conditions (breakfast with moderate fat content);

Treatment C: Diazepam Buccal Film under fed conditions (breakfast with high fat content).

Data source: Listing 16.2.7-2

28-Jun-2019 (Final 1.0) 



**Aquestive Therapeutics** 

Table 14.3.1-4 Frequency of Subjects Experiencing Treatment-Emergent Adverse Events Summarized per Treatment and Relationship – Safety Population

| MedDRA® System Organ Class MedDRA® Preferred Term | | Treatment B (N=XX) | | | | | | |
|---|---|---|---|---|---|---|---|---|
| n (%) | Unrelated | Unlikely | Possible | Probable | Unrelated | Unlikely | Possible | Probable |
| MedDRA® System Organ Class 1 MedDRA® Preferred Term 1 MedDRA® Preferred Term 2 | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) |
| | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) |
| | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) |
| MedDRA® System Organ Class 2 MedDRA® Preferred Term 1 MedDRA® Preferred Term 2 | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) |
| | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) |
| | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) |

#### Programming Notes:

- 1) SOC will be presented in descending order of overall incidence rate in terms of frequency of subjects and then in frequency of events (alphabetical order will be used in case of equal rates). For each SOC, PT will be presented the same way.
- 2) If the distribution of treatments is presented on more than one page, preserve the order of the SOC and PT as defined in the generation of the global table without relationship.
- *3)* Refer to footnotes for additional instructions.

N: Number of subjects dosed; n (%): Number and percent of subjects with treatment-emergent adverse event; MedDRA®: Medical Dictionary for Regulatory Activities, version 21.1.

Each subject could only contribute once to each of the incidence rates, regardless of the number of occurrence; the highest relationship is presented.

Overall: Included results from all treatment groups.

Treatment A: Diazepam Buccal Film under fed conditions (breakfast with moderate fat content);

Treatment B: Diastat® AcuDial<sup>TM</sup> rectal gel under fed conditions (breakfast with moderate fat content);

Treatment C: Diazepam Buccal Film under fed conditions (breakfast with high fat content).

Data source: Listing 16.2.7-2

28-Jun-2019 (Final 1.0) 



Aquestive Therapeutics

Table 14.3.1-4 Frequency of Subjects Experiencing Treatment-Emergent Adverse Events Summarized per Treatment and Relationship – Safety Population

| MedDRA® System Organ Class MedDRA® Preferred Term | | Overall (N=XX) | | | | | | |
|---|---|---|---|---|---|---|---|---|
| n (%) | Unrelated | Unlikely | Possible | Probable | Unrelated | Unlikely | Possible | Probable |
| MedDRA® System Organ Class 1 MedDRA® Preferred Term 1 MedDRA® Preferred Term 2 | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) |
| | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) |
| | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) |
| MedDRA® System Organ Class 2 MedDRA® Preferred Term 1 MedDRA® Preferred Term 2 | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) |
| | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) |
| | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) | x ( xx.x) |

#### Programming Notes:

- 1) SOC will be presented in descending order of overall incidence rate in terms of frequency of subjects and then in frequency of events (alphabetical order will be used in case of equal rates). For each SOC, PT will be presented the same way.
- 2) If the distribution of treatments is presented on more than one page, preserve the order of the SOC and PT as defined in the generation of the global table without relationship.
- 3) Refer to footnotes for additional instructions.

N: Number of subjects dosed; n (%): Number and percent of subjects with treatment-emergent adverse event; MedDRA®: Medical Dictionary for Regulatory Activities, version 21.1.

Each subject could only contribute once to each of the incidence rates, regardless of the number of occurrence; the highest relationship is presented.

Overall: Included results from all treatment groups.

Treatment A: Diazepam Buccal Film under fed conditions (breakfast with moderate fat content);

Treatment B: Diastat® AcuDial<sup>TM</sup> rectal gel under fed conditions (breakfast with moderate fat content);

Treatment C: Diazepam Buccal Film under fed conditions (breakfast with high fat content).

Data source: Listing 16.2.7-2

28-Jun-2019 (Final 1.0) 



**Aquestive Therapeutics** 

Table 14.3.1-5 Number of Treatment-Emergent Adverse Events Summarized per Treatment and Relationship – Safety Population

| MedDRA® System Organ Class MedDRA® Preferred Term | | | Treatment (N=XX) | | | | Treatmo<br>(N=X | | |
|---|---|---|---|---|---|---|---|---|---|
| | Е | Unrelated | Unlikely | Possible | Probable | Unrelated | Unlikely | Possible | Probable |
| MedDRA® System Organ Class 1 | | x | x | x | x | x | X | x | x |
| MedDRA® Preferred Term 1 | | x | x | x | x | x | X | x | x |
| MedDRA® Preferred Term 2 | | x | x | x | x | x | X | x | x |
| MedDRA® System Organ Class 2 | | x | x | x | x | x | x | x | x |
| MedDRA® Preferred Term 1 | | x | x | x | x | x | x | x | x |
| MedDRA® Preferred Term 2 | | x | x | x | x | x | x | x | x |

#### Programming Notes:

E: Number of treatment-emergent adverse event; N: Number of subjects dosed; MedDRA®: Medical Dictionary for Regulatory Activities, version 21.1.

Overall: Included results from all treatment groups.

Treatment A: Diazepam Buccal Film under fed conditions (breakfast with moderate fat content);

Treatment B: Diastat® AcuDial<sup>TM</sup> rectal gel under fed conditions (breakfast with moderate fat content);

Treatment C: Diazepam Buccal Film under fed conditions (breakfast with high fat content).

Data source: Listing 16.2.7-2

28-Jun-2019 (Final 1.0) 

<sup>4)</sup> SOC will be presented in descending order of overall incidence rate in terms of frequency of subjects and then in frequency of events (alphabetical order will be used in case of equal rates). For each SOC, PT will be presented the same way.

<sup>5)</sup> If the distribution of treatments is presented on more than one page, preserve the order of the SOC and PT as defined in the generation of the global table without relationship.



**Aquestive Therapeutics** 

Table 14.3.1-5 Number of Treatment-Emergent Adverse Events Summarized per Treatment and Relationship – Safety Population

| MedDRA® System Organ Class<br>MedDRA® Preferred Term | | | Treatment C (N=XX) | | | Overall (N=XX) | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Е | Unrelated | Unlikely | Possible | Probable | Unrelated | Unlikely | Possible | Probable |
| MedDRA® System Organ Class 1<br>MedDRA® Preferred Term 1 | | x<br>x | x<br>x | x<br>x | x<br>x | x<br>x | x<br>x | x<br>x | x<br>x |
| MedDRA® Preferred Term 2 | | X | X | X | x | X | X | X | X |
| MedDRA <sup>®</sup> System Organ Class 2<br>MedDRA <sup>®</sup> Preferred Term 1<br>MedDRA <sup>®</sup> Preferred Term 2 | | x<br>x<br>x | x<br>x<br>x | x<br>x<br>x | X<br>X<br>X | x<br>x<br>x | x<br>x<br>x | x<br>x<br>x | x<br>x<br>x |

#### Programming Notes:

E: Number of treatment-emergent adverse event; N: Number of subjects dosed; MedDRA®: Medical Dictionary for Regulatory Activities, version 21.1.

Overall: Included results from all treatment groups.

Treatment A: Diazepam Buccal Film under fed conditions (breakfast with moderate fat content);

Treatment B: Diastat® AcuDial<sup>TM</sup> rectal gel under fed conditions (breakfast with moderate fat content);

Treatment C: Diazepam Buccal Film under fed conditions (breakfast with high fat content).

Data source: Listing 16.2.7-2

28-Jun-2019 (Final 1.0) 

<sup>1)</sup> SOC will be presented in descending order of overall incidence rate in terms of frequency of subjects and then in frequency of events (alphabetical order will be used in case of equal rates). For each SOC, PT will be presented the same way.

<sup>2)</sup> If the distribution of treatments is presented on more than one page, preserve the order of the SOC and PT as defined in the generation of the global table without relationship.



Aquestive Therapeutics

Table 14.3.4-1 Biochemistry Summary Descriptive Statistics and Change from Screening to Study Exit – Safety Population

| Parameter (unit)<br>Normal Range | Visit | Statistic | Overall (N=XX) |
|---|---|---|---|
| | | | (0 : 2 = 2 = 5) |
| Parameter 1 (xxx) | Screening | n | XX |
| XX-XX | C | Mean | xx.x |
| | | SD | XX.X |
| | | Median | XX.X |
| | | Min, Max | XX, XX |
| | Study Exit | n | xx |
| | - | Mean | XX.X |
| | | SD | XX.X |
| | | Median | XX.X |
| | | Min, Max | XX, XX |
| | Study Exit - CFS | n | xx |
| | • | Mean | XX.X |
| | | SD | xx.x |
| | | Median | XX.X |
| | | Min, Max | xx, xx |

•••

#### Programming Notes:

- 1) Refer to study protocol for laboratory tests to be presented.
- 2) Urinalysis parameters (quantitative results) expected and sorted as: pH (PH) and Specific Gravity(SPGRAV).
- 3) For each parameter provide normal range of primary facility and, for gender specific parameters, use the same sorting of sex from demographic table.
- 4) If multiple laboratories involved, refer to the SAP instructions for results normalization.
- 5) Evaluate individually for each table if some standard results were not quantifiable and, if applicable, add footnote: Not quantifiable values outside of limit of quantitation (<x or >y) will be set to missing for calculation of summary statistics.
- 6) Refer to footnotes for additional instructions.
- 7) Adapt Data Source to the appropriate laboratory category listing.

CFS: Change from screening; N: Number of subjects dossed; n: number of subjects; SD: Standard Deviation. Screening is defined as the last screening results (scheduled or unscheduled).

Data source: Listing 16.2.8-1

Note: This table will be repeated for Tables 14.3.4-3, 14.3.4-5 and Table 14.3.4-10. Please adapt title and data source footnote accordingly.



Aquestive Therapeutics

# Table 14.3.4-2 Frequency of Subjects – Biochemistry Shifts from Screening to Study Exit – Safety Population

| | | | Study Exit | |
|-------------------|-----------|-----------|------------|----------|
| Parameter (unit) | Screening | Low | Normal | High |
| | | n (%) | n (%) | n (%) |
| Parameter 1 (xxx) | Low | x(xx.x) | x(xx.x) | x(xx.x) |
| | Normal | x(xx.x) | x(xx.x) | x(xx.x) |
| | High | x ( xx.x) | x ( xx.x) | x (xx.x) |
| | _ | , | | |
| Parameter 2 (xxx) | Low | x (xx.x) | x (xx.x) | x (xx.x) |
| | Normal | x(xx.x) | x(xx.x) | x (xx.x) |
| | High | x(xx.x) | x(xx.x) | x(xx.x) |

#### Programming Notes:

- 1) Refer to study protocol for parameters to be presented.
- 2) Preserve parameters and sorting defined in Summary Descriptive Statistics Table
- 3) Refer to footnotes for additional instructions.
- 4) Adapt Data Source to the appropriate laboratory category listing.

#### n (%): Number and percentage of subjects.

Percentage based on the number of subjects having available results at screening and at study exit.

Screening is defined as the last screening results (scheduled or unscheduled).

Data source: Listing 16.2.8-1

Note: This table will be repeated for Tables 14.3.4-4, and 14.3.4-6. Please adapt title and data source accordingly.

Aquestive Therapeutics

Table 14.3.4-7 Urinalysis Frequency Summary: Categorical Results – Safety Population

| | <i>J</i> 1 <i>J</i> | | <i>U</i> 1 |
|---|---|---|---|
| Parameter (unit) Normal range | Visit | Result | Overall<br>n (%) |
| Parameter 1 (xxx) | Screening | Clear | x ( xx.x) |
| [Normal range] | | Cloudy | x ( xx.x) |
| | | Turbid | x ( xx.x) |
| | Study Exit | Clear | x ( xx.x) |
| | | Cloudy | x ( xx.x) |
| | | Turbid | x(xx.x) |
| Parameter 2 (xxx) | Screening | + | x ( xx.x) |
| [Normal range] | C | Negative | x ( xx.x) |
| | Study Exit | Negative | x ( xx.x) |
| Parameter 3 (xxx)) | Screening | + | x ( xx.x) |
| [Normal range] | C | Negative | x ( xx.x) |
| | | Trace | x ( xx.x) |
| | Study Exit | + | x ( xx.x) |
| | • | Negative | x ( xx.x) |
| | | Trace | x ( xx.x) |

#### Programming Notes:

- 1) Refer to study protocol for parameters to be presented.
- 2) Urine Microscopy parameters will not presented in this table.
- 3) Evaluate if the units must be added to parameter name if a numeric result was observed. Remove (Units) from column header if no numeric results were observed.
- 4) For each parameter provide normal range of primary facility and, for gender specific parameters, use the same sorting of sex from demographic table.
- 5) Independently for each parameter test, sort results by gradation.
- 6) Refer to footnotes for additional instructions.

#### n (%): Number and percentage of subjects.

Percentage based on the number of subjects having available results at screening and at study exit.

Data source: Listing 16.2.8-3



Aquestive Therapeutics

| Table 14.3.4-8 Frequency of Subjects - Urinalysis Shifts from Screening to Study Exit: Categorical Results – Safety Population |
|---|
|---|

| Parameter | Screening | Study Exit | |
|--------------------|-----------|------------|----------|
| | | Normal | Abnormal |
| | | n (%) | n (%) |
| Parameter 1 | | | |
| | M1 | () | () |
| | Normal | x (xx.x) | x (xx.x) |
| | Abnormal | x (xx.x) | x(xx.x) |
| Parameter 2 | | | |
| | Normal | x (xx.x) | x (xx.x) |
| | Abnormal | x (xx.x) | x(xx.x) |
| Parameter 3 | | | |
| | Normal | x (xx.x) | x (xx.x) |
| | Abnormal | x (xx.x) | x(xx.x) |
| Programming Notes: | | | |

- 1) Refer to study protocol for parameters to be presented.
- 2) Preserve parameters and sorting defined in Summary Descriptive Statistics Table
- 3) Refer to footnotes for additional instructions.

### n (%): Number and percentage of subjects.

Percentage based on the number of subjects having available results at screening and at study exit.

Screening is defined as the last screening results (scheduled or unscheduled).

Data source: Listing 16.2.8-3

28-Jun-2019 (Final 1.0) 



Aquestive Therapeutics

**Table 14.3.4-9 Vital Signs Summary Descriptive Statistics - Safety Population** 

| Timepoint Screening | Statistic n Mean | (N=XX) | Treatment B (N=XX) | Treatment C (N=XX) | (N=XX) |
|---|---|---|---|---|---|
| Screening | | _ | | | |
| Screening | | _ | | | |
| | wiean | | <del>-</del> | - | XX |
| | SD | - | - | - | XX.X |
| | Median | _ | - | - | XX.X<br>XX.X |
| | Min, Max | <del>-</del> | - | - | |
| | IVIIII, IVIAX | - | - | - | XX, XX |
| Pre-dose | n | XX | XX | XX | - |
| | Mean | XX.X | XX.X | XX.X | - |
| | SD | XX.X | XX.X | XX.X | - |
| | Median | XX.X | XX.X | XX.X | - |
| | Min, Max | XX, XX | XX, XX | XX, XX | - |
| Baseline | n | XX | XX | XX | - |
| | Mean | XX.X | XX.X | XX.X | - |
| | SD | XX.X | XX.X | XX.X | - |
| | Median | XX.X | XX.X | XX.X | - |
| | Min, Max | xx, xx | XX, XX | xx, xx | - |
| 0.5H Post-Dose | n | XX | XX | XX | - |
| | | XX.X | XX.X | | - |
| | SD | | | | - |
| | Median | | xx.x | XX.X | - |
| | Min, Max | XX, XX | XX, XX | xx, xx | - |
| 0 5H Post-Dose – CFR | n | YY | XX | YY | _ |
| O.S.I.I.OSI DOSC OID | | | | | _ |
| | | | | | - |
| | | | | | - |
| | | XX | XX | XX | - |
| | 0.5H Post-Dose 0.5H Post-Dose – CFB | Median Min, Max 0.5H Post-Dose n Mean SD Median Min, Max 0.5H Post-Dose – CFB n Mean SD Median SD Median | Median Min, Max xx.x Min, Max xx, xx 0.5H Post-Dose n xx.x Mean xx.x xx.x Median xx.x xx.x Min, Max xx, xx 0.5H Post-Dose – CFB n xx xx Mean xx xx Median xx xx Median xx xx Median xx xx | Median Min, Max XX.X XX.X XX.X 0.5H Post-Dose n XX XX.X Mean Mean Median Median Median Median Mean Mean Mean Mean Mean Mean Mean Me | Median xx.x xx.x xx.x xx.x Min, Max xx, xx xx, xx xx, xx 0.5H Post-Dose n xx xx xx.x Mean xx.x xx.x xx.x xx.x SD xx.x xx.x xx.x xx.x Median xx.x xx, xx xx, xx Min, Max xx, xx xx xx, xx 0.5H Post-Dose – CFB n xx xx xx Mean xx xx xx xx SD xx xx xx xx |

28-Jun-2019 (Final 1.0)



Aquestive Therapeutics

| 1.00H Post-Dose | n | XX | XX | XX | - |
|-----------------------|----------|--------|--------|--------|--------|
| | Mean | XX.X | XX.X | XX.X | - |
| | SD | XX.X | XX.X | XX.X | - |
| | Median | XX.X | XX.X | XX.X | - |
| | Min, Max | XX, XX | XX, XX | XX, XX | - |
| 1.00H Post-Dose – CFB | N | XX | XX | XX | - |
| | Mean | XX | XX | XX | - |
| | SD | XX | XX | XX | - |
| | Median | XX | XX | XX | - |
| | Min, Max | XX, XX | XX, XX | xx, xx | - |
| Study Exit | n | - | - | - | XX |
| | Mean | - | - | - | XX.X |
| | SD | - | - | - | XX.X |
| | Median | - | - | - | XX.X |
| | Min, Max | - | - | - | XX, XX |
| Study Exit - CFS | n | - | - | - | XX |
| · | Mean | - | - | - | XX.X |
| | SD | - | - | - | xx.x |
| | Median | - | - | - | xx.x |

#### Programming Notes:

1) Preserve parameters and sorting defined in Summary Descriptive Statistics Table

CFB: Change from Baseline; CFS: Change from Screening; N: Number of subjects dosed; n: Number of subjects; SD: Standard Deviation.

Screening is defined as the last screening results (scheduled or unscheduled).

Baseline is defined as the last results (scheduled or unscheduled) obtained prior to drug administration in each period.

Data source: Listing 16.2.8-4

28-Jun-2019 (Final 1.0)

<sup>2)</sup> Independently for each parameter, if Baseline assessment is composed by the same visit and timepoint for all subjects, identify this timepoint with Baseline between parentheses. ex. Day 1 Pre-Dose (Baseline)

*Refer to footnotes for additional instructions.* 

Aquestive Therapeutics

# 5. Figures

Syneos Healt Statistical Analysis Plan (Table/Figure/Listing Shells)

Project 180323

Figure 14.2.2-1a: Plasma Concentrations of Diazepam for Subject XX - Linear Scale



Treatment A: Diazepam Buccal Film under fed conditions (breakfast with moderate fat content);

Treatment B: Diastat® AcuDial<sup>TM</sup> rectal gel under fed conditions (breakfast with moderate fat content);

Treatment C: Diazepam Buccal Film under fed conditions (breakfast with high fat content).

Note: This figure will be repeated for each subject included in the PK population, and for nordiazepam.



Figure 14.2.2-1b: Plasma Concentrations of Diazepam for Subject XX – Semi-Log Scale



Treatment B: Diastat® AcuDial<sup>TM</sup> rectal gel under fed conditions (breakfast with moderate fat content);

Treatment C: Diazepam Buccal Film under fed conditions (breakfast with high fat content).

Note: This figure will be repeated for each subject included in the PK population, and for nordiazepam.



Figure 14.2.2-33a: Mean (± SD) Plasma Concentrations of Diazepam - Linear Scale



Treatment B: Diastat® AcuDial<sup>TM</sup> rectal gel under fed conditions (breakfast with moderate fat content);

Treatment C: Diazepam Buccal Film under fed conditions (breakfast with high fat content).



Figure 14.2.2-33b: Mean (± SD) Plasma Concentrations of Diazepam - Semi-Log Scale



Treatment B: Diastat® AcuDial<sup>TM</sup> rectal gel under fed conditions (breakfast with moderate fat content);

Treatment C: Diazepam Buccal Film under fed conditions (breakfast with high fat content).

Figure 14.2.2-34a: Overlay of Individual and Mean Plasma Concentrations of Diazepam by Treatment - Linear Scale



Treatment B: Diastat® AcuDial<sup>TM</sup> rectal gel under fed conditions (breakfast with moderate fat content);

Treatment C: Diazepam Buccal Film under fed conditions (breakfast with high fat content).

Figure 14.2.2-34b: Overlay of Individual and Mean Plasma Concentrations of Diazepam by Treatment - Semi-Log Scale



Treatment B: Diastat® AcuDial<sup>TM</sup> rectal gel under fed conditions (breakfast with moderate fat content);

Treatment C: Diazepam Buccal Film under fed conditions (breakfast with high fat content).
Aquestive Therapeutics

## 6. Listings

Aquestive Therapeutics

## **Listing 16.1.9-1 ANOVA for Treatment Comparison of Diazepam – PK Population**

Comparison: A vs B Dependent Variable: xxx

| PERIOD TRT SUBJECT (SEQ) Source DF Type II SS Mean Square F Value Pr > F SEQ PERIOD TRT SUBJECT (SEQ) Source DF Type III SS Mean Square F Value Pr > F SEQ PERIOD TRT SUBJECT (SEQ) SEQ PERIOD TRT SUBJECT (SEQ) Source DF Type IV SS Mean Square F Value Pr > F SEQ PERIOD TRT SUBJECT (SEQ) | Source | DF | Sum of Squares | Mean Square | F Value | Pr > F | |
|---|---|---|---|---|---|---|---|
| R-Square Coeff Var Root MSE VAR Mean | Model | | | | | • | |
| R-Square Coeff Var Root MSE VAR Mean | Error | | | | | | |
| Source | Corrected | d Total | | | | | |
| SEQ PERIOD TRT SUBJECT (SEQ) Source DF Type II SS Mean Square F Value Pr > F SEQ PERIOD TRT SUBJECT (SEQ) Source DF Type III SS Mean Square F Value Pr > F SEQ PERIOD TRT SUBJECT (SEQ) Source DF Type III SS Mean Square F Value Pr > F SEQ PERIOD TRT SUBJECT (SEQ) | | R-Square | e Coeff Var | Root MSE | VAR Mean | | |
| SEQ PERIOD TRT SUBJECT (SEQ) Source DF Type II SS Mean Square F Value Pr > F SEQ PERIOD TRT SUBJECT (SEQ) Source DF Type III SS Mean Square F Value Pr > F SEQ PERIOD TRT SUBJECT (SEQ) Source DF Type III SS Mean Square F Value Pr > F SEQ PERIOD TRT SUBJECT (SEQ) | | - | | | | | |
| PERIOD TRT SUBJECT (SEQ) Source DF Type II SS Mean Square F Value Pr > F SEQ PERIOD TRT SUBJECT (SEQ) Source DF Type III SS Mean Square F Value Pr > F SEQ PERIOD TRT SUBJECT (SEQ) SEQ PERIOD TRT SUBJECT (SEQ) Source DF Type IV SS Mean Square F Value Pr > F SEQ PERIOD TRT SUBJECT (SEQ) | | DF Typ | e I SS N | Mean Square | F Valu | e Pr > I | F |
| Source DF Type II SS Mean Square F Value Pr > F SEQ PERIOD TRT SUBJECT (SEQ) Source DF Type III SS Mean Square F Value Pr > F SEQ PERIOD TRT SUBJECT (SEQ) Source DF Type III SS Mean Square F Value Pr > F SEQ PERIOD TRT SUBJECT (SEQ) Source DF Type IV SS Mean Square F Value Pr > F SEQ PERIOD TRT SUBJECT (SEQ) | SEQ | | | | | | |
| SOURCE DF Type II SS Mean Square F Value Pr > F SEQ PERIOD TRT SUBJECT (SEQ) Source DF Type III SS Mean Square F Value Pr > F SEQ PERIOD TRT SUBJECT (SEQ) SEQ PERIOD TRT SUBJECT (SEQ) SOURCE DF Type IV SS Mean Square F Value Pr > F SEQ PERIOD TRT SUBJECT (SEQ) | PERIOD | | | | | | |
| Source DF Type II SS Mean Square F Value Pr > F SEQ PERIOD TRT SUBJECT (SEQ) Source DF Type III SS Mean Square F Value Pr > F SEQ PERIOD TRT SUBJECT (SEQ) SEQ PERIOD TRT SUBJECT (SEQ) Source DF Type IV SS Mean Square F Value Pr > F SEQ PERIOD TRT SUBJECT (SEQ) | TRT | | | | | | |
| SEQ PERIOD TRT SUBJECT (SEQ) Source DF Type III SS Mean Square F Value Pr > F SEQ PERIOD TRT SUBJECT (SEQ) Source DF Type IV SS Mean Square F Value Pr > F SEQ PERIOD TRT SUBJECT (SEQ) | SUBJECT (SEQ) | | | | | | |
| SEQ PERIOD TRT SUBJECT (SEQ) Source DF Type III SS Mean Square F Value Pr > F SEQ PERIOD TRT SUBJECT (SEQ) Source DF Type IV SS Mean Square F Value Pr > F SEQ PERIOD TRT SUBJECT (SEQ) | Course | DE True | a II CC N | Ason Sayons | E Waln | | |
| PERIOD TRT SUBJECT (SEQ) Source DF Type III SS Mean Square F Value Pr > F SEQ PERIOD TRT SUBJECT (SEQ) Source DF Type IV SS Mean Square F Value Pr > F SEQ PERIOD TRT TRT SUBJECT (SEQ) | | Dr Typ | e 11 55 r | viean Square | r valu | e Pr > I | r |
| Source DF Type III SS Mean Square F Value Pr > F SEQ PERIOD TRT SUBJECT (SEQ) Source DF Type IV SS Mean Square F Value Pr > F SEQ PERIOD TRT SUBJECT (SEQ) FROM Type IV SS Mean Square F Value Pr > F SEQ PERIOD TRT | | | | | | | |
| Source DF Type III SS Mean Square F Value Pr > F SEQ PERIOD TRT SUBJECT (SEQ) Source DF Type IV SS Mean Square F Value Pr > F SEQ PERIOD TRT SEQ PERIOD TRT | | | | | | | |
| Source DF Type III SS Mean Square F Value Pr > F SEQ PERIOD TRT SUBJECT (SEQ) Source DF Type IV SS Mean Square F Value Pr > F SEQ PERIOD TRT | | | | | | | |
| SEQ PERIOD TRT SUBJECT (SEQ) Source DF Type IV SS Mean Square F Value Pr > F SEQ PERIOD TRT | SUBJECT (SEQ) | | | | | | |
| PERIOD TRT SUBJECT (SEQ) Source DF Type IV SS Mean Square F Value Pr > F SEQ PERIOD TRT | Source | DF Typ | e III SS N | Mean Square | F Valu | e Pr > I | F |
| SOURCE DF Type IV SS Mean Square F Value Pr > F SEQ PERIOD TRT | SEQ | | | | | | |
| SUBJECT (SEQ) Source DF Type IV SS Mean Square F Value Pr > F SEQ PERIOD TRT | PERIOD | | | | | | |
| Source DF Type IV SS Mean Square F Value Pr > F SEQ PERIOD TRT | TRT | | | | | | |
| SEQ<br>PERIOD<br>TRT | SUBJECT (SEQ) | | | | | | |
| SEQ<br>PERIOD<br>TRT | Source | DF Tyn | e IV SS M | Mean Square | F Value | e Pr > 1 | —<br>F |
| PERIOD<br>TRT | | Бі Тур | 517 DD 1 | | 1 valu | | |
| TRT | | | | | | | |
| | SUBJECT (SEQ) | | | | | | |



**Aquestive Therapeutics** 

| ource | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| SEQ | | •• | • | | |
| | | Level of TRT N Mean | Std Dev | | |
| | | A N Wear | Sid Dev | | |
| | | В | | | |
| | | TRT VAR LSMEAN | Standard Error $Pr > t $ | | |
| | | A | • | | |
| | | В | | | |
| Pa | rameter | Estimate Standard Error | t Value $Pr > t $ | 90% Confidence Li | mits |
| | A - B | | | | |

Treatment A: Diazepam Buccal Film under fed conditions (breakfast with moderate fat content)

Treatment B: Diastat® AcuDial<sup>TM</sup> rectal gel under fed conditions (breakfast with moderate fat content)

Note 1: For each comparison, all ANOVA results for ln-transformed AUC $_{0\text{-t}}$ , AUC $_{0\text{-inf}}$ ,  $C_{max}$ , Cl/F, Cl/F/kg, Vd/F, Vd/F/kg and untransformed,  $K_{el}$ , and  $T_{\frac{1}{2}el}$  for plasma concentration will be presented in this listing.

Note 2: For B vs C comparison, PERIOD will not be included in the model.

Note: Similar layout will be used for listing 16.1.9-2. Please adapt title and footnotes accordingly.



**Aquestive Therapeutics** 

## Listing 16.1.9-3 Wilcoxon Signed-Rank Test for $T_{max}$ for Treatment Comparison of Diazepam – PK Population

Comparison: A vs B

| Difference | Statistic | Value |
|------------------|-----------|-------|
| A - B | n | |
| | Mean | |
| | Median | |
| | SD | |
| Wilcoxon | S | |
| Signed-rank Test | p-value | |

n: Number of subjects; SD: Standard Deviation.

Treatment A: Diazepam Buccal Film under fed conditions (breakfast with moderate fat content)

Treatment B: Diastat® AcuDial<sup>TM</sup> rectal gel under fed conditions (breakfast with moderate fat content)

Treatment C: Diazepam Buccal Film under fed conditions (breakfast with high fat content)

Note 1: For each comparison Wilcoxon Signed-Rank Test for  $T_{\text{max}}$  will be presented in this listing.

Note2: Similar layout will be used for listing 16.1.9-4. Please adapt title and footnotes accordingly.



Aquestive Therapeutics

**Listing 16.2.1-1 Subjects Completion and Discontinuation Information** 

| | 5 100201 1 2002 | J • | STEETOTE WITH 2 ISCOTT | | ***** | | |
|---|---|---|---|---|---|---|---|
| Subject | Treatment | | Last Treatment Received | Last Period Prior to | Completion/ Discontinuation | Primary Reason for | |
| Number | Sequence | Period | Prior to Discontinuation | Discontinuation | Date and Time | Discontinuation | Comment |
| | ABC | 1 | A | 2 | DD-MM-YYYY/HH:MM | XXX | XXX |
| | | 2. | В | 3 | | | |

Treatment A: Diazepam Buccal Film under fed conditions (breakfast with moderate fat content);

Treatment B: Diastat® AcuDial<sup>TM</sup> rectal gel under fed conditions (breakfast with moderate fat content);

Treatment C: Diazepam Buccal Film under fed conditions (breakfast with high fat content).

28-Jun-2019 (Final 1.0) 



Aquestive Therapeutics

## **Listing 16.2.2-1 Protocol Deviations**

| Subject | Treatment Sequence | Period | Category | Deviation |
|---------|--------------------|--------|----------|-----------|

Treatment A: Diazepam Buccal Film under fed conditions (breakfast with moderate fat content);

Treatment B: Diastat® AcuDial<sup>TM</sup> rectal gel under fed conditions (breakfast with moderate fat content);

Treatment C: Diazepam Buccal Film under fed conditions (breakfast with high fat content).

28-Jun-2019 (Final 1.0) 



Aquestive Therapeutics

#### **Listing 16.2.4-1 Demographics**

| Subject | Treatment Sequence | Age (years) | Gender | Race | Ethnicity | BMI (kg/m <sup>2</sup> ) | Height (cm) | Weight (kg) |
|---|---|---|---|---|---|---|---|---|
| | ABC | | | | | | | |

BMI: Body Mass Index.

Last results (scheduled or unscheduled) obtained at screening were used to generate this table.

Treatment A: Diazepam Buccal Film under fed conditions (breakfast with moderate fat content);

Treatment B: Diastat® AcuDial<sup>TM</sup> rectal gel under fed conditions (breakfast with moderate fat content);

Treatment C: Diazepam Buccal Film under fed conditions (breakfast with high fat content).

28-Jun-2019 (Final 1.0) 



Aquestive Therapeutics

Listing 16.2.4-2 Medical History Findings at Screening

| Subject | Treatment<br>Sequence | Finding | MedDRA® Preferred Term | MedDRA® System Organ Class | Onset Date | Resolution Date<br>(or Ongoing) |
|---|---|---|---|---|---|---|
| | | FINDING 1 | Preferred Term 1 | SOC 1 | YYYY-MM-DDTHH:MM | YYYY-MM-DDTHH:MM |
| | | FINDING 2 | Preferred Term 2 | SOC 2 | YYYY-MM-DDTHH:MM | ONGOING |

#### Programming Notes:

- 1) SOC and Finding will be presented in uppercase. The Preferred Term will be presented in "propage". The SAS coding "/~n" between terms will generate the break line.
- 2) The SAS coding "/~n" between dates will generate the break line.
- 3) If finding is ongoing, replace missing resolution date per ONGOING.
- 4) Sort events per Subject, Start Date, Stop Date, SOC and PT.
- 5) For incomplete date display, refer to CDISC SDTM Implementation Guide according to ISO 8601 format.

MedDRA®: Medical Dictionary for Regulatory Activities; MedDRA® Version 21.1.

Treatment A: Diazepam Buccal Film under fed conditions (breakfast with moderate fat content);

Treatment B: Diastat® AcuDial<sup>TM</sup> rectal gel under fed conditions (breakfast with moderate fat content);

Treatment C: Diazepam Buccal Film under fed conditions (breakfast with high fat content).

28-Jun-2019 (Final 1.0) 



Aquestive Therapeutics

**Listing 16.2.4-3 Prior and Concomitant Medications** 

| | Treatment Sequence/ | Prior/ | WHO DDE ATC / WHO DDE Preferred Term / | Dose (unit)/ | | Onset Date and Time/<br>Resolution Date and Time | Indication |
|---|---|---|---|---|---|---|---|
| Subject | Treatment | Concomitant | Medication | Frequency | Route | (or Ongoing) | (Condition or AE No.) |
| | ABC | Prior | ATC 1/ | 20 (mg) | ORAL | YYYY-MM-DDTHH:MM/ | |
| | | | Preferred Term 1/ | QID | | YYYY-MM-DDTHH:MM | |
| | | | MEDICATION 1/ | | | | |
| | BAC/ | Concomitant | ATC 2/ | | | YYYY-MM-DDTHH:MM/ | |
| | В | | Preferred Term 2/ | | | ONGOING | |
| | | | MEDICATION 2/ | | | | |

#### Programming Notes:

- 1) ATC and Medication will be presented in uppercase. The Preferred Term will be presented in "propage". The SAS coding "/~n" between terms will generate the break line.
- 2) The SAS coding "/~n" will generate the break line between treatment sequence and treatment, dose with units and frequency. In the same way apply a break line between dates.
- 3) If medication is ongoing, replace missing resolution date per ONGOING.
- 4) Sort events per Subject, Onset Date, Resolution Date, ATC and PT.
- 5) For incomplete date display, refer to CDISC SDTM Implementation Guide according to ISO 8601 format.

ATC: Anatomic Therapeutic Chemical; WHO DDE: World Health Organization Drug Dictionary Enhanced Version Sep2018, format B.

Treatment A: Diazepam Buccal Film under fed conditions (breakfast with moderate fat content);

Treatment B: Diastat® AcuDial<sup>TM</sup> rectal gel under fed conditions (breakfast with moderate fat content);

Treatment C: Diazepam Buccal Film under fed conditions (breakfast with high fat content).

28-Jun-2019 (Final 1.0) 



Aquestive Therapeutics

**Listing 16.2.4-4 Study Drug Administration** 

| Subject | Treatment<br>Sequence | Period | Treatment | Total Dose | Units | Start Date and Time | End Date and Time |
|---|---|---|---|---|---|---|---|
| | | | | | | YYYY-MM-DDTHH:MM:SS | YYYY-MM-DDTHH:MM:SS |

Treatment A: Diazepam Buccal Film under fed conditions (breakfast with moderate fat content);

Treatment B: Diastat® AcuDial<sup>TM</sup> rectal gel under fed conditions (breakfast with moderate fat content);

Treatment C: Diazepam Buccal Film under fed conditions (breakfast with high fat content).



Aquestive Therapeutics

### **Listing 16.2.4-5 Assignment to Analysis Populations**

| Listing | 0.2. i 5 rassignment to rai | |
|---------|-----------------------------|----------------------------|
| | | Included in |
| Subject | Safety Population | Pharmacokinetic Population |
| 101 | Y | N |

Y: Yes; N: No



Aquestive Therapeutics

Listing 16.2.6-1 Listing of Individual Actual Sampling Times and Pharmacokinetic Concentrations

| | | | | Nominal | Time | Actual | | | | Dose Date and | PK Sampling Date and |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Analyte | Subject | Period | Treatment | Time | Unit | Time | Concentration Concentration Unit | Excluded flag | Reason | Time | Time |
| Diazepam | 001 | 01 | A | 0.500 | h | 0.450 | ng/mL | N | | DDMMMYYYY/<br>HH:MM:SS | DDMMMYYYY/<br>HH:MM:SS |
| | | | | 1.00 | h | 1.00 | ng /mL | N | | | |
| | | | | 2.00 | h | 2.01 | ng /mL | Y | inconclusive | 2 | |
| | 001 | 02 | В | 0.500 | h | 0.450 | ng /mL | N | | | |
| | | | | 1.00 | h | 1.00 | ng /mL | N | | | |
| | | | | 2.00 | h | 2.01 | ng /mL | Y | inconclusive | 2 | |
| | 002 | 02 | В | 0.500 | h | 0.450 | ng /mL | | | | |
| | | | | 1.00 | h | 1.00 | ng /mL | | | | |
| | | | | 2.00 | h | 2.01 | ng /mL | | | | |

Treatment A: Diazepam Buccal Film under fed conditions (breakfast with moderate fat content);

Treatment B: Diastat® AcuDial<sup>TM</sup> rectal gel under fed conditions (breakfast with moderate fat content);

Treatment C: Diazepam Buccal Film under fed conditions (breakfast with high fat content).



Aquestive Therapeutics

Listing 16.2.6-2 Listing of Individual Pharmacokinetic Parameters

| nalyte | Subject | Period | Treatment | Parameter | Results | Unit | Excluding flag | Reason |
|---|---|---|---|---|---|---|---|---|
| iazepam | 001 | 01 | A | $\mathrm{AUC}_{0	ext{-t}}$ | | | N | |
| | | | | $\mathrm{AUC}_{0	ext{-inf}}$ | | | N | |
| | | | | $C_{max}$ | | | Y | Not Estimable |
| | | | | Residual area | | | Y | Not Estimable |
| | | | | ••• | | | | |
| | | 02 | В | $\mathrm{AUC}_{0	ext{-t}}$ | | | N | |
| | | | | $\mathrm{AUC}_{0	ext{-inf}}$ | | | N | |
| | | | | $C_{max}$ | | | Y | Not Estimable |
| | | | | Residual area | | | Y | Not Estimable |

 28-Jun-2019 (Final 1.0)

<sup>...</sup>Treatment A: Diazepam Buccal Film under fed conditions (breakfast with moderate fat content);

Treatment B: Diastat® AcuDial<sup>TM</sup> rectal gel under fed conditions (breakfast with moderate fat content);

Treatment C: Diazepam Buccal Film under fed conditions (breakfast with high fat content).



Aquestive Therapeutics

## Listing 16.2.6-3 Listing of Individual Ratios or Differences between Treatment for Pharmacokinetic Parameters

| Analyte | Subject | Parameter (unit) | Treatment A | Treatment B | Treatment C | A/B | C/B | Unit |
|---|---|---|---|---|---|---|---|---|
| Diazepam | 001 | AUC <sub>0-t</sub> (h*ng/mL) | | | | | | % |
| | | $AUC_{0-inf}(h*ng/mL)$ | | | | | | % |
| | | Residual Area(%) | | | | | | % |
| | | $C_{max}(ng/mL)$ | | | | | | % |
| | | $T_{max}(h)$ | | | | | | h |
| | | $T_{\frac{1}{2} \text{ el}}(h)$ | | | | | | % |
| | | $K_{el}(/h)$ | | | | | | % |

Differences are presented for Residual area and T<sub>max</sub>.

Treatment A: Diazepam Buccal Film under fed conditions (breakfast with moderate fat content);

Treatment B: Diastat® AcuDial<sup>TM</sup> rectal gel under fed conditions (breakfast with moderate fat content);

Treatment C: Diazepam Buccal Film under fed conditions (breakfast with high fat content).



**Aquestive Therapeutics** 

| | | MedDRA® System Organ Class/ | Onset Date and Time/ | | | Actio | n taken | |
|---|---|---|---|---|---|---|---|---|
| | AΕ | MedDRA® Preferred Term/ | Resolution Date and Time | Severity/ | Serious | | | |
| Subject | Number | Adverse Event Description | (or Ongoing) | Relationship | (Yes/No) | Study Drug | Other | Outcome |
| | | SOC 1/ | YYYY-MM-DDTHH:MM/ | Severe/ | Yes | | | |
| | | | | | 1 68 | | | |
| | | Preferred Term 1/ | YYYY-MM-DDTHH:MM | Unrelated | | | | |
| | | DESCRIPTION 1 | | | | | | |
| | | SOC 2/ | YYYY-MM-DDTHH:MM/ | Mild/ | No | | | |
| | | Preferred Term 2/ | ONGOING | | | | | |
| | | DESCRIPTION 2 | | | | | | |

#### Programming Notes:

- 1) SOC and AE Description will be presented in uppercase. The Preferred Term will be presented in "propercase". The SAS coding "/~n" between terms will generate the break line.
- 2) The SAS coding "/~n" will generate the break line between dates and between Severity and Relationship.
- 3) If needed, hardcode OUTCOME and ACTIONS in order to introduce break line (~n) between answer elements.
- 4) If medication is ongoing, replace missing resolution date per ONGOING.
- 5) Sort events per Subject, Onset Date/time, Resolution Date/time, SOC and PT.
- 6) For incomplete date display, refer to CDISC SDTM Implementation Guide according to ISO 8601 format.
- 7) Please update' MedDRA® System Organ Class' footnote by keeping only those SOC terms referred in table.

MedDRA®: Medical Dictionary for Regulatory Activities (MedDRA®); MedDRA® Version 21.1.

MedDRA® System Organ Class (SOC): Cardiac disorders (Card); Eye disorders (Eye); Gastrointestinal disorders (Gastr); General disorders and administration site conditions (Genrl); Infections and infestations (Infec); Injury, poisoning and procedural complications (Inj&P); Investigations (Inv); Musculoskeletal and connective tissue disorders (Musc); Nervous system disorders (Nerv); Psychiatric disorders (Psych); Respiratory, thoracic and mediastinal disorders (Resp); Skin and subcutaneous tissue disorders (Skin) Vascular disorders (Vasc).

Note: The list of MedDRA® SOC will be updated according to the AEs observed for the study.

28-Jun-2019 (Final 1.0) 



Aquestive Therapeutics

| <b>Listing 16.2.7-2 Treatment-Emergent Adverse Ev</b> | ents |
|-------------------------------------------------------|------|
|-------------------------------------------------------|------|

| | | | MedDRA® System Organ Class/ | Onset Date and Time/ | | | Action | ı taken | |
|---|---|---|---|---|---|---|---|---|---|
| | | AΕ | MedDRA® Preferred Term/ | Resolution Date and Time | Severity/ | Serious | | | |
| Subject | Treatment | Number | Adverse Event Description | (or Ongoing) | Relationship | (Yes/No) | Study Drug | Other | Outcome |
| 001 | | | SOC 1/<br>Preferred Term 1/<br>DESCRIPTION 1 | YYYY-MM-DDTHH:MM/<br>YYYY-MM-DDTHH:MM | Severe/<br>Unrelated | Yes | | | |
| | | | SOC 2/<br>Preferred Term 2/<br>DESCRIPTION 2 | YYYY-MM-DDTHH:MM/<br>ONGOING | Mild/ | No | | | |

#### Programming Notes:

- 1) SOC and AE Description will be presented in uppercase. The Preferred Term will be presented in "propage". The SAS coding "/~n" between terms will generate the break line.
- 2) The SAS coding "/-n" will generate the break line between dates and between Severity and Relationship.
- 3) If needed, hardcode OUTCOME and ACTIONS in order to introduce break line (~n) between answer elements.
- 4) If medication is ongoing, replace missing resolution date per ONGOING.
- 5) Sort events per Subject, Onset Date/time, Resolution Date/time, SOC and PT.
- 6) For incomplete date display, refer to CDISC SDTM Implementation Guide according to ISO 8601 format.
- 7) Please update' MedDRA® System Organ Class' footnote by keeping only those SOC terms referred in table.

### MedDRA®: Medical Dictionary for Regulatory Activities (MedDRA®); MedDRA® Version 21.1.

MedDRA® System Organ Class (SOC): Cardiac disorders (Card); Eye disorders (Eye); Gastrointestinal disorders (Gastr); General disorders and administration site conditions (Genrl); Infections and infestations (Infec); Injury, poisoning and procedural complications (Inj&P); Investigations (Inv); Musculoskeletal and connective tissue disorders (Musc); Nervous system disorders (Nerv); Psychiatric disorders (Psych); Respiratory, thoracic and mediastinal disorders (Resp); Skin and subcutaneous tissue disorders (Skin) Vascular disorders (Vasc).

Treatment A: Diazepam Buccal Film under fed conditions (breakfast with moderate fat content);

Treatment B: Diastat® AcuDial™ rectal gel under fed conditions (breakfast with moderate fat content);

Treatment C: Diazepam Buccal Film under fed conditions (breakfast with high fat content).

Note: The list of MedDRA® SOC will be updated according to the AEs observed for the study.

Note: Similar layout will be used for Listings 16.2.7-3 and 16.2.7-4, please adapt title and footnotes accordingly.

28-Jun-2019 (Final 1.0) 



**Aquestive Therapeutics** 

**Listing 16.2.8-1 Clinical Laboratory - Biochemistry** 

| | 101210 1 | JIIII BUN | | -10 C11 C11115 C1 J | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Subject | Period | Treatment | Laboratory | Visit | Collection Date and Time | Parameter(unit) | Result | Flag | Normal Range |
| 001 | | | | | YYYY-MM-DDTHH:MM | | | Н | XX.X-XX.X |

#### Programming Notes:

- 1) Sort assessments per Subject, Timepoint/Date and parameters. Sorting for parameter should be as defined in Summary Descriptive Statistics Table.
- 2) For each parameter provide normal range of primary facility and, for gender specific parameters, use the same sorting of gender from demographic table.
- 3) If multiple laboratories involved, display standard and normalised results. Display the ranges in the same way. The SAS coding "/~n" between results or ranges will generate the break line.
  - Take care to use the same precision of both, standard and normalised results/ranges.
- A) Adapt flag footnote for Urinalysis listing per
  - N: Normal result; A: Abnormal result; H: Above normal range; L: Below normal range.
- 5) Laboratory facilities could be abbreviated with appropriation description on footnote (iHC: inVentiv Health Clinical Laboratory; BML: Biron Medical Laboratory).

H: Above normal range; L: Below normal range; N: Normal Range.

Treatment A: Diazepam Buccal Film under fed conditions (breakfast with moderate fat content);

Treatment B: Diastat® AcuDial<sup>TM</sup> rectal gel under fed conditions (breakfast with moderate fat content);

Treatment C: Diazepam Buccal Film under fed conditions (breakfast with high fat content).

Note: Similar layout will be used for Listing 16.2.8-2 and 16.2.8-3. Please adapt title and footnotes accordingly.

28-Jun-2019 (Final 1.0)




Aquestive Therapeutics

#### **Listing 16.2.8-4 Vital Signs Result**

| Subject Period Treatment Time point Measurement Date and Time Parameter(unit) Result |
|---|
|---|

YYYY-MM-DDTHH:MM

#### Programming Notes:

1) Sort assessments per Subject, Timepoint/Date and parameter. Parameters for each subject to be sorted as defined in Summary Descriptive Statistics Table.

Treatment A: Diazepam Buccal Film under fed conditions (breakfast with moderate fat content);

Treatment B: Diastat® AcuDial<sup>TM</sup> rectal gel under fed conditions (breakfast with moderate fat content);

Treatment C: Diazepam Buccal Film under fed conditions (breakfast with high fat content).



Aquestive Therapeutics

## **Listing 16.2.8-5 Electrocardiogram Result**

| Subject | Period | Treatment | Visit | Measurement Date and Time | Parameter(unit) | Result/ Interpretation* |
|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|

YYYY-MM-DDTHH:MM

#### Programming Notes:

1) Sort assessments per Subject, timepoint/Date and parameter. Parameters for each subject to be sorted as defined in Summary Descriptive Statistics Table.

\*The medical judgement for abnormal ECG interpretation is also presented in this column as CS: Clinically significant or NCS: Not clinically significant.

Treatment A: Diazepam Buccal Film under fed conditions (breakfast with moderate fat content);

Treatment B: Diastat® AcuDial<sup>TM</sup> rectal gel under fed conditions (breakfast with moderate fat content);

Treatment C: Diazepam Buccal Film under fed conditions (breakfast with high fat content).



Aquestive Therapeutics

| <b>Listing 16.2.8-6 DBF</b> | <b>Application Site</b> | Visual Inspection |
|-----------------------------|-------------------------|-------------------|
|-----------------------------|-------------------------|-------------------|

| Subject | Time point | Inspection Date and Time | Result | Abnormality |
|---|---|---|---|---|
| | | YYYY-MM-DDTHH:MM | Normal<br>Abnormal | |

DBF: Diazepam Buccal Film

# Listing 16.1.9-1 ANOVA for Treatment Comparison of Diazepam - PK Population Comparison: A $vs\ B$

Dependent Variable: AUC<sub>0-t</sub> (h\*ng/mL)

## The GLM Procedure

| Class Le | vel In | formation | |
|---|---|---|---|
| Class | Class Levels Values | | |
| subject | 6 407 408 409 | | |
| - | | 410 411 412 413 414 501 502 503 505 507 508 | |
| sequence 2 AB BA | | | |
| period | 2 | 1 2 | |
| trt | 2 | A B | |
| Number | of Ob | oservations Read | 54 |
| Number | Number of Observations Used 5 | | |

Comparison: A vs B

Dependent Variable: AUC<sub>0-t</sub> (h\*ng/mL)

## The GLM Procedure

| R-Square | Coeff Var | Root MSE | | LN_AUCI | LST Mean |
|---|---|---|---|---|---|
| 0.695214 | 7.128689 | 0.625101 | 8.768809 | | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.03076554 | 0.03076554 | 0.08 | 0.7813 |
| period | 1 | 0.00220583 | 0.00220583 | 0.01 | 0.9407 |
| trt | 1 | 0.83747933 | 0.83747933 | 2.14 | 0.1557 |
| subject(sequence | ce) 25 | 21.41205990 | 0.85648240 | 2.19 | 0.0275 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.03076554 | 0.03076554 | 0.08 | 0.7813 |
| period | 1 | 0.00653318 | 0.00653318 | 0.02 | 0.8982 |
| trt | 1 | 0.83747933 | 0.83747933 | 2.14 | 0.1557 |
| subject(sequence | ce) 25 | 21.41205990 | 0.85648240 | 2.19 | 0.0275 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.03076554 | 0.03076554 | 0.08 | 0.7813 |
| period | 1 | 0.00653318 | 0.00653318 | 0.02 | 0.8982 |
| trt | 1 | 0.83747933 | 0.83747933 | 2.14 | 0.1557 |
| subject(sequence | ce) 25 | 21.41205990 | 0.85648240 | 2.19 | 0.0275 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.03076554 | 0.03076554 | 0.08 | 0.7813 |
| period | 1 | 0.00653318 | 0.00653318 | 0.02 | 0.8982 |
| trt | 1 | 0.83747933 | 0.83747933 | 2.14 | 0.1557 |
| subject(sequence | ce) 25 | 21.41205990 | 0.85648240 | 2.19 | 0.0275 |

Comparison: A vs B

Dependent Variable: AUC<sub>0-t</sub> (h\*ng/mL)

## The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_AUCLST

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.030766 | 0.030766 | 0.04 | 0.8512 |
| Error | 25 | 21.412060 | 0.856482 | | _ |
| Error: MS(s | Error: MS(subject(sequence)) | | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| *period | 1 | 0.002206 | 0.002206 | 0.01 | 0.9407 |
| trt | 1 | 0.837479 | 0.837479 | 2.14 | 0.1557 |
| subject(sequence) | 25 | 21.412060 | 0.856482 | 2.19 | 0.0275 |
| Error: MS(Error) | 25 | 9.768787 | 0.390751 | | |
| * This test assumes one or m | ore othe | er fixed effects | are zero. | | |

## Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------|----------|------------|-------------|---------|--------|
| sequence | 1 | 0.030766 | 0.030766 | 0.04 | 0.8512 |
| Error | 25 | 21.412060 | 0.856482 | | |
| Frror: MS(s | uhiect(s | equence)) | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.006533 | 0.006533 | 0.02 | 0.8982 |
| trt | 1 | 0.837479 | 0.837479 | 2.14 | 0.1557 |
| subject(sequence) | 25 | 21.412060 | 0.856482 | 2.19 | 0.0275 |
| Error: MS(Error) | 25 | 9.768787 | 0.390751 | | |

Comparison: A vs B

Dependent Variable: AUC<sub>0-t</sub> (h\*ng/mL)

## Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_AUCLST

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.030766 | 0.030766 | 0.04 | 0.8512 |
| Error | 25 | 21.412060 | 0.856482 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 0.006533 | 0.006533 | 0.02 | 0.8982 |
| trt | 1 | 0.837479 | 0.837479 | 2.14 | 0.1557 |
| subject(sequence) | 25 | 21.412060 | 0.856482 | 2.19 | 0.0275 |
| Error: MS(Error) | 25 | 9.768787 | 0.390751 | | |

## Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.030766 | 0.030766 | 0.04 | 0.8512 |
| Error | 25 | 21.412060 | 0.856482 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.006533 | 0.006533 | 0.02 | 0.8982 |
| trt | 1 | 0.837479 | 0.837479 | 2.14 | 0.1557 |
| subject(sequence) | 25 | 21.412060 | 0.856482 | 2.19 | 0.0275 |
| Error: MS(Error) | 25 | 9.768787 | 0.390751 | | |

Comparison: A vs B

Dependent Variable: AUC<sub>0-t</sub> (h\*ng/mL)

## Least Squares Means

| | | H0: | LSMean1=LSMean2 | |
|---|---|---|---|---|
| trt | LN AUCLST LSMEAN | | | Pr > t |
| A | 8.89431407 | | | 0.1557 |
| В | 8.64507378 | | | |
| trt | LN_AUCLST LSMEAN | Ç | 90% Confidence Limits | |
| A | 8.894314 | 8.688682 | 9.099946 | |
| В | 8.645074 | 8.439442 | 8.850706 | |
| Lea | ast Squares Means for Effec | t trt | | |
| | Difference Between | | | |
| i | j Means | 90% Confidence I | Limits for LSMean(i)-LSMe | ean(j) |
| 1 | 2 0.249240 | -0.041567 | 0.540047 | |

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confid | dence Limits |
| A - B | 0.24924028 | 0.17024780 | 1.46 | 0.1557-0 | 0.04156692 | 0.54004749 |

# Listing 16.1.9-1 ANOVA for Treatment Comparison of Diazepam - PK Population Comparison: A $vs\ B$

Dependent Variable: AUC<sub>0-inf</sub> (h\*ng/mL)

## The GLM Procedure

| Class Le | evel In | formation | |
|---|---|---|---|
| Class | Leve | ls Values | |
| subject | 27 | 101 201 202 203 204 205 301 302 303 304 402 40 | 4 406 407 408 409 |
| | | 410 411 412 413 414 501 502 503 505 507 508 | |
| sequenc | e 2 | AB BA | |
| period | 2 | 1 2 | |
| trt | 2 | A B | |
| , | | | |
| Number | of Ob | servations Read | 54 |
| Number of Observations Used | | | |

Comparison: A vs B

Dependent Variable: AUC<sub>0-inf</sub> (h\*ng/mL)

The GLM Procedure

| R-Square | Coeff Var | Root MSE | | LN_AUC | IFO Mean |
|---|---|---|---|---|---|
| 0.845550 | 4.690616 | 0.419817 | 8.950149 | _ | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.16367800 | 0.16367800 | 0.93 | 0.3444 |
| period | 1 | 0.11005743 | 0.11005743 | 0.62 | 0.4368 |
| trt | 1 | 0.72158060 | 0.72158060 | 4.09 | 0.0538 |
| subject(sequence | e) 25 | 23.12666887 | 0.92506675 | 5.25 | <.0001 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.16367800 | 0.16367800 | 0.93 | 0.3444 |
| period | 1 | 0.09003600 | 0.09003600 | 0.51 | 0.4814 |
| trt | 1 | 0.72158060 | 0.72158060 | 4.09 | 0.0538 |
| subject(sequence | e) 25 | 23.12666887 | 0.92506675 | 5.25 | <.0001 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.16367800 | 0.16367800 | 0.93 | 0.3444 |
| period | 1 | 0.09003600 | 0.09003600 | 0.51 | 0.4814 |
| trt | 1 | 0.72158060 | 0.72158060 | 4.09 | 0.0538 |
| subject(sequence | e) 25 | 23.12666887 | 0.92506675 | 5.25 | <.0001 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.16367800 | 0.16367800 | 0.93 | 0.3444 |
| period | 1 | 0.09003600 | 0.09003600 | 0.51 | 0.4814 |
| trt | 1 | 0.72158060 | 0.72158060 | 4.09 | 0.0538 |
| subject(sequence | e) 25 | 23.12666887 | 0.92506675 | 5.25 | <.0001 |

Comparison: A vs B

Dependent Variable: AUC<sub>0-inf</sub> (h\*ng/mL)

## The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_AUCIFO

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.163678 | 0.163678 | 0.18 | 0.6776 |
| Error | 25 | 23.126669 | 0.925067 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| *period | 1 | 0.110057 | 0.110057 | 0.62 | 0.4368 |
| trt | 1 | 0.721581 | 0.721581 | 4.09 | 0.0538 |
| subject(sequence) | 25 | 23.126669 | 0.925067 | 5.25 | <.0001 |
| Error: MS(Error) | 25 | 4.406161 | 0.176246 | | |
| * This test assumes one or m | ore oth | er fixed effects | are zero. | | |

## Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------|----------|------------|-------------|---------|--------|
| sequence | 1 | 0.163678 | 0.163678 | 0.18 | 0.6776 |
| Error | 25 | 23.126669 | 0.925067 | | |
| Error: MS(s | uhiect(s | equence)) | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.090036 | 0.090036 | 0.51 | 0.4814 |
| trt | 1 | 0.721581 | 0.721581 | 4.09 | 0.0538 |
| subject(sequence) | 25 | 23.126669 | 0.925067 | 5.25 | <.0001 |
| Error: MS(Error) | 25 | 4.406161 | 0.176246 | | |

Comparison: A vs B

Dependent Variable: AUC<sub>0-inf</sub> (h\*ng/mL)

## Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.163678 | 0.163678 | 0.18 | 0.6776 |
| Error | 25 | 23.126669 | 0.925067 | | _ |
| Error: MS(s | Error: MS(subject(sequence)) | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 0.090036 | 0.090036 | 0.51 | 0.4814 |
| trt | 1 | 0.721581 | 0.721581 | 4.09 | 0.0538 |
| subject(sequence) | 25 | 23.126669 | 0.925067 | 5.25 | <.0001 |
| Error: MS(Error) | 25 | 4.406161 | 0.176246 | | |

Comparison: A vs B

Dependent Variable: AUC<sub>0-inf</sub> (h\*ng/mL)

## Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.163678 | 0.163678 | 0.18 | 0.6776 |
| Error | 25 | 23.126669 | 0.925067 | | |
| Error: MS(s | Error: MS(subject(sequence)) | | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.090036 | 0.090036 | 0.51 | 0.4814 |
| trt | 1 | 0.721581 | 0.721581 | 4.09 | 0.0538 |
| subject(sequence) | 25 | 23.126669 | 0.925067 | 5.25 | <.0001 |
| Error: MS(Error) | 25 | 4.406161 | 0.176246 | | |

Comparison: A vs B

Dependent Variable: AUC<sub>0-inf</sub> (h\*ng/mL)

## Least Squares Means

| | | H0:LS | SMean1=LSMean2 | |
|---|---|---|---|---|
| trt | LN_AUCIFO LSMEAN | | | Pr > t |
| A | 9.06786545 | | | 0.0538 |
| В | 8.83651326 | | | |
| trt | LN_AUCIFO LSMEAN | 90 | % Confidence Limits | |
| A | 9.067865 | 8.929763 | 9.205967 | |
| В | 8.836513 | 8.698411 | 8.974615 | |
| Lea | ast Squares Means for Effec | et trt | | |
| | Difference Between | | | |
| i | j Means | 90% Confidence Li | mits for LSMean(i)-LSN | Aean(j) |
| 1 | 2 0.231352 | 0.036046 | 0.426658 | |

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Conf | idence Limits |
| A - B | 0.23135219 | 0.11433820 | 2.02 | 0.05380 | .03604644 | 0.42665794 |

# Listing 16.1.9-1 ANOVA for Treatment Comparison of Diazepam - PK Population Comparison: A $vs\ B$

Dependent Variable: C<sub>max</sub> (ng/mL)

## The GLM Procedure

| Class Le | vel Inf | Cormation | |
|---|---|---|---|
| Class | Level | s Values | |
| subject | 28 | 101 201 202 203 204 205 301 302 303 304 402 404 406 407 408 4 410 411 412 413 414 501 502 503 505 506 507 508 | 09 |
| sequence | 2 | AB BA | |
| period | 2 | 1 2 | |
| trt | 2 | A B | |
| Number | of Obs | servations Read 56 | |
| Number | Number of Observations Used 56 | | |

Comparison: A vs B

Dependent Variable: C<sub>max</sub> (ng/mL)

The GLM Procedure

Dependent Variable: LN\_CMAX

| 0.507826 12 | 07076 | | | | AX Mean |
|-------------------|---------|-------------|-------------|---------|---------|
| 0.00,0=0 | 2.97276 | 0.692244 | 5.336136 | | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.04753083 | 0.04753083 | 0.10 | 0.7553 |
| period | 1 | 0.03349429 | 0.03349429 | 0.07 | 0.7936 |
| trt | 1 | 0.01574029 | 0.01574029 | 0.03 | 0.8576 |
| subject(sequence) | 26 | 12.75869056 | 0.49071887 | 1.02 | 0.4761 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.04753083 | 0.04753083 | 0.10 | 0.7553 |
| period | 1 | 0.03349429 | 0.03349429 | 0.07 | 0.7936 |
| trt | 1 | 0.01574029 | 0.01574029 | 0.03 | 0.8576 |
| subject(sequence) | 26 | 12.75869056 | 0.49071887 | 1.02 | 0.4761 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.04753083 | 0.04753083 | 0.10 | 0.7553 |
| period | 1 | 0.03349429 | 0.03349429 | 0.07 | 0.7936 |
| trt | 1 | 0.01574029 | 0.01574029 | 0.03 | 0.8576 |
| subject(sequence) | 26 | 12.75869056 | 0.49071887 | 1.02 | 0.4761 |
| subject(sequence) | 20 | 12.73007030 | 0.17071007 | 1.02 | 0.1701 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.04753083 | 0.04753083 | 0.10 | 0.7553 |
| period | 1 | 0.03349429 | 0.03349429 | 0.07 | 0.7936 |
| trt | 1 | 0.01574029 | 0.01574029 | 0.03 | 0.8576 |
| subject(sequence) | 26 | 12.75869056 | 0.49071887 | 1.02 | 0.4761 |

Comparison: A vs B

Dependent Variable: C<sub>max</sub> (ng/mL)

## The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_CMAX

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.047531 | 0.047531 | 0.10 | 0.7581 |
| Error | 26 | 12.758691 | 0.490719 | | _ |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-------------------|----|-----------|-------------|---------|--------|
| period | 1 | 0.033494 | 0.033494 | 0.07 | 0.7936 |
| trt | 1 | 0.015740 | 0.015740 | 0.03 | 0.8576 |
| subject(sequence) | 26 | 12.758691 | 0.490719 | 1.02 | 0.4761 |
| Error: MS(Error) | 26 | 12.459242 | 0.479202 | | |

## Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_CMAX

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.047531 | 0.047531 | 0.10 | 0.7581 |
| Error | 26 | 12.758691 | 0.490719 | | _ |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.033494 | 0.033494 | 0.07 | 0.7936 |
| trt | 1 | 0.015740 | 0.015740 | 0.03 | 0.8576 |
| subject(sequence) | 26 | 12.758691 | 0.490719 | 1.02 | 0.4761 |
| Error: MS(Error) | 26 | 12.459242 | 0.479202 | | |

Comparison: A vs B

Dependent Variable: C<sub>max</sub> (ng/mL)

## Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_CMAX

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.047531 | 0.047531 | 0.10 | 0.7581 |
| Error | 26 | 12.758691 | 0.490719 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|----------|
| period | 1 | 0.033494 | 0.033494 | 0.07 | 0.7936 |
| trt | 1 | 0.015740 | 0.015740 | 0.03 | 0.8576 |
| subject(sequence) | 26 | 12.758691 | 0.490719 | 1.02 | 0.4761 |
| Error: MS(Error) | 26 | 12.459242 | 0.479202 | | <u> </u> |

## Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_CMAX

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.047531 | 0.047531 | 0.10 | 0.7581 |
| Error | 26 | 12.758691 | 0.490719 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.033494 | 0.033494 | 0.07 | 0.7936 |
| trt | 1 | 0.015740 | 0.015740 | 0.03 | 0.8576 |
| subject(sequence) | 26 | 12.758691 | 0.490719 | 1.02 | 0.4761 |
| Error: MS(Error) | 26 | 12.459242 | 0.479202 | | |
Comparison: A vs B

Dependent Variable: C<sub>max</sub> (ng/mL)

## Least Squares Means

| | | | H0:I | LSMean1=LSMean2 |
|---|---|---|---|---|
| trt | L | N_CMAX LSMEAN | | Pr > t |
| A | 5 | .31937021 | | 0.8576 |
| В | 5 | .35290089 | | |
| trt | | LN_CMAX LSMEAN | 9 | 0% Confidence Limits |
| A | | 5.319370 | 5.096238 | 5.542502 |
| В | | 5.352901 | 5.129769 | 5.576033 |
| Le | ast | Squares Means for Effec | et trt | |
| | | Difference Between | | |
| i | j | Means | 90% Confidence | Limits for LSMean(i)-LSMean(j) |
| 1 | 2 | -0.033531 | -0.349087 | 0.282026 |

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confi | dence Limits |
| A - B | -0.03353068 | 0.18500996 | -0.18 | 0.8576-0 | 0.34908699 | 0.28202562 |

# Listing 16.1.9-1 ANOVA for Treatment Comparison of Diazepam - PK Population Comparison: A $vs\ B$

Dependent Variable: Cl/F/kg ((L/h)/kg)

## The GLM Procedure

| vel In | Formation | |
|---|---|---|
| Leve | s Values | |
| 28 | 101 201 202 203 204 205 301 302 303 304 402 404 | 406 407 408 409 |
| | 410 411 412 413 414 501 502 503 505 506 507 508 | |
| 2 | AB BA | |
| 2 | 1 2 | |
| 2 | AB | |
| of Ob | servations Read | 55 |
| Number of Observations Used 55 | | |
| , | Level 28 2 2 2 2 of Obs | 410 411 412 413 414 501 502 503 505 506 507 508 2 AB BA 2 1 2 2 A B of Observations Read |

Comparison: A vs B

Dependent Variable: Cl/F/kg ((L/h)/kg)

The GLM Procedure

| R-Square | Coeff Var | Root MSE | | LN_CLF | OW Mean |
|------------------|-----------|-------------|-------------|---------|---------|
| 0.855739 | -11.79232 | 0.435284 | -3.691249 | | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.40957690 | 0.40957690 | 2.16 | 0.1540 |
| period | 1 | 0.04998166 | 0.04998166 | 0.26 | 0.6120 |
| trt | 1 | 1.58691124 | 1.58691124 | 8.38 | 0.0078 |
| subject(sequence | e) 26 | 26.05157410 | 1.00198362 | 5.29 | <.0001 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.38456027 | 0.38456027 | 2.03 | 0.1666 |
| period | 1 | 0.07279375 | 0.07279375 | 0.38 | 0.5410 |
| trt | 1 | 1.38322100 | 1.38322100 | 7.30 | 0.0122 |
| subject(sequence | e) 26 | 26.05157410 | 1.00198362 | 5.29 | <.0001 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.47095872 | 0.47095872 | 2.49 | 0.1275 |
| period | 1 | 0.07279375 | 0.07279375 | 0.38 | 0.5410 |
| trt | 1 | 1.38322100 | 1.38322100 | 7.30 | 0.0122 |
| subject(sequence | e) 26 | 26.05157410 | 1.00198362 | 5.29 | <.0001 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.47095872 | 0.47095872 | 2.49 | 0.1275 |
| period | 1 | 0.07279375 | 0.07279375 | 0.38 | 0.5410 |
| trt | 1 | 1.38322100 | 1.38322100 | 7.30 | 0.0122 |
| subject(sequence | e) 26 | 26.05157410 | 1.00198362 | 5.29 | <.0001 |

Comparison: A vs B

Dependent Variable: Cl/F/kg ((L/h)/kg)

## The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_CLFOW

| | | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|----------|--------|-----------|-------------|---------|--------|
| * | sequence | 1 | 0.409577 | 0.409577 | 0.41 | 0.5299 |
| | Error | 25.903 | 26.164431 | 1.010105 | | |

Error: 1.01\*MS(subject(sequence)) - 0.01\*MS(Error)

<sup>\*</sup> This test assumes one or more other fixed effects are zero.

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---------|--------|-----------|-------------|---------|--------|
| *period | 1 | 0.049982 | 0.049982 | 0.25 | 0.6185 |
| Error | 27.469 | 5.411267 | 0.196998 | | |

Error: 0.0093\*MS(subject(sequence)) + 0.9907\*MS(Error)

<sup>\*</sup> This test assumes one or more other fixed effects are zero.

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| trt | 1 | 1.586911 | 1.586911 | 8.04 | 0.0085 |
| Error | 27.564 | 5.438057 | 0.197288 | | |
| Error: 0.0 | 096*MS(sub | ject(sequence)) | + 0.9904*MS(Erro | or) | |

| Source | DF Type | I SS Mean Square | F Value | Pr > F |
|-------------------|-----------|------------------|---------|--------|
| subject(sequence) | 26 26.05 | 1574 1.001984 | 5.29 | <.0001 |
| Error: MS(Error) | 25 4.7368 | 300 0.189472 | | |

Comparison: A vs B

Dependent Variable: Cl/F/kg ((L/h)/kg)

## Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_CLFOW

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.384560 | 0.384560 | 0.38 | 0.5426 |
| Error 25.903 26.164357 1.010100 | | | | | |
| Error: 1.01*MS(subject(sequence)) - 0.01*MS(Error) | | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|----------|
| period | 1 | 0.072794 | 0.072794 | 0.38 | 0.5410 |
| trt | 1 | 1.383221 | 1.383221 | 7.30 | 0.0122 |
| subject(sequence) | 26 | 26.051574 | 1.001984 | 5.29 | <.0001 |
| Error: MS(Error) | 25 | 4.736800 | 0.189472 | | <u>_</u> |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN CLFOW

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.470959 | 0.470959 | 0.48 | 0.4958 |
| Error | 26.182 | 25.847523 | 0.987232 | | |
| Error: 0.9818*MS(subject(sequence)) + 0.0182*MS(Error) | | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 0.072794 | 0.072794 | 0.38 | 0.5410 |
| trt | 1 | 1.383221 | 1.383221 | 7.30 | 0.0122 |
| subject(sequence) | 26 | 26.051574 | 1.001984 | 5.29 | <.0001 |
| Error: MS(Error) | 25 | 4.736800 | 0.189472 | | |

Comparison: A vs B

Dependent Variable: Cl/F/kg ((L/h)/kg)

## Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.470959 | 0.470959 | 0.48 | 0.4958 |
| Error | 26.182 | 25.847523 | 0.987232 | | |
| Error: 0.9818*MS(subject(sequence)) + 0.0182*MS(Error) | | | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.072794 | 0.072794 | 0.38 | 0.5410 |
| trt | 1 | 1.383221 | 1.383221 | 7.30 | 0.0122 |
| subject(sequence) | 26 | 26.051574 | 1.001984 | 5.29 | <.0001 |
| Error: MS(Error) | 25 | 4.736800 | 0.189472 | · | |

Comparison: A vs B

Dependent Variable: Cl/F/kg ((L/h)/kg)

## Least Squares Means

| | | Н | I0:LSMean1=LSMean2 | |
|---|---|---|---|---|
| trt | LN_CLFOW LSMEAN | | | Pr > t |
| A | -3.86011863 | | | 0.0122 |
| В | -3.53980386 | | | |
| trt | LN_CLFOW LSMEAN | | 90% Confidence Limits | |
| A | -3.860119 | -4.000632 | -3.719605 | |
| В | -3.539804 | -3.685621 | -3.393986 | |
| Lea | ast Squares Means for Effec | t trt | | |
| | Difference Between | | | |
| i | j Means | 90% Confiden | ce Limits for LSMean(i)-LS | Mean(j) |
| 1 | 2 -0.320315 | -0.522816 | -0.117814 | |

| | | Standard | | | |
|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confidence Limits |
| A - B | -0.32031478 | 0.11855059 | -2.70 | 0.0122-0 | .52281587 -0.11781369 |

# **Listing 16.1.9-1 ANOVA for Treatment Comparison of Diazepam - PK Population** Comparison: A vs B

Dependent Variable: Cl/F (L/h)

## The GLM Procedure

| Class Le | evel In | formation | |
|---|---|---|---|
| Class | Leve | els Values | |
| subject | 28 | 101 201 202 203 204 205 301 302 303 304 402 404 40 | 6 407 408 409 |
| · | | 410 411 412 413 414 501 502 503 505 506 507 508 | |
| sequence | e 2 | AB BA | |
| period | 2 | 1 2 | |
| trt | 2 | A B | |
| Number | of Ot | oservations Read | 55 |
| Number of Observations Used 55 | | | |

Comparison: A vs B

Dependent Variable: Cl/F (L/h)

## The GLM Procedure

| R-Square | Coeff Var | Root MSE | | LN_CI | LFO Mean |
|---|---|---|---|---|---|
| 0.853402 | 60.55102 | 0.435284 | 0.718871 | | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.10625215 | 0.10625215 | 0.56 | 0.4609 |
| period | 1 | 0.04807082 | 0.04807082 | 0.25 | 0.6189 |
| trt | 1 | 1.59800963 | 1.59800963 | 8.43 | 0.0076 |
| subject(sequence | ) 26 | 25.82232211 | 0.99316624 | 5.24 | <.0001 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.09367124 | 0.09367124 | 0.49 | 0.4885 |
| period | 1 | 0.07279375 | 0.07279375 | 0.38 | 0.5410 |
| trt | 1 | 1.38322100 | 1.38322100 | 7.30 | 0.0122 |
| subject(sequence | ) 26 | 25.82232211 | 0.99316624 | 5.24 | <.0001 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.14399810 | 0.14399810 | 0.76 | 0.3916 |
| period | 1 | 0.07279375 | 0.07279375 | 0.38 | 0.5410 |
| trt | 1 | 1.38322100 | 1.38322100 | 7.30 | 0.0122 |
| subject(sequence | ) 26 | 25.82232211 | 0.99316624 | 5.24 | <.0001 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.14399810 | 0.14399810 | 0.76 | 0.3916 |
| period | 1 | 0.07279375 | 0.07279375 | 0.38 | 0.5410 |
| trt | 1 | 1.38322100 | 1.38322100 | 7.30 | 0.0122 |
| subject(sequence | ) 26 | 25.82232211 | 0.99316624 | 5.24 | <.0001 |

Comparison: A vs B

Dependent Variable: Cl/F (L/h)

## The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_CLFO

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-----------|--------|-----------|-------------|---------|--------|
| *sequence | 1 | 0.106252 | 0.106252 | 0.11 | 0.7472 |
| Error | 25.902 | 25.932889 | 1.001199 | | |

Error: 1.01\*MS(subject(sequence)) - 0.01\*MS(Error)

<sup>\*</sup> This test assumes one or more other fixed effects are zero.

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---------|--------|-----------|-------------|---------|--------|
| *period | 1 | 0.048071 | 0.048071 | 0.24 | 0.6252 |
| Error | 27.447 | 5.404762 | 0.196916 | | |

Error: 0.0093\*MS(subject(sequence)) + 0.9907\*MS(Error)

<sup>\*</sup> This test assumes one or more other fixed effects are zero.

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| trt | 1 | 1.598010 | 1.598010 | 8.10 | 0.0083 |
| Error | 27.542 | 5.431288 | 0.197203 | | |
| Error: 0.0096*MS(subject(sequence)) + 0.9904*MS(Error) | | | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-------------------|----|-----------|-------------|---------|--------|
| subject(sequence) | 26 | 25.822322 | 0.993166 | 5.24 | <.0001 |
| Error: MS(Error) | 25 | 4.736800 | 0.189472 | | |

Comparison: A vs B

Dependent Variable: Cl/F (L/h)

## Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_CLFO

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.093671 | 0.093671 | 0.09 | 0.7621 |
| Error | 25.902 | 25.932817 | 1.001194 | | |
| Error: 1.01 | Error: 1.01*MS(subject(sequence)) - 0.01*MS(Error) | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|----------|
| period | 1 | 0.072794 | 0.072794 | 0.38 | 0.5410 |
| trt | 1 | 1.383221 | 1.383221 | 7.30 | 0.0122 |
| subject(sequence) | 26 | 25.822322 | 0.993166 | 5.24 | <.0001 |
| Error: MS(Error) | 25 | 4.736800 | 0.189472 | | <u>_</u> |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN CLFO

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.143998 | 0.143998 | 0.15 | 0.7044 |
| Error | 26.183 | 25.622439 | 0.978575 | | |
| Error: 0.9818*MS(subject(sequence)) + 0.0182*MS(Error) | | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 0.072794 | 0.072794 | 0.38 | 0.5410 |
| trt | 1 | 1.383221 | 1.383221 | 7.30 | 0.0122 |
| subject(sequence) | 26 | 25.822322 | 0.993166 | 5.24 | <.0001 |
| Error: MS(Error) | 25 | 4.736800 | 0.189472 | | |

Comparison: A vs B

Dependent Variable: Cl/F (L/h)

## Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.143998 | 0.143998 | 0.15 | 0.7044 |
| Error | 26.183 | 25.622439 | 0.978575 | | _ |
| Error: 0.9818*MS(subject(sequence)) + 0.0182*MS(Error) | | | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.072794 | 0.072794 | 0.38 | 0.5410 |
| trt | 1 | 1.383221 | 1.383221 | 7.30 | 0.0122 |
| subject(sequence) | 26 | 25.822322 | 0.993166 | 5.24 | <.0001 |
| Error: MS(Error) | 25 | 4.736800 | 0.189472 | | |

Comparison: A vs B

Dependent Variable: Cl/F (L/h)

## Least Squares Means

| | | 110 | I CM 1 I CM 2 | |
|---|---|---|---|---|
| | | H0: | LSMean1=LSMean2 | |
| trt | LN_CLFO LSMEAN | | | Pr > t |
| A | 0.55019981 | | | 0.0122 |
| В | 0.87051459 | | | |
| trt | LN_CLFO LSMEAN | Ç | 0% Confidence Limits | |
| A | 0.550200 | 0.409687 | 0.690713 | |
| В | 0.870515 | 0.724697 | 1.016332 | |
| Lea | ast Squares Means for Effective | et trt | | |
| | Difference Between | | | |
| i | j Means | 90% Confidenc | e Limits for LSMean(i)-LS | SMean(j) |
| 1 | 2 -0.320315 | -0.522816 | -0.117814 | |

| | | Standard | | | |
|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confidence Limits |
| A - B | -0.32031478 | 0.11855059 | -2.70 | 0.0122-0 | .52281587 -0.11781369 |

# Listing 16.1.9-1 ANOVA for Treatment Comparison of Diazepam - PK Population Comparison: A $vs\ B$

Dependent Variable: V<sub>d</sub>/F/kg (L/kg)

## The GLM Procedure

| Class Le | vel In | formation | |
|---|---|---|---|
| Class | Leve | ls Values | |
| subject | 28 | 101 201 202 203 204 205 301 302 303 304 402 404 406 407 | 7 408 409 |
| | | 410 411 412 413 414 501 502 503 505 506 507 508 | |
| sequence | e 2 | AB BA | |
| period | 2 | 1 2 | |
| trt | 2 | AB | |
| Number | of Ob | servations Read | 55 |
| Number of Observations Used 55 | | | |

Comparison: A vs B

Dependent Variable: V<sub>d</sub>/F/kg (L/kg)

The GLM Procedure

| R-Square | Coeff Var | Root MSE | | LN_VZF0 | OW Mean |
|------------------|-----------|-------------|-------------|---------|---------|
| 0.632660 | 86.92906 | 0.774751 | 0.891245 | | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.47432211 | 0.47432211 | 0.79 | 0.3825 |
| period | 1 | 0.06567700 | 0.06567700 | 0.11 | 0.7436 |
| trt | 1 | 1.61360452 | 1.61360452 | 2.69 | 0.1136 |
| subject(sequence | e) 26 | 23.69080306 | 0.91118473 | 1.52 | 0.1502 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.51435042 | 0.51435042 | 0.86 | 0.3635 |
| period | 1 | 0.03845720 | 0.03845720 | 0.06 | 0.8022 |
| trt | 1 | 1.38527031 | 1.38527031 | 2.31 | 0.1413 |
| subject(sequence | e) 26 | 23.69080306 | 0.91118473 | 1.52 | 0.1502 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.39567269 | 0.39567269 | 0.66 | 0.4245 |
| period | 1 | 0.03845720 | 0.03845720 | 0.06 | 0.8022 |
| trt | 1 | 1.38527031 | 1.38527031 | 2.31 | 0.1413 |
| subject(sequence | e) 26 | 23.69080306 | 0.91118473 | 1.52 | 0.1502 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.39567269 | 0.39567269 | 0.66 | 0.4245 |
| period | 1 | 0.03845720 | 0.03845720 | 0.06 | 0.8022 |
| trt | 1 | 1.38527031 | 1.38527031 | 2.31 | 0.1413 |
| subject(sequence | e) 26 | 23.69080306 | 0.91118473 | 1.52 | 0.1502 |

Comparison: A vs B

Dependent Variable: V<sub>d</sub>/F/kg (L/kg)

## The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN VZFOW

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-----------|--------|-----------|-------------|---------|--------|
| *sequence | 1 | 0.474322 | 0.474322 | 0.52 | 0.4779 |
| Error | 25.661 | 23.461639 | 0.914293 | | |

Error: 1.01\*MS(subject(sequence)) - 0.01\*MS(Error)

<sup>\*</sup> This test assumes one or more other fixed effects are zero.

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---------|-------|-----------|-------------|---------|--------|
| *period | 1 | 0.065677 | 0.065677 | 0.11 | 0.7441 |
| Error | 25.71 | 15.505995 | 0.603119 | | |

Error: 0.0093\*MS(subject(sequence)) + 0.9907\*MS(Error)

<sup>\*</sup> This test assumes one or more other fixed effects are zero.

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| trt | 1 | 1.613605 | 1.613605 | 2.67 | 0.1141 |
| Error | 25.737 | 15.525466 | 0.603230 | | |
| Error: 0.0096*MS(subject(sequence)) + 0.9904*MS(Error) | | | | | |

| Source | DF Type I SS | Mean Square | F Value | Pr > F |
|-------------------|--------------|-------------|---------|--------|
| subject(sequence) | 26 23.690803 | 0.911185 | 1.52 | 0.1502 |
| Error: MS(Error) | 25 15.005966 | 0.600239 | | |

Comparison: A vs B

Dependent Variable: V<sub>d</sub>/F/kg (L/kg)

## Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_VZFOW

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.514350 | 0.514350 | 0.56 | 0.4600 |
| Error 25.661 23.461786 0.914291 | | | | | |
| Error: 1.01 | Error: 1.01*MS(subject(sequence)) - 0.01*MS(Error) | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|----------|----------|
| period | 1 | 0.038457 | 0.038457 | 0.06 | 0.8022 |
| trt | 1 | 1.385270 | 1.385270 | 2.31 | 0.1413 |
| subject(sequence) | 26 | 23.690803 | 0.911185 | 1.52 | 0.1502 |
| Error: MS(Error) | 25 | 15.005966 | 0.600239 | <u> </u> | <u> </u> |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.395673 | 0.395673 | 0.44 | 0.5143 |
| Error | 26.633 | 24.117372 | 0.905539 | | |
| Error: 0.9818*MS(subject(sequence)) + 0.0182*MS(Error) | | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 0.038457 | 0.038457 | 0.06 | 0.8022 |
| trt | 1 | 1.385270 | 1.385270 | 2.31 | 0.1413 |
| subject(sequence) | 26 | 23.690803 | 0.911185 | 1.52 | 0.1502 |
| Error: MS(Error) | 25 | 15.005966 | 0.600239 | | |

Comparison: A vs B

Dependent Variable: V<sub>d</sub>/F/kg (L/kg)

## Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.395673 | 0.395673 | 0.44 | 0.5143 |
| Error 26.633 24.117372 0.905539 | | | | | |
| Error: 0.98 | Error: 0.9818*MS(subject(sequence)) + 0.0182*MS(Error) | | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.038457 | 0.038457 | 0.06 | 0.8022 |
| trt | 1 | 1.385270 | 1.385270 | 2.31 | 0.1413 |
| subject(sequence) | 26 | 23.690803 | 0.911185 | 1.52 | 0.1502 |
| Error: MS(Error) | 25 | 15.005966 | 0.600239 | | |

Comparison: A vs B

Dependent Variable: V<sub>d</sub>/F/kg (L/kg)

## Least Squares Means

| | | H0 | :LSMean1=LSMean2 | |
|---|---|---|---|---|
| trt | LN_VZFOW LSMEAN | | | Pr > t |
| A | 0.72543476 | | | 0.1413 |
| В | 1.04598673 | | | |
| trt | LN_VZFOW LSMEAN | | 90% Confidence Limits | |
| A | 0.725435 | 0.475339 | 0.975531 | |
| В | 1.045987 | 0.786450 | 1.305524 | |
| Lea | ast Squares Means for Effec | t trt | | |
| | Difference Between | | | |
| i | j Means | 90% Confidence | Limits for LSMean(i)-LSM | Mean(j) |
| 1 | 2 -0.320552 | -0.680979 | 0.039875 | |

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confi | dence Limits |
| A - B | -0.32055197 | 0.21100520 | -1.52 | 0.1413-0 | 0.68097856 | 0.03987461 |

# **Listing 16.1.9-1 ANOVA for Treatment Comparison of Diazepam - PK Population** Comparison: A vs B

Dependent Variable: V<sub>d</sub>/F (L)

## The GLM Procedure

| Class Le | vel In | Cormation | |
|---|---|---|---|
| Class | Leve | s Values | |
| subject | 28 | 101 201 202 203 204 205 301 302 303 304 402 404 410 411 412 413 414 501 502 503 505 506 507 508 | 406 407 408 409 |
| sequence | e 2 | AB BA | |
| period | 2 | 1 2 | |
| trt | 2 | AB | |
| Number | of Ob | servations Read | 55 |
| Number of Observations Used | | | |

Comparison: A vs B

Dependent Variable: V<sub>d</sub>/F (L)

## The GLM Procedure

| R-Square | Coeff Var | Root MSE | | LN_ | VZFO Mean |
|---|---|---|---|---|---|
| 0.717804 | 14.61417 | 0.774751 | 5.301365 | | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 1.00546546 | 1.00546546 | 1.68 | 0.2074 |
| period | 1 | 0.06790738 | 0.06790738 | 0.11 | 0.7394 |
| trt | 1 | 1.62479570 | 1.62479570 | 2.71 | 0.1124 |
| subject(sequence | ) 26 | 35.47146425 | 1.36428709 | 2.27 | 0.0218 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 1.06348469 | 1.06348469 | 1.77 | 0.1952 |
| period | 1 | 0.03845720 | 0.03845720 | 0.06 | 0.8022 |
| trt | 1 | 1.38527031 | 1.38527031 | 2.31 | 0.1413 |
| subject(sequence | ) 26 | 35.47146425 | 1.36428709 | 2.27 | 0.0218 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.87575663 | 0.87575663 | 1.46 | 0.2384 |
| period | 1 | 0.03845720 | 0.03845720 | 0.06 | 0.8022 |
| trt | 1 | 1.38527031 | 1.38527031 | 2.31 | 0.1413 |
| subject(sequence | ) 26 | 35.47146425 | 1.36428709 | 2.27 | 0.0218 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.87575663 | 0.87575663 | 1.46 | 0.2384 |
| period | 1 | 0.03845720 | 0.03845720 | 0.06 | 0.8022 |
| trt | 1 | 1.38527031 | 1.38527031 | 2.31 | 0.1413 |
| subject(sequence | ) 26 | 35.47146425 | 1.36428709 | 2.27 | 0.0218 |

Comparison: A vs B

Dependent Variable: V<sub>d</sub>/F (L)

## The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_VZFO

| ********** | | | | | |
|------------|--------|-----------|----------|------|--------|
| *sequen | nce I | 1.005465 | 1.005465 | 0.73 | 0.3998 |
| Error | 25.774 | 35.359383 | 1.371924 | | |

Error: 1.01\*MS(subject(sequence)) - 0.01\*MS(Error)

<sup>\*</sup> This test assumes one or more other fixed effects are zero.

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---------|--------|-----------|-------------|---------|--------|
| *period | 1 | 0.067907 | 0.067907 | 0.11 | 0.7408 |
| Error | 26.062 | 15.828153 | 0.607316 | | |

Error: 0.0093\*MS(subject(sequence)) + 0.9907\*MS(Error)

<sup>\*</sup> This test assumes one or more other fixed effects are zero.

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| trt | 1 | 1.624796 | 1.624796 | 2.67 | 0.1140 |
| Error | 26.104 | 15.860304 | 0.607588 | | |
| Error: 0.0 | Error: 0.0096*MS(subject(sequence)) + 0.9904*MS(Error) | | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-------------------|----|-----------|-------------|---------|--------|
| subject(sequence) | 26 | 35.471464 | 1.364287 | 2.27 | 0.0218 |
| Error: MS(Error) | 25 | 15.005966 | 0.600239 | | |

Comparison: A vs B

Dependent Variable: V<sub>d</sub>/F (L)

## Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_VZFO

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 1.063485 | 1.063485 | 0.78 | 0.3868 |
| Error | Error 25.774 35.359454 1.371919 | | | | |
| Error: 1.01 | Error: 1.01*MS(subject(sequence)) - 0.01*MS(Error) | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.038457 | 0.038457 | 0.06 | 0.8022 |
| trt | 1 | 1.385270 | 1.385270 | 2.31 | 0.1413 |
| subject(sequence) | 26 | 35.471464 | 1.364287 | 2.27 | 0.0218 |
| Error: MS(Error) | 25 | 15.005966 | 0.600239 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.875757 | 0.875757 | 0.65 | 0.4278 |
| Error | 26.423 | 35.681954 | 1.350415 | | |
| Error: 0.9818*MS(subject(sequence)) + 0.0182*MS(Error) | | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 0.038457 | 0.038457 | 0.06 | 0.8022 |
| trt | 1 | 1.385270 | 1.385270 | 2.31 | 0.1413 |
| subject(sequence) | 26 | 35.471464 | 1.364287 | 2.27 | 0.0218 |
| Error: MS(Error) | 25 | 15.005966 | 0.600239 | | |

Comparison: A vs B

Dependent Variable: V<sub>d</sub>/F (L)

## Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.875757 | 0.875757 | 0.65 | 0.4278 |
| Error | 26.423 | 35.681954 | 1.350415 | | |
| Error: 0.98 | Error: 0.9818*MS(subject(sequence)) + 0.0182*MS(Error) | | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.038457 | 0.038457 | 0.06 | 0.8022 |
| trt | 1 | 1.385270 | 1.385270 | 2.31 | 0.1413 |
| subject(sequence) | 26 | 35.471464 | 1.364287 | 2.27 | 0.0218 |
| Error: MS(Error) | 25 | 15.005966 | 0.600239 | · | |

Comparison: A vs B

Dependent Variable: V<sub>d</sub>/F (L)

## Least Squares Means

| | | | НО | LSMean1=LSMean2 | |
|---|---|---|---|---|---|
| trt | L | N VZFO LSMEAN | 110 | | > t |
| A | 5 | 1.13575320 | | 0.1 | 413 |
| В | 5 | .45630517 | | | |
| trt | | LN_VZFO LSMEAN | <u> </u> | 00% Confidence Limits | |
| A | | 5.135753 | 4.885657 | 5.385849 | |
| В | | 5.456305 | 5.196768 | 5.715842 | |
| Le | ast | Squares Means for Effect | et trt | | |
| | | Difference Between | | | |
| i | j | Means | 90% Confidenc | e Limits for LSMean(i)-LSMean( | (j) |
| 1 | 2 | -0.320552 | -0.680979 | 0.039875 | |

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confid | dence Limits |
| A - B | -0.32055197 | 0.21100520 | -1.52 | 0.1413-0 | 0.68097856 | 0.03987461 |

# Listing 16.1.9-1 ANOVA for Treatment Comparison of Diazepam - PK Population Comparison: A $vs\ B$

Dependent Variable: T<sub>max</sub> (h)

## The GLM Procedure

| Class Le | evel In | formation | |
|---|---|---|---|
| Class | Leve | els Values | |
| subject | 28 | 101 201 202 203 204 205 301 302 303 304 402 404 4 | 06 407 408 409 |
| | | 410 411 412 413 414 501 502 503 505 506 507 508 | |
| sequenc | e 2 | AB BA | |
| period | 2 | 1 2 | |
| trt | 2 | A B | |
| Number | of Ob | oservations Read | 56 |
| Number of Observations Used 56 | | | |

Comparison: A vs B

Dependent Variable: T<sub>max</sub> (h)

## The GLM Procedure

| R-Square | Coeff Var | Root 1 | MSE | TN | MAX Mean |
|---|---|---|---|---|---|
| 0.501084 | 86.12793 | 0.961: | 541 1. | .116411 | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.04855716 | 0.04855716 | 0.05 | 0.8205 |
| period | 1 | 0.16973016 | 0.16973016 | 0.18 | 0.6718 |
| trt | 1 | 7.32326787 | 7.32326787 | 7.92 | 0.0092 |
| subject(sequence) | 26 | 16.60152389 | 0.63852015 | 0.69 | 0.8244 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.04855716 | 0.04855716 | 0.05 | 0.8205 |
| period | 1 | 0.16973016 | 0.16973016 | 0.18 | 0.6718 |
| trt | 1 | 7.32326787 | 7.32326787 | 7.92 | 0.0092 |
| subject(sequence) | 26 | 16.60152389 | 0.63852015 | 0.69 | 0.8244 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.04855716 | 0.04855716 | 0.05 | 0.8205 |
| period | 1 | 0.16973016 | 0.16973016 | 0.18 | 0.6718 |
| trt | 1 | 7.32326787 | 7.32326787 | 7.92 | 0.0092 |
| subject(sequence) | 26 | 16.60152389 | 0.63852015 | 0.69 | 0.8244 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.04855716 | 0.04855716 | 0.05 | 0.8205 |
| period | 1 | 0.16973016 | 0.16973016 | 0.18 | 0.6718 |
| trt | 1 | 7.32326787 | 7.32326787 | 7.92 | 0.0092 |
| subject(sequence) | 26 | 16.60152389 | 0.63852015 | 0.69 | 0.8244 |

Comparison: A vs B

Dependent Variable: T<sub>max</sub> (h)

## The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: TMAX

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-------------|----------|-----------|-------------|---------|--------|
| sequence | 1 | 0.048557 | 0.048557 | 0.08 | 0.7849 |
| Error | 26 | 16.601524 | 0.638520 | | _ |
| Error: MS(s | ubject(s | equence)) | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-------------------|----|-----------|-------------|---------|--------|
| period | 1 | 0.169730 | 0.169730 | 0.18 | 0.6718 |
| trt | 1 | 7.323268 | 7.323268 | 7.92 | 0.0092 |
| subject(sequence) | 26 | 16.601524 | 0.638520 | 0.69 | 0.8244 |
| Error: MS(Error) | 26 | 24.038608 | 0.924562 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.048557 | 0.048557 | 0.08 | 0.7849 |
| Error | 26 | 16.601524 | 0.638520 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.169730 | 0.169730 | 0.18 | 0.6718 |
| trt | 1 | 7.323268 | 7.323268 | 7.92 | 0.0092 |
| subject(sequence) | 26 | 16.601524 | 0.638520 | 0.69 | 0.8244 |
| Error: MS(Error) | 26 | 24.038608 | 0.924562 | | |

Comparison: A vs B

Dependent Variable: T<sub>max</sub> (h)

## Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: TMAX

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.048557 | 0.048557 | 0.08 | 0.7849 |
| Error | 26 | 16.601524 | 0.638520 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|-----------|
| period | 1 | 0.169730 | 0.169730 | 0.18 | 0.6718 |
| trt | 1 | 7.323268 | 7.323268 | 7.92 | 0.0092 |
| subject(sequence) | 26 | 16.601524 | 0.638520 | 0.69 | 0.8244 |
| Error: MS(Error) | 26 | 24.038608 | 0.924562 | | <u></u> ; |

## Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.048557 | 0.048557 | 0.08 | 0.7849 |
| Error | 26 | 16.601524 | 0.638520 | | |
| Error: MS(s | Error: MS(subject(sequence)) | | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.169730 | 0.169730 | 0.18 | 0.6718 |
| trt | 1 | 7.323268 | 7.323268 | 7.92 | 0.0092 |
| subject(sequence) | 26 | 16.601524 | 0.638520 | 0.69 | 0.8244 |
| Error: MS(Error) | 26 | 24.038608 | 0.924562 | | |

Comparison: A vs B

Dependent Variable: T<sub>max</sub> (h)

## Least Squares Means

| - | | | H0:LSN | Mean1=LSMean2 | |
|---|---|---|---|---|---|
| trt | TMAX LSMEAN | | | | Pr > t |
| A | 1.47803571 | | | | 0.0092 |
| В | 0.75478571 | | | | |
| trt | TMAX LSMEAN | | 90% | Confidence Limits | |
| A | 1.478036 | 1 | .168101 | 1.787971 | |
| В | 0.754786 | 0 | .444851 | 1.064721 | |
| Le | ast Squares Means for Effec | t trt | | | |
| | Difference Between | | | | |
| i | j Means | 90% Confid | ence Limits | for LSMean(i)-LSM | Iean(j) |
| 1 | 2 0.723250 | 0.284936 | | 1.161564 | |

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confi | dence Limits |
| A - B | 0.72325000 | 0.25698275 | 2.81 | 0.00920 | .28493562 | 1.16156438 |

# Listing 16.1.9-1 ANOVA for Treatment Comparison of Diazepam - PK Population Comparison: A $vs\ B$

Dependent Variable: K<sub>el</sub> (/h)

## The GLM Procedure

| vel In | Formation | |
|---|---|---|
| Leve | s Values | |
| 28 | 101 201 202 203 204 205 301 302 303 304 402 404 | 406 407 408 409 |
| | 410 411 412 413 414 501 502 503 505 506 507 508 | |
| 2 | AB BA | |
| 2 | 1 2 | |
| 2 | AB | |
| of Ob | servations Read | 55 |
| Number of Observations Used | | |
| , | Level 28 2 2 2 2 of Obs | 410 411 412 413 414 501 502 503 505 506 507 508 2 AB BA 2 1 2 2 A B of Observations Read |

Comparison: A vs B

Dependent Variable: K<sub>el</sub> (/h)

## The GLM Procedure

| R-Square | Coeff Var | Root | Root MSE | | LAMZ Mean |
|---|---|---|---|---|---|
| 0.946551 | 25.74042 | 0.003 | 3426 | 0.013309 | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.00056954 | 0.00056954 | 48.53 | <.0001 |
| period | 1 | 0.00000351 | 0.00000351 | 0.30 | 0.5896 |
| trt | 1 | 0.00000846 | 0.00000846 | 0.72 | 0.4039 |
| subject(sequence) | 26 | 0.00461412 | 0.00017747 | 15.12 | <.0001 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.00057011 | 0.00057011 | 48.58 | <.0001 |
| period | 1 | 0.00000301 | 0.00000301 | 0.26 | 0.6167 |
| trt | 1 | 0.00000867 | 0.00000867 | 0.74 | 0.3981 |
| subject(sequence) | 26 | 0.00461412 | 0.00017747 | 15.12 | <.0001 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.00056257 | 0.00056257 | 47.94 | <.0001 |
| period | 1 | 0.00000301 | 0.00000301 | 0.26 | 0.6167 |
| trt | 1 | 0.00000867 | 0.00000867 | 0.74 | 0.3981 |
| subject(sequence) | 26 | 0.00461412 | 0.00017747 | 15.12 | <.0001 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.00056257 | 0.00056257 | 47.94 | <.0001 |
| period | 1 | 0.00000301 | 0.00000301 | 0.26 | 0.6167 |
| trt | 1 | 0.00000867 | 0.00000867 | 0.74 | 0.3981 |
| subject(sequence) | 26 | 0.00461412 | 0.00017747 | 15.12 | <.0001 |

Comparison: A vs B

Dependent Variable: K<sub>el</sub> (/h)

## The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LAMZ

| Source | e DF | Type I SS | Mean Square | F Value | Pr > F |
|--------|--------|-----------|-------------|---------|--------|
| *seque | nce 1 | 0.000570 | 0.000570 | 3.18 | 0.0863 |
| Error | 25.966 | 0.004651 | 0.000179 | | |

Error: 1.01\*MS(subject(sequence)) - 0.01\*MS(Error)

<sup>\*</sup> This test assumes one or more other fixed effects are zero.

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---------|--------|-------------|-------------|---------|--------|
| *period | 1 | 0.000003505 | 0.000003505 | 0.26 | 0.6108 |
| Error | 31.955 | 0.000424 | 0.000013270 | | |

Error: 0.0093\*MS(subject(sequence)) + 0.9907\*MS(Error)

<sup>\*</sup> This test assumes one or more other fixed effects are zero.

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| trt | 1 | 0.000008459 | 0.000008459 | 0.63 | 0.4315 |
| Error | Error 32.215 0.000429 0.000013329 | | | | |
| Error: 0.0 | Error: 0.0096*MS(subject(sequence)) + 0.9904*MS(Error) | | | | |

| Source | DF Typ | e I SS Mean Square | F Value | Pr > F |
|-------------------|---------|--------------------|---------|--------|
| subject(sequence) | 26 0.00 | 0.000177 | 15.12 | <.0001 |
| Error: MS(Error) | 25 0.00 | 0.000011735 | ,<br>I | |

Comparison: A vs B

Dependent Variable: K<sub>el</sub> (/h)

## Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LAMZ

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.000570 | 0.000570 | 3.18 | 0.0861 |
| Error | | | | | |
| Error: 1.01*MS(subject(sequence)) - 0.01*MS(Error) | | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 0.000003015 | 0.000003015 | 0.26 | 0.6167 |
| trt | 1 | 0.000008674 | 0.000008674 | 0.74 | 0.3981 |
| subject(sequence) | 26 | 0.004614 | 0.000177 | 15.12 | <.0001 |
| Error: MS(Error) | 25 | 0.000293 | 0.000011735 | | |

## Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.000563 | 0.000563 | 3.22 | 0.0841 |
| Error | | | | | |
| Error: 0.98 | Error: 0.9818*MS(subject(sequence)) + 0.0182*MS(Error) | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 0.000003015 | 0.000003015 | 0.26 | 0.6167 |
| trt | 1 | 0.000008674 | 0.000008674 | 0.74 | 0.3981 |
| subject(sequence) | 26 | 0.004614 | 0.000177 | 15.12 | <.0001 |
| Error: MS(Error) | 25 | 0.000293 | 0.000011735 | | |

Comparison: A vs B

Dependent Variable: K<sub>el</sub> (/h)

## Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.000563 | 0.000563 | 3.22 | 0.0841 |
| Error | Error 26.064 0.004547 0.000174 | | | | |
| Error: 0.9818*MS(subject(sequence)) + 0.0182*MS(Error) | | | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 0.000003015 | 0.000003015 | 0.26 | 0.6167 |
| trt | 1 | 0.000008674 | 0.000008674 | 0.74 | 0.3981 |
| subject(sequence) | 26 | 0.004614 | 0.000177 | 15.12 | <.0001 |
| Error: MS(Error) | 25 | 0.000293 | 0.000011735 | | |

Comparison: A vs B

Dependent Variable: K<sub>el</sub> (/h)

## Least Squares Means

| | | | H0·LS | Mean1=LSMean2 | |
|---|---|---|---|---|---|
| trt | LAMZ LSMEAN | | 110.25 | Micani Estileanz | Pr > t |
| A | 0.01363966 | | | | 0.3981 |
| В | 0.01283753 | | | | |
| trt | LAMZ LSMEAN | | 90% | 6 Confidence Limits | |
| A | 0.013640 | | 0.012534 | 0.014745 | |
| В | 0.012838 | | 0.011690 | 0.013985 | |
| Le | ast Squares Means for Effec | et trt | | | |
| | Difference Between | | | | |
| i | j Means | 90% Conf | idence Limit | s for LSMean(i)-LSM | 1ean(j) |
| 1 | 2 0.000802 | -0.000792 | | 0.002396 | |

| | | Standard | | | | _ |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confid | dence Limits |
| A - B | 0.00080213 | 0.00093299 | 0.86 | 0.3981-0 | 0.00079154 | 0.00239581 |
# Listing 16.1.9-1 ANOVA for Treatment Comparison of Diazepam - PK Population Comparison: A $vs\ B$

Dependent Variable: T<sub>1/2 el</sub> (h)

#### The GLM Procedure

| Class Le | evel In | formation | |
|---|---|---|---|
| Class | Leve | els Values | |
| subject | 28 | 101 201 202 203 204 205 301 302 303 304 402 404 40 | 6 407 408 409 |
| · | | 410 411 412 413 414 501 502 503 505 506 507 508 | |
| sequence | e 2 | AB BA | |
| period | 2 | 1 2 | |
| trt | 2 | A B | |
| Number | of Ot | oservations Read | 55 |
| Number of Observations Used 55 | | | |

Comparison: A vs B

Dependent Variable: T<sub>1/2 el</sub> (h)

#### The GLM Procedure

| R-Square | Coeff Var | r Root MSE | | LAMZHL Mean | |
|---|---|---|---|---|---|
| 0.606732 | 108.1335 | 103.9234 | 96.1066 | 0 | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 4800.1835 | 4800.1835 | 0.44 | 0.5111 |
| period | 1 | 25036.9728 | 25036.9728 | 2.32 | 0.1404 |
| trt | 1 | 15.8745 | 15.8745 | 0.00 | 0.9697 |
| subject(sequence | ) 26 | 386704.1776 | 14873.2376 | 1.38 | 0.2134 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 5200.3781 | 5200.3781 | 0.48 | 0.4941 |
| period | 1 | 23912.6921 | 23912.6921 | 2.21 | 0.1493 |
| trt | 1 | 35.5975 | 35.5975 | 0.00 | 0.9547 |
| subject(sequence | ) 26 | 386704.1776 | 14873.2376 | 1.38 | 0.2134 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 4819.6458 | 4819.6458 | 0.45 | 0.5102 |
| period | 1 | 23912.6921 | 23912.6921 | 2.21 | 0.1493 |
| trt | 1 | 35.5975 | 35.5975 | 0.00 | 0.9547 |
| subject(sequence | ) 26 | 386704.1776 | 14873.2376 | 1.38 | 0.2134 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 4819.6458 | 4819.6458 | 0.45 | 0.5102 |
| period | 1 | 23912.6921 | 23912.6921 | 2.21 | 0.1493 |
| trt | 1 | 35.5975 | 35.5975 | 0.00 | 0.9547 |
| subject(sequence | ) 26 | 386704.1776 | 14873.2376 | 1.38 | 0.2134 |

Comparison: A vs B

Dependent Variable: T<sub>1/2 el</sub> (h)

# The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LAMZHL

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-----------|--------|-------------|-------------|---------|--------|
| *sequence | 1 | 4800.183539 | 4800.183539 | 0.32 | 0.5754 |
| Error | 25.626 | 382189 | 14914 | | |

Error: 1.01\*MS(subject(sequence)) - 0.01\*MS(Error)

<sup>\*</sup> This test assumes one or more other fixed effects are zero.

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---------|--------|-----------|-------------|---------|--------|
| *period | 1 | 25037 | 25037 | 2.31 | 0.1408 |
| Error | 25.644 | 277923 | 10838 | | |

Error: 0.0093\*MS(subject(sequence)) + 0.9907\*MS(Error)

<sup>\*</sup> This test assumes one or more other fixed effects are zero.

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| trt | 1 | 15.874529 | 15.874529 | 0.00 | 0.9698 |
| Error | 25.669 | 278231 | 10839 | | |
| Error: 0.0 | Error: 0.0096*MS(subject(sequence)) + 0.9904*MS(Error) | | | | |

| Source | DF Type I SS | Mean Square | F Value | Pr > F |
|-------------------|--------------|-------------|---------|--------|
| subject(sequence) | 26 386704 | 14873 | 1.38 | 0.2134 |
| Error: MS(Error) | 25 270002 | 10800 | | |

Comparison: A vs B

Dependent Variable: T<sub>1/2 el</sub> (h)

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LAMZHL

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 5200.378088 | 5200.378088 | 0.35 | 0.5600 |
| Error | 25.627 | 382192 | 14914 | | |
| Error: 1.01*MS(subject(sequence)) - 0.01*MS(Error) | | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 23913 | 23913 | 2.21 | 0.1493 |
| trt | 1 | 35.597453 | 35.597453 | 0.00 | 0.9547 |
| subject(sequence) | 26 | 386704 | 14873 | 1.38 | 0.2134 |
| Error: MS(Error) | 25 | 270002 | 10800 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 4819.645818 | 4819.645818 | 0.33 | 0.5730 |
| Error | 26.698 | 395110 | 14799 | | |
| Error: 0.98 | Error: 0.9818*MS(subject(sequence)) + 0.0182*MS(Error) | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 23913 | 23913 | 2.21 | 0.1493 |
| trt | 1 | 35.597453 | 35.597453 | 0.00 | 0.9547 |
| subject(sequence) | 26 | 386704 | 14873 | 1.38 | 0.2134 |
| Error: MS(Error) | 25 | 270002 | 10800 | | |

Comparison: A vs B

Dependent Variable: T<sub>1/2 el</sub> (h)

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 4819.645818 | 4819.645818 | 0.33 | 0.5730 |
| Error | 26.698 | 395110 | 14799 | | |
| Error: 0.98 | Error: 0.9818*MS(subject(sequence)) + 0.0182*MS(Error) | | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 23913 | 23913 | 2.21 | 0.1493 |
| trt | 1 | 35.597453 | 35.597453 | 0.00 | 0.9547 |
| subject(sequence) | 26 | 386704 | 14873 | 1.38 | 0.2134 |
| Error: MS(Error) | 25 | 270002 | 10800 | - | |

Comparison: A vs B

Dependent Variable: T<sub>1/2 el</sub> (h)

#### Least Squares Means

| | | | H0:LSMean1=LSMean2 | |
|---|---|---|---|---|
| | | | HU.LSIVIEAIII-LSIVIEAIIZ | |
| trt | LAMZHL LSMEAN | | | Pr > t |
| Α | 97.1991044 | | | 0.9547 |
| В | 95.5741519 | | | |
| trt | LAMZHL LSMEAN | | 90% Confidence Limits | |
| A | 97.199104 | 63.651764 | 130.746444 | |
| В | 95.574152 | 60.760432 | 130.387872 | |
| Lea | ast Squares Means for Effe | ect trt | | |
| | Difference Between | | | |
| i | j Means | 90% Confid | dence Limits for LSMean(i)-L | SMean(j) |
| 1 | 2 1.624952 | -46.721910 | 49.971815 | <u> </u> |

| _ | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confi | dence Limits |
| A - B | 1.62495244 | 28.3037931 | 0.06 | 0.9547-4 | 6.72191032 | 49.97181521 |

# **Listing 16.1.9-1 ANOVA for Treatment Comparison of Diazepam - PK Population** Comparison: C vs B

Dependent Variable: AUC<sub>0-t</sub> (h\*ng/mL)

#### The GLM Procedure

| Class | Levels | Values |
|----------|--------|-------------------------------------|
| subject | 9 | 101 201 202 203 204 301 402 404 406 |
| sequence | 2 | ABC BAC |
| trt | 2 | ВС |

Comparison: C vs B

Dependent Variable: AUC<sub>0-t</sub> (h\*ng/mL)

#### The GLM Procedure

| R-Square | Coeff Var | Root MSE | | LN_AUC | LST Mean |
|---|---|---|---|---|---|
| 0.756552 | 3.539328 | 0.317973 | 8.983989 | | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.00053007 | 0.00053007 | 0.01 | 0.9441 |
| trt | 1 | 0.02765765 | 0.02765765 | 0.27 | 0.6151 |
| subject(sequence | e) 7 | 2.48544900 | 0.35506414 | 3.51 | 0.0496 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.00053007 | 0.00053007 | 0.01 | 0.9441 |
| trt | 1 | 0.02765765 | 0.02765765 | 0.27 | 0.6151 |
| subject(sequence | e) 7 | 2.48544900 | 0.35506414 | 3.51 | 0.0496 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.00053007 | 0.00053007 | 0.01 | 0.9441 |
| trt | 1 | 0.02765765 | 0.02765765 | 0.27 | 0.6151 |
| subject(sequence | e) 7 | 2.48544900 | 0.35506414 | 3.51 | 0.0496 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.00053007 | 0.00053007 | 0.01 | 0.9441 |
| trt | 1 | 0.02765765 | 0.02765765 | 0.27 | 0.6151 |
| subject(sequence | e) 7 | 2.48544900 | 0.35506414 | 3.51 | 0.0496 |

Comparison: C vs B

Dependent Variable: AUC<sub>0-t</sub> (h\*ng/mL)

# The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_AUCLST

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.000530 | 0.000530 | 0.00 | 0.9703 |
| Error | 7 | 2.485449 | 0.355064 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-------------------|----|-----------|-------------|---------|--------|
| trt | 1 | 0.027658 | 0.027658 | 0.27 | 0.6151 |
| subject(sequence) | 7 | 2.485449 | 0.355064 | 3.51 | 0.0496 |
| Error: MS(Error) | 8 | 0.808854 | 0.101107 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.000530 | 0.000530 | 0.00 | 0.9703 |
| Error | 7 | 2.485449 | 0.355064 | | |
| Error: MS(s | ubject(s | equence)) | Error: MS(subject(sequence)) | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| trt | 1 | 0.027658 | 0.027658 | 0.27 | 0.6151 |
| subject(sequence) | 7 | 2.485449 | 0.355064 | 3.51 | 0.0496 |
| Error: MS(Error) | 8 | 0.808854 | 0.101107 | | - |

Comparison: C vs B

Dependent Variable: AUC<sub>0-t</sub> (h\*ng/mL)

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_AUCLST

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.000530 | 0.000530 | 0.00 | 0.9703 |
| Error | 7 | 2.485449 | 0.355064 | | |
| Error: MS(s | Error: MS(subject(sequence)) | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| trt | 1 | 0.027658 | 0.027658 | 0.27 | 0.6151 |
| subject(sequence) | 7 | 2.485449 | 0.355064 | 3.51 | 0.0496 |
| Error: MS(Error) | 8 | 0.808854 | 0.101107 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.000530 | 0.000530 | 0.00 | 0.9703 |
| Error | 7 | 2.485449 | 0.355064 | | |
| Error: MS(s | Error: MS(subject(sequence)) | | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| trt | 1 | 0.027658 | 0.027658 | 0.27 | 0.6151 |
| subject(sequence) | 7 | 2.485449 | 0.355064 | 3.51 | 0.0496 |
| Error: MS(Error) | 8 | 0.808854 | 0.101107 | | |

Comparison: C vs B

Dependent Variable: AUC<sub>0-t</sub> (h\*ng/mL)

#### Least Squares Means

| | | H0:1 | LSMean1=LSMean2 | |
|---|---|---|---|---|
| trt | LN_AUCLST LSMEA | N | | Pr > t |
| В | 8.94418393 | | | 0.6151 |
| C | 9.02258127 | | | |
| trt | LN_AUCLST LSMEA | AN 9 | 0% Confidence Limits | |
| В | 8.944184 | 8.746474 | 9.141894 | |
| C | 9.022581 | 8.824871 | 9.220291 | |
| Lea | ast Squares Means for Ef | fect trt | | |
| | Difference Between | | | |
| i | j Means | 90% Confidence I | Limits for LSMean(i)-LSM | Iean(j) |
| 1 | 2 -0.078397 | -0.357132 | 0.200337 | |

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confidence | ce Limits |
| C - B | 0.07839735 | 0.14989384 | 0.52 | 0.6151-0 | 0.20033744 0.3 | 35713214 |

# **Listing 16.1.9-1 ANOVA for Treatment Comparison of Diazepam - PK Population** Comparison: C vs B

Dependent Variable: AUC<sub>0-inf</sub> (h\*ng/mL)

#### The GLM Procedure

| Class Level | Information | n | |
|---|---|---|---|
| Class | Levels | Values | |
| subject | 9 | 101 201 202 203 204 301 402 404 406 | |
| sequence | 2 | ABC BAC | |
| trt | 2 | BC | |
| Number of | Observation | ns Read | 18 |
| Number of Observations Used 18 | | | |

Comparison: C vs B

Dependent Variable: AUC<sub>0-inf</sub> (h\*ng/mL)

#### The GLM Procedure

| R-Square | Coeff Var | Root MSE | | LN_AUC | IFO Mean |
|---|---|---|---|---|---|
| 0.808882 | 3.355740 | 0.305435 | 9.101874 | | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| | | 0.01021615 | 0.01021615 | 0.11 | |
| sequence | 1 | **** | ****** | | 0.7492 |
| trt | 1 | 0.06391088 | 0.06391088 | 0.69 | 0.4318 |
| subject(sequence | ee) 7 | 3.08458984 | 0.44065569 | 4.72 | 0.0222 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.01021615 | 0.01021615 | 0.11 | 0.7492 |
| trt | 1 | 0.06391088 | 0.06391088 | 0.69 | 0.4318 |
| subject(sequence | e) 7 | 3.08458984 | 0.44065569 | 4.72 | 0.0222 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.01021615 | 0.01021615 | 0.11 | 0.7492 |
| trt | 1 | 0.06391088 | 0.06391088 | 0.69 | 0.4318 |
| subject(sequence | e) 7 | 3.08458984 | 0.44065569 | 4.72 | 0.0222 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.01021615 | 0.01021615 | 0.11 | 0.7492 |
| trt | 1 | 0.06391088 | 0.06391088 | 0.11 | 0.7432 |
| subject(sequence | - | 3.08458984 | 0.44065569 | 4.72 | 0.4318 |
| <u>subject(sequence</u> | ,,, , | J.00-J070- | 0.77003307 | 7.72 | 0.0222 |

Comparison: C vs B

Dependent Variable: AUC<sub>0-inf</sub> (h\*ng/mL)

# The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_AUCIFO

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.010216 | 0.010216 | 0.02 | 0.8833 |
| Error | 7 | 3.084590 | 0.440656 | | _ |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-------------------|----|-----------|-------------|---------|--------|
| trt | 1 | 0.063911 | 0.063911 | 0.69 | 0.4318 |
| subject(sequence) | 7 | 3.084590 | 0.440656 | 4.72 | 0.0222 |
| Error: MS(Error) | 8 | 0.746325 | 0.093291 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.010216 | 0.010216 | 0.02 | 0.8833 |
| Error | 7 | 3.084590 | 0.440656 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| trt | 1 | 0.063911 | 0.063911 | 0.69 | 0.4318 |
| subject(sequence) | 7 | 3.084590 | 0.440656 | 4.72 | 0.0222 |
| Error: MS(Error) | 8 | 0.746325 | 0.093291 | | |

Comparison: C vs B

Dependent Variable: AUC<sub>0-inf</sub> (h\*ng/mL)

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_AUCIFO

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.010216 | 0.010216 | 0.02 | 0.8833 |
| Error | 7 | 3.084590 | 0.440656 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| trt | 1 | 0.063911 | 0.063911 | 0.69 | 0.4318 |
| subject(sequence) | 7 | 3.084590 | 0.440656 | 4.72 | 0.0222 |
| Error: MS(Error) | 8 | 0.746325 | 0.093291 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.010216 | 0.010216 | 0.02 | 0.8833 |
| Error | 7 | 3.084590 | 0.440656 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| trt | 1 | 0.063911 | 0.063911 | 0.69 | 0.4318 |
| subject(sequence) | 7 | 3.084590 | 0.440656 | 4.72 | 0.0222 |
| Error: MS(Error) | 8 | 0.746325 | 0.093291 | | |

Comparison: C vs B

Dependent Variable: AUC<sub>0-inf</sub> (h\*ng/mL)

2 -0.119174

#### Least Squares Means

| | | H0:LSN | Mean1=LSMean2 | |
|---|---|---|---|---|
| trt | LN_AUCIFO LSMEAN | | | Pr > t |
| В | 9.03962326 | | | 0.4318 |
| C | 9.15879716 | | | |
| trt | LN_AUCIFO LSMEAN | 90% | Confidence Limits | |
| В | 9.039623 | 8.849709 | 9.229538 | |
| C | 9.158797 | 8.968883 | 9.348712 | |
| Lea | ast Squares Means for Effect | trt | | |
| | Difference Between | | | |
| i | j Means | 90% Confidence Lim | its for LSMean(i)-LSI | Mean(j) |

#### Dependent Variable: LN\_AUCIFO

-0.386918 0.148570

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confi | dence Limits |
| C - B | 0.11917390 | 0.14398354 | 0.83 | 0.4318-0 | 0.14857041 | 0.38691820 |

# **Listing 16.1.9-1 ANOVA for Treatment Comparison of Diazepam - PK Population** Comparison: C vs B

Dependent Variable: C<sub>max</sub> (ng/mL)

#### The GLM Procedure

| Class | Levels | Values |
|----------|--------|-------------------------------------|
| subject | 9 | 101 201 202 203 204 301 402 404 406 |
| sequence | 2 | ABC BAC |
| trt | 2 | ВС |

Comparison: C vs B

Dependent Variable: C<sub>max</sub> (ng/mL)

#### The GLM Procedure

Dependent Variable: LN\_CMAX

| R-Square | Coeff Var | Root MSE | | LN_C | CMAX Mean |
|---|---|---|---|---|---|
| 0.611429 | 8.546452 | 0.452382 | 5.293215 | _ | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.02048684 | 0.02048684 | 0.10 | 0.7598 |
| trt | 1 | 0.16288431 | 0.16288431 | 0.80 | 0.3984 |
| subject(sequence | ce) 7 | 2.39281131 | 0.34183019 | 1.67 | 0.2436 |
| <u> </u> | DE | T. H.GG | ) | D 1 / 1 | D . E |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.02048684 | 0.02048684 | 0.10 | 0.7598 |
| trt | 1 | 0.16288431 | 0.16288431 | 0.80 | 0.3984 |
| subject(sequence | ce) 7 | 2.39281131 | 0.34183019 | 1.67 | 0.2436 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.02048684 | 0.02048684 | 0.10 | 0.7598 |
| trt | 1 | 0.16288431 | 0.16288431 | 0.80 | 0.3984 |
| subject(sequence | ce) 7 | 2.39281131 | 0.34183019 | 1.67 | 0.2436 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.02048684 | 0.02048684 | 0.10 | 0.7598 |
| trt | 1 | 0.16288431 | 0.16288431 | 0.80 | 0.3984 |
| subject(sequence | ce) 7 | 2.39281131 | 0.34183019 | 1.67 | 0.2436 |

Comparison: C vs B

Dependent Variable: C<sub>max</sub> (ng/mL)

# The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_CMAX

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.020487 | 0.020487 | 0.06 | 0.8136 |
| Error | 7 | 2.392811 | 0.341830 | | _ |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-------------------|----|-----------|-------------|---------|--------|
| trt | 1 | 0.162884 | 0.162884 | 0.80 | 0.3984 |
| subject(sequence) | 7 | 2.392811 | 0.341830 | 1.67 | 0.2436 |
| Error: MS(Error) | 8 | 1.637197 | 0.204650 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_CMAX

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.020487 | 0.020487 | 0.06 | 0.8136 |
| Error | 7 | 2.392811 | 0.341830 | | |
| Error: MS(s | Error: MS(subject(sequence)) | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| trt | 1 | 0.162884 | 0.162884 | 0.80 | 0.3984 |
| subject(sequence) | 7 | 2.392811 | 0.341830 | 1.67 | 0.2436 |
| Error: MS(Error) | 8 | 1.637197 | 0.204650 | | |

Comparison: C vs B

Dependent Variable: C<sub>max</sub> (ng/mL)

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_CMAX

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.020487 | 0.020487 | 0.06 | 0.8136 |
| Error | 7 | 2.392811 | 0.341830 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| trt | 1 | 0.162884 | 0.162884 | 0.80 | 0.3984 |
| subject(sequence) | 7 | 2.392811 | 0.341830 | 1.67 | 0.2436 |
| Error: MS(Error) | 8 | 1.637197 | 0.204650 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_CMAX

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.020487 | 0.020487 | 0.06 | 0.8136 |
| Error | 7 | 2.392811 | 0.341830 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| trt | 1 | 0.162884 | 0.162884 | 0.80 | 0.3984 |
| subject(sequence) | 7 | 2.392811 | 0.341830 | 1.67 | 0.2436 |
| Error: MS(Error) | 8 | 1.637197 | 0.204650 | | |

Comparison: C vs B

Dependent Variable: C<sub>max</sub> (ng/mL)

j Means 2 0.190254

#### Least Squares Means

| | | H0: | LSMean1=LSMean2 | |
|---|---|---|---|---|
| trt | LN_CMAX LSMEAN | | | Pr > t |
| В | 5.39211392 | | | 0.3984 |
| C | 5.20186011 | | | |
| trt | LN CMAX LSMEAN | Ç | 90% Confidence Limits | |
| В | 5.392114 | 5.110830 | 5.673398 | |
| C | 5.201860 | 4.920576 | 5.483144 | |
| Lea | ast Squares Means for Effect trt | | | |
| | Difference Between | | | |

#### Dependent Variable: LN\_CMAX

-0.206304

90% Confidence Limits for LSMean(i)-LSMean(j)

0.586812

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confid | dence Limits |
| C - B | -0.19025381 | 0.21325497 | -0.89 | 0.3984-0 | 0.58681167 | 0.20630405 |

# **Listing 16.1.9-1 ANOVA for Treatment Comparison of Diazepam - PK Population** Comparison: C vs B

Dependent Variable: Cl/F/kg ((L/h)/kg)

#### The GLM Procedure

| Class Level | Information | n | |
|---|---|---|---|
| Class | Levels | Values | |
| subject | 9 | 101 201 202 203 204 301 402 404 406 | |
| sequence | 2 | ABC BAC | |
| trt | 2 | BC | |
| Number of | Observation | ns Read | 18 |
| Number of Observations Read 18<br>Number of Observations Used 18 | | | |

Comparison: C vs B

Dependent Variable: Cl/F/kg ((L/h)/kg)

#### The GLM Procedure

| R-Square | Coeff Var | Root MSE | | LN_CLF | OW Mean |
|------------------|-----------|-------------|-------------|---------|---------|
| 0.830934 | -8.026668 | 0.309145 | -3.851478 | | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.10324202 | 0.10324202 | 1.08 | 0.3290 |
| trt | 1 | 0.20373302 | 0.20373302 | 2.13 | 0.1824 |
| subject(sequence | e) 7 | 3.45075985 | 0.49296569 | 5.16 | 0.0172 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.10324202 | 0.10324202 | 1.08 | 0.3290 |
| trt | 1 | 0.20373302 | 0.20373302 | 2.13 | 0.1824 |
| subject(sequence | e) 7 | 3.45075985 | 0.49296569 | 5.16 | 0.0172 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.10324202 | 0.10324202 | 1.08 | 0.3290 |
| trt | 1 | 0.20373302 | 0.20373302 | 2.13 | 0.1824 |
| subject(sequence | e) 7 | 3.45075985 | 0.49296569 | 5.16 | 0.0172 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.10324202 | 0.10324202 | 1.08 | 0.3290 |
| trt | 1 | 0.20373302 | 0.20373302 | 2.13 | 0.1824 |
| subject(sequence | e) 7 | 3.45075985 | 0.49296569 | 5.16 | 0.0172 |

Comparison: C vs B

Dependent Variable: Cl/F/kg ((L/h)/kg)

# The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_CLFOW

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.103242 | 0.103242 | 0.21 | 0.6611 |
| Error | 7 | 3.450760 | 0.492966 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-------------------|----|-----------|-------------|---------|--------|
| trt | 1 | 0.203733 | 0.203733 | 2.13 | 0.1824 |
| subject(sequence) | 7 | 3.450760 | 0.492966 | 5.16 | 0.0172 |
| Error: MS(Error) | 8 | 0.764567 | 0.095571 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.103242 | 0.103242 | 0.21 | 0.6611 |
| Error | 7 | 3.450760 | 0.492966 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| trt | 1 | 0.203733 | 0.203733 | 2.13 | 0.1824 |
| subject(sequence) | 7 | 3.450760 | 0.492966 | 5.16 | 0.0172 |
| Error: MS(Error) | 8 | 0.764567 | 0.095571 | | |

Comparison: C vs B

Dependent Variable: Cl/F/kg ((L/h)/kg)

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_CLFOW

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.103242 | 0.103242 | 0.21 | 0.6611 |
| Error | 7 | 3.450760 | 0.492966 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| trt | 1 | 0.203733 | 0.203733 | 2.13 | 0.1824 |
| subject(sequence) | 7 | 3.450760 | 0.492966 | 5.16 | 0.0172 |
| Error: MS(Error) | 8 | 0.764567 | 0.095571 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.103242 | 0.103242 | 0.21 | 0.6611 |
| Error | 7 | 3.450760 | 0.492966 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| trt | 1 | 0.203733 | 0.203733 | 2.13 | 0.1824 |
| subject(sequence) | 7 | 3.450760 | 0.492966 | 5.16 | 0.0172 |
| Error: MS(Error) | 8 | 0.764567 | 0.095571 | | |

Comparison: C vs B

Dependent Variable: Cl/F/kg ((L/h)/kg)

#### Least Squares Means

| | | F | H0:LSMean1=LSMean2 |
|---|---|---|---|
| trt | LN_CLFOW LSMEAN | | Pr > |
| В | -3.73662235 | | 0.182 |
| C | -3.94939924 | | |
| trt | LN_CLFOW LSMEAN | | 90% Confidence Limits |
| В | -3.736622 | -3.928844 | -3.544401 |
| C | -3.949399 | -4.141621 | -3.757178 |
| Lea | ast Squares Means for Effec | t trt | |
| | Difference Between | | |
| i | j Means | 90% Confiden | ce Limits for LSMean(i)-LSMean(j) |
| 1 | 2 0.212777 | -0.058220 | 0.483774 |

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confi | dence Limits |
| C - B | -0.21277689 | 0.14573253 | -1.46 | 0.1824-0 | 0.48377353 | 0.05821975 |

Comparison: C vs B

Dependent Variable: Cl/F (L/h)

#### The GLM Procedure

| Class | Levels | Values |
|----------|--------|-------------------------------------|
| subject | 9 | 101 201 202 203 204 301 402 404 406 |
| sequence | 2 | ABC BAC |
| trt | 2 | BC |

Comparison: C vs B

Dependent Variable: Cl/F (L/h)

#### The GLM Procedure

| R-Square | Coeff Var | Root MSE | E | LN_ | CLFO Mean |
|---|---|---|---|---|---|
| 0.836327 | 52.51067 | 0.309145 | 0.588729 | _ | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.06051145 | 0.06051145 | 0.63 | 0.4492 |
| trt | 1 | 0.20373302 | 0.20373302 | 2.13 | 0.1824 |
| subject(sequence | 2) 7 | 3.64249195 | 0.52035599 | 5.44 | 0.0147 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.06051145 | 0.06051145 | 0.63 | 0.4492 |
| trt | 1 | 0.20373302 | 0.20373302 | 2.13 | 0.1824 |
| subject(sequence | 2) 7 | 3.64249195 | 0.52035599 | 5.44 | 0.0147 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.06051145 | 0.06051145 | 0.63 | 0.4492 |
| trt | 1 | 0.20373302 | 0.20373302 | 2.13 | 0.1824 |
| subject(sequence | 2) 7 | 3.64249195 | 0.52035599 | 5.44 | 0.0147 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.06051145 | 0.06051145 | 0.63 | 0.4492 |
| trt | 1 | 0.20373302 | 0.20373302 | 2.13 | 0.1824 |
| subject(sequence | ) 7 | 3.64249195 | 0.52035599 | 5.44 | 0.0147 |

Comparison: C vs B

Dependent Variable: Cl/F (L/h)

# The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_CLFO

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.060511 | 0.060511 | 0.12 | 0.7431 |
| Error 7 3.642492 | | | 0.520356 | | _ |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-------------------|----|-----------|-------------|---------|--------|
| trt | 1 | 0.203733 | 0.203733 | 2.13 | 0.1824 |
| subject(sequence) | 7 | 3.642492 | 0.520356 | 5.44 | 0.0147 |
| Error: MS(Error) | 8 | 0.764567 | 0.095571 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.060511 | 0.060511 | 0.12 | 0.7431 |
| Error | 7 | 3.642492 | 0.520356 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| trt | 1 | 0.203733 | 0.203733 | 2.13 | 0.1824 |
| subject(sequence) | 7 | 3.642492 | 0.520356 | 5.44 | 0.0147 |
| Error: MS(Error) | 8 | 0.764567 | 0.095571 | | - |

Comparison: C vs B

Dependent Variable: Cl/F (L/h)

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_CLFO

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.060511 | 0.060511 | 0.12 | 0.7431 |
| Error | 7 | 3.642492 | 0.520356 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| trt | 1 | 0.203733 | 0.203733 | 2.13 | 0.1824 |
| subject(sequence) | 7 | 3.642492 | 0.520356 | 5.44 | 0.0147 |
| Error: MS(Error) | 8 | 0.764567 | 0.095571 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.060511 | 0.060511 | 0.12 | 0.7431 |
| Error | 7 | 3.642492 | 0.520356 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| trt | 1 | 0.203733 | 0.203733 | 2.13 | 0.1824 |
| subject(sequence) | 7 | 3.642492 | 0.520356 | 5.44 | 0.0147 |
| Error: MS(Error) | 8 | 0.764567 | 0.095571 | | |

Comparison: C vs B

Dependent Variable: Cl/F (L/h)

#### Least Squares Means

| | | 110.1 | CM 1 - I CM 2 | |
|---|---|---|---|---|
| | | HU:L | SMean1=LSMean2 | |
| trt | LN_CLFO LSMEAN | | Pr | > t |
| В | 0.68863474 | | 0.1 | 824 |
| <u>C</u> | 0.47585785 | | | |
| trt | LN_CLFO LSMEAN | 90 | % Confidence Limits | |
| В | 0.688635 | 0.496413 | 0.880856 | |
| C | 0.475858 | 0.283636 | 0.668079 | |
| Lea | ast Squares Means for Eff | ect trt | | |
| | Difference Between | | | |
| i | j Means | 90% Confidence | Limits for LSMean(i)-LSMean | (j) |
| 1 | 2 0.212777 | -0.058220 | 0.483774 | |

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confid | dence Limits |
| C - B | -0.21277689 | 0.14573253 | -1.46 | 0.1824-0 | 0.48377353 | 0.05821975 |

# **Listing 16.1.9-1 ANOVA for Treatment Comparison of Diazepam - PK Population** Comparison: C vs B

Dependent Variable: V<sub>d</sub>/F/kg (L/kg)

#### The GLM Procedure

| Class | Levels | Values |
|----------|--------|-------------------------------------|
| subject | 9 | 101 201 202 203 204 301 402 404 406 |
| sequence | 2 | ABC BAC |
| trt | 2 | BC |

Comparison: C vs B

Dependent Variable: V<sub>d</sub>/F/kg (L/kg)

#### The GLM Procedure

| R-Square | Coeff Var | Root MSE | | LN_VZF | OW Mean |
|------------------|-----------|-------------|-------------|---------|---------|
| 0.476731 | 65.76292 | 0.488595 | 0.742964 | | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.29614945 | 0.29614945 | 1.24 | 0.2977 |
| trt | 1 | 0.00000581 | 0.00000581 | 0.00 | 0.9962 |
| subject(sequence | - | 1.44379145 | 0.20625592 | 0.86 | 0.5700 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.29614945 | 0.29614945 | 1.24 | 0.2977 |
| trt | 1 | 0.00000581 | 0.00000581 | 0.00 | 0.9962 |
| subject(sequence | ce) 7 | 1.44379145 | 0.20625592 | 0.86 | 0.5700 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.29614945 | 0.29614945 | 1.24 | 0.2977 |
| trt | 1 | 0.00000581 | 0.00000581 | 0.00 | 0.9962 |
| subject(sequence | ce) 7 | 1.44379145 | 0.20625592 | 0.86 | 0.5700 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.29614945 | 0.29614945 | 1.24 | 0.2977 |
| trt | 1 | 0.00000581 | 0.00000581 | 0.00 | 0.9962 |
| subject(sequence | ce) 7 | 1.44379145 | 0.20625592 | 0.86 | 0.5700 |

Comparison: C vs B

Dependent Variable: V<sub>d</sub>/F/kg (L/kg)

# The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_VZFOW

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.296149 | 0.296149 | 1.44 | 0.2698 |
| Error | 7 | 1.443791 | 0.206256 | | _ |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| trt | 1 | 0.000005808 | 0.000005808 | 0.00 | 0.9962 |
| subject(sequence) | 7 | 1.443791 | 0.206256 | 0.86 | 0.5700 |
| Error: MS(Error) | 8 | 1.909799 | 0.238725 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.296149 | 0.296149 | 1.44 | 0.2698 |
| Error | 7 | 1.443791 | 0.206256 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| trt | 1 | 0.000005808 | 0.000005808 | 0.00 | 0.9962 |
| subject(sequence) | 7 | 1.443791 | 0.206256 | 0.86 | 0.5700 |
| Error: MS(Error) | 8 | 1.909799 | 0.238725 | · | · |

Comparison: C vs B

Dependent Variable: V<sub>d</sub>/F/kg (L/kg)

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_VZFOW

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.296149 | 0.296149 | 1.44 | 0.2698 |
| Error | 7 | 1.443791 | 0.206256 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| trt | 1 | 0.000005808 | 0.000005808 | 0.00 | 0.9962 |
| subject(sequence) | 7 | 1.443791 | 0.206256 | 0.86 | 0.5700 |
| Error: MS(Error) | 8 | 1.909799 | 0.238725 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.296149 | 0.296149 | 1.44 | 0.2698 |
| Error | 7 | 1.443791 | 0.206256 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| trt | 1 | 0.000005808 | 0.000005808 | 0.00 | 0.9962 |
| subject(sequence) | 7 | 1.443791 | 0.206256 | 0.86 | 0.5700 |
| Error: MS(Error) | 8 | 1.909799 | 0.238725 | | |

Comparison: C vs B

Dependent Variable: V<sub>d</sub>/F/kg (L/kg)

2 0.001136

#### Least Squares Means

| | | H0:LSMean1=LSMean2 | | |
|---|---|---|---|---|
| trt | LN_VZFOW LSMEAN | | | Pr > t |
| В | 0.72919115 | | | 0.9962 |
| C | 0.72805507 | | | |
| trt | LN VZFOW LSMEAN | 90% Confidence Limits | | |
| В | 0.729191 | 0.425391 | 1.032991 | |
| C | 0.728055 | 0.424255 | 1.031855 | |
| Lea | ast Squares Means for Effect | trt | | |
| | Difference Between | | | |
| i | j Means | 90% Confidence Limits for LSMean(i)-LSMean(j) | | |

## Dependent Variable: LN\_VZFOW

-0.427166

0.429438

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confid | dence Limits |
| C - B | -0.00113608 | 0.23032577 | -0.00 | 0.9962-0 | 0.42943792 | 0.42716576 |
# $\begin{tabular}{ll} \textbf{Listing 16.1.9-1 ANOVA for Treatment Comparison of Diazepam - PK Population} \\ \textbf{Comparison: C vs B} \\ \textbf{Dependent Variable: $V_d/F(L)$} \end{tabular}$

#### The GLM Procedure

| | Levels | Values |
|----------|--------|-------------------------------------|
| subject | 9 | 101 201 202 203 204 301 402 404 406 |
| sequence | 2 | ABC BAC |
| trt | 2 | BC |

Comparison: C vs B

Dependent Variable: V<sub>d</sub>/F (L)

#### The GLM Procedure

| R-Square | Coeff Var | Root MSE | Ε | LN | VZFO Mean |
|---|---|---|---|---|---|
| 0.671281 | 9.426561 | 0.488595 | 5.183171 | | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 1.23543199 | 1.23543199 | 5.18 | 0.0525 |
| trt | 1 | 0.00000581 | 0.00000581 | 0.00 | 0.9962 |
| subject(sequence | e) 7 | 2.66458657 | 0.38065522 | 1.59 | 0.2632 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 1.23543199 | 1.23543199 | 5.18 | 0.0525 |
| trt | 1 | 0.00000581 | 0.00000581 | 0.00 | 0.9962 |
| subject(sequence | e) 7 | 2.66458657 | 0.38065522 | 1.59 | 0.2632 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 1.23543199 | 1.23543199 | 5.18 | 0.0525 |
| trt | 1 | 0.00000581 | 0.00000581 | 0.00 | 0.9962 |
| subject(sequence | e) 7 | 2.66458657 | 0.38065522 | 1.59 | 0.2632 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 1.23543199 | 1.23543199 | 5.18 | 0.0525 |
| trt | 1 | 0.00000581 | 0.00000581 | 0.00 | 0.9962 |
| subject(sequence | e) 7 | 2.66458657 | 0.38065522 | 1.59 | 0.2632 |

Comparison: C vs B

Dependent Variable: V<sub>d</sub>/F (L)

## The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_VZFO

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 1.235432 | 1.235432 | 3.25 | 0.1146 |
| Error | 7 | 2.664587 | 0.380655 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| trt | 1 | 0.000005808 | 0.000005808 | 0.00 | 0.9962 |
| subject(sequence) | 7 | 2.664587 | 0.380655 | 1.59 | 0.2632 |
| Error: MS(Error) | 8 | 1.909799 | 0.238725 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 1.235432 | 1.235432 | 3.25 | 0.1146 |
| Error | 7 | 2.664587 | 0.380655 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| trt | 1 | 0.000005808 | 0.000005808 | 0.00 | 0.9962 |
| subject(sequence) | 7 | 2.664587 | 0.380655 | 1.59 | 0.2632 |
| Error: MS(Error) | 8 | 1.909799 | 0.238725 | | |

Comparison: C vs B

Dependent Variable: V<sub>d</sub>/F (L)

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_VZFO

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 1.235432 | 1.235432 | 3.25 | 0.1146 |
| Error | 7 | 2.664587 | 0.380655 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| trt | 1 | 0.000005808 | 0.000005808 | 0.00 | 0.9962 |
| subject(sequence) | 7 | 2.664587 | 0.380655 | 1.59 | 0.2632 |
| Error: MS(Error) | 8 | 1.909799 | 0.238725 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 1.235432 | 1.235432 | 3.25 | 0.1146 |
| Error | 7 | 2.664587 | 0.380655 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| trt | 1 | 0.000005808 | 0.000005808 | 0.00 | 0.9962 |
| subject(sequence) | 7 | 2.664587 | 0.380655 | 1.59 | 0.2632 |
| Error: MS(Error) | 8 | 1.909799 | 0.238725 | | |

Comparison: C vs B

Dependent Variable: V<sub>d</sub>/F (L)

#### Least Squares Means

| | | Н | 0:LSMean1=LSMean2 | |
|-----|----------------|----------|-----------------------|---------|
| trt | LN_VZFO LSMEAN | | | Pr > t |
| В | 5.15444823 | | | 0.9962 |
| C | 5.15331216 | | | |
| trt | LN_VZFO LSMEAN | | 90% Confidence Limits | |
| В | 5.154448 | 4.850648 | 5.458248 | |
| C | 5.153312 | 4.849512 | 5.457112 | |

| Le | Least Squares Means for Effect trt | | | |
|---|---|---|---|---|
| | | Difference Between | | |
| i | j | Means | 90% Confider | nce Limits for LSMean(i)-LSMean(j) |
| 1 | 2 | 0.001136 | -0.427166 | 0.429438 |

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confid | dence Limits |
| C - B | -0.00113608 | 0.23032577 | -0.00 | 0.9962-0 | 0.42943792 | 0.42716576 |

# **Listing 16.1.9-1 ANOVA for Treatment Comparison of Diazepam - PK Population** Comparison: C vs B

Dependent Variable: T<sub>max</sub> (h)

#### The GLM Procedure

| Class Level | Information | n | |
|-------------|-------------|-------------------------------------|----|
| Class | Levels | Values | |
| subject | 9 | 101 201 202 203 204 301 402 404 406 | |
| sequence | 2 | ABC BAC | |
| trt | 2 | BC | |
| Number of | Observation | ns Read | 18 |

Comparison: C vs B

Dependent Variable: T<sub>max</sub> (h)

#### The GLM Procedure

| R-Square | Coeff Var | Root | MSE | T | MAX Mean |
|---|---|---|---|---|---|
| 0.631705 | 72.78556 | 0.933 | 434 1. | 282444 | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.35576247 | 0.35576247 | 0.41 | 0.5407 |
| trt | 1 | 7.32679200 | 7.32679200 | 8.41 | 0.0199 |
| subject(sequence) | 7 | 4.27317898 | 0.61045414 | 0.70 | 0.6739 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.35576247 | 0.35576247 | 0.41 | 0.5407 |
| trt | 1 | 7.32679200 | 7.32679200 | 8.41 | 0.0199 |
| subject(sequence) | 7 | 4.27317898 | 0.61045414 | 0.70 | 0.6739 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.35576247 | 0.35576247 | 0.41 | 0.5407 |
| trt | 1 | 7.32679200 | 7.32679200 | 8.41 | 0.0199 |
| subject(sequence) | 7 | 4.27317898 | 0.61045414 | 0.70 | 0.6739 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.35576247 | 0.35576247 | 0.41 | 0.5407 |
| trt | 1 | 7.32679200 | 7.32679200 | 8.41 | 0.0199 |
| <pre>subject(sequence)</pre> | 7 | 4.27317898 | 0.61045414 | 0.70 | 0.6739 |

Comparison: C vs B

Dependent Variable: T<sub>max</sub> (h)

## The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: TMAX

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-------------|----------|-----------|-------------|---------|--------|
| sequence | 1 | 0.355762 | 0.355762 | 0.58 | 0.4702 |
| Error | 7 | 4.273179 | 0.610454 | | |
| Error: MS(s | ubject(s | equence)) | | | _ |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-------------------|----|-----------|-------------|---------|--------|
| trt | 1 | 7.326792 | 7.326792 | 8.41 | 0.0199 |
| subject(sequence) | 7 | 4.273179 | 0.610454 | 0.70 | 0.6739 |
| Error: MS(Error) | 8 | 6.970397 | 0.871300 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------|-----------|------------|-------------|---------|--------|
| sequence | 1 | 0.355762 | 0.355762 | 0.58 | 0.4702 |
| Error | 7 | 4.273179 | 0.610454 | | |
| Error: MS(s | subject(s | equence)) | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| trt | 1 | 7.326792 | 7.326792 | 8.41 | 0.0199 |
| subject(sequence) | 7 | 4.273179 | 0.610454 | 0.70 | 0.6739 |
| Error: MS(Error) | 8 | 6.970397 | 0.871300 | | |

Comparison: C vs B

Dependent Variable: T<sub>max</sub> (h)

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: TMAX

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------|-----------|-------------|-------------|---------|--------|
| sequence | 1 | 0.355762 | 0.355762 | 0.58 | 0.4702 |
| Error | 7 | 4.273179 | 0.610454 | | |
| Error: MS(s | subject(s | sequence)) | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| trt | 1 | 7.326792 | 7.326792 | 8.41 | 0.0199 |
| subject(sequence) | 7 | 4.273179 | 0.610454 | 0.70 | 0.6739 |
| Error: MS(Error) | 8 | 6.970397 | 0.871300 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------|-----------|------------|-------------|---------|--------|
| sequence | 1 | 0.355762 | 0.355762 | 0.58 | 0.4702 |
| Error | 7 | 4.273179 | 0.610454 | | |
| Error: MS(s | subject(s | sequence)) | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| trt | 1 | 7.326792 | 7.326792 | 8.41 | 0.0199 |
| subject(sequence) | 7 | 4.273179 | 0.610454 | 0.70 | 0.6739 |
| Error: MS(Error) | 8 | 6.970397 | 0.871300 | | |

Comparison: C vs B

Dependent Variable: T<sub>max</sub> (h)

#### Least Squares Means

| | | H0:LSM | ean1=LSMean2 |
|----------|-------------------------|--------|----------------------------|
| trt | TMAX LSMEAN | | $P_{r} > $ |
| В | 0.66016250 | | 0.019 |
| C | 1.93616250 | | |
| trt | TMAX LSMEAN | 90% ( | Confidence Limits |
| trt<br>B | TMAX LSMEAN<br>0.660162 | 90% ( | Confidence Limits 1.240556 |

Least Squares Means for Effect trt

Difference Between

i j Means 90% Confidence Limits for LSMean(i)-LSMean(j)

1 2 -1.276000 -2.094248 -0.457752

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confi | idence Limits |
| C - B | 1.27600000 | 0.44002516 | 2.90 | 0.01990 | .45775208 | 2.09424792 |

# **Listing 16.1.9-1 ANOVA for Treatment Comparison of Diazepam - PK Population** Comparison: C vs B

Dependent Variable: K<sub>el</sub> (/h)

#### The GLM Procedure

| Class | Levels | Values |
|----------|--------|-------------------------------------|
| subject | 9 | 101 201 202 203 204 301 402 404 406 |
| sequence | 2 | ABC BAC |
| trt | 2 | ВС |

Comparison: C vs B

Dependent Variable: K<sub>el</sub> (/h)

#### The GLM Procedure

| | 0.012217<br>n Square F Val | |
|---|---|---|
| | n Square F Val | |
| | n Square F Val | |
| | n Square - F van | |
| 24799 0 000 | | |
| | 024799 34.99 | 0.0004 |
| | 001316 1.86 | 0.2100 |
| 26274 0.000 | 018039 25.45 | <.0001 |
| ISS Mea | n Square — F Vali | ${\text{ue}} \text{Pr} > \text{F}$ |
| | | 0.0004 |
| | | 0.2100 |
| 202/4 0.000 | 018039 23.43 | <.0001 |
| II SS Mean | n Square F Val | $\overline{ue}$ $Pr > F$ |
| 4799 0.000 | 024799 34.99 | 0.0004 |
| 0.000 | 001316 1.86 | 0.2100 |
| 26274 0.000 | 018039 25.45 | <.0001 |
| VICC M | C EVI | D > E |
| | | 0.0004 |
| | | 0.2100 |
| 26274 0.000 | 018039 25.45 | <.0001 |
| | II SS Mea 24799 0.00 01316 0.00 026274 0.00 III SS Mea 24799 0.00 01316 0.00 026274 0.00 IV SS Mea 24799 0.00 01316 0.00 01316 0.00 01316 0.00 | ISS Mean Square F Value Value |

Comparison: C vs B

Dependent Variable: Kel (/h)

## The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LAMZ

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.000248 | 0.000248 | 1.37 | 0.2793 |
| Error | 7 | 0.001263 | 0.000180 | | _ |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| trt | 1 | 0.000013165 | 0.000013165 | 1.86 | 0.2100 |
| subject(sequence) | 7 | 0.001263 | 0.000180 | 25.45 | <.0001 |
| Error: MS(Error) | 8 | 0.000056699 | 0.000007087 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.000248 | 0.000248 | 1.37 | 0.2793 |
| Error | 7 | 0.001263 | 0.000180 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| trt | 1 | 0.000013165 | 0.000013165 | 1.86 | 0.2100 |
| subject(sequence) | 7 | 0.001263 | 0.000180 | 25.45 | <.0001 |
| Error: MS(Error) | 8 | 0.000056699 | 0.000007087 | · | · |

Comparison: C vs B

Dependent Variable: K<sub>el</sub> (/h)

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LAMZ

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.000248 | 0.000248 | 1.37 | 0.2793 |
| Error | 7 | 0.001263 | 0.000180 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| trt | 1 | 0.000013165 | 0.000013165 | 1.86 | 0.2100 |
| subject(sequence) | 7 | 0.001263 | 0.000180 | 25.45 | <.0001 |
| Error: MS(Error) | 8 | 0.000056699 | 0.000007087 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.000248 | 0.000248 | 1.37 | 0.2793 |
| Error | 7 | 0.001263 | 0.000180 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| trt | 1 | 0.000013165 | 0.000013165 | 1.86 | 0.2100 |
| subject(sequence) | 7 | 0.001263 | 0.000180 | 25.45 | <.0001 |
| Error: MS(Error) | 8 | 0.000056699 | 0.000007087 | | |

Comparison: C vs B

Dependent Variable: K<sub>el</sub> (/h)

#### Least Squares Means

| _ | | H0·LSMea | n1=LSMean2 | |
|-----|-------------|-----------------------|----------------|---------|
| trt | LAMZ LSMEAN | 110.1251/104 | III ESIVICAIIE | Pr > t |
| В | 0.01348751 | | | 0.2100 |
| C | 0.01177711 | | | |
| trt | LAMZ LSMEAN | 90% Confidence Limits | | |
| В | 0.013488 | 0.011832 | 0.015143 | |
| C | 0.011777 | 0.010122 | 0.013432 | |

| Le | Least Squares Means for Effect trt | | | |
|---|---|---|---|---|
| Difference Between | | | | |
| i | j | Means | 90% Confide | ence Limits for LSMean(i)-LSMean(j) |
| 1 | 2 | 0.001710 | -0.000623 | 0.004044 |

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confid | dence Limits |
| C - B | -0.00171041 | 0.00125498 | -1.36 | 0.2100-0 | 0.00404409 | 0.00062328 |

# **Listing 16.1.9-1 ANOVA for Treatment Comparison of Diazepam - PK Population** Comparison: C vs B

Dependent Variable: T<sub>1/2 el</sub> (h)

#### The GLM Procedure

| Class Level | Information | n | |
|---|---|---|---|
| Class | Levels | Values | |
| subject | 9 | 101 201 202 203 204 301 402 404 406 | |
| sequence | 2 | ABC BAC | |
| trt | 2 | ВС | |
| Number of | Observation | ns Read | 18 |
| Number of | Number of Observations Used 18 | | |

Comparison: C vs B

Dependent Variable: T<sub>1/2 el</sub> (h)

#### The GLM Procedure

| R-Square | Coeff Var | Root MSE | | LAMZ | HL Mean |
|------------------|-----------|-------------|-------------|---------|---------|
| 0.678170 | 39.06391 | 30.52961 | 78.15299 | | |
| | | | 1. | | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 1843.72360 | 1843.72360 | 1.98 | 0.1972 |
| trt | 1 | 1955.28434 | 1955.28434 | 2.10 | 0.1855 |
| subject(sequence | e) 7 | 11913.47712 | 1701.92530 | 1.83 | 0.2085 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 1843.72360 | 1843.72360 | 1.98 | 0.1972 |
| trt | 1 | 1955.28434 | 1955.28434 | 2.10 | 0.1855 |
| subject(sequence | e) 7 | 11913.47712 | 1701.92530 | 1.83 | 0.2085 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 1843.72360 | 1843.72360 | 1.98 | 0.1972 |
| trt | 1 | 1955.28434 | 1955.28434 | 2.10 | 0.1855 |
| subject(sequence | e) 7 | 11913.47712 | 1701.92530 | 1.83 | 0.2085 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 1843.72360 | 1843.72360 | 1.98 | 0.1972 |
| trt | 1 | 1955.28434 | 1955.28434 | 2.10 | 0.1855 |
| subject(sequence | e) 7 | 11913.47712 | 1701.92530 | 1.83 | 0.2085 |

Comparison: C vs B

Dependent Variable: T<sub>1/2 el</sub> (h)

## The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LAMZHL

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 1843.723597 | 1843.723597 | 1.08 | 0.3326 |
| Error | 7 | 11913 | 1701.925303 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| trt | 1 | 1955.284335 | 1955.284335 | 2.10 | 0.1855 |
| subject(sequence) | 7 | 11913 | 1701.925303 | 1.83 | 0.2085 |
| Error: MS(Error) | 8 | 7456.458594 | 932.057324 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 1843.723597 | 1843.723597 | 1.08 | 0.3326 |
| Error | 7 | 11913 | 1701.925303 | | |
| Error: MS(s | Error: MS(subject(sequence)) | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| trt | 1 | 1955.284335 | 1955.284335 | 2.10 | 0.1855 |
| subject(sequence) | 7 | 11913 | 1701.925303 | 1.83 | 0.2085 |
| Error: MS(Error) | 8 | 7456.458594 | 932.057324 | | |

Comparison: C vs B

Dependent Variable: T<sub>1/2 el</sub> (h)

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LAMZHL

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 1843.723597 | 1843.723597 | 1.08 | 0.3326 |
| Error | 7 | 11913 | 1701.925303 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| trt | 1 | 1955.284335 | 1955.284335 | 2.10 | 0.1855 |
| subject(sequence) | 7 | 11913 | 1701.925303 | 1.83 | 0.2085 |
| Error: MS(Error) | 8 | 7456.458594 | 932.057324 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 1843.723597 | 1843.723597 | 1.08 | 0.3326 |
| Error | 7 | 11913 | 1701.925303 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| trt | 1 | 1955.284335 | 1955.284335 | 2.10 | 0.1855 |
| subject(sequence) | 7 | 11913 | 1701.925303 | 1.83 | 0.2085 |
| Error: MS(Error) | 8 | 7456.458594 | 932.057324 | | |

Comparison: C vs B

Dependent Variable: T<sub>1/2 el</sub> (h)

2 -20.844847

#### Least Squares Means

| | | | H0:LSMean1=LSMean2 | |
|---|---|---|---|---|
| trt | LAMZHL LSMEAN | | | Pr > t |
| В | 66.5990342 | | | 0.1855 |
| C | 87.4438808 | | | |
| trt | LAMZHL LSMEAN | | 90% Confidence Limits | |
| В | 66.599034 | 47.616228 | 85.581840 | |
| C | 87.443881 | 68.461075 | 106.426687 | |
| Lea | ast Squares Means for Effe | ect trt | | |
| | Difference Between | | | |
| i | j Means | 90% Confi | dence Limits for LSMean(i)-I | LSMean(j) |

#### Dependent Variable: LAMZHL

-47.607086

5.917393

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Conf | idence Limits |
| C - B | 20.8448466 | 14.3917980 | 1.45 | 0.1855- | 5.9173931 | 47.6070863 |

# Listing 16.1.9-2 ANOVA for Treatment Comparison of Nordiazepam - PK Population Comparison: A vs ${\bf B}$

Dependent Variable: AUC<sub>0-t</sub> (h\*pg/mL)

#### The GLM Procedure

| | | formation | |
|---|---|---|---|
| Class | Leve | ls Values | |
| subject | 27 | 101 201 202 203 204 205 301 302 303 304 402 | 404 406 407 408 409 |
| | | 410 411 412 413 414 501 502 503 505 507 508 | |
| sequenc | e 2 | AB BA | |
| period | 2 | 1 2 | |
| trt | 2 | A B | |
| Number | r of Ol | oservations Read | 54 |
| Marianta | of Ol | oservations Used | 54 |

Comparison: A vs B

Dependent Variable: AUC<sub>0-t</sub> (h\*pg/mL)

#### The GLM Procedure

| R-Square | Coeff Var | Root MSE | | LN_AUCI | LST Mean |
|---|---|---|---|---|---|
| 0.598953 | 3.509791 | 0.548042 | 15.61468 | | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.19341151 | 0.19341151 | 0.64 | 0.4298 |
| period | 1 | 0.10547371 | 0.10547371 | 0.35 | 0.5588 |
| trt | 1 | 0.58421444 | 0.58421444 | 1.95 | 0.1754 |
| subject(sequence | ce) 25 | 10.33106002 | 0.41324240 | 1.38 | 0.2153 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.19341151 | 0.19341151 | 0.64 | 0.4298 |
| period | 1 | 0.12450538 | 0.12450538 | 0.41 | 0.5255 |
| trt | 1 | 0.58421444 | 0.58421444 | 1.95 | 0.1754 |
| subject(sequence | ce) 25 | 10.33106002 | 0.41324240 | 1.38 | 0.2153 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.19341151 | 0.19341151 | 0.64 | 0.4298 |
| period | 1 | 0.12450538 | 0.12450538 | 0.41 | 0.5255 |
| trt | 1 | 0.58421444 | 0.58421444 | 1.95 | 0.1754 |
| subject(sequence | ce) 25 | 10.33106002 | 0.41324240 | 1.38 | 0.2153 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.19341151 | 0.19341151 | 0.64 | 0.4298 |
| period | 1 | 0.12450538 | 0.12450538 | 0.41 | 0.5255 |
| trt | 1 | 0.58421444 | 0.58421444 | 1.95 | 0.1754 |
| subject(sequence | ce) 25 | 10.33106002 | 0.41324240 | 1.38 | 0.2153 |

Comparison: A vs B

Dependent Variable: AUC<sub>0-t</sub> (h\*pg/mL)

## The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_AUCLST

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.193412 | 0.193412 | 0.47 | 0.5002 |
| Error 25 10.331060 | | 10.331060 | 0.413242 | | _ |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| *period | 1 | 0.105474 | 0.105474 | 0.35 | 0.5588 |
| trt | 1 | 0.584214 | 0.584214 | 1.95 | 0.1754 |
| subject(sequence) | 25 | 10.331060 | 0.413242 | 1.38 | 0.2153 |
| Error: MS(Error) | 25 | 7.508763 | 0.300351 | | |
| * This test assumes one or more other fixed effects are zero. | | | | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.193412 | 0.193412 | 0.47 | 0.5002 |
| Error | 25 | 10.331060 | 0.413242 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.124505 | 0.124505 | 0.41 | 0.5255 |
| trt | 1 | 0.584214 | 0.584214 | 1.95 | 0.1754 |
| subject(sequence) | 25 | 10.331060 | 0.413242 | 1.38 | 0.2153 |
| Error: MS(Error) | 25 | 7.508763 | 0.300351 | | |

Comparison: A vs B

Dependent Variable: AUC<sub>0-t</sub> (h\*pg/mL)

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_AUCLST

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.193412 | 0.193412 | 0.47 | 0.5002 |
| Error | 25 | 10.331060 | 0.413242 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 0.124505 | 0.124505 | 0.41 | 0.5255 |
| trt | 1 | 0.584214 | 0.584214 | 1.95 | 0.1754 |
| subject(sequence) | 25 | 10.331060 | 0.413242 | 1.38 | 0.2153 |
| Error: MS(Error) | 25 | 7.508763 | 0.300351 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.193412 | 0.193412 | 0.47 | 0.5002 |
| Error 25 10.331060 | | 10.331060 | 0.413242 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|-------------|
| period | 1 | 0.124505 | 0.124505 | 0.41 | 0.5255 |
| trt | 1 | 0.584214 | 0.584214 | 1.95 | 0.1754 |
| subject(sequence) | 25 | 10.331060 | 0.413242 | 1.38 | 0.2153 |
| Error: MS(Error) | 25 | 7.508763 | 0.300351 | · | <del></del> |

Comparison: A vs B

Dependent Variable: AUC<sub>0-t</sub> (h\*pg/mL)

#### Least Squares Means

| | | H0:I | LSMean1=LSMean2 | |
|---|---|---|---|---|
| trt | LN_AUCLST LSMEAN | | Pr | > t |
| A | 15.7165433 | | 0.1 | 1754 |
| В | 15.5083737 | | | |
| trt | LN_AUCLST LSMEAN | 90 | % Confidence Limits | |
| A | 15.716543 | 15.536261 | 15.896826 | |
| В | 15.508374 | 15.328091 | 15.688656 | |
| Lea | ast Squares Means for Effec | t trt | | |
| | Difference Between | | | |
| i | j Means | 90% Confidence L | imits for LSMean(i)-LSMean | ı(j) |
| 1 | 2 0.208170 | -0.046789 | 0.463128 | |

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confi | dence Limits |
| A - B | 0.20816961 | 0.14926067 | 1.39 | 0.1754-0 | 0.04678862 | 0.46312785 |

# Listing 16.1.9-2 ANOVA for Treatment Comparison of Nordiazepam - PK Population Comparison: A vs ${\bf B}$

Dependent Variable: AUC<sub>0-inf</sub> (h\*pg/mL)

#### The GLM Procedure

| Class Le | vel In | formation | |
|---|---|---|---|
| Class | Leve | ls Values | |
| subject | 23 | 101 201 202 203 204 205 301 302 303 304 404 407 408 | 410 411 412 |
| | | 413 414 501 502 503 505 507 | |
| sequence | e 2 | AB BA | |
| period | 2 | 1 2 | |
| trt | 2 | A B | |
| · | | | |
| Number | of Ob | servations Read | 38 |
| Number | Number of Observations Used 38 | | |

Comparison: A vs B

Dependent Variable: AUC<sub>0-inf</sub> (h\*pg/mL)

#### The GLM Procedure

Dependent Variable: LN\_AUCIFO

| R-Square | Coeff Var | Root MSE | | LN_AUC | IFO Mean |
|---|---|---|---|---|---|
| 0.798291 | 2.274302 | 0.367814 | 16.17260 | | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.03357891 | 0.03357891 | 0.25 | 0.6267 |
| period | 1 | 0.07277073 | 0.07277073 | 0.54 | 0.4763 |
| trt | 1 | 0.27876163 | 0.27876163 | 2.06 | 0.1748 |
| subject(sequence | e) 21 | 6.57528343 | 0.31310873 | 2.31 | 0.0612 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.01837981 | 0.01837981 | 0.14 | 0.7184 |
| period | 1 | 0.18098559 | 0.18098559 | 1.34 | 0.2682 |
| trt | 1 | 0.14121341 | 0.14121341 | 1.04 | 0.3256 |
| subject(sequence | e) 21 | 6.57528343 | 0.31310873 | 2.31 | 0.0612 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.02101493 | 0.02101493 | 0.16 | 0.6999 |
| period | 1 | 0.18098559 | 0.18098559 | 1.34 | 0.2682 |
| trt | 1 | 0.14121341 | 0.14121341 | 1.04 | 0.3256 |
| subject(sequence | e) 21 | 6.57528343 | 0.31310873 | 2.31 | 0.0612 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.02101493 | 0.02101493 | 0.16 | 0.6999 |
| period | 1 | 0.18098559 | 0.18098559 | 1.34 | 0.2682 |
| trt | 1 | 0.14121341 | 0.14121341 | 1.04 | 0.3256 |
| subject(sequence | e) 21 | 6.57528343 | 0.31310873 | 2.31 | 0.0612 |

Comparison: A vs B

Dependent Variable: AUC<sub>0-inf</sub> (h\*pg/mL)

## The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_AUCIFO

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| *sequence | 1 | 0.033579 | 0.033579 | 0.10 | 0.7532 |
| Error | 19.404 | 6.404979 | 0.330078 | | |
| E 1,007,4\$\(\frac{1}{2}\) \(\frac{1}{2}\) \(\frac{1}\) \(\frac{1}2\) \(\frac{1}2\) \(\frac{1}\) \(\frac{1}2\) \(\frac{1}2\) \( | | | | | |

Error: 1.0954\*MS(subject(sequence)) - 0.0954\*MS(Error)

<sup>\*</sup> This test assumes one or more other fixed effects are zero.

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---------|--------|-----------|-------------|---------|--------|
| *period | 1 | 0.072771 | 0.072771 | 0.46 | 0.5049 |
| Error | 21.876 | 3.462747 | 0.158289 | | |

Error: 0.1294\*MS(subject(sequence)) + 0.8706\*MS(Error)

<sup>\*</sup> This test assumes one or more other fixed effects are zero.

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| trt | 1 | 0.278762 | 0.278762 | 1.74 | 0.2004 |
| Error | 22.69 | 3.636742 | 0.160278 | | |
| Error: 0.1 | Error: 0.1405*MS(subject(sequence)) + 0.8595*MS(Error) | | | | |

| Source | DF Type I SS | Mean Square | F Value | Pr > F |
|-------------------|--------------|-------------|---------|--------|
| subject(sequence) | 21 6.575283 | 0.313109 | 2.31 | 0.0612 |
| Error: MS(Error) | 13 1.758730 | 0.135287 | | |

Comparison: A vs B

Dependent Variable: AUC<sub>0-inf</sub> (h\*pg/mL)

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_AUCIFO

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.018380 | 0.018380 | 0.06 | 0.8159 |
| Error | 19.415 | 6.406079 | 0.329958 | | |
| Error: 1.0948*MS(subject(sequence)) - 0.0948*MS(Error) | | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.180986 | 0.180986 | 1.34 | 0.2682 |
| trt | 1 | 0.141213 | 0.141213 | 1.04 | 0.3256 |
| subject(sequence) | 21 | 6.575283 | 0.313109 | 2.31 | 0.0612 |
| Error: MS(Error) | 13 | 1.758730 | 0.135287 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN AUCIFO

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.021015 | 0.021015 | 0.07 | 0.7896 |
| Error | 23.811 | 6.873102 | 0.288651 | | |
| Error: 0.8625*MS(subject(sequence)) + 0.1375*MS(Error) | | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 0.180986 | 0.180986 | 1.34 | 0.2682 |
| trt | 1 | 0.141213 | 0.141213 | 1.04 | 0.3256 |
| subject(sequence) | 21 | 6.575283 | 0.313109 | 2.31 | 0.0612 |
| Error: MS(Error) | 13 | 1.758730 | 0.135287 | | |

Comparison: A vs B

Dependent Variable: AUC<sub>0-inf</sub> (h\*pg/mL)

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_AUCIFO

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.021015 | 0.021015 | 0.07 | 0.7896 |
| Error | 23.811 | 6.873102 | 0.288651 | | |
| Error: 0.86 | Error: 0.8625*MS(subject(sequence)) + 0.1375*MS(Error) | | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.180986 | 0.180986 | 1.34 | 0.2682 |
| trt | 1 | 0.141213 | 0.141213 | 1.04 | 0.3256 |
| subject(sequence) | 21 | 6.575283 | 0.313109 | 2.31 | 0.0612 |
| Error: MS(Error) | 13 | 1.758730 | 0.135287 | · | |

Comparison: A vs B

Dependent Variable: AUC<sub>0-inf</sub> (h\*pg/mL)

#### Least Squares Means

| | | 110 | 1.01. | |
|---|---|---|---|---|
| | | H0: | LSMean1=LSMean2 | |
| trt | LN_AUCIFO LSMEAN | | Pr > | > t |
| A | 16.3376718 | | 0.32 | 256 |
| В | 16.1976255 | | | |
| trt | LN AUCIFO LSMEAN | 9 | 0% Confidence Limits | |
| A | 16.337672 | 16.182337 | 16.493007 | |
| В | 16.197625 | 16.019279 | 16.375972 | |
| Lea | ast Squares Means for Effec | t trt | | — |
| | Difference Between | | | |
| i | j Means | 90% Confidence | Limits for LSMean(i)-LSMean( | j) |
| 1 | 2 0.140046 | -0.102706 | 0.382799 | |

#### Dependent Variable: LN\_AUCIFO

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confi | dence Limits |
| A - B | 0.14004633 | 0.13707607 | 1.02 | 0.3256-0 | 0.10270627 | 0.38279892 |

# Listing 16.1.9-2 ANOVA for Treatment Comparison of Nordiazepam - PK Population Comparison: A vs ${\bf B}$

Dependent Variable: C<sub>max</sub> (pg/mL)

#### The GLM Procedure

| Class Le | evel In | formation | |
|---|---|---|---|
| Class | Leve | els Values | |
| subject | 28 | 101 201 202 203 204 205 301 302 303 304 402 404 406 407 | 408 409 |
| v | | 410 411 412 413 414 501 502 503 505 506 507 508 | |
| sequenc | e 2 | AB BA | |
| period | 2 | 1 2 | |
| trt | 2 | A B | |
| Number | of Ob | oservations Read | 56 |
| Number | Number of Observations Used 56 | | |

Comparison: A vs B

Dependent Variable: C<sub>max</sub> (pg/mL)

#### The GLM Procedure

| R-Square | Coeff Var | Root MSE | | LN_CM | AX Mean |
|------------------|-----------|-------------|-------------|---------|---------|
| 0.652247 | 5.248044 | 0.551299 | 10.50485 | | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 1.00601538 | 1.00601538 | 3.31 | 0.0804 |
| period | 1 | 0.05642288 | 0.05642288 | 0.19 | 0.6701 |
| trt | 1 | 0.63660316 | 0.63660316 | 2.09 | 0.1598 |
| subject(sequence | e) 26 | 13.12238367 | 0.50470706 | 1.66 | 0.1013 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 1.00601538 | 1.00601538 | 3.31 | 0.0804 |
| period | 1 | 0.05642288 | 0.05642288 | 0.19 | 0.6701 |
| trt | 1 | 0.63660316 | 0.63660316 | 2.09 | 0.1598 |
| subject(sequence | e) 26 | 13.12238367 | 0.50470706 | 1.66 | 0.1013 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 1.00601538 | 1.00601538 | 3.31 | 0.0804 |
| period | 1 | 0.05642288 | 0.05642288 | 0.19 | 0.6701 |
| trt | 1 | 0.63660316 | 0.63660316 | 2.09 | 0.1598 |
| subject(sequence | e) 26 | 13.12238367 | 0.50470706 | 1.66 | 0.1013 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 1.00601538 | 1.00601538 | 3.31 | 0.0804 |
| period | 1 | 0.05642288 | 0.05642288 | 0.19 | 0.6701 |
| trt | 1 | 0.63660316 | 0.63660316 | 2.09 | 0.1598 |
| subject(sequence | e) 26 | 13.12238367 | 0.50470706 | 1.66 | 0.1013 |

Comparison: A vs B

Dependent Variable: C<sub>max</sub> (pg/mL)

## The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_CMAX

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 1.006015 | 1.006015 | 1.99 | 0.1699 |
| Error | 26 | 13.122384 | 0.504707 | | _ |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-------------------|----|-----------|-------------|---------|--------|
| period | 1 | 0.056423 | 0.056423 | 0.19 | 0.6701 |
| trt | 1 | 0.636603 | 0.636603 | 2.09 | 0.1598 |
| subject(sequence) | 26 | 13.122384 | 0.504707 | 1.66 | 0.1013 |
| Error: MS(Error) | 26 | 7.902201 | 0.303931 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------|-----------|------------|-------------|---------|--------|
| sequence | 1 | 1.006015 | 1.006015 | 1.99 | 0.1699 |
| Error | 26 | 13.122384 | 0.504707 | | |
| Error: MS(s | subject(s | equence)) | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.056423 | 0.056423 | 0.19 | 0.6701 |
| trt | 1 | 0.636603 | 0.636603 | 2.09 | 0.1598 |
| subject(sequence) | 26 | 13.122384 | 0.504707 | 1.66 | 0.1013 |
| Error: MS(Error) | 26 | 7.902201 | 0.303931 | | - |

Comparison: A vs B

Dependent Variable: C<sub>max</sub> (pg/mL)

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_CMAX

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 1.006015 | 1.006015 | 1.99 | 0.1699 |
| Error | 26 | 13.122384 | 0.504707 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 0.056423 | 0.056423 | 0.19 | 0.6701 |
| trt | 1 | 0.636603 | 0.636603 | 2.09 | 0.1598 |
| subject(sequence) | 26 | 13.122384 | 0.504707 | 1.66 | 0.1013 |
| Error: MS(Error) | 26 | 7.902201 | 0.303931 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------|-----------|------------|-------------|---------|--------|
| sequence | 1 | 1.006015 | 1.006015 | 1.99 | 0.1699 |
| Error | 26 | 13.122384 | 0.504707 | | |
| Error: MS(s | subject(s | sequence)) | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.056423 | 0.056423 | 0.19 | 0.6701 |
| trt | 1 | 0.636603 | 0.636603 | 2.09 | 0.1598 |
| subject(sequence) | 26 | 13.122384 | 0.504707 | 1.66 | 0.1013 |
| Error: MS(Error) | 26 | 7.902201 | 0.303931 | | |
Comparison: A vs B

Dependent Variable: C<sub>max</sub> (pg/mL)

2 0.213241

#### Least Squares Means

| | | H0:L9 | SMean1=LSMean2 | |
|---|---|---|---|---|
| trt | LN_CMAX LSMEAN | | | Pr > t |
| A | 10.6114713 | | | 0.1598 |
| В | 10.3982305 | | | |
| trt | LN_CMAX LSMEAN | 90% | 6 Confidence Limits | |
| A | 10.611471 | 10.433770 | 10.789172 | |
| В | 10.398230 | 10.220529 | 10.575932 | |
| Lea | ast Squares Means for Effect | trt | | |
| | Difference Between | | | |
| i | j Means | 90% Confidence I | Limits for LSMean(i)-LS | Mean(j) |

#### Dependent Variable: LN\_CMAX

0.464548

-0.038066

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confi | dence Limits |
| A - B | 0.21324084 | 0.14734091 | 1.45 | 0.1598-0 | 0.03806646 | 0.46454814 |

Comparison: A vs B

Dependent Variable: Cl/F/kg ((L/h)/kg)

#### The GLM Procedure

| Class Le | evel In | nformation | |
|---|---|---|---|
| Class | Leve | els Values | |
| subject | 23 | 101 201 202 203 204 205 301 302 303 304 404 407 408 41 | 0 411 412 |
| - | | 413 414 501 502 503 505 507 | |
| sequenc | e 2 | AB BA | |
| period | 2 | 1 2 | |
| trt | 2 | A B | |
| Number | of Ob | oservations Read | 38 |
| Number | of Ob | oservations Used | 38 |

Comparison: A vs B

Dependent Variable: Cl/F/kg ((L/h)/kg)

The GLM Procedure

| R-Square | Coeff Var | Root MSE | | LN_CLF | OW Mean |
|------------------|-----------|-------------|-------------|---------|---------|
| 0.809488 | -9.734415 | 0.385756 | -3.962809 | | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.08291686 | 0.08291686 | 0.56 | 0.4687 |
| period | 1 | 0.03561332 | 0.03561332 | 0.24 | 0.6328 |
| trt | 1 | 0.70236923 | 0.70236923 | 4.72 | 0.0489 |
| subject(sequence | e) 21 | 7.39881399 | 0.35232448 | 2.37 | 0.0564 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.03880462 | 0.03880462 | 0.26 | 0.6182 |
| period | 1 | 0.16754588 | 0.16754588 | 1.13 | 0.3080 |
| trt | 1 | 0.31055767 | 0.31055767 | 2.09 | 0.1722 |
| subject(sequence | e) 21 | 7.39881399 | 0.35232448 | 2.37 | 0.0564 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.05903403 | 0.05903403 | 0.40 | 0.5397 |
| period | 1 | 0.16754588 | 0.16754588 | 1.13 | 0.3080 |
| trt | 1 | 0.31055767 | 0.31055767 | 2.09 | 0.1722 |
| subject(sequence | e) 21 | 7.39881399 | 0.35232448 | 2.37 | 0.0564 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.05903403 | 0.05903403 | 0.40 | 0.5397 |
| period | 1 | 0.16754588 | 0.16754588 | 1.13 | 0.3080 |
| trt | 1 | 0.31055767 | 0.31055767 | 2.09 | 0.1722 |
| subject(sequence | 21 | 7.39881399 | 0.35232448 | 2.37 | 0.0564 |

Comparison: A vs B

Dependent Variable: Cl/F/kg ((L/h)/kg)

# The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN CLFOW

| Sourc | ee DF | Type I SS | Mean Square | F Value | Pr > F |
|--------|--------|-----------|-------------|---------|--------|
| *seque | ence 1 | 0.082917 | 0.082917 | 0.22 | 0.6420 |
| Error | 19.441 | 7.226947 | 0.371746 | | |

Error: 1.0954\*MS(subject(sequence)) - 0.0954\*MS(Error)

<sup>\*</sup> This test assumes one or more other fixed effects are zero.

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---------|--------|-----------|-------------|---------|--------|
| *period | 1 | 0.035613 | 0.035613 | 0.20 | 0.6564 |
| Error | 22.064 | 3.864214 | 0.175134 | | |

Error: 0.1294\*MS(subject(sequence)) + 0.8706\*MS(Error)

<sup>\*</sup> This test assumes one or more other fixed effects are zero.

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| trt | 1 | 0.702369 | 0.702369 | 3.96 | 0.0587 |
| Error | 22.891 | 4.061091 | 0.177411 | | |
| Error: 0.1405*MS(subject(sequence)) + 0.8595*MS(Error) | | | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-------------------|----|-----------|-------------|---------|--------|
| subject(sequence) | 21 | 7.398814 | 0.352324 | 2.37 | 0.0564 |
| Error: MS(Error) | 13 | 1.934503 | 0.148808 | | |

Comparison: A vs B

Dependent Variable: Cl/F/kg ((L/h)/kg)

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_CLFOW

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.038805 | 0.038805 | 0.10 | 0.7500 |
| Error | 19.451 | 7.228050 | 0.371608 | | |
| Error: 1.0948*MS(subject(sequence)) - 0.0948*MS(Error) | | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.167546 | 0.167546 | 1.13 | 0.3080 |
| trt | 1 | 0.310558 | 0.310558 | 2.09 | 0.1722 |
| subject(sequence) | 21 | 7.398814 | 0.352324 | 2.37 | 0.0564 |
| Error: MS(Error) | 13 | 1.934503 | 0.148808 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.059034 | 0.059034 | 0.18 | 0.6735 |
| Error | 23.75 | 7.702956 | 0.324333 | | |
| Error: 0.8625*MS(subject(sequence)) + 0.1375*MS(Error) | | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 0.167546 | 0.167546 | 1.13 | 0.3080 |
| trt | 1 | 0.310558 | 0.310558 | 2.09 | 0.1722 |
| subject(sequence) | 21 | 7.398814 | 0.352324 | 2.37 | 0.0564 |
| Error: MS(Error) | 13 | 1.934503 | 0.148808 | | |

Comparison: A vs B

Dependent Variable: Cl/F/kg ((L/h)/kg)

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.059034 | 0.059034 | 0.18 | 0.6735 |
| Error | 23.75 | 7.702956 | 0.324333 | | |
| Error: 0.8625*MS(subject(sequence)) + 0.1375*MS(Error) | | | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.167546 | 0.167546 | 1.13 | 0.3080 |
| trt | 1 | 0.310558 | 0.310558 | 2.09 | 0.1722 |
| subject(sequence) | 21 | 7.398814 | 0.352324 | 2.37 | 0.0564 |
| Error: MS(Error) | 13 | 1.934503 | 0.148808 | - | |

Comparison: A vs B

Dependent Variable: Cl/F/kg ((L/h)/kg)

#### Least Squares Means

| | | Н | 0:LSMean1=LSMean2 | |
|---|---|---|---|---|
| trt | LN_CLFOW LSMEAN | | | Pr > t |
| A | -4.17286608 | | | 0.1722 |
| В | -3.96518120 | | | |
| trt | LN CLFOW LSMEAN | | 90% Confidence Limits | |
| A | -4.172866 | -4.335778 | -4.009954 | |
| В | -3.965181 | -4.152228 | -3.778135 | |
| Le | ast Squares Means for Effec | t trt | | |
| | Difference Between | | | |
| i | j Means | 90% Confidence | ce Limits for LSMean(i)-LS | Mean(j) |
| 1 | 2 -0.207685 | -0.462279 | 0.046910 | <u>.</u> |

| | | Standard | | |
|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t 90% Confidence Limits |
| A - B | -0.20768488 | 0.14376288 | -1.44 | 0.1722-0.46227937 |

# Listing 16.1.9-2 ANOVA for Treatment Comparison of Nordiazepam - PK Population Comparison: A vs ${\bf B}$

Dependent Variable: Cl/F (L/h)

#### The GLM Procedure

| Class Le | evel Ir | formation | |
|---|---|---|---|
| Class | Leve | els Values | |
| subject | 23 | 101 201 202 203 204 205 301 302 303 304 404 407 | 7 408 410 411 412 |
| | | 413 414 501 502 503 505 507 | |
| sequence | e 2 | AB BA | |
| period | 2 | 1 2 | |
| trt | 2 | A B | |
| Number | of Ob | oservations Read | 38 |
| Number of Observations Used 38 | | | |

Comparison: A vs B

Dependent Variable: Cl/F (L/h)

#### The GLM Procedure

| R-Square | Coeff Var | Root MSE | 3 | LN_C | LFO Mean |
|---|---|---|---|---|---|
| 0.772445 | 101.1422 | 0.385756 | 0.381400 | | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.01820094 | 0.01820094 | 0.12 | 0.7321 |
| period | 1 | 0.15040156 | 0.15040156 | 1.01 | 0.3331 |
| trt | 1 | 0.36542174 | 0.36542174 | 2.46 | 0.1411 |
| subject(sequence | ) 21 | 6.03273972 | 0.28727332 | 1.93 | 0.1119 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.00740836 | 0.00740836 | 0.05 | 0.8269 |
| period | 1 | 0.16754588 | 0.16754588 | 1.13 | 0.3080 |
| trt | 1 | 0.31055767 | 0.31055767 | 2.09 | 0.1722 |
| subject(sequence | ) 21 | 6.03273972 | 0.28727332 | 1.93 | 0.1119 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.00335522 | 0.00335522 | 0.02 | 0.8829 |
| period | 1 | 0.16754588 | 0.16754588 | 1.13 | 0.3080 |
| trt | 1 | 0.31055767 | 0.31055767 | 2.09 | 0.1722 |
| subject(sequence | ) 21 | 6.03273972 | 0.28727332 | 1.93 | 0.1119 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.00335522 | 0.00335522 | 0.02 | 0.8829 |
| period | 1 | 0.16754588 | 0.16754588 | 1.13 | 0.3080 |
| trt | 1 | 0.31055767 | 0.31055767 | 2.09 | 0.1722 |
| subject(sequence | 21 | 6.03273972 | 0.28727332 | 1.93 | 0.1119 |

Comparison: A vs B

Dependent Variable: Cl/F (L/h)

# The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_CLFO

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| *sequence | 1 | 0.018201 | 0.018201 | 0.06 | 0.8082 |
| Error | 19.085 | 5.734701 | 0.300487 | | |
| E-man, 1 005 4*MC(a.l.i.a.t/a.a.u.a.a.)) 0 005 4*MC(E-man) | | | | | |

Error: 1.0954\*MS(subject(sequence)) - 0.0954\*MS(Error)

<sup>\*</sup> This test assumes one or more other fixed effects are zero.

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---------|--------|-----------|-------------|---------|--------|
| *period | 1 | 0.150402 | 0.150402 | 0.90 | 0.3533 |
| Error | 20.484 | 3.414999 | 0.166719 | | |

Error: 0.1294\*MS(subject(sequence)) + 0.8706\*MS(Error)

<sup>\*</sup> This test assumes one or more other fixed effects are zero.

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| trt | 1 | 0.365422 | 0.365422 | 2.17 | 0.1553 |
| Error | 21.196 | 3.566563 | 0.168268 | | |
| Error: 0.1405*MS(subject(sequence)) + 0.8595*MS(Error) | | | | | |

| Source | DF Type I SS | Mean Square | F Value | Pr > F |
|-------------------|--------------|-------------|---------|--------|
| subject(sequence) | 21 6.032740 | 0.287273 | 1.93 | 0.1119 |
| Error: MS(Error) | 13 1.934503 | 0.148808 | | |

Comparison: A vs B

Dependent Variable: Cl/F (L/h)

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_CLFO

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.007408 | 0.007408 | 0.02 | 0.8769 |
| Error | 19.097 | 5.736667 | 0.300393 | | |
| Error: 1.0948*MS(subject(sequence)) - 0.0948*MS(Error) | | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|-----------|
| period | 1 | 0.167546 | 0.167546 | 1.13 | 0.3080 |
| trt | 1 | 0.310558 | 0.310558 | 2.09 | 0.1722 |
| subject(sequence) | 21 | 6.032740 | 0.287273 | 1.93 | 0.1119 |
| Error: MS(Error) | 13 | 1.934503 | 0.148808 | | <u></u> ; |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------|------------|-------------|-------------|---------|--------|
| sequence | 1 | 0.003355 | 0.003355 | 0.01 | 0.9119 |
| Error | 24.345 | 6.529893 | 0.268229 | | |
| Error: 0.86 | 525*MS(sub | .) | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 0.167546 | 0.167546 | 1.13 | 0.3080 |
| trt | 1 | 0.310558 | 0.310558 | 2.09 | 0.1722 |
| subject(sequence) | 21 | 6.032740 | 0.287273 | 1.93 | 0.1119 |
| Error: MS(Error) | 13 | 1.934503 | 0.148808 | | |

Comparison: A vs B

Dependent Variable: Cl/F (L/h)

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.003355 | 0.003355 | 0.01 | 0.9119 |
| Error | 24.345 | 6.529893 | 0.268229 | | |
| Error: 0.86 | 25*MS(sub | ject(sequence)) + | 0.1375*MS(Error | ) | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.167546 | 0.167546 | 1.13 | 0.3080 |
| trt | 1 | 0.310558 | 0.310558 | 2.09 | 0.1722 |
| subject(sequence) | 21 | 6.032740 | 0.287273 | 1.93 | 0.1119 |
| Error: MS(Error) | 13 | 1.934503 | 0.148808 | · | |

Comparison: A vs B

Dependent Variable: Cl/F (L/h)

#### Least Squares Means

| | | I | H0:LSMean1=LSMean2 | |
|---|---|---|---|---|
| trt | LN_CLFO LSMEAN | | | Pr > t |
| A | 0.18972659 | | | 0.1722 |
| В | 0.39741148 | | | |
| trt | LN_CLFO LSMEAN | | 90% Confidence Limits | |
| A | 0.189727 | 0.026814 | 0.352639 | |
| В | 0.397411 | 0.210365 | 0.584458 | |
| Lea | ast Squares Means for Effect | et trt | | |
| | Difference Between | | | |
| i | j Means | 90% Confide | nce Limits for LSMean(i)-LS | SMean(j) |
| 1 | 2 -0.207685 | -0 462279 | 0.046910 | |

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confid | dence Limits |
| A - B | -0.20768488 | 0.14376288 | -1.44 | 0.1722-0 | 0.46227937 | 0.04690961 |

Comparison: A vs B

Dependent Variable: V<sub>d</sub>/F/kg (L/kg)

#### The GLM Procedure

| Class Le | evel In | nformation | |
|---|---|---|---|
| Class | Leve | els Values | |
| subject | 23 | 101 201 202 203 204 205 301 302 303 304 404 407 408 41 | 0 411 412 |
| - | | 413 414 501 502 503 505 507 | |
| sequenc | e 2 | AB BA | |
| period | 2 | 1 2 | |
| trt | 2 | A B | |
| Number | of Ob | oservations Read | 38 |
| Number of Observations Used 38 | | | |

Comparison: A vs B

Dependent Variable: V<sub>d</sub>/F/kg (L/kg)

The GLM Procedure

| R-Square | Coeff Var | Root MSE | | LN_VZF0 | OW Mean |
|------------------|-----------|-------------|-------------|---------|---------|
| 0.868076 | 29.95886 | 0.380787 | 1.271034 | | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.17703292 | 0.17703292 | 1.22 | 0.2892 |
| period | 1 | 0.35833365 | 0.35833365 | 2.47 | 0.1400 |
| trt | 1 | 0.53284924 | 0.53284924 | 3.67 | 0.0775 |
| subject(sequence | e) 21 | 11.33526148 | 0.53977436 | 3.72 | 0.0091 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.21714612 | 0.21714612 | 1.50 | 0.2428 |
| period | 1 | 0.10125275 | 0.10125275 | 0.70 | 0.4184 |
| trt | 1 | 0.23872722 | 0.23872722 | 1.65 | 0.2219 |
| subject(sequence | e) 21 | 11.33526148 | 0.53977436 | 3.72 | 0.0091 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.01415919 | 0.01415919 | 0.10 | 0.7596 |
| period | 1 | 0.10125275 | 0.10125275 | 0.70 | 0.4184 |
| trt | 1 | 0.23872722 | 0.23872722 | 1.65 | 0.2219 |
| subject(sequence | e) 21 | 11.33526148 | 0.53977436 | 3.72 | 0.0091 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.01415919 | 0.01415919 | 0.10 | 0.7596 |
| period | 1 | 0.10125275 | 0.10125275 | 0.70 | 0.4184 |
| trt | 1 | 0.23872722 | 0.23872722 | 1.65 | 0.2219 |
| subject(sequence | e) 21 | 11.33526148 | 0.53977436 | 3.72 | 0.0091 |

Comparison: A vs B

Dependent Variable: V<sub>d</sub>/F/kg (L/kg)

# The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN VZFOW

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-----------|--------|-----------|-------------|---------|--------|
| *sequence | 1 | 0.177033 | 0.177033 | 0.31 | 0.5859 |
| Error | 20.011 | 11.555255 | 0.577447 | | |

Error: 1.0954\*MS(subject(sequence)) - 0.0954\*MS(Error)

<sup>\*</sup> This test assumes one or more other fixed effects are zero.

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---------|--------|-----------|-------------|---------|--------|
| *period | 1 | 0.358334 | 0.358334 | 1.83 | 0.1879 |
| Error | 26.364 | 5.169085 | 0.196065 | | |

Error: 0.1294\*MS(subject(sequence)) + 0.8706\*MS(Error)

<sup>\*</sup> This test assumes one or more other fixed effects are zero.

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| trt | 1 | 0.532849 | 0.532849 | 2.66 | 0.1145 |
| Error | 27.367 | 5.486520 | 0.200482 | | |
| Error: 0.1405*MS(subject(sequence)) + 0.8595*MS(Error) | | | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-------------------|----|-----------|-------------|---------|--------|
| subject(sequence) | 21 | 11.335261 | 0.539774 | 3.72 | 0.0091 |
| Error: MS(Error) | 13 | 1.884985 | 0.144999 | | |

Comparison: A vs B

Dependent Variable: V<sub>d</sub>/F/kg (L/kg)

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_VZFOW

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.217146 | 0.217146 | 0.38 | 0.5465 |
| Error | 20.017 | 11.553626 | 0.577180 | | |
| Error: 1.09 | Error: 1.0948*MS(subject(sequence)) - 0.0948*MS(Error) | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|----------|--------|
| period | 1 | 0.101253 | 0.101253 | 0.70 | 0.4184 |
| trt | 1 | 0.238727 | 0.238727 | 1.65 | 0.2219 |
| subject(sequence) | 21 | 11.335261 | 0.539774 | 3.72 | 0.0091 |
| Error: MS(Error) | 13 | 1.884985 | 0.144999 | <u> </u> | · |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.014159 | 0.014159 | 0.03 | 0.8659 |
| Error | 22.77 | 11.054446 | 0.485476 | | |
| Error: 0.8625*MS(subject(sequence)) + 0.1375*MS(Error) | | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 0.101253 | 0.101253 | 0.70 | 0.4184 |
| trt | 1 | 0.238727 | 0.238727 | 1.65 | 0.2219 |
| subject(sequence) | 21 | 11.335261 | 0.539774 | 3.72 | 0.0091 |
| Error: MS(Error) | 13 | 1.884985 | 0.144999 | | |

Comparison: A vs B

Dependent Variable: V<sub>d</sub>/F/kg (L/kg)

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.014159 | 0.014159 | 0.03 | 0.8659 |
| Error | 22.77 | 11.054446 | 0.485476 | | |
| Error: 0.86 | Error: 0.8625*MS(subject(sequence)) + 0.1375*MS(Error) | | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.101253 | 0.101253 | 0.70 | 0.4184 |
| trt | 1 | 0.238727 | 0.238727 | 1.65 | 0.2219 |
| subject(sequence) | 21 | 11.335261 | 0.539774 | 3.72 | 0.0091 |
| Error: MS(Error) | 13 | 1.884985 | 0.144999 | - | |

Comparison: A vs B

Dependent Variable: V<sub>d</sub>/F/kg (L/kg)

#### Least Squares Means

| | | H0:L | SMean1=LSMean2 |
|---|---|---|---|
| trt | LN_VZFOW LSMEAN | | $\Pr > t $ |
| A | 1.20517079 | | 0.2219 |
| В | 1.38726022 | | |
| trt | LN VZFOW LSMEAN | 90 | 0% Confidence Limits |
| Ā | 1.205171 | 1.044357 | 1.365984 |
| В | 1.387260 | 1.202623 | 1.571897 |
| Le | ast Squares Means for Effec | t trt | |
| | Difference Between | | |
| i | j Means | 90% Confidence L | Limits for LSMean(i)-LSMean(j) |
| 1 | 2 -0.182089 | -0 433404 | 0.069225 |

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confi | dence Limits |
| A - B | -0.18208942 | 0.14191099 | -1.28 | 0.2219-0 | 0.43340434 | 0.06922549 |

Comparison: A vs B

Dependent Variable: V<sub>d</sub>/F (L)

#### The GLM Procedure

| Class Le | vel In | formation | |
|---|---|---|---|
| Class | Leve | ls Values | |
| subject | 23 | 101 201 202 203 204 205 301 302 303 304 404 407 408 | 410 411 412 |
| | | 413 414 501 502 503 505 507 | |
| sequence | e 2 | AB BA | |
| period | 2 | 1 2 | |
| trt | 2 | A B | |
| · | | | |
| Number | of Ob | servations Read | 38 |
| Number | Number of Observations Used 38 | | |

Comparison: A vs B

Dependent Variable: V<sub>d</sub>/F (L)

#### The GLM Procedure

| R-Square | Coeff Var | Root MSE | | LN_ | VZFO Mean |
|---|---|---|---|---|---|
| 0.913813 | 6.781312 | 0.380787 | 5.615243 | | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.32924050 | 0.32924050 | 2.27 | 0.1558 |
| period | 1 | 0.63634324 | 0.63634324 | 4.39 | 0.0563 |
| trt | 1 | 0.24640477 | 0.24640477 | 1.70 | 0.2150 |
| subject(sequence | e) 21 | 18.77380507 | 0.89399072 | 6.17 | 0.0008 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.33282108 | 0.33282108 | 2.30 | 0.1537 |
| period | 1 | 0.10125275 | 0.10125275 | 0.70 | 0.4184 |
| trt | 1 | 0.23872722 | 0.23872722 | 1.65 | 0.2219 |
| subject(sequence | e) 21 | 18.77380507 | 0.89399072 | 6.17 | 0.0008 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.09243872 | 0.09243872 | 0.64 | 0.4390 |
| period | 1 | 0.10125275 | 0.10125275 | 0.70 | 0.4184 |
| trt | 1 | 0.23872722 | 0.23872722 | 1.65 | 0.2219 |
| subject(sequence | e) 21 | 18.77380507 | 0.89399072 | 6.17 | 0.0008 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.09243872 | 0.09243872 | 0.64 | 0.4390 |
| period | 1 | 0.10125275 | 0.10125275 | 0.70 | 0.4184 |
| trt | 1 | 0.23872722 | 0.23872722 | 1.65 | 0.2219 |
| subject(sequence | e) 21 | 18.77380507 | 0.89399072 | 6.17 | 0.0008 |

Comparison: A vs B

Dependent Variable: V<sub>d</sub>/F (L)

# The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_VZFO

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| *sequence | 1 | 0.329240 | 0.329240 | 0.34 | 0.5656 |
| Error | 20.404 | 19.699538 | 0.965466 | | |
| Eman: 1 005 4*MC(a) | Empty 1 005.4*MS(gubioct(gaguanas)) 0 005.4*MS(Empty) | | | | |

Error: 1.0954\*MS(subject(sequence)) - 0.0954\*MS(Error)

<sup>\*</sup> This test assumes one or more other fixed effects are zero.

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---------|--------|-----------|-------------|---------|--------|
| *period | 1 | 0.636343 | 0.636343 | 2.63 | 0.1148 |
| Error | 31.409 | 7.597440 | 0.241884 | | |

Error: 0.1294\*MS(subject(sequence)) + 0.8706\*MS(Error)

<sup>\*</sup> This test assumes one or more other fixed effects are zero.

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| trt | 1 | 0.246405 | 0.246405 | 0.98 | 0.3285 |
| Error | 32.179 | 8.053252 | 0.250264 | | |
| Error: 0.1405*MS(subject(sequence)) + 0.8595*MS(Error) | | | | | |

| Source | DF Type I SS | Mean Square | F Value | Pr > F |
|-------------------|--------------|-------------|---------|--------|
| subject(sequence) | 21 18.773805 | 0.893991 | 6.17 | 0.0008 |
| Error: MS(Error) | 13 1.884985 | 0.144999 | | |

Comparison: A vs B

Dependent Variable: V<sub>d</sub>/F (L)

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_VZFO

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.332821 | 0.332821 | 0.34 | 0.5635 |
| Error 20.408 19.692930 0.964959 | | | | | |
| Error: 1.0948*MS(subject(sequence)) - 0.0948*MS(Error) | | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.101253 | 0.101253 | 0.70 | 0.4184 |
| trt | 1 | 0.238727 | 0.238727 | 1.65 | 0.2219 |
| subject(sequence) | 21 | 18.773805 | 0.893991 | 6.17 | 0.0008 |
| Error: MS(Error) | 13 | 1.884985 | 0.144999 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.092439 | 0.092439 | 0.12 | 0.7357 |
| Error | 22.077 | 17.461966 | 0.790973 | | |
| Error: 0.8625*MS(subject(sequence)) + 0.1375*MS(Error) | | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 0.101253 | 0.101253 | 0.70 | 0.4184 |
| trt | 1 | 0.238727 | 0.238727 | 1.65 | 0.2219 |
| subject(sequence) | 21 | 18.773805 | 0.893991 | 6.17 | 0.0008 |
| Error: MS(Error) | 13 | 1.884985 | 0.144999 | | - |

Comparison: A vs B

Dependent Variable: V<sub>d</sub>/F (L)

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.092439 | 0.092439 | 0.12 | 0.7357 |
| Error | 22.077 | 17.461966 | 0.790973 | | |
| Error: 0.8625*MS(subject(sequence)) + 0.1375*MS(Error) | | | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.101253 | 0.101253 | 0.70 | 0.4184 |
| trt | 1 | 0.238727 | 0.238727 | 1.65 | 0.2219 |
| subject(sequence) | 21 | 18.773805 | 0.893991 | 6.17 | 0.0008 |
| Error: MS(Error) | 13 | 1.884985 | 0.144999 | | |

Comparison: A vs B

Dependent Variable: V<sub>d</sub>/F (L)

#### Least Squares Means

| | | Н | 0:LSMean1=LSMean2 | |
|---|---|---|---|---|
| trt | LN_VZFO LSMEAN | | | Pr > t |
| A | 5.56776347 | | | 0.2219 |
| В | 5.74985289 | | | |
| trt | LN_VZFO LSMEAN | | 90% Confidence Limits | |
| A | 5.567763 | 5.406950 | 5.728577 | |
| В | 5.749853 | 5.565216 | 5.934490 | |
| Lea | st Squares Means for Effec | et trt | | |
| | Difference Between | | | |
| i | j Means | 90% Confider | nce Limits for LSMean(i)-LS | SMean(j) |
| 1 | 2 -0.182089 | -0.433404 | 0.069225 | |

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confi | dence Limits |
| A - B | -0.18208942 | 0.14191099 | -1.28 | 0.2219-0 | 0.43340434 | 0.06922549 |

# Listing 16.1.9-2 ANOVA for Treatment Comparison of Nordiazepam - PK Population Comparison: A $\ensuremath{\mathsf{vs}}\ \ensuremath{\mathsf{B}}$

Dependent Variable: T<sub>max</sub> (h)

#### The GLM Procedure

| 7 408 409 |
|--------------------------------|
| 7 408 409 |
| 56 |
| Number of Observations Used 56 |
| _ |

Comparison: A vs B

Dependent Variable: T<sub>max</sub> (h)

#### The GLM Procedure

| R-Square | Coeff Var | Root | MSE | TI | MAX Mean |
|---|---|---|---|---|---|
| 0.862069 | 30.47680 | 34.15 | 705 11 | 12.0756 | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 17217.7568 | 17217.7568 | 14.76 | 0.0007 |
| period | 1 | 1236.4385 | 1236.4385 | 1.06 | 0.3127 |
| trt | 1 | 679.7005 | 679.7005 | 0.58 | 0.4522 |
| subject(sequence) | 26 | 170454.9347 | 6555.9590 | 5.62 | <.0001 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 17217.7568 | 17217.7568 | 14.76 | 0.0007 |
| period | 1 | 1236.4385 | 1236.4385 | 1.06 | 0.3127 |
| trt | 1 | 679.7005 | 679.7005 | 0.58 | 0.4522 |
| subject(sequence) | 26 | 170454.9347 | 6555.9590 | 5.62 | <.0001 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 17217.7568 | 17217.7568 | 14.76 | 0.0007 |
| period | 1 | 1236.4385 | 1236.4385 | 1.06 | 0.3127 |
| trt | 1 | 679.7005 | 679.7005 | 0.58 | 0.4522 |
| subject(sequence) | 26 | 170454.9347 | 6555.9590 | 5.62 | <.0001 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 17217.7568 | 17217.7568 | 14.76 | 0.0007 |
| period | 1 | 1236.4385 | 1236.4385 | 1.06 | 0.3127 |
| trt | 1 | 679.7005 | 679.7005 | 0.58 | 0.4522 |
| subject(sequence) | 26 | 170454.9347 | 6555.9590 | 5.62 | <.0001 |

Comparison: A vs B

Dependent Variable: T<sub>max</sub> (h)

# The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: TMAX

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 17218 | 17218 | 2.63 | 0.1172 |
| Error | 26 | 170455 | 6555.959028 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 1236.438473 | 1236.438473 | 1.06 | 0.3127 |
| trt | 1 | 679.700529 | 679.700529 | 0.58 | 0.4522 |
| subject(sequence) | 26 | 170455 | 6555.959028 | 5.62 | <.0001 |
| Error: MS(Error) | 26 | 30334 | 1166.704165 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 17218 | 17218 | 2.63 | 0.1172 |
| Error | 26 | 170455 | 6555.959028 | | _ |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 1236.438473 | 1236.438473 | 1.06 | 0.3127 |
| trt | 1 | 679.700529 | 679.700529 | 0.58 | 0.4522 |
| subject(sequence) | 26 | 170455 | 6555.959028 | 5.62 | <.0001 |
| Error: MS(Error) | 26 | 30334 | 1166.704165 | | |

Comparison: A vs B

Dependent Variable: T<sub>max</sub> (h)

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: TMAX

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 17218 | 17218 | 2.63 | 0.1172 |
| Error | 26 | 170455 | 6555.959028 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|-------------|
| period | 1 | 1236.438473 | 1236.438473 | 1.06 | 0.3127 |
| trt | 1 | 679.700529 | 679.700529 | 0.58 | 0.4522 |
| subject(sequence) | 26 | 170455 | 6555.959028 | 5.62 | <.0001 |
| Error: MS(Error) | 26 | 30334 | 1166.704165 | | <del></del> |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 17218 | 17218 | 2.63 | 0.1172 |
| Error | 26 | 170455 | 6555.959028 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 1236.438473 | 1236.438473 | 1.06 | 0.3127 |
| trt | 1 | 679.700529 | 679.700529 | 0.58 | 0.4522 |
| subject(sequence) | 26 | 170455 | 6555.959028 | 5.62 | <.0001 |
| Error: MS(Error) | 26 | 30334 | 1166.704165 | | |

Comparison: A vs B

Dependent Variable: T<sub>max</sub> (h)

#### Least Squares Means

| | | Н | 0:LSMean1=LSMean2 |
|---|---|---|---|
| trt | TMAX LSMEAN | | Pr > t |
| A | 115.559464 | | 0.4522 |
| В | 108.591679 | | |
| trt | TMAX LSMEAN | 9 | 00% Confidence Limits |
| A | 115.559464 | 104.549571 | 126.569358 |
| В | 108.591679 | 97.581785 | 119.601572 |
| Le | ast Squares Means for Effec | t trt | |
| | Difference Between | | |
| i | j Means | 90% Confidence I | Limits for LSMean(i)-LSMean(j) |
| 1 | 2 6.967786 | -8.602555 | 22.538126 |

| | | Standard | | | | _ |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Conf | idence Limits |
| A - B | 6.96778571 | 9.12885599 | 0.76 | 0.4522-8 | .60255466 | 22.53812609 |

# Listing 16.1.9-2 ANOVA for Treatment Comparison of Nordiazepam - PK Population Comparison: A vs ${\bf B}$

Dependent Variable: K<sub>el</sub> (/h)

#### The GLM Procedure

| Class Le | evel In | nformation | |
|---|---|---|---|
| Class | Leve | els Values | |
| subject | 23 | 101 201 202 203 204 205 301 302 303 304 404 407 408 41 | 0 411 412 |
| - | | 413 414 501 502 503 505 507 | |
| sequenc | e 2 | AB BA | |
| period | 2 | 1 2 | |
| trt | 2 | A B | |
| Number | of Ob | oservations Read | 38 |
| Number of Observations Used 38 | | | |
| Number of Observations Read<br>Number of Observations Used | | | |

Comparison: A vs B

Dependent Variable: K<sub>el</sub> (/h)

#### The GLM Procedure

| R-Square | Coeff Var | Root | t MSE | | LAMZ Mean |
|---|---|---|---|---|---|
| 0.982877 | 17.62657 | 0.00 | 1282 | 0.007272 | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.00012625 | 0.00012625 | 76.83 | <.0001 |
| period | 1 | 0.000012023 | 0.000012023 | 4.13 | 0.0631 |
| trt | 1 | 0.000000075 | 0.000000075 | 0.04 | 0.8537 |
| subject(sequence) | 21 | 0.00109304 | 0.00005205 | 31.68 | <.0001 |
| <u>subject(sequence)</u> | 21 | 0.00109301 | 0.00003203 | 31.00 | 0001 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.00011961 | 0.00011961 | 72.79 | <.0001 |
| period | 1 | 0.00000016 | 0.00000016 | 0.10 | 0.7608 |
| trt | 1 | 0.00000000 | 0.00000000 | 0.00 | 0.9849 |
| <pre>subject(sequence)</pre> | 21 | 0.00109304 | 0.00005205 | 31.68 | <.0001 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.00007798 | 0.00007798 | 47.46 | <.0001 |
| period | 1 | 0.00000016 | 0.00000016 | 0.10 | 0.7608 |
| trt | 1 | 0.00000000 | 0.00000000 | 0.00 | 0.9849 |
| subject(sequence) | 21 | 0.00109304 | 0.00005205 | 31.68 | <.0001 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.00007798 | 0.00007798 | 47.46 | <.0001 |
| period | 1 | 0.000007736 | 0.000007736 | 0.10 | 0.7608 |
| trt | 1 | 0.00000000 | 0.00000000 | 0.00 | 0.9849 |
| subject(sequence) | 21 | 0.00109304 | 0.00005205 | 31.68 | <.0001 |
| zazjece(zequence) | | | 3.00002202 | 21.00 | .0001 |

Comparison: A vs B

Dependent Variable: K<sub>el</sub> (/h)

# The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LAMZ

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| *sequence | 1 | 0.000126 | 0.000126 | 2.22 | 0.1511 |
| Error | 20.884 | 0.001187 | 0.000056860 | | |
| E 1 005 4*MC(a | [ | | | | |

Error: 1.0954\*MS(subject(sequence)) - 0.0954\*MS(Error)

<sup>\*</sup> This test assumes one or more other fixed effects are zero.

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---------|--------|-------------|-------------|---------|--------|
| *period | 1 | 0.000006786 | 0.000006786 | 0.83 | 0.3695 |
| Error | 28.774 | 0.000235 | 0.000008163 | | |

Error: 0.1294\*MS(subject(sequence)) + 0.8706\*MS(Error)

<sup>\*</sup> This test assumes one or more other fixed effects are zero.

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| trt | 1 | 5.810284E-8 | 5.810284E-8 | 0.01 | 0.9355 |
| Error | 28.194 | 0.000246 | 0.000008727 | | |
| Error: 0.1 | 405*MS(sub | oject(sequence)) + | 0.8595*MS(Error) | | |

| Source | DF Type I SS | Mean Square | F Value | Pr > F |
|-------------------|----------------|-------------|---------|--------|
| subject(sequence) | 21 0.001093 | 0.000052050 | 31.68 | <.0001 |
| Error: MS(Error) | 13 0.000021361 | 0.000001643 | | |

Comparison: A vs B

Dependent Variable: K<sub>el</sub> (/h)

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LAMZ

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.000120 | 0.000120 | 2.10 | 0.1617 |
| Error | 20.885 | 0.001187 | 0.000056826 | | |
| Error: 1.09 | Error: 1.0948*MS(subject(sequence)) - 0.0948*MS(Error) | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|--------------|--------------|-------------|--------|
| period | 1 | 0.000000159 | 0.000000159 | 0.10 | 0.7608 |
| trt | 1 | 6.101771E-10 | 6.101771E-10 | 0.00 | 0.9849 |
| subject(sequence) | 21 | 0.001093 | 0.000052050 | 31.68 | <.0001 |
| Error: MS(Error) | 13 | 0.000021361 | 0.000001643 | <del></del> | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.000077983 | 0.000077983 | 1.73 | 0.2026 |
| Error | 21.211 | 0.000957 | 0.000045117 | | |
| Error: 0.86 | Error: 0.8625*MS(subject(sequence)) + 0.1375*MS(Error) | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|--------------|--------------|---------|--------|
| period | 1 | 0.000000159 | 0.000000159 | 0.10 | 0.7608 |
| trt | 1 | 6.101771E-10 | 6.101771E-10 | 0.00 | 0.9849 |
| subject(sequence) | 21 | 0.001093 | 0.000052050 | 31.68 | <.0001 |
| Error: MS(Error) | 13 | 0.000021361 | 0.000001643 | | |

Comparison: A vs B

Dependent Variable: K<sub>el</sub> (/h)

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.000077983 | 0.000077983 | 1.73 | 0.2026 |
| Error | 21.211 | 0.000957 | 0.000045117 | | |
| Error: 0.86 | 625*MS(sub | oject(sequence)) + | 0.1375*MS(Error) | | |

| Source | DI | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|--------------|--------------|---------|--------|
| period | 1 | 0.000000159 | 0.000000159 | 0.10 | 0.7608 |
| trt | 1 | 6.101771E-10 | 6.101771E-10 | 0.00 | 0.9849 |
| subject(sequence) | 21 | 0.001093 | 0.000052050 | 31.68 | <.0001 |
| Error: MS(Error) | 13 | 0.000021361 | 0.000001643 | | |

Comparison: A vs B

Dependent Variable: K<sub>el</sub> (/h)

#### Least Squares Means

| | | H0:I | SMean1=LSMean2 | |
|---|---|---|---|---|
| trt | LAMZ LSMEAN | | | Pr > t |
| A | 0.00646826 | | | 0.9849 |
| В | 0.00647746 | | | |
| trt | LAMZ LSMEAN | 9 | 0% Confidence Limits | |
| A | 0.006468 | 0.005927 | 0.007010 | |
| В | 0.006477 | 0.005856 | 0.007099 | |
| Lea | ast Squares Means for Effect trt | | | |
| | | 90% C | onfidence Limits for | |
| i | j Difference Between Means | LSM | Iean(i)-LSMean(j) | |
| 1 | 2 -0.000009206 | -0.000855 | 0.000837 | |

| <u> </u> | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confi | dence Limits |
| A - B | -9.205803E-6 | 0.00047772 | -0.02 | 0.9849-0. | 000855215 | 0.0008368035 |
# Listing 16.1.9-2 ANOVA for Treatment Comparison of Nordiazepam - PK Population Comparison: A vs ${\bf B}$

Dependent Variable: T<sub>1/2 el</sub> (h)

### The GLM Procedure

| Class Le | evel In | nformation | |
|---|---|---|---|
| Class | Leve | els Values | |
| subject | 23 | 101 201 202 203 204 205 301 302 303 304 404 407 408 41 | 0 411 412 |
| - | | 413 414 501 502 503 505 507 | |
| sequenc | e 2 | AB BA | |
| period | 2 | 1 2 | |
| trt | 2 | A B | |
| Number | of Ob | oservations Read | 38 |
| Number | Number of Observations Used 38 | | |

Comparison: A vs B

Dependent Variable: T<sub>1/2 el</sub> (h)

### The GLM Procedure

| R-Square | Coeff Var | Root MSE | | LAMZ | ZHL Mean |
|---|---|---|---|---|---|
| 0.824637 | 77.23745 | 146.9343 | 190.237 | 1 | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 14942.202 | 14942.202 | 0.69 | 0.4205 |
| period | 1 | 3473.904 | 3473.904 | 0.16 | 0.6948 |
| trt | 1 | 29.534 | 29.534 | 0.00 | 0.9711 |
| subject(sequence | 21 | 1301373.296 | 61970.157 | 2.87 | 0.0272 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 15431.968 | 15431.968 | 0.71 | 0.4132 |
| period | 1 | 7687.035 | 7687.035 | 0.36 | 0.5610 |
| trt | 1 | 1577.042 | 1577.042 | 0.07 | 0.7912 |
| subject(sequence | 21 | 1301373.296 | 61970.157 | 2.87 | 0.0272 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 42212.895 | 42212.895 | 1.96 | 0.1854 |
| period | 1 | 7687.035 | 7687.035 | 0.36 | 0.5610 |
| trt | 1 | 1577.042 | 1577.042 | 0.07 | 0.7912 |
| subject(sequence | 21 | 1301373.296 | 61970.157 | 2.87 | 0.0272 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 42212.895 | 42212.895 | 1.96 | 0.1854 |
| period | 1 | 7687.035 | 7687.035 | 0.36 | 0.5610 |
| trt | 1 | 1577.042 | 1577.042 | 0.07 | 0.7912 |
| subject(sequence | 21 | 1301373.296 | 61970.157 | 2.87 | 0.0272 |

Comparison: A vs B

Dependent Variable: T<sub>1/2 el</sub> (h)

# The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LAMZHL

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-----------|--------|-----------|-------------|---------|--------|
| *sequence | 1 | 14942 | 14942 | 0.23 | 0.6390 |
| Error | 19.715 | 1297733 | 65824 | | |

Error: 1.0954\*MS(subject(sequence)) - 0.0954\*MS(Error)

<sup>\*</sup> This test assumes one or more other fixed effects are zero.

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---------|--------|-------------|-------------|---------|--------|
| *period | 1 | 3473.903776 | 3473.903776 | 0.13 | 0.7221 |
| Error | 23.775 | 637490 | 26813 | | |

Error: 0.1294\*MS(subject(sequence)) + 0.8706\*MS(Error)

<sup>\*</sup> This test assumes one or more other fixed effects are zero.

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| trt | 1 | 29.534427 | 29.534427 | 0.00 | 0.9740 |
| Error | 24.699 | 673421 | 27265 | | _ |
| Error: 0.1 | Error: 0.1405*MS(subject(sequence)) + 0.8595*MS(Error) | | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-------------------|----|-----------|-------------|---------|--------|
| subject(sequence) | 21 | 1301373 | 61970 | 2.87 | 0.0272 |
| Error: MS(Error) | 13 | 280666 | 21590 | | |

Comparison: A vs B

Dependent Variable: T<sub>1/2 el</sub> (h)

### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LAMZHL

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 15432 | 15432 | 0.23 | 0.6335 |
| Error | 19.724 | 1297745 | 65796 | | |
| Error: 1.0948*MS(subject(sequence)) - 0.0948*MS(Error) | | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 7687.035147 | 7687.035147 | 0.36 | 0.5610 |
| trt | 1 | 1577.042328 | 1577.042328 | 0.07 | 0.7912 |
| subject(sequence) | 21 | 1301373 | 61970 | 2.87 | 0.0272 |
| Error: MS(Error) | 13 | 280666 | 21590 | | |

### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------|------------|-------------|-------------|---------|--------|
| sequence | 1 | 42213 | 42213 | 0.75 | 0.3959 |
| Error | 23.282 | 1313494 | 56416 | | _ |
| Error: 0.86 | 525*MS(sub | r) | _ | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 7687.035147 | 7687.035147 | 0.36 | 0.5610 |
| trt | 1 | 1577.042328 | 1577.042328 | 0.07 | 0.7912 |
| subject(sequence) | 21 | 1301373 | 61970 | 2.87 | 0.0272 |
| Error: MS(Error) | 13 | 280666 | 21590 | | |

Comparison: A vs B

Dependent Variable: T<sub>1/2 el</sub> (h)

### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 42213 | 42213 | 0.75 | 0.3959 |
| Error | 23.282 | 1313494 | 56416 | | _ |
| Error: 0.86 | Error: 0.8625*MS(subject(sequence)) + 0.1375*MS(Error) | | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 7687.035147 | 7687.035147 | 0.36 | 0.5610 |
| trt | 1 | 1577.042328 | 1577.042328 | 0.07 | 0.7912 |
| subject(sequence) | 21 | 1301373 | 61970 | 2.87 | 0.0272 |
| Error: MS(Error) | 13 | 280666 | 21590 | | |

Comparison: A vs B

Dependent Variable: T<sub>1/2 el</sub> (h)

### Least Squares Means

| | | H0 | LSMean1=LSMean2 | |
|---|---|---|---|---|
| trt | LAMZHL LSMEAN | | P | r > t |
| A | 223.656359 | | 0 | .7912 |
| В | 208.856574 | | | |
| | I AMERICA CONTRACT | 0.0 | 0/ 0 01 1: ' | |
| trt | LAMZHL LSMEAN | 90 | % Confidence Limits | |
| Α | 223.656359 | 161.603193 | 285.709526 | |
| В | 208.856574 | 137.610653 | 280.102495 | |
| T | С М С Б.С. | -4.44 | | |
| Lea | ast Squares Means for Effe | ct trt | | |
| | Difference Between | | | |
| i | j Means | 90% Confidence | e Limits for LSMean(i)-LSMea | n(j) |
| 1 | 2 14.799786 | -82.175073 | 111.774644 | |

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Conf | idence Limits |
| A - B | 14.7997857 | 54.7591787 | 0.27 | 0.7912-8 | 2.1750725 | 111.7746439 |

# Listing 16.1.9-2 ANOVA for Treatment Comparison of Nordiazepam - PK Population Comparison: C vs B

Dependent Variable: AUC<sub>0-t</sub> (h\*pg/mL)

### The GLM Procedure

| Class Level | Information | n |
|---|---|---|
| Class | Levels | Values |
| subject | 9 | 101 201 202 203 204 301 402 404 406 |
| sequence | 2 | ABC BAC |
| trt | 2 | ВС |
| ' | | |
| Number of | Number of Observations Read 18 | |
| Number of Observations Used 18 | | |

Comparison: C vs B

Dependent Variable: AUC<sub>0-t</sub> (h\*pg/mL)

### The GLM Procedure

Dependent Variable: LN\_AUCLST

| R-Square | Coeff Var | Root MSE | | LN_AUC | LST Mean |
|---|---|---|---|---|---|
| 0.724163 | 2.081304 | 0.328591 | 15.78774 | | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.05754936 | 0.05754936 | 0.53 | 0.4862 |
| trt | 1 | 0.17097803 | 0.17097803 | 1.58 | 0.2437 |
| subject(sequence | ee) 7 | 2.03916611 | 0.29130944 | 2.70 | 0.0939 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.05754936 | 0.05754936 | 0.53 | 0.4862 |
| trt | 1 | 0.17097803 | 0.17097803 | 1.58 | 0.2437 |
| subject(sequence | ee) 7 | 2.03916611 | 0.29130944 | 2.70 | 0.0939 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.05754936 | 0.05754936 | 0.53 | 0.4862 |
| trt | 1 | 0.17097803 | 0.17097803 | 1.58 | 0.2437 |
| subject(sequence | e) 7 | 2.03916611 | 0.29130944 | 2.70 | 0.0939 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.05754936 | 0.05754936 | 0.53 | 0.4862 |
| trt | 1 | 0.17097803 | 0.17097803 | 1.58 | 0.2437 |
| subject(sequence | ce) 7 | 2.03916611 | 0.29130944 | 2.70 | 0.0939 |

Comparison: C vs B

Dependent Variable: AUC<sub>0-t</sub> (h\*pg/mL)

# The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_AUCLST

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.057549 | 0.057549 | 0.20 | 0.6701 |
| Error 7 2.039166 | | | 0.291309 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-------------------|----|-----------|-------------|---------|--------|
| trt | 1 | 0.170978 | 0.170978 | 1.58 | 0.2437 |
| subject(sequence) | 7 | 2.039166 | 0.291309 | 2.70 | 0.0939 |
| Error: MS(Error) | 8 | 0.863775 | 0.107972 | | |

### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN AUCLST

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.057549 | 0.057549 | 0.20 | 0.6701 |
| Error | 7 | 2.039166 | 0.291309 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| trt | 1 | 0.170978 | 0.170978 | 1.58 | 0.2437 |
| subject(sequence) | 7 | 2.039166 | 0.291309 | 2.70 | 0.0939 |
| Error: MS(Error) | 8 | 0.863775 | 0.107972 | | |

Comparison: C vs B

Dependent Variable: AUC<sub>0-t</sub> (h\*pg/mL)

### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_AUCLST

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.057549 | 0.057549 | 0.20 | 0.6701 |
| Error | 7 | 2.039166 | 0.291309 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| trt | 1 | 0.170978 | 0.170978 | 1.58 | 0.2437 |
| subject(sequence) | 7 | 2.039166 | 0.291309 | 2.70 | 0.0939 |
| Error: MS(Error) | 8 | 0.863775 | 0.107972 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_AUCLST

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.057549 | 0.057549 | 0.20 | 0.6701 |
| Error | 7 | 2.039166 | 0.291309 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| trt | 1 | 0.170978 | 0.170978 | 1.58 | 0.2437 |
| subject(sequence) | 7 | 2.039166 | 0.291309 | 2.70 | 0.0939 |
| Error: MS(Error) | 8 | 0.863775 | 0.107972 | | |

Comparison: C vs B

Dependent Variable: AUC<sub>0-t</sub> (h\*pg/mL)

### Least Squares Means

| | | H0:L | SMean1=LSMean2 |
|---|---|---|---|
| trt | LN AUCLST LSMEAN | | Pr > t |
| В | 15.6965982 | | 0.2437 |
| C | 15.8915216 | | |
| trt | LN AUCLST LSMEAN | 900 | % Confidence Limits |
| В | 15.696598 | 15.492286 | 15.900911 |
| C | 15.891522 | 15.687209 | 16.095834 |
| Le | ast Squares Means for Effect | trt | |
| | Difference Between | | |
| i | j Means | 90% Confidence Li | imits for LSMean(i)-LSMean(j) |
| 1 | 2 -0.194923 | -0.482966 | 0.093119 |

### Dependent Variable: LN\_AUCLST

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confi | dence Limits |
| C - B | 0.19492337 | 0.15489919 | 1.26 | 0.2437-0 | 0.09311913 | 0.48296586 |

# Listing 16.1.9-2 ANOVA for Treatment Comparison of Nordiazepam - PK Population Comparison: C vs B

Dependent Variable: AUC<sub>0-inf</sub> (h\*pg/mL)

### The GLM Procedure

| Class Level | Class Level Information | |
|---|---|---|
| Class | Levels | Values |
| subject | 8 | 101 201 202 203 204 301 404 406 |
| sequence | 2 | ABC BAC |
| trt | 2 | ВС |
| Number of C | Number of Observations Read 11 | |
| Number of Observations Used 11 | | |

Comparison: C vs B

Dependent Variable: AUC<sub>0-inf</sub> (h\*pg/mL)

#### The GLM Procedure

| R-Square | Coeff Var | Root MSE | | LN_AUC | IFO Mean |
|---|---|---|---|---|---|
| 0.904625 | 2.451480 | 0.399149 | 16.28198 | | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.07415386 | 0.07415386 | 0.47 | 0.5655 |
| trt | 1 | 0.36277910 | 0.36277910 | 2.28 | 0.2704 |
| subject(sequence | e) 6 | 2.58535267 | 0.43089211 | 2.70 | 0.2944 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.04440121 | 0.04440121 | 0.28 | 0.6503 |
| trt | 1 | 0.35468757 | 0.35468757 | 2.23 | 0.2742 |
| subject(sequence | e) 6 | 2.58535267 | 0.43089211 | 2.70 | 0.2944 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.02708903 | 0.02708903 | 0.17 | 0.7201 |
| trt | 1 | 0.35468757 | 0.35468757 | 2.23 | 0.2742 |
| subject(sequenc | e) 6 | 2.58535267 | 0.43089211 | 2.70 | 0.2944 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.02708903 | 0.02708903 | 0.17 | 0.7201 |
| trt | 1 | 0.35468757 | 0.35468757 | 2.23 | 0.2742 |
| subject(sequence | e) 6 | 2.58535267 | 0.43089211 | 2.70 | 0.2944 |

Comparison: C vs B

Dependent Variable: AUC<sub>0-inf</sub> (h\*pg/mL)

# The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_AUCIFO

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-----------|--------|-----------|-------------|---------|--------|
| *sequence | 1 | 0.074154 | 0.074154 | 0.15 | 0.7130 |
| Error | 5.1578 | 2.530606 | 0.490633 | | |

Error: 1.22\*MS(subject(sequence)) - 0.22\*MS(Error)

<sup>\*</sup> This test assumes one or more other fixed effects are zero.

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| trt | 1 | 0.362779 | 0.362779 | 1.41 | 0.2731 |
| Error | 7.2018 | 1.856133 | 0.257731 | | |
| Error: 0.3 | 624*MS(sub | iect(sequence)) | + 0.6376*MS(Erro | or) | |

Error: 0.3624\*MS(subject(sequence)) + 0.63/6\*MS(Error)

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-------------------|----|-----------|-------------|---------|--------|
| subject(sequence) | 6 | 2.585353 | 0.430892 | 2.70 | 0.2944 |
| Error: MS(Error) | 2 | 0.318641 | 0.159320 | | |

Comparison: C vs B

Dependent Variable: AUC<sub>0-inf</sub> (h\*pg/mL)

### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_AUCIFO

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.044401 | 0.044401 | 0.09 | 0.7752 |
| Error | 5.1649 | 2.531028 | 0.490046 | | _ |
| Error: 1.21 | Error: 1.2178*MS(subject(sequence)) - 0.2178*MS(Error) | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| trt | 1 | 0.354688 | 0.354688 | 2.23 | 0.2742 |
| subject(sequence) | 6 | 2.585353 | 0.430892 | 2.70 | 0.2944 |
| Error: MS(Error) | 2 | 0.318641 | 0.159320 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.027089 | 0.027089 | 0.06 | 0.8079 |
| Error | 6.1708 | 2.595918 | 0.420675 | | |
| Error: 0.96 | Error: 0.9624*MS(subject(sequence)) + 0.0376*MS(Error) | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| trt | 1 | 0.354688 | 0.354688 | 2.23 | 0.2742 |
| subject(sequence) | 6 | 2.585353 | 0.430892 | 2.70 | 0.2944 |
| Error: MS(Error) | 2 | 0.318641 | 0.159320 | | |

Comparison: C vs B

Dependent Variable: AUC<sub>0-inf</sub> (h\*pg/mL)

### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.027089 | 0.027089 | 0.06 | 0.8079 |
| Error | 6.1708 | 2.595918 | 0.420675 | | |
| Error: 0.96 | Error: 0.9624*MS(subject(sequence)) + 0.0376*MS(Error) | | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| trt | 1 | 0.354688 | 0.354688 | 2.23 | 0.2742 |
| subject(sequence) | 6 | 2.585353 | 0.430892 | 2.70 | 0.2944 |
| Error: MS(Error) | 2 | 0.318641 | 0.159320 | | |

Comparison: C vs B

Dependent Variable: AUC<sub>0-inf</sub> (h\*pg/mL)

### Least Squares Means

| | | H0:L | SMean1=LSMean2 |
|---|---|---|---|
| trt | LN_AUCIFO LSMEAN | | Pr > |
| В | 16.1264488 | | 0.274 |
| C | 16.6127187 | | |
| trt | LN_AUCIFO LSMEAN | 90% | % Confidence Limits |
| В | 16.126449 | 15.474909 | 16.777989 |
| C | 16.612719 | 16.054773 | 17.170664 |
| Le | ast Squares Means for Effec | t trt | |
| | Difference Between | | |
| i | j Means | 90% Confidence L | imits for LSMean(i)-LSMean(j) |
| 1 | 2 -0.486270 | -1.437905 | 0.465366 |

| | | Standard | | | | _ |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confi | dence Limits |
| C - B | 0.48626987 | 0.32590416 | 1.49 | 0.2742-0 | 0.46536558 | 1.43790531 |

# **Listing 16.1.9-2 ANOVA for Treatment Comparison of Nordiazepam - PK Population** Comparison: C vs B

Dependent Variable: C<sub>max</sub> (pg/mL)

### The GLM Procedure

| Class | Levels | Values |
|----------|--------|-------------------------------------|
| subject | 9 | 101 201 202 203 204 301 402 404 406 |
| sequence | 2 | ABC BAC |
| trt | 2 | ВС |

Comparison: C vs B

Dependent Variable: C<sub>max</sub> (pg/mL)

## The GLM Procedure

Dependent Variable: LN\_CMAX

| R-Square | Coeff Var | Root MSE | | LN_C | MAX Mean |
|---|---|---|---|---|---|
| 0.742680 | 3.444682 | 0.366647 | 10.64385 | | _ |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.19249555 | 0.19249555 | 1.43 | 0.2657 |
| trt | 1 | 0.14829852 | 0.14829852 | 1.10 | 0.3243 |
| subject(sequence | e) 7 | 2.76314852 | 0.39473550 | 2.94 | 0.0771 |
| | | | | | _ |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.19249555 | 0.19249555 | 1.43 | 0.2657 |
| trt | 1 | 0.14829852 | 0.14829852 | 1.10 | 0.3243 |
| subject(sequence | e) 7 | 2.76314852 | 0.39473550 | 2.94 | 0.0771 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.19249555 | 0.19249555 | 1.43 | 0.2657 |
| trt | 1 | 0.14829852 | 0.14829852 | 1.10 | 0.3243 |
| subject(sequence | e) 7 | 2.76314852 | 0.39473550 | 2.94 | 0.0771 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.19249555 | 0.19249555 | 1.43 | 0.2657 |
| trt | 1 | 0.14829852 | 0.14829852 | 1.10 | 0.3243 |
| subject(sequence | e) 7 | 2.76314852 | 0.39473550 | 2.94 | 0.0771 |

Comparison: C vs B

Dependent Variable: C<sub>max</sub> (pg/mL)

# The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_CMAX

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.192496 | 0.192496 | 0.49 | 0.5075 |
| Error | 7 | 2.763149 | 0.394736 | | _ |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-------------------|----|-----------|-------------|---------|--------|
| trt | 1 | 0.148299 | 0.148299 | 1.10 | 0.3243 |
| subject(sequence) | 7 | 2.763149 | 0.394736 | 2.94 | 0.0771 |
| Error: MS(Error) | 8 | 1.075439 | 0.134430 | | |

### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_CMAX

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.192496 | 0.192496 | 0.49 | 0.5075 |
| Error | 7 | 2.763149 | 0.394736 | | _ |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| trt | 1 | 0.148299 | 0.148299 | 1.10 | 0.3243 |
| subject(sequence) | 7 | 2.763149 | 0.394736 | 2.94 | 0.0771 |
| Error: MS(Error) | 8 | 1.075439 | 0.134430 | | |

Comparison: C vs B

Dependent Variable: C<sub>max</sub> (pg/mL)

### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_CMAX

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.192496 | 0.192496 | 0.49 | 0.5075 |
| Error | 7 | 2.763149 | 0.394736 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| trt | 1 | 0.148299 | 0.148299 | 1.10 | 0.3243 |
| subject(sequence) | 7 | 2.763149 | 0.394736 | 2.94 | 0.0771 |
| Error: MS(Error) | 8 | 1.075439 | 0.134430 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_CMAX

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.192496 | 0.192496 | 0.49 | 0.5075 |
| Error | 7 | 2.763149 | 0.394736 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| trt | 1 | 0.148299 | 0.148299 | 1.10 | 0.3243 |
| subject(sequence) | 7 | 2.763149 | 0.394736 | 2.94 | 0.0771 |
| Error: MS(Error) | 8 | 1.075439 | 0.134430 | | |

Comparison: C vs B

Dependent Variable: C<sub>max</sub> (pg/mL)

2 -0.181536

### Least Squares Means

| | | H0:L9 | SMean1=LSMean2 | |
|---|---|---|---|---|
| trt | LN CMAX LSMEAN | | | Pr > t |
| В | 10.5646446 | | | 0.3243 |
| C | 10.7461803 | | | |
| trt | LN_CMAX LSMEAN | 90% | 6 Confidence Limits | |
| В | 10.564645 | 10.336670 | 10.792619 | |
| C | 10.746180 | 10.518205 | 10.974155 | |
| Lea | ast Squares Means for Effect | trt | | |
| | Difference Between | | | |
| i | j Means | 90% Confidence I | Limits for LSMean(i)-LS | SMean(j) |

### Dependent Variable: LN\_CMAX

0.139867

-0.502938

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confi | dence Limits |
| C - B | 0.18153574 | 0.17283895 | 1.05 | 0.3243-0 | .13986659 | 0.50293808 |

# Listing 16.1.9-2 ANOVA for Treatment Comparison of Nordiazepam - PK Population Comparison: C vs B

Dependent Variable: Cl/F/kg ((L/h)/kg)

### The GLM Procedure

| Class Level | Information | | |
|---|---|---|---|
| Class | Levels | Values | |
| subject | 8 | 101 201 202 203 204 301 404 406 | |
| sequence | 2 | ABC BAC | |
| trt | 2 | ВС | |
| Number of ( | Observations | Read | 11 |
| Number of C | Number of Observations Used 11 | | |

Comparison: C vs B

Dependent Variable: Cl/F/kg ((L/h)/kg)

### The GLM Procedure

| R-Square | Coeff Var | Root MSE | | LN_CL | FOW Mean |
|-----------------|-----------|-------------|-------------|---------|----------|
| 0.902109 | -10.77248 | 0.443098 | -4.113246 | | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.16198223 | 0.16198223 | 0.83 | 0.4596 |
| trt | 1 | 0.73224034 | 0.73224034 | 3.73 | 0.1932 |
| subject(sequenc | e) 6 | 2.72441644 | 0.45406941 | 2.31 | 0.3323 |
| <u>C</u> | DE | Т Ц СС | Man Carre | F W-1 | D. S. F. |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.09915049 | 0.09915049 | 0.51 | 0.5510 |
| trt | 1 | 0.50837219 | 0.50837219 | 2.59 | 0.2489 |
| subject(sequenc | e) 6 | 2.72441644 | 0.45406941 | 2.31 | 0.3323 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.00445321 | 0.00445321 | 0.02 | 0.8941 |
| trt | 1 | 0.50837219 | 0.50837219 | 2.59 | 0.2489 |
| subject(sequenc | e) 6 | 2.72441644 | 0.45406941 | 2.31 | 0.3323 |
| <u> </u> | DE | T. W.CC | M C | F 37 1 | D . F |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.00445321 | 0.00445321 | 0.02 | 0.8941 |
| trt | 1 | 0.50837219 | 0.50837219 | 2.59 | 0.2489 |
| subject(sequenc | e) 6 | 2.72441644 | 0.45406941 | 2.31 | 0.3323 |

Comparison: C vs B

Dependent Variable: Cl/F/kg ((L/h)/kg)

# The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_CLFOW

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-----------|--------|-----------|-------------|---------|--------|
| *sequence | 1 | 0.161982 | 0.161982 | 0.32 | 0.5976 |
| Error | 5.0095 | 2.558688 | 0.510766 | | |

Error: 1.22\*MS(subject(sequence)) - 0.22\*MS(Error)

<sup>\*</sup> This test assumes one or more other fixed effects are zero.

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| trt | 1 | 0.732240 | 0.732240 | 2.53 | 0.1572 |
| Error | 6.798 | 1.969591 | 0.289733 | | |
| Error: 0.3 | Error: 0.3624*MS(subject(sequence)) + 0.6376*MS(Error) | | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-------------------|----|-----------|-------------|---------|--------|
| subject(sequence) | 6 | 2.724416 | 0.454069 | 2.31 | 0.3323 |
| Error: MS(Error) | 2 | 0.392672 | 0.196336 | | |

Comparison: C vs B

Dependent Variable: Cl/F/kg ((L/h)/kg)

### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_CLFOW

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.099150 | 0.099150 | 0.19 | 0.6777 |
| Error | 5.0178 | 2.560122 | 0.510209 | | |
| Error: 1.21 | Error: 1.2178*MS(subject(sequence)) - 0.2178*MS(Error) | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| trt | 1 | 0.508372 | 0.508372 | 2.59 | 0.2489 |
| subject(sequence) | 6 | 2.724416 | 0.454069 | 2.31 | 0.3323 |
| Error: MS(Error) | 2 | 0.392672 | 0.196336 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.004453 | 0.004453 | 0.01 | 0.9234 |
| Error | 6.1993 | 2.754777 | 0.444373 | | _ |
| Error: 0.96 | Error: 0.9624*MS(subject(sequence)) + 0.0376*MS(Error) | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| trt | 1 | 0.508372 | 0.508372 | 2.59 | 0.2489 |
| subject(sequence) | 6 | 2.724416 | 0.454069 | 2.31 | 0.3323 |
| Error: MS(Error) | 2 | 0.392672 | 0.196336 | | |

Comparison: C vs B

Dependent Variable: Cl/F/kg ((L/h)/kg)

### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------|-----------|------------|-------------|---------|--------|
| sequence | 1 | 0.004453 | 0.004453 | 0.01 | 0.9234 |
| Error | 6.1993 | 2.754777 | 0.444373 | | |
| Error: 0.96 | 24*MS(sub | ) | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| trt | 1 | 0.508372 | 0.508372 | 2.59 | 0.2489 |
| subject(sequence) | 6 | 2.724416 | 0.454069 | 2.31 | 0.3323 |
| Error: MS(Error) | 2 | 0.392672 | 0.196336 | | |

Comparison: C vs B

Dependent Variable: Cl/F/kg ((L/h)/kg)

2 0.582164

### Least Squares Means

| | | H0:L | SMean1=LSMean2 | |
|---|---|---|---|---|
| trt | LN_CLFOW LSMEAN | | | Pr > t |
| В | -3.91316447 | | | 0.2489 |
| C | -4.49532836 | | | |
| trt | LN_CLFOW LSMEAN | 900 | % Confidence Limits | |
| В | -3.913164 | -4.636444 | -3.189885 | |
| C | -4.495328 | -5.114708 | -3.875949 | |
| Lea | ast Squares Means for Effect | trt | | |
| | Difference Between | | | |
| i | j Means | 90% Confidence L | imits for LSMean(i)-LS | Mean(j) |

### Dependent Variable: LN\_CLFOW

1.638581

-0.474253

| | | Standard | | | |
|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confidence Limits |
| C - B | -0.58216389 | 0.36178831 | -1.61 | 0.2489-1 | 1.63858054 0.47425276 |

# Listing 16.1.9-2 ANOVA for Treatment Comparison of Nordiazepam - PK Population Comparison: C vs B

Dependent Variable: Cl/F (L/h)

### The GLM Procedure

| Class Level | | V-1 | |
|---|---|---|---|
| Class | Levels | Values | |
| subject | 8 | 101 201 202 203 204 301 404 406 | |
| sequence | 2 | ABC BAC | |
| trt | 2 | ВС | |
| Number of 0 | Observations | Read | 11 |
| Number of Observations Used | | | |

Comparison: C vs B

Dependent Variable: Cl/F (L/h)

### The GLM Procedure

| R-Square | Coeff Var | Root MSE | B | LN_ | CLFO Mean |
|---|---|---|---|---|---|
| 0.911563 | 161.6764 | 0.443098 | 0.274065 | | |
| Source | DF | Type I SS | Mean Square | F Value | |
| sequence | 1 | 0.00821426 | 0.00821426 | 0.04 | 0.8569 |
| trt | 1 | 0.32342250 | 0.32342250 | 1.65 | 0.3280 |
| subject(sequence | e) 6 | 3.71584302 | 0.61930717 | 3.15 | 0.2602 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| | 1 | 0.00110942 | 0.00110942 | 0.01 | 0.9469 |
| sequence<br>trt | 1 | 0.50837219 | 0.50837219 | 2.59 | 0.2489 |
| subject(sequence | - | 3.71584302 | 0.61930717 | 3.15 | 0.2489 |
| subject(sequence | <i>5)</i> 0 | 3./1364302 | 0.01930717 | 3.13 | 0.2002 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.15060463 | 0.15060463 | 0.77 | 0.4735 |
| trt | 1 | 0.50837219 | 0.50837219 | 2.59 | 0.2489 |
| subject(sequence | e) 6 | 3.71584302 | 0.61930717 | 3.15 | 0.2602 |
| Source | DF | Tyma IV CC | Maan Sauara | F Value | Pr > F |
| | | Type IV SS | Mean Square | | |
| sequence | 1 | 0.15060463 | 0.15060463 | 0.77 | 0.4735 |
| trt | 1 | 0.50837219 | 0.50837219 | 2.59 | 0.2489 |
| subject(sequence | e) 6 | 3.71584302 | 0.61930717 | 3.15 | 0.2602 |

Comparison: C vs B

Dependent Variable: Cl/F (L/h)

# The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_CLFO

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-----------|--------|-----------|-------------|---------|--------|
| *sequence | 1 | 0.008214 | 0.008214 | 0.01 | 0.9184 |
| Error | 5.2819 | 3.762543 | 0.712353 | | |

Error: 1.22\*MS(subject(sequence)) - 0.22\*MS(Error)

<sup>\*</sup> This test assumes one or more other fixed effects are zero.

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| trt | 1 | 0.323422 | 0.323422 | 0.93 | 0.3660 |
| Error | 7.5308 | 2.632859 | 0.349611 | | |
| Error: 0.3 | 624*MS(sub | iect(sequence)) | + 0.6376*MS(Erro | or) | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-------------------|----|-----------|-------------|---------|--------|
| subject(sequence) | 6 | 3.715843 | 0.619307 | 3.15 | 0.2602 |
| Error: MS(Error) | 2 | 0.392672 | 0.196336 | | |

Comparison: C vs B

Dependent Variable: Cl/F (L/h)

### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_CLFO

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------|-----------|------------|-------------|---------|--------|
| sequence | 1 | 0.001109 | 0.001109 | 0.00 | 0.9699 |
| Error | 5.2878 | 3.761979 | 0.711439 | | |
| Error: 1.21 | 78*MS(sub | ) | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| trt | 1 | 0.508372 | 0.508372 | 2.59 | 0.2489 |
| subject(sequence) | 6 | 3.715843 | 0.619307 | 3.15 | 0.2602 |
| Error: MS(Error) | 2 | 0.392672 | 0.196336 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------|-----------|-------------|-------------|---------|--------|
| sequence | 1 | 0.150605 | 0.150605 | 0.25 | 0.6347 |
| Error | 6.1468 | 3.708949 | 0.603393 | | |
| Error: 0.96 | 24*MS(sub | ) | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| trt | 1 | 0.508372 | 0.508372 | 2.59 | 0.2489 |
| subject(sequence) | 6 | 3.715843 | 0.619307 | 3.15 | 0.2602 |
| Error: MS(Error) | 2 | 0.392672 | 0.196336 | | |

Comparison: C vs B

Dependent Variable: Cl/F (L/h)

### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.150605 | 0.150605 | 0.25 | 0.6347 |
| Error | 6.1468 | 3.708949 | 0.603393 | | |
| Error: 0.9624*MS(subject(sequence)) + 0.0376*MS(Error) | | | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| trt | 1 | 0.508372 | 0.508372 | 2.59 | 0.2489 |
| subject(sequence) | 6 | 3.715843 | 0.619307 | 3.15 | 0.2602 |
| Error: MS(Error) | 2 | 0.392672 | 0.196336 | | |

Comparison: C vs B

Dependent Variable: Cl/F (L/h)

2 0.582164

### Least Squares Means

| | | H0:L | SMean1=LSMean2 |
|---|---|---|---|
| trt | LN CLFO LSMEAN | | Pr > t |
| В | 0.48125860 | | 0.2489 |
| C | -0.10090529 | | |
| trt | LN_CLFO LSMEAN | 90% | 6 Confidence Limits |
| В | 0.481259 | -0.242020 | 1.204538 |
| C | -0.100905 | -0.720284 | 0.518474 |
| Lea | ast Squares Means for Effec | t trt | |
| | Difference Between | | |
| i | j Means | 90% Confidence L | imits for LSMean(i)-LSMean(j) |

Dependent Variable: LN\_CLFO

-0.474253

1.638581

| | Standard | | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confid | ence Limits |
| C - B | -0.58216389 | 0.36178831 | -1.61 | 0.2489-1 | .63858054 | 0.47425276 |

# Listing 16.1.9-2 ANOVA for Treatment Comparison of Nordiazepam - PK Population Comparison: C vs B

Dependent Variable: V<sub>d</sub>/F/kg (L/kg)

### The GLM Procedure

| Class Level | Information | |
|---|---|---|
| Class | Levels | Values |
| subject | 8 | 101 201 202 203 204 301 404 406 |
| sequence | 2 | ABC BAC |
| trt | 2 | ВС |
| Number of Observations Read | | |
| Number of Observations Used 11 | | |

Comparison: C vs B

Dependent Variable: V<sub>d</sub>/F/kg (L/kg)

### The GLM Procedure

Dependent Variable: LN\_VZFOW

| R-Square | Coeff Var | Root MSE | | LN_VZ | FOW Mean |
|---|---|---|---|---|---|
| 0.770703 | 58.09245 | 0.685302 | 1.179674 | _ | |
| | | | | | _ |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.00961309 | 0.00961309 | 0.02 | 0.8993 |
| trt | 1 | 0.23838114 | 0.23838114 | 0.51 | 0.5501 |
| subject(sequence | e) 6 | 2.90905346 | 0.48484224 | 1.03 | 0.5680 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.02142687 | 0.02142687 | 0.05 | 0.8507 |
| trt | 1 | 0.46004136 | 0.46004136 | 0.98 | 0.4266 |
| subject(sequence | e) 6 | 2.90905346 | 0.48484224 | 1.03 | 0.5680 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.04288477 | 0.04288477 | 0.09 | 0.7910 |
| trt | 1 | 0.46004136 | 0.46004136 | 0.98 | 0.4266 |
| subject(sequence | e) 6 | 2.90905346 | 0.48484224 | 1.03 | 0.5680 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.04288477 | 0.04288477 | 0.09 | 0.7910 |
| trt | 1 | 0.46004136 | 0.46004136 | 0.98 | 0.4266 |
| subject(sequence | e) 6 | 2.90905346 | 0.48484224 | 1.03 | 0.5680 |
Comparison: C vs B

Dependent Variable: V<sub>d</sub>/F/kg (L/kg)

## The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_VZFOW

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-----------|--------|-----------|-------------|---------|--------|
| *sequence | 1 | 0.009613 | 0.009613 | 0.02 | 0.8956 |
| Error | 3.7444 | 1.827974 | 0.488187 | | |

Error: 1.22\*MS(subject(sequence)) - 0.22\*MS(Error)

<sup>\*</sup> This test assumes one or more other fixed effects are zero.

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| trt | 1 | 0.238381 | 0.238381 | 0.50 | 0.5136 |
| Error | 4.5171 | 2.146267 | 0.475148 | | _ |
| Error: 0.3 | 624*MS(sub | iect(sequence)) | + 0.6376*MS(Erro | or) | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-------------------|----|-----------|-------------|---------|--------|
| subject(sequence) | 6 | 2.909053 | 0.484842 | 1.03 | 0.5680 |
| Error: MS(Error) | 2 | 0.939277 | 0.469638 | | |

Comparison: C vs B

Dependent Variable: V<sub>d</sub>/F/kg (L/kg)

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_VZFOW

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.021427 | 0.021427 | 0.04 | 0.8449 |
| Error | 3.7623 | 1.836568 | 0.488154 | | |
| Error: 1.21 | Error: 1.2178*MS(subject(sequence)) - 0.2178*MS(Error) | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| trt | 1 | 0.460041 | 0.460041 | 0.98 | 0.4266 |
| subject(sequence) | 6 | 2.909053 | 0.484842 | 1.03 | 0.5680 |
| Error: MS(Error) | 2 | 0.939277 | 0.469638 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.042885 | 0.042885 | 0.09 | 0.7754 |
| Error | 6.4353 | 3.116445 | 0.484270 | | _ |
| Error: 0.96 | 24*MS(sub | ject(sequence)) + | 0.0376*MS(Error | ) | _ |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| trt | 1 | 0.460041 | 0.460041 | 0.98 | 0.4266 |
| subject(sequence) | 6 | 2.909053 | 0.484842 | 1.03 | 0.5680 |
| Error: MS(Error) | 2 | 0.939277 | 0.469638 | | |

Comparison: C vs B

Dependent Variable: V<sub>d</sub>/F/kg (L/kg)

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.042885 | 0.042885 | 0.09 | 0.7754 |
| Error | 6.4353 | 3.116445 | 0.484270 | | _ |
| Error: 0.96 | 524*MS(sub | ject(sequence)) + | 0.0376*MS(Error | •) | _ |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| trt | 1 | 0.460041 | 0.460041 | 0.98 | 0.4266 |
| subject(sequence) | 6 | 2.909053 | 0.484842 | 1.03 | 0.5680 |
| Error: MS(Error) | 2 | 0.939277 | 0.469638 | | |

Comparison: C vs B

Dependent Variable: V<sub>d</sub>/F/kg (L/kg)

2 0.553800

#### Least Squares Means

| | | H0:LSMean1=LSMean2 | | |
|---|---|---|---|---|
| trt | LN_VZFOW LSMEAN | | Pr > | · t |
| В | 1.48139692 | | 0.42 | 66 |
| C | 0.92759710 | | | |
| trt | LN_VZFOW LSMEAN | 90% | Confidence Limits | |
| В | 1.481397 | 0.362764 | 2.600030 | |
| C | 0.927597 | -0.030343 | 1.885537 | |
| Lag | not Squarag Manna for Effort | tvt | | |
| Lea | ast Squares Means for Effect Difference Between | uı | | |
| | i Means | 000/ Confidence Lim | its for LSMean(i)-LSMean(i | |

#### Dependent Variable: LN\_VZFOW

2.187667

-1.080068

| | | Standard | | | |
|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confidence Limits |
| C - B | -0.55379982 | 0.55954645 | -0.99 | 0.4266-2 | 2.18766737 1.08006773 |

# Listing 16.1.9-2 ANOVA for Treatment Comparison of Nordiazepam - PK Population Comparison: C vs B

Dependent Variable: V<sub>d</sub>/F (L)

#### The GLM Procedure

| Class Level | Information | | |
|---|---|---|---|
| Class | Levels | Values | |
| subject | 8 | 101 201 202 203 204 301 404 406 | |
| sequence | 2 | ABC BAC | |
| trt | 2 | ВС | |
| Number of C | Observations | Read | 11 |
| Number of Observations Used | | | |

Comparison: C vs B

Dependent Variable: V<sub>d</sub>/F (L)

#### The GLM Procedure

| R-Square | Coeff Var | Root MSE | 3 | LN | VZFO Mean |
|---|---|---|---|---|---|
| 0.855335 | 12.31010 | 0.685302 | 5.566985 | _ | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.16800486 | 0.16800486 | 0.36 | 0.6105 |
| trt | 1 | 0.04049550 | 0.04049550 | 0.09 | 0.7967 |
| subject(sequence | ) 6 | 5.34497302 | 0.89082884 | 1.90 | 0.3847 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.18314367 | 0.18314367 | 0.39 | 0.5961 |
| trt | 1 | 0.46004136 | 0.46004136 | 0.98 | 0.4266 |
| subject(sequence | ) 6 | 5.34497302 | 0.89082884 | 1.90 | 0.3847 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.27924049 | 0.27924049 | 0.59 | 0.5213 |
| trt | 1 | 0.46004136 | 0.46004136 | 0.98 | 0.4266 |
| subject(sequence | ) 6 | 5.34497302 | 0.89082884 | 1.90 | 0.3847 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.27924049 | 0.27924049 | 0.59 | 0.5213 |
| trt | 1 | 0.46004136 | 0.46004136 | 0.98 | 0.4266 |
| subject(sequence | ) 6 | 5.34497302 | 0.89082884 | 1.90 | 0.3847 |

Comparison: C vs B

Dependent Variable: V<sub>d</sub>/F (L)

## The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_VZFO

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-----------|--------|-----------|-------------|---------|--------|
| *sequence | 1 | 0.168005 | 0.168005 | 0.17 | 0.6972 |
| Error | 4.7838 | 4.704785 | 0.983483 | | |

Error: 1.22\*MS(subject(sequence)) - 0.22\*MS(Error)

<sup>\*</sup> This test assumes one or more other fixed effects are zero.

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| trt | 1 | 0.040496 | 0.040496 | 0.07 | 0.8069 |
| Error | 6.2249 | 3.873577 | 0.622268 | | |
| Error: 0.3 | 624*MS(sub | iect(sequence)) | + 0.6376*MS(Erro | or) | |

| C | DE T 100 | M C | Г 17-1 | г |
|---|----------|-----|--------|---|

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-------------------|----|-----------|-------------|---------|--------|
| subject(sequence) | 6 | 5.344973 | 0.890829 | 1.90 | 0.3847 |
| Error: MS(Error) | 2 | 0.939277 | 0.469638 | | |

Comparison: C vs B

Dependent Variable: V<sub>d</sub>/F (L)

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_VZFO

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.183144 | 0.183144 | 0.19 | 0.6847 |
| Error | 4.7939 | 4.710396 | 0.982573 | | |
| Error: 1.21 | Error: 1.2178*MS(subject(sequence)) - 0.2178*MS(Error) | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| trt | 1 | 0.460041 | 0.460041 | 0.98 | 0.4266 |
| subject(sequence) | 6 | 5.344973 | 0.890829 | 1.90 | 0.3847 |
| Error: MS(Error) | 2 | 0.939277 | 0.469638 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.279240 | 0.279240 | 0.32 | 0.5918 |
| Error | 6.2419 | 5.461567 | 0.874982 | | |
| Error: 0.96 | 524*MS(sub | ject(sequence)) + | 0.0376*MS(Error | ) | _ |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| trt | 1 | 0.460041 | 0.460041 | 0.98 | 0.4266 |
| subject(sequence) | 6 | 5.344973 | 0.890829 | 1.90 | 0.3847 |
| Error: MS(Error) | 2 | 0.939277 | 0.469638 | | |

Comparison: C vs B

Dependent Variable: V<sub>d</sub>/F (L)

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.279240 | 0.279240 | 0.32 | 0.5918 |
| Error | 6.2419 | 5.461567 | 0.874982 | | |
| Error: 0.96 | 524*MS(sub | ject(sequence)) + | 0.0376*MS(Error | .) | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| trt | 1 | 0.460041 | 0.460041 | 0.98 | 0.4266 |
| subject(sequence) | 6 | 5.344973 | 0.890829 | 1.90 | 0.3847 |
| Error: MS(Error) | 2 | 0.939277 | 0.469638 | | |

Comparison: C vs B

Dependent Variable: V<sub>d</sub>/F (L)

#### Least Squares Means

| | | H0:L | SMean1=LSMean2 |
|---|---|---|---|
| trt | LN VZFO LSMEAN | | Pr > |
| В | 5.87582000 | | 0.426 |
| C | 5.32202018 | | |
| trt | LN VZFO LSMEAN | 90 | % Confidence Limits |
| В | 5.875820 | 4.757187 | 6.994453 |
| C | 5.322020 | 4.364080 | 6.279960 |
| Lea | ast Squares Means for Effec | et trt | |
| | Difference Between | | |
| i | j Means | 90% Confidence | Limits for LSMean(i)-LSMean(j) |
| 1 | 2 0.553800 | -1.080068 | 2.187667 |

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confid | dence Limits |
| C - B | -0.55379982 | 0.55954645 | -0.99 | 0.4266-2 | 2.18766737 | 1.08006773 |

# Listing 16.1.9-2 ANOVA for Treatment Comparison of Nordiazepam - PK Population Comparison: C vs B

Dependent Variable: T<sub>max</sub> (h)

#### The GLM Procedure

| Class Level | Information | n | |
|---|---|---|---|
| Class | Levels | Values | |
| subject | 9 | 101 201 202 203 204 301 402 404 406 | |
| sequence | 2 | ABC BAC | |
| trt | 2 | ВС | |
| ' | | | |
| Number of | Observation | ns Read | 18 |
| Number of | Number of Observations Used 18 | | |

Comparison: C vs B

Dependent Variable: T<sub>max</sub> (h)

### The GLM Procedure

| R-Square | Coeff Var | Root 1 | MSE | TM | IAX Mean |
|---|---|---|---|---|---|
| 0.709476 | 32.06432 | 33.76 | 521 10: | 5.3046 | |
| | | | | | _ |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 1284.96583 | 1284.96583 | 1.13 | 0.3194 |
| trt | 1 | 1546.58827 | 1546.58827 | 1.36 | 0.2777 |
| subject(sequence) | 7 | 19441.71556 | 2777.38794 | 2.44 | 0.1178 |
| | | | | | _ |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 1284.96583 | 1284.96583 | 1.13 | 0.3194 |
| trt | 1 | 1546.58827 | 1546.58827 | 1.36 | 0.2777 |
| subject(sequence) | 7 | 19441.71556 | 2777.38794 | 2.44 | 0.1178 |
| | | | | | _ |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 1284.96583 | 1284.96583 | 1.13 | 0.3194 |
| trt | 1 | 1546.58827 | 1546.58827 | 1.36 | 0.2777 |
| subject(sequence) | 7 | 19441.71556 | 2777.38794 | 2.44 | 0.1178 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 1284.96583 | 1284.96583 | 1.13 | 0.3194 |
| trt | 1 | 1546.58827 | 1546.58827 | 1.36 | 0.2777 |
| subject(sequence) | 7 | 19441.71556 | 2777.38794 | 2.44 | 0.1178 |

Comparison: C vs B

Dependent Variable: T<sub>max</sub> (h)

## The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: TMAX

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-------------|----------|-------------|-------------|---------|--------|
| sequence | 1 | 1284.965831 | 1284.965831 | 0.46 | 0.5182 |
| Error | 7 | 19442 | 2777.387937 | | |
| Error: MS(s | subiect( | sequence)) | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| trt | 1 | 1546.588267 | 1546.588267 | 1.36 | 0.2777 |
| subject(sequence) | 7 | 19442 | 2777.387937 | 2.44 | 0.1178 |
| Error: MS(Error) | 8 | 9120.713962 | 1140.089245 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------|----------|-------------|-------------|---------|--------|
| sequence | 1 | 1284.965831 | 1284.965831 | 0.46 | 0.5182 |
| Error | 7 | 19442 | 2777.387937 | | |
| Error: MS(s | subject( | sequence)) | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| trt | 1 | 1546.588267 | 1546.588267 | 1.36 | 0.2777 |
| subject(sequence) | 7 | 19442 | 2777.387937 | 2.44 | 0.1178 |
| Error: MS(Error) | 8 | 9120.713962 | 1140.089245 | | |

Comparison: C vs B

Dependent Variable: T<sub>max</sub> (h)

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: TMAX

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 1284.965831 | 1284.965831 | 0.46 | 0.5182 |
| Error | 7 | 19442 | 2777.387937 | | |
| Error: MS(s | Error: MS(subject(sequence)) | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| trt | 1 | 1546.588267 | 1546.588267 | 1.36 | 0.2777 |
| subject(sequence) | 7 | 19442 | 2777.387937 | 2.44 | 0.1178 |
| Error: MS(Error) | 8 | 9120.713962 | 1140.089245 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 1284.965831 | 1284.965831 | 0.46 | 0.5182 |
| Error | 7 | 19442 | 2777.387937 | | |
| Error: MS(s | Error: MS(subject(sequence)) | | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| trt | 1 | 1546.588267 | 1546.588267 | 1.36 | 0.2777 |
| subject(sequence) | 7 | 19442 | 2777.387937 | 2.44 | 0.1178 |
| Error: MS(Error) | 8 | 9120.713962 | 1140.089245 | | |

Comparison: C vs B

Dependent Variable: T<sub>max</sub> (h)

#### Least Squares Means

| | | | H0: | LSMean1=LSMean2 |
|---|---|---|---|---|
| trt | TI | MAX LSMEAN | | Pr > t |
| В | 11 | 3.629364 | | 0.2777 |
| C | 95 | 5.090586 | | |
| trt | T | MAX LSMEAN | 90 | % Confidence Limits |
| В | 11 | 13.629364 | 92.634720 | 134.624008 |
| C | 95 | 5.090586 | 74.095942 | 116.085230 |
| Le | ast | Squares Means for Effec | et trt | |
| | | Difference Between | | |
| i | j | Means | 90% Confidence Lir | nits for LSMean(i)-LSMean(j) |
| 1 | 2 | 18.538778 | -11.059781 | 48.137337 |

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confi | dence Limits |
| C - B | -18.5387778 | 15.9170715 | -1.16 | 0.2777-4 | 18.1373369 | 11.0597813 |

# Listing 16.1.9-2 ANOVA for Treatment Comparison of Nordiazepam - PK Population Comparison: C vs B

Dependent Variable: K<sub>el</sub> (/h)

#### The GLM Procedure

| Class Level | | V-1 |
|---|---|---|
| Class | Levels | Values |
| subject | 8 | 101 201 202 203 204 301 404 406 |
| sequence | 2 | ABC BAC |
| trt | 2 | ВС |
| Number of 0 | Number of Observations Read 11 | |
| Number of Observations Used 1 | | |

Comparison: C vs B

Dependent Variable: K<sub>el</sub> (/h)

#### The GLM Procedure

| R-Square | Coeff Var | Root | MSE | | LAMZ Mean |
|---|---|---|---|---|---|
| 0.979044 | 25.02204 | 0.00 | 1571 | 0.006279 | |
| Source | DF | Type I SS | Mean Square | e F Valu | e Pr > F |
| sequence | 1 | 0.00002833 | 0.00002833 | 11.48 | 0.0772 |
| trt | 1 | 0.00000170 | 0.00000170 | 0.69 | 0.4941 |
| subject(sequence) | 6 | 0.00020060 | 0.00003343 | 13.55 | 0.0703 |
| Source | DF | Type II SS | Mean Square | F Value | e $Pr > F$ |
| sequence | 1 | 0.00002668 | 0.00002668 | 10.81 | 0.0814 |
| trt | 1 | 0.00000001 | 0.00000001 | 0.01 | 0.9482 |
| subject(sequence) | 6 | 0.00020060 | 0.00003343 | 13.55 | 0.0703 |
| Source | DF | Type III SS | Mean Square | F Valu | e Pr > F |
| sequence | 1 | 0.00000850 | 0.00000850 | 3.44 | 0.2046 |
| trt | 1 | 0.00000001 | 0.00000001 | 0.01 | 0.9482 |
| subject(sequence) | 6 | 0.00020060 | 0.00003343 | 13.55 | 0.0703 |
| Source | DF | Type IV SS | Mean Square | F Valu | e Pr > F |
| sequence | 1 | 0.00000850 | 0.00000850 | 3.44 | 0.2046 |
| trt | 1 | 0.00000001 | 0.00000001 | 0.01 | 0.9482 |
| subject(sequence) | 6 | 0.00020060 | 0.00003343 | 13.55 | 0.0703 |

Comparison: C vs B

Dependent Variable: K<sub>el</sub> (/h)

## The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LAMZ

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-----------|--------|-------------|-------------|---------|--------|
| *sequence | 1 | 0.000028326 | 0.000028326 | 0.70 | 0.4345 |
| Error | 5.8382 | 0.000235 | 0.000040245 | | |

Error: 1.22\*MS(subject(sequence)) - 0.22\*MS(Error)

<sup>\*</sup> This test assumes one or more other fixed effects are zero.

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| trt | 1 | 0.000001698 | 0.000001698 | 0.12 | 0.7347 |
| Error | 7.2909 | 0.000099806 | 0.000013689 | | |
| Error: 0.3 | 3624*MS(sul | oject(sequence)) + | 0.6376*MS(Error) | | _ |

| Source | D | F Type I SS | Mean Square | F Value | Pr > F |
|-------------------|---|-------------|-------------|---------|--------|
| subject(sequence) | 6 | 0.000201 | 0.000033433 | 13.55 | 0.0703 |
| Error: MS(Error) | 2 | 0.000004936 | 0.000002468 | | |

Comparison: C vs B

Dependent Variable: K<sub>el</sub> (/h)

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LAMZ

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.000026680 | 0.000026680 | 0.66 | 0.4471 |
| Error | 5.8395 | 0.000235 | 0.000040178 | | |
| Error: 1.21 | 78*MS(sub | oject(sequence)) - 0 | .2178*MS(Error) | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|--------------|--------------|---------|--------|
| trt | 1 | 1.3259677E-8 | 1.3259677E-8 | 0.01 | 0.9482 |
| subject(sequence) | 6 | 0.000201 | 0.000033433 | 13.55 | 0.0703 |
| Error: MS(Error) | 2 | 0.000004936 | 0.000002468 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.000008502 | 0.000008502 | 0.26 | 0.6260 |
| Error | 6.0345 | 0.000195 | 0.000032268 | | |
| Error: 0.96 | 524*MS(sub | oject(sequence)) + ( | 0.0376*MS(Error) | | _ |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|--------------|--------------|---------|--------|
| trt | 1 | 1.3259677E-8 | 1.3259677E-8 | 0.01 | 0.9482 |
| subject(sequence) | 6 | 0.000201 | 0.000033433 | 13.55 | 0.0703 |
| Error: MS(Error) | 2 | 0.000004936 | 0.000002468 | | |

Comparison: C vs B

Dependent Variable: K<sub>el</sub> (/h)

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.000008502 | 0.000008502 | 0.26 | 0.6260 |
| Error | 6.0345 | 0.000195 | 0.000032268 | | |
| Error: 0.96 | 524*MS(sub | pject(sequence)) + | 0.0376*MS(Error) | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|--------------|--------------|---------|--------|
| trt | 1 | 1.3259677E-8 | 1.3259677E-8 | 0.01 | 0.9482 |
| subject(sequence) | 6 | 0.000201 | 0.000033433 | 13.55 | 0.0703 |
| Error: MS(Error) | 2 | 0.000004936 | 0.000002468 | | |

Comparison: C vs B

Dependent Variable: K<sub>el</sub> (/h)

#### Least Squares Means

| | | I | H0:LSMean1=LSMean2 | 2 |
|---|---|---|---|---|
| trt | LAMZ LSMEAN | | | Pr > t |
| В | 0.00555261 | | | 0.9482 |
| C | 0.00545859 | | | |
| trt | LAMZ LSMEAN | | 90% Confidence Lin | nits |
| В | 0.005553 | 0.0029 | 0.008117 | 7 |
| C | 0.005459 | 0.0032 | 263 0.007655 | 5 |
| Lea | ast Squares Means for Effect trt | | | |
| | | 90% | 6 Confidence Limits for | r |
| i | j Difference Between Means | I | SMean(i)-LSMean(j) | |
| 1 | 2 0.000094020 | -0.003652 | 0.003840 | |

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confid | dence Limits |
| C - B | -0.00009402 | 0.00128273 | -0.07 | 0.9482-0 | 0.00383959 | 0.00365155 |

# Listing 16.1.9-2 ANOVA for Treatment Comparison of Nordiazepam - PK Population Comparison: C vs B

Dependent Variable: T<sub>1/2 el</sub> (h)

#### The GLM Procedure

| Class Level | Information | |
|---|---|---|
| Class | Levels | Values |
| subject | 8 | 101 201 202 203 204 301 404 406 |
| sequence | 2 | ABC BAC |
| trt | 2 | ВС |
| Number of ( | Number of Observations Read 11 | |
| Number of Observations Used 11 | | |

Comparison: C vs B

Dependent Variable: T<sub>1/2 el</sub> (h)

#### The GLM Procedure

| R-Square | Coeff Var | Root MSE | , | LAMZ | ZHL Mean |
|---|---|---|---|---|---|
| 0.936339 | 32.11823 | 52.93033 | 164.7984 | | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 781.19473 | 781.19473 | 0.28 | 0.6502 |
| trt | 1 | 6489.38122 | 6489.38122 | 2.32 | 0.2674 |
| subject(sequence | ) 6 | 75143.68682 | 12523.94780 | 4.47 | 0.1941 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 390.22411 | 390.22411 | 0.14 | 0.7448 |
| trt | 1 | 78.94660 | 78.94660 | 0.03 | 0.8821 |
| subject(sequence | ) 6 | 75143.68682 | 12523.94780 | 4.47 | 0.1941 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 455.07734 | 455.07734 | 0.16 | 0.7259 |
| trt | 1 | 78.94660 | 78.94660 | 0.03 | 0.8821 |
| subject(sequence | ) 6 | 75143.68682 | 12523.94780 | 4.47 | 0.1941 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 455.07734 | 455.07734 | 0.16 | 0.7259 |
| trt | 1 | 78.94660 | 78.94660 | 0.03 | 0.8821 |
| subject(sequence | ) 6 | 75143.68682 | 12523.94780 | 4.47 | 0.1941 |

Comparison: C vs B

Dependent Variable: T<sub>1/2 el</sub> (h)

## The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LAMZHL

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-----------|--------|------------|-------------|---------|--------|
| *sequence | 1 | 781.194725 | 781.194725 | 0.05 | 0.8258 |
| Error | 5.4989 | 80628 | 14663 | | |

Error: 1.22\*MS(subject(sequence)) - 0.22\*MS(Error)

<sup>\*</sup> This test assumes one or more other fixed effects are zero.

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| trt | 1 | 6489.381224 | 6489.381224 | 1.03 | 0.3409 |
| Error | 7.9553 | 50316 | 6324.760478 | | |
| Error: 0.3 | Error: 0.3624*MS(subject(sequence)) + 0.6376*MS(Error) | | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| subject(sequence) | 6 | 75144 | 12524 | 4.47 | 0.1941 |
| Error: MS(Error) | 2 | 5603.239711 | 2801.619856 | | |

Comparison: C vs B

Dependent Variable: T<sub>1/2 el</sub> (h)

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LAMZHL

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 390.224108 | 390.224108 | 0.03 | 0.8761 |
| Error | 5.503 | 80574 | 14642 | | |
| Error: 1.2178*MS(subject(sequence)) - 0.2178*MS(Error) | | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| trt | 1 | 78.946602 | 78.946602 | 0.03 | 0.8821 |
| subject(sequence) | 6 | 75144 | 12524 | 4.47 | 0.1941 |
| Error: MS(Error) | 2 | 5603.239711 | 2801.619856 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 455.077342 | 455.077342 | 0.04 | 0.8529 |
| Error | 6.104 | 74213 | 12158 | | _ |
| Error: 0.9624*MS(subject(sequence)) + 0.0376*MS(Error) | | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| trt | 1 | 78.946602 | 78.946602 | 0.03 | 0.8821 |
| subject(sequence) | 6 | 75144 | 12524 | 4.47 | 0.1941 |
| Error: MS(Error) | 2 | 5603.239711 | 2801.619856 | | |

Comparison: C vs B

Dependent Variable: T<sub>1/2 el</sub> (h)

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 455.077342 | 455.077342 | 0.04 | 0.8529 |
| Error | 6.104 | 74213 | 12158 | | |
| Error: 0.96 | Error: 0.9624*MS(subject(sequence)) + 0.0376*MS(Error) | | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| trt | 1 | 78.946602 | 78.946602 | 0.03 | 0.8821 |
| subject(sequence) | 6 | 75144 | 12524 | 4.47 | 0.1941 |
| Error: MS(Error) | 2 | 5603.239711 | 2801.619856 | | |

Comparison: C vs B

Dependent Variable: T<sub>1/2 el</sub> (h)

#### Least Squares Means

| | | H | 0:LSMean1=LSMean2 |
|---|---|---|---|
| trt | LAMZHL LSMEAN | | Pr > t |
| В | 177.749549 | | 0.8821 |
| <u>C</u> | 185.004276 | | |
| trt | LAMZHL LSMEAN | 9 | 0% Confidence Limits |
| В | 177.749549 | 91.350230 | 264.148869 |
| C | 185.004276 | 111.016320 | 258.992233 |
| Lea | ast Squares Means for Effe | ect trt | |
| | Difference Between | | |
| i | j Means | 90% Confidence | ee Limits for LSMean(i)-LSMean(j) |
| 1 | 2 -7.254727 | -133.449010 | 118.939556 |

| | | Standard | | | | _ |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confi | dence Limits |
| C - B | 7.25472729 | 43.2174336 | 0.17 | 0.8821-1 | 18.9395558 | 133.44901033 |

Listing 16.1.9-3 Wilcoxon Signed-Rank Test for  $T_{max}$  for Treatment Comparison of Diazepam – PK Population

Listing 16.1.9-3 Wilcoxon Signed-Rank Test for T<sub>max</sub> for Treatment Comparison of Diazepam - PK Population

| 0 | | |
|------------------|-----------|--------|
| Difference | Statistic | Value |
| A - B | n | 28 |
| | Mean | 0.723 |
| | Median | 0.367 |
| | SD | 1.339 |
| Wilcoxon | S | 116.5 |
| Signed-rank Test | p-value | 0.0015 |
| C - B | n | 9 |
| | Mean | 1.276 |
| | Median | 1.017 |
| | SD | 1.320 |
| Wilcoxon | S | 16 |
| Signed-rank Test | p-value | 0.0234 |

n: Number of subjects; SD: Standard Deviation.

Treatment A: Diazepam Buccal Film under fed conditions (breakfast with moderate fat content);

Treatment B: Diastat® AcuDial<sup>TM</sup> rectal gel under fed conditions (breakfast with moderate fat content);

Treatment C: Diazepam Buccal Film under fed conditions (breakfast with high fat content).

Listing 16.1.9-4 Wilcoxon Signed-Rank Test for  $T_{\text{max}}$  for Treatment Comparison of Nordiazepam – PK Population

Listing 16.1.9-4 Wilcoxon Signed-Rank Test for T<sub>max</sub> for Treatment Comparison of Nordiazepam - PK Population

| Difference | Statistic | Value |
|------------------|-----------|---------|
| A - B | n | 28 |
| | Mean | 6.968 |
| | Median | 0.192 |
| | SD | 48.359 |
| Wilcoxon | S | 36 |
| Signed-rank Test | p-value | 0.4223 |
| C - B | n | 9 |
| | Mean | -18.539 |
| | Median | -23.083 |
| | SD | 47.751 |
| Wilcoxon | S | -7.5 |
| Signed-rank Test | p-value | 0.4258 |

n: Number of subjects; SD: Standard Deviation.

Treatment A: Diazepam Buccal Film under fed conditions (breakfast with moderate fat content);

Treatment B: Diastat® AcuDial<sup>TM</sup> rectal gel under fed conditions (breakfast with moderate fat content);

Treatment C: Diazepam Buccal Film under fed conditions (breakfast with high fat content).

Listing 16.1.9-5 ANOVA for Treatment Comparison of Diazepam for Weight Group 51-62 kg - PK Population

## Listing 16.1.9-5 ANOVA for Treatment Comparison of Diazepam for Weight Group 51-62 kg - PK Population

Comparison: A vs B

Dependent Variable: AUC<sub>0-t</sub> (h\*ng/mL) Weight Group: 51-62

#### The GLM Procedure

| Class Level In | Class Level Information | |
|---|---|---|
| Class | Levels | Values |
| subject | 6 | 101 201 302 412 414 503 |
| sequence | 2 | AB BA |
| period | 2 | 1 2 |
| trt | 2 | AΒ |
| Number of Observations Read | | |
| Number of Ob | Number of Observations Used | |

## Listing 16.1.9-5 ANOVA for Treatment Comparison of Diazepam for Weight Group $51\text{-}62~\mathrm{kg}$ - PK Population

Comparison: A vs B

Dependent Variable: AUC<sub>0-t</sub> (h\*ng/mL) Weight Group: 51-62

#### The GLM Procedure

Dependent Variable: LN\_AUCLST

| R-Square | Coeff Var | Root MSE | | LN_AUC | LST Mean |
|---|---|---|---|---|---|
| 0.989131 | 1.149609 | 0.104716 | 9.108814 | | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.87353230 | 0.87353230 | 79.66 | 0.0009 |
| period | 1 | 0.02943586 | 0.02943586 | 2.68 | 0.1767 |
| trt | 1 | 0.00942171 | 0.00942171 | 0.86 | 0.4064 |
| subject(sequence | e) 4 | 3.07934290 | 0.76983573 | 70.21 | 0.0006 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.87353230 | 0.87353230 | 79.66 | 0.0009 |
| period | 1 | 0.03767939 | 0.03767939 | 3.44 | 0.1374 |
| trt | 1 | 0.00942171 | 0.00942171 | 0.86 | 0.4064 |
| subject(sequence | e) 4 | 3.07934290 | 0.76983573 | 70.21 | 0.0006 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.87353230 | 0.87353230 | 79.66 | 0.0009 |
| period | 1 | 0.03767939 | 0.03767939 | 3.44 | 0.1374 |
| trt | 1 | 0.00942171 | 0.00942171 | 0.86 | 0.4064 |
| subject(sequence | e) 4 | 3.07934290 | 0.76983573 | 70.21 | 0.0006 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.87353230 | 0.87353230 | 79.66 | 0.0009 |
| period | 1 | 0.03767939 | 0.03767939 | 3.44 | 0.1374 |
| trt | 1 | 0.00942171 | 0.00942171 | 0.86 | 0.4064 |
| subject(sequence | e) 4 | 3.07934290 | 0.76983573 | 70.21 | 0.0006 |

## Listing 16.1.9-5 ANOVA for Treatment Comparison of Diazepam for Weight Group 51-62 kg - PK Population

Comparison: A vs B

Dependent Variable: AUC<sub>0-t</sub> (h\*ng/mL) Weight Group: 51-62

## The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_AUCLST

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.873532 | 0.873532 | 1.13 | 0.3468 |
| Error | 4 | 3.079343 | 0.769836 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| *period | 1 | 0.029436 | 0.029436 | 2.68 | 0.1767 |
| trt | 1 | 0.009422 | 0.009422 | 0.86 | 0.4064 |
| subject(sequence) | 4 | 3.079343 | 0.769836 | 70.21 | 0.0006 |
| Error: MS(Error) | 4 | 0.043862 | 0.010965 | | |
| * This test assumes one or m | ore ot | her fixed effects | are zero. | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_AUCLST

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.873532 | 0.873532 | 1.13 | 0.3468 |
| Error | 4 | 3.079343 | 0.769836 | | _ |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.037679 | 0.037679 | 3.44 | 0.1374 |
| trt | 1 | 0.009422 | 0.009422 | 0.86 | 0.4064 |
| subject(sequence) | 4 | 3.079343 | 0.769836 | 70.21 | 0.0006 |
| Error: MS(Error) | 4 | 0.043862 | 0.010965 | | |

## Listing 16.1.9-5 ANOVA for Treatment Comparison of Diazepam for Weight Group 51-62 kg - PK Population

Comparison: A vs B

Dependent Variable: AUC<sub>0-t</sub> (h\*ng/mL) Weight Group: 51-62

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_AUCLST

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.873532 | 0.873532 | 1.13 | 0.3468 |
| Error | 4 | 3.079343 | 0.769836 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 0.037679 | 0.037679 | 3.44 | 0.1374 |
| trt | 1 | 0.009422 | 0.009422 | 0.86 | 0.4064 |
| subject(sequence) | 4 | 3.079343 | 0.769836 | 70.21 | 0.0006 |
| Error: MS(Error) | 4 | 0.043862 | 0.010965 | | - |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_AUCLST

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.873532 | 0.873532 | 1.13 | 0.3468 |
| Error | 4 | 3.079343 | 0.769836 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.037679 | 0.037679 | 3.44 | 0.1374 |
| trt | 1 | 0.009422 | 0.009422 | 0.86 | 0.4064 |
| subject(sequence) | 4 | 3.079343 | 0.769836 | 70.21 | 0.0006 |
| Error: MS(Error) | 4 | 0.043862 | 0.010965 | | |
Comparison: A vs B

Dependent Variable: AUC<sub>0-t</sub> (h\*ng/mL) Weight Group: 51-62

#### Least Squares Means

| | | H0:LSMean1=LSMean2 | |
|-----|------------------|--------------------|---------|
| trt | LN_AUCLST LSMEAN | | Pr > t |
| A | 9.23392481 | | 0.4064 |
| В | 9.17448459 | | |

| trt | LN_AUCLST LSMEAN | 90% Confidence Limits | |
|-----|------------------|-----------------------|----------|
| A | 9.233925 | 9.137260 | 9.330590 |
| В | 9.174485 | 9.077820 | 9.271149 |

| Le | Least Squares Means for Effect trt | | | |
|---|---|---|---|---|
| Difference Between | | | | |
| i | j | Means | 90% Confide | ence Limits for LSMean(i)-LSMean(j) |
| 1 | 2 | 0.059440 | -0.077265 | 0.196145 |

Dependent Variable: LN\_AUCLST

| | | Standard | | | |
|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confidence Limits |
| A - B | 0.05944022 | 0.06412503 | 0.93 | 0.4064-0 | 0.07726452 0.19614497 |

Comparison: A vs B

Dependent Variable: AUC<sub>0-inf</sub> (h\*ng/mL) Weight Group: 51-62

#### The GLM Procedure

| Class Level In | nformation | |
|---|---|---|
| Class | Levels | Values |
| subject | 6 | 101 201 302 412 414 503 |
| sequence | 2 | AB BA |
| period | 2 | 1 2 |
| trt | 2 | AΒ |
| Number of Observations Read 12 | | |
| Number of Ob | Number of Observations Used 12 | |

Comparison: A vs B

Dependent Variable: AUC<sub>0-inf</sub> (h\*ng/mL) Weight Group: 51-62

#### The GLM Procedure

| R-Square | Coeff Var | Root MSE | | LN_AUC | IFO Mean |
|---|---|---|---|---|---|
| 0.995963 | 0.748004 | 0.068472 | 9.154019 | | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 1.05980441 | 1.05980441 | 226.04 | 0.0001 |
| period | 1 | 0.04650127 | 0.04650127 | 9.92 | 0.0345 |
| trt | 1 | 0.02448664 | 0.02448664 | 5.22 | 0.0843 |
| subject(sequence | e) 4 | 3.49588930 | 0.87397232 | 186.41 | <.0001 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 1.05980441 | 1.05980441 | 226.04 | 0.0001 |
| period | 1 | 0.06526465 | 0.06526465 | 13.92 | 0.0203 |
| trt | 1 | 0.02448664 | 0.02448664 | 5.22 | 0.0843 |
| subject(sequence | e) 4 | 3.49588930 | 0.87397232 | 186.41 | <.0001 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 1.05980441 | 1.05980441 | 226.04 | 0.0001 |
| period | 1 | 0.06526465 | 0.06526465 | 13.92 | 0.0203 |
| trt | 1 | 0.02448664 | 0.02448664 | 5.22 | 0.0843 |
| subject(sequence | e) 4 | 3.49588930 | 0.87397232 | 186.41 | <.0001 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 1.05980441 | 1.05980441 | 226.04 | 0.0001 |
| period | 1 | 0.06526465 | 0.06526465 | 13.92 | 0.0203 |
| trt | 1 | 0.02448664 | 0.02448664 | 5.22 | 0.0843 |
| subject(sequence | e) 4 | 3.49588930 | 0.87397232 | 186.41 | <.0001 |

Comparison: A vs B

Dependent Variable: AUC<sub>0-inf</sub> (h\*ng/mL) Weight Group: 51-62

# The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN AUCIFO

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 1.059804 | 1.059804 | 1.21 | 0.3326 |
| Error | 4 | 3.495889 | 0.873972 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| *period | 1 | 0.046501 | 0.046501 | 9.92 | 0.0345 |
| trt | 1 | 0.024487 | 0.024487 | 5.22 | 0.0843 |
| subject(sequence) | 4 | 3.495889 | 0.873972 | 186.41 | <.0001 |
| Error: MS(Error) 4 0.018754 0.004688 | | | | | |
| * This test assumes one or more other fixed effects are zero. | | | | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 1.059804 | 1.059804 | 1.21 | 0.3326 |
| Error | 4 | 3.495889 | 0.873972 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.065265 | 0.065265 | 13.92 | 0.0203 |
| trt | 1 | 0.024487 | 0.024487 | 5.22 | 0.0843 |
| subject(sequence) | 4 | 3.495889 | 0.873972 | 186.41 | <.0001 |
| Error: MS(Error) | 4 | 0.018754 | 0.004688 | | |

Comparison: A vs B

Dependent Variable: AUC<sub>0-inf</sub> (h\*ng/mL) Weight Group: 51-62

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_AUCIFO

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 1.059804 | 1.059804 | 1.21 | 0.3326 |
| Error | 4 | 3.495889 | 0.873972 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 0.065265 | 0.065265 | 13.92 | 0.0203 |
| trt | 1 | 0.024487 | 0.024487 | 5.22 | 0.0843 |
| subject(sequence) | 4 | 3.495889 | 0.873972 | 186.41 | <.0001 |
| Error: MS(Error) | 4 | 0.018754 | 0.004688 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 1.059804 | 1.059804 | 1.21 | 0.3326 |
| Error | 4 | 3.495889 | 0.873972 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.065265 | 0.065265 | 13.92 | 0.0203 |
| trt | 1 | 0.024487 | 0.024487 | 5.22 | 0.0843 |
| subject(sequence) | 4 | 3.495889 | 0.873972 | 186.41 | <.0001 |
| Error: MS(Error) | 4 | 0.018754 | 0.004688 | | |

Comparison: A vs B

Dependent Variable: AUC<sub>0-inf</sub> (h\*ng/mL) Weight Group: 51-62

#### Least Squares Means

| - | | H0:LSMean1=LSMean2 | |
|-----|------------------|--------------------|---------|
| trt | LN_AUCIFO LSMEAN | | Pr > t |
| A | 9.30700089 | | 0.0843 |
| В | 9.21117558 | | |

| trt | LN_AUCIFO LSMEAN | 90% Confidence Limits | |
|-----|------------------|-----------------------|----------|
| A | 9.307001 | 9.243793 | 9.370209 |
| В | 9.211176 | 9.147968 | 9.274384 |

| Le | Least Squares Means for Effect trt | | | |
|---|---|---|---|---|
| | | Difference Between | | |
| i | j | Means | 90% Confider | nce Limits for LSMean(i)-LSMean(j) |
| 1 | 2 | 0.095825 | 0.006436 | 0.185215 |

| | | Standard | | | |
|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confidence Limits |
| A - B | 0.09582531 | 0.04193065 | 2.29 | 0.08430 | .00643560 0.18521503 |

Comparison: A vs B

Dependent Variable: C<sub>max</sub> (ng/mL) Weight Group: 51-62

#### The GLM Procedure

| Class Level In | formation | |
|---|---|---|
| Class | Levels | Values |
| subject | 6 | 101 201 302 412 414 503 |
| sequence | 2 | AB BA |
| period | 2 | 1 2 |
| trt | 2 | AΒ |
| Number of Observations Read 12 | | |
| Number of Ob | Number of Observations Used 12 | |

Comparison: A vs B

Dependent Variable:  $C_{max}$  (ng/mL) Weight Group: 51-62

#### The GLM Procedure

| R-Square | Coeff Var | Root MSE | | LN_CM | IAX Mean |
|---|---|---|---|---|---|
| 0.825032 | 4.588682 | 0.263298 | 5.737989 | | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.04000138 | 0.04000138 | 0.58 | 0.4898 |
| period | 1 | 0.20877172 | 0.20877172 | 3.01 | 0.1577 |
| trt | 1 | 0.28386147 | 0.28386147 | 4.09 | 0.1130 |
| subject(sequence | e) 4 | 0.77494679 | 0.19373670 | 2.79 | 0.1717 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.04000138 | 0.04000138 | 0.58 | 0.4898 |
| period | 1 | 0.06410442 | 0.06410442 | 0.92 | 0.3907 |
| trt | 1 | 0.28386147 | 0.28386147 | 4.09 | 0.1130 |
| subject(sequence | e) 4 | 0.77494679 | 0.19373670 | 2.79 | 0.1717 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.04000138 | 0.04000138 | 0.58 | 0.4898 |
| period | 1 | 0.06410442 | 0.06410442 | 0.92 | 0.3907 |
| trt | 1 | 0.28386147 | 0.28386147 | 4.09 | 0.1130 |
| subject(sequence | e) 4 | 0.77494679 | 0.19373670 | 2.79 | 0.1717 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.04000138 | 0.04000138 | 0.58 | 0.4898 |
| period | 1 | 0.06410442 | 0.06410442 | 0.92 | 0.3907 |
| trt | 1 | 0.28386147 | 0.28386147 | 4.09 | 0.1130 |
| subject(sequence | e) 4 | 0.77494679 | 0.19373670 | 2.79 | 0.1717 |

Comparison: A vs B

Dependent Variable: C<sub>max</sub> (ng/mL) Weight Group: 51-62

# The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_CMAX

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.040001 | 0.040001 | 0.21 | 0.6731 |
| Error | 4 | | | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| *period | 1 | 0.208772 | 0.208772 | 3.01 | 0.1577 |
| trt | 1 | 0.283861 | 0.283861 | 4.09 | 0.1130 |
| subject(sequence) | 4 | 0.774947 | 0.193737 | 2.79 | 0.1717 |
| Error: MS(Error) | 4 | 0.277304 | 0.069326 | | |
| * This test assumes one or m | ore oth | er fixed effects | are zero. | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.040001 | 0.040001 | 0.21 | 0.6731 |
| Error | 4 | 0.774947 | 0.193737 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.064104 | 0.064104 | 0.92 | 0.3907 |
| trt | 1 | 0.283861 | 0.283861 | 4.09 | 0.1130 |
| subject(sequence) | 4 | 0.774947 | 0.193737 | 2.79 | 0.1717 |
| Error: MS(Error) | 4 | 0.277304 | 0.069326 | | |

Comparison: A vs B

Dependent Variable: C<sub>max</sub> (ng/mL) Weight Group: 51-62

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_CMAX

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.040001 | 0.040001 | 0.21 | 0.6731 |
| Error | 4 | 0.774947 | 0.193737 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 0.064104 | 0.064104 | 0.92 | 0.3907 |
| trt | 1 | 0.283861 | 0.283861 | 4.09 | 0.1130 |
| subject(sequence) | 4 | 0.774947 | 0.193737 | 2.79 | 0.1717 |
| Error: MS(Error) | 4 | 0.277304 | 0.069326 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.040001 | 0.040001 | 0.21 | 0.6731 |
| Error | 4 | 0.774947 | 0.193737 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.064104 | 0.064104 | 0.92 | 0.3907 |
| trt | 1 | 0.283861 | 0.283861 | 4.09 | 0.1130 |
| subject(sequence) | 4 | 0.774947 | 0.193737 | 2.79 | 0.1717 |
| Error: MS(Error) | 4 | 0.277304 | 0.069326 | | |

Comparison: A vs B

Dependent Variable: C<sub>max</sub> (ng/mL) Weight Group: 51-62

-0.326264

#### Least Squares Means

| | | H0:LSMean1=LSMean2 | | |
|---|---|---|---|---|
| trt | LN_CMAX LSMEAN | | | Pr > t |
| A | 5.55444448 | | | 0.1130 |
| В | 5.88070825 | | | |
| trt | LN_CMAX LSMEAN | 90% | 6 Confidence Limits | |
| A | 5.554444 | 5.311390 | 5.797499 | |
| В | 5.880708 | 5.637653 | 6.123763 | |
| Lea | ast Squares Means for Effect | trt | | |
| | Difference Between | | | |
| i | j Means | 90% Confidence Li | mits for LSMean(i)-LS | Mean(j) |

#### Dependent Variable: LN\_CMAX

0.017468

-0.669995

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confid | dence Limits |
| A - B | -0.32626377 | 0.16123650 | -2.02 | 0.1130-0 | ).66999529 | 0.01746774 |

Comparison: A vs B

Dependent Variable: Cl/F/kg ((L/h)/kg) Weight Group: 51-62

#### The GLM Procedure

| Class Level In | nformation | |
|---|---|---|
| Class | Levels | Values |
| subject | 6 | 101 201 302 412 414 503 |
| sequence | 2 | AB BA |
| period | 2 | 1 2 |
| trt | 2 | AΒ |
| Number of Ob | Number of Observations Read 12 | |
| Number of Ob | Number of Observations Used 12 | |

Comparison: A vs B

Dependent Variable: Cl/F/kg ((L/h)/kg) Weight Group: 51-62

#### The GLM Procedure

| R-Square | Coeff Var | Root MSE | | LN_CLF | OW Mean |
|------------------|-----------|-------------|-------------|---------|---------|
| 0.995684 | -1.805055 | 0.068472 | -3.793372 | | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.82529228 | 0.82529228 | 176.03 | 0.0002 |
| period | 1 | 0.04650127 | 0.04650127 | 9.92 | 0.0345 |
| trt | 1 | 0.02448664 | 0.02448664 | 5.22 | 0.0843 |
| subject(sequence | e) 4 | 3.42986729 | 0.85746682 | 182.89 | <.0001 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.82529228 | 0.82529228 | 176.03 | 0.0002 |
| period | 1 | 0.06526465 | 0.06526465 | 13.92 | 0.0203 |
| trt | 1 | 0.02448664 | 0.02448664 | 5.22 | 0.0843 |
| subject(sequence | e) 4 | 3.42986729 | 0.85746682 | 182.89 | <.0001 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.82529228 | 0.82529228 | 176.03 | 0.0002 |
| period | 1 | 0.06526465 | 0.06526465 | 13.92 | 0.0203 |
| trt | 1 | 0.02448664 | 0.02448664 | 5.22 | 0.0843 |
| subject(sequence | e) 4 | 3.42986729 | 0.85746682 | 182.89 | <.0001 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.82529228 | 0.82529228 | 176.03 | 0.0002 |
| period | 1 | 0.06526465 | 0.06526465 | 13.92 | 0.0203 |
| trt | 1 | 0.02448664 | 0.02448664 | 5.22 | 0.0843 |
| subject(sequence | e) 4 | 3.42986729 | 0.85746682 | 182.89 | <.0001 |

Comparison: A vs B

Dependent Variable: Cl/F/kg ((L/h)/kg) Weight Group: 51-62

# The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_CLFOW

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.825292 | 0.825292 | 0.96 | 0.3821 |
| Error | 4 | 3.429867 | 0.857467 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| *period | 1 | 0.046501 | 0.046501 | 9.92 | 0.0345 |
| trt | 1 | 0.024487 | 0.024487 | 5.22 | 0.0843 |
| subject(sequence) | 4 | 3.429867 | 0.857467 | 182.89 | <.0001 |
| Error: MS(Error) | 4 | 0.018754 | 0.004688 | | |
| * This test assumes one or more other fixed effects are zero. | | | | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.825292 | 0.825292 | 0.96 | 0.3821 |
| Error | 4 | 3.429867 | 0.857467 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.065265 | 0.065265 | 13.92 | 0.0203 |
| trt | 1 | 0.024487 | 0.024487 | 5.22 | 0.0843 |
| subject(sequence) | 4 | 3.429867 | 0.857467 | 182.89 | <.0001 |
| Error: MS(Error) | 4 | 0.018754 | 0.004688 | | |

Comparison: A vs B

Dependent Variable: Cl/F/kg ((L/h)/kg) Weight Group: 51-62

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_CLFOW

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.825292 | 0.825292 | 0.96 | 0.3821 |
| Error | 4 | 3.429867 | 0.857467 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 0.065265 | 0.065265 | 13.92 | 0.0203 |
| trt | 1 | 0.024487 | 0.024487 | 5.22 | 0.0843 |
| subject(sequence) | 4 | 3.429867 | 0.857467 | 182.89 | <.0001 |
| Error: MS(Error) | 4 | 0.018754 | 0.004688 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.825292 | 0.825292 | 0.96 | 0.3821 |
| Error | 4 | 3.429867 | 0.857467 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.065265 | 0.065265 | 13.92 | 0.0203 |
| trt | 1 | 0.024487 | 0.024487 | 5.22 | 0.0843 |
| subject(sequence) | 4 | 3.429867 | 0.857467 | 182.89 | <.0001 |
| Error: MS(Error) | 4 | 0.018754 | 0.004688 | | |

Comparison: A vs B

Dependent Variable: Cl/F/kg ((L/h)/kg) Weight Group: 51-62

-0.095825

#### Least Squares Means

| | | H0:LS | Mean1=LSMean2 | |
|---|---|---|---|---|
| trt | LN_CLFOW LSMEAN | | | Pr > t |
| A | -3.93400394 | | | 0.0843 |
| В | -3.83817863 | | | |
| trt | LN_CLFOW LSMEAN | 90% | Confidence Limits | |
| A | -3.934004 | -3.997212 | -3.870796 | |
| В | -3.838179 | -3.901387 | -3.774971 | |
| Lea | st Squares Means for Effect | trt | | |
| | Difference Between | | | |
| i | j Means | 90% Confidence Lin | mits for LSMean(i)-LS | Mean(j) |

#### Dependent Variable: LN\_CLFOW

-0.006436

-0.185215

| | | Standard | | | |
|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confidence Limits |
| A - B | -0.09582531 | 0.04193065 | -2.29 | 0.0843-0 | .18521503 -0.00643560 |

Comparison: A vs B

Dependent Variable: Cl/F (L/h) Weight Group: 51-62

#### The GLM Procedure

| Class Level In | nformation | |
|---|---|---|
| Class | Levels | Values |
| subject | 6 | 101 201 302 412 414 503 |
| sequence | 2 | AB BA |
| period | 2 | 1 2 |
| trt | 2 | AΒ |
| Number of Ob | Number of Observations Read 12 | |
| Number of Ob | Number of Observations Used 12 | |

Comparison: A vs B

Dependent Variable: Cl/F (L/h) Weight Group: 51-62

#### The GLM Procedure

| R-Square | Coeff Var | Root MSE | • | LN_ | CLFO Mean |
|---|---|---|---|---|---|
| 0.995963 | 24.50124 | 0.068472 | 0.279465 | | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 1.05980441 | 1.05980441 | 226.04 | 0.0001 |
| period | 1 | 0.04650127 | 0.04650127 | 9.92 | 0.0345 |
| trt | 1 | 0.02448664 | 0.02448664 | 5.22 | 0.0843 |
| subject(sequence | ) 4 | 3.49588930 | 0.87397232 | 186.41 | <.0001 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 1.05980441 | 1.05980441 | 226.04 | 0.0001 |
| period | 1 | 0.06526465 | 0.06526465 | 13.92 | 0.0203 |
| trt | 1 | 0.02448664 | 0.02448664 | 5.22 | 0.0843 |
| subject(sequence | ) 4 | 3.49588930 | 0.87397232 | 186.41 | <.0001 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 1.05980441 | 1.05980441 | 226.04 | 0.0001 |
| period | 1 | 0.06526465 | 0.06526465 | 13.92 | 0.0203 |
| trt | 1 | 0.02448664 | 0.02448664 | 5.22 | 0.0843 |
| subject(sequence | ) 4 | 3.49588930 | 0.87397232 | 186.41 | <.0001 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 1.05980441 | 1.05980441 | 226.04 | 0.0001 |
| period | 1 | 0.06526465 | 0.06526465 | 13.92 | 0.0203 |
| trt | 1 | 0.02448664 | 0.02448664 | 5.22 | 0.0843 |
| subject(sequence | ) 4 | 3.49588930 | 0.87397232 | 186.41 | <.0001 |

Comparison: A vs B

Dependent Variable: Cl/F (L/h) Weight Group: 51-62

# The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN CLFO

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 1.059804 | 1.059804 | 1.21 | 0.3326 |
| Error | 4 | 3.495889 | 0.873972 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| *period | 1 | 0.046501 | 0.046501 | 9.92 | 0.0345 |
| trt | 1 | 0.024487 | 0.024487 | 5.22 | 0.0843 |
| subject(sequence) | 4 | 3.495889 | 0.873972 | 186.41 | <.0001 |
| Error: MS(Error) 4 0.018754 0.004688 | | | | | |
| * This test assumes one or more other fixed effects are zero. | | | | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 1.059804 | 1.059804 | 1.21 | 0.3326 |
| Error | 4 | 3.495889 | 0.873972 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.065265 | 0.065265 | 13.92 | 0.0203 |
| trt | 1 | 0.024487 | 0.024487 | 5.22 | 0.0843 |
| subject(sequence) | 4 | 3.495889 | 0.873972 | 186.41 | <.0001 |
| Error: MS(Error) | 4 | 0.018754 | 0.004688 | | |

Comparison: A vs B

Dependent Variable: Cl/F (L/h) Weight Group: 51-62

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_CLFO

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 1.059804 | 1.059804 | 1.21 | 0.3326 |
| Error | 4 | 3.495889 | 0.873972 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 0.065265 | 0.065265 | 13.92 | 0.0203 |
| trt | 1 | 0.024487 | 0.024487 | 5.22 | 0.0843 |
| subject(sequence) | 4 | 3.495889 | 0.873972 | 186.41 | <.0001 |
| Error: MS(Error) | 4 | 0.018754 | 0.004688 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 1.059804 | 1.059804 | 1.21 | 0.3326 |
| Error | 4 | 3.495889 | 0.873972 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.065265 | 0.065265 | 13.92 | 0.0203 |
| trt | 1 | 0.024487 | 0.024487 | 5.22 | 0.0843 |
| subject(sequence) | 4 | 3.495889 | 0.873972 | 186.41 | <.0001 |
| Error: MS(Error) | 4 | 0.018754 | 0.004688 | | |

Comparison: A vs B

Dependent Variable: Cl/F (L/h) Weight Group: 51-62

#### Least Squares Means

| | | H0:LSMean1=LSMean2 | |
|-----|----------------|--------------------|---------|
| trt | LN_CLFO LSMEAN | | Pr > t |
| A | 0.12648303 | | 0.0843 |
| В | 0.22230834 | | |

| trt | LN_CLFO LSMEAN | | 90% Confidence Limits |
|-----|----------------|----------|-----------------------|
| A | 0.126483 | 0.063275 | 0.189691 |
| В | 0.222308 | 0.159100 | 0.285516 |

| Le | ast S | Squares Means for Effec | t trt | |
|---|---|---|---|---|
| | | Difference Between | | |
| i | j | Means | 90% Confide | ence Limits for LSMean(i)-LSMean(j) |
| 1 | 2 | -0.095825 | -0.185215 | -0.006436 |

| | | Standard | | | |
|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confidence Limits |
| A - B | -0.09582531 | 0.04193065 | -2.29 | 0.0843-0 | .18521503 -0.00643560 |

Comparison: A vs B

Dependent Variable: V<sub>d</sub>/F/kg (L/kg) Weight Group: 51-62

#### The GLM Procedure

| Class Level In | formation | |
|---|---|---|
| Class | Levels | Values |
| subject | 6 | 101 201 302 412 414 503 |
| sequence | 2 | AB BA |
| period | 2 | 1 2 |
| trt | 2 | AΒ |
| Number of Observations Read 12 | | |
| Number of Ob | Number of Observations Used 12 | |

Comparison: A vs B

Dependent Variable: V<sub>d</sub>/F/kg (L/kg) Weight Group: 51-62

#### The GLM Procedure

| R-Square | Coeff Var | Root MSE | | LN_VZF | OW Mean |
|------------------|-----------|-------------|-------------|---------|---------|
| 0.850422 | 149.0144 | 0.249852 | 0.167670 | | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.06679525 | 0.06679525 | 1.07 | 0.3594 |
| period | 1 | 0.00364857 | 0.00364857 | 0.06 | 0.8209 |
| trt | 1 | 0.00056004 | 0.00056004 | 0.01 | 0.9291 |
| subject(sequence | e) 4 | 1.34868165 | 0.33717041 | 5.40 | 0.0656 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.06679525 | 0.06679525 | 1.07 | 0.3594 |
| period | 1 | 0.00420387 | 0.00420387 | 0.07 | 0.8081 |
| trt | 1 | 0.00056004 | 0.00056004 | 0.01 | 0.9291 |
| subject(sequence | e) 4 | 1.34868165 | 0.33717041 | 5.40 | 0.0656 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.06679525 | 0.06679525 | 1.07 | 0.3594 |
| period | 1 | 0.00420387 | 0.00420387 | 0.07 | 0.8081 |
| trt | 1 | 0.00056004 | 0.00056004 | 0.01 | 0.9291 |
| subject(sequence | e) 4 | 1.34868165 | 0.33717041 | 5.40 | 0.0656 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.06679525 | 0.06679525 | 1.07 | 0.3594 |
| period | 1 | 0.00420387 | 0.00420387 | 0.07 | 0.8081 |
| trt | 1 | 0.00056004 | 0.00056004 | 0.01 | 0.9291 |
| subject(sequence | e) 4 | 1.34868165 | 0.33717041 | 5.40 | 0.0656 |

Comparison: A vs B

Dependent Variable: V<sub>d</sub>/F/kg (L/kg) Weight Group: 51-62

# The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN VZFOW

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.066795 | 0.066795 | 0.20 | 0.6793 |
| Error | 4 | 1.348682 | 0.337170 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| *period | 1 | 0.003649 | 0.003649 | 0.06 | 0.8209 |
| trt | 1 | 0.000560 | 0.000560 | 0.01 | 0.9291 |
| subject(sequence) | 4 | 1.348682 | 0.337170 | 5.40 | 0.0656 |
| Error: MS(Error) | 4 | 0.249704 | 0.062426 | | |
| * This test assumes one or more other fixed effects are zero. | | | | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.066795 | 0.066795 | 0.20 | 0.6793 |
| Error | | | | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.004204 | 0.004204 | 0.07 | 0.8081 |
| trt | 1 | 0.000560 | 0.000560 | 0.01 | 0.9291 |
| subject(sequence) | 4 | 1.348682 | 0.337170 | 5.40 | 0.0656 |
| Error: MS(Error) | 4 | 0.249704 | 0.062426 | | |

Comparison: A vs B

Dependent Variable: V<sub>d</sub>/F/kg (L/kg) Weight Group: 51-62

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_VZFOW

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.066795 | 0.066795 | 0.20 | 0.6793 |
| Error | 4 | 1.348682 | 0.337170 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 0.004204 | 0.004204 | 0.07 | 0.8081 |
| trt | 1 | 0.000560 | 0.000560 | 0.01 | 0.9291 |
| subject(sequence) | 4 | 1.348682 | 0.337170 | 5.40 | 0.0656 |
| Error: MS(Error) | 4 | 0.249704 | 0.062426 | | - |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.066795 | 0.066795 | 0.20 | 0.6793 |
| Error | 4 | 1.348682 | 0.337170 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.004204 | 0.004204 | 0.07 | 0.8081 |
| trt | 1 | 0.000560 | 0.000560 | 0.01 | 0.9291 |
| subject(sequence) | 4 | 1.348682 | 0.337170 | 5.40 | 0.0656 |
| Error: MS(Error) | 4 | 0.249704 | 0.062426 | | |

Comparison: A vs B

Dependent Variable: V<sub>d</sub>/F/kg (L/kg) Weight Group: 51-62

#### Least Squares Means

| Pr > t |
|---------|
| 0.9291 |
| _ |

| trt | LN_VZFOW LSMEAN | 90% | Confidence Limits |
|-----|-----------------|-----------|-------------------|
| A | 0.201293 | -0.029349 | 0.431936 |
| В | 0.186802 | -0.043841 | 0.417444 |

| Le | Least Squares Means for Effect trt | | | |
|---|---|---|---|---|
| | | Difference Between | | |
| i | j | Means | 90% Confide | nce Limits for LSMean(i)-LSMean(j) |
| 1 | 2 | 0.014492 | -0.311686 | 0.340670 |

| • | | Standard | | | |
|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confidence Limits |
| A - B | 0.01449185 | 0.15300260 | 0.09 | 0.9291-0 | 0.31168624 |

Comparison: A vs B

Dependent Variable: V<sub>d</sub>/F (L) Weight Group: 51-62

#### The GLM Procedure

| Class Level In | nformation | |
|-----------------------------|------------|-------------------------|
| Class | Levels | Values |
| subject | 6 | 101 201 302 412 414 503 |
| sequence | 2 | AB BA |
| period | 2 | 1 2 |
| trt | 2 | AΒ |
| Number of Ob | 12 | |
| Number of Observations Used | | |

Comparison: A vs B

Dependent Variable: V<sub>d</sub>/F (L) Weight Group: 51-62

#### The GLM Procedure

| R-Square | Coeff Var | Root MSF | E | LN | VZFO Mean |
|---|---|---|---|---|---|
| 0.847614 | 5.892035 | 0.249852 | 4.240507 | | |
| <u></u> | DE | T. 100 | N. C | E 17.1 | D . D |
| Source | DF | Type I SS | Mean Square | F Value | |
| sequence | 1 | 0.01888858 | 0.01888858 | 0.30 | 0.6115 |
| period | 1 | 0.00364857 | 0.00364857 | 0.06 | 0.8209 |
| trt | 1 | 0.00056004 | 0.00056004 | 0.01 | 0.9291 |
| subject(sequence | 2) 4 | 1.36582781 | 0.34145695 | 5.47 | 0.0643 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| | 1 | 0.01888858 | 0.01888858 | 0.30 | 0.6115 |
| sequence | 1 | 0.01888838 | 0.01888838 | 0.30 | 0.8081 |
| period | _ | | | | |
| trt | 1 | 0.00056004 | 0.00056004 | 0.01 | 0.9291 |
| subject(sequence | e) 4 | 1.36582781 | 0.34145695 | 5.47 | 0.0643 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.01888858 | 0.01888858 | 0.30 | 0.6115 |
| period | 1 | 0.00420387 | 0.00420387 | 0.07 | 0.8081 |
| trt | 1 | 0.00056004 | 0.00056004 | 0.01 | 0.9291 |
| subject(sequence | e) 4 | 1.36582781 | 0.34145695 | 5.47 | 0.0643 |
| | , | | | | |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.01888858 | 0.01888858 | 0.30 | 0.6115 |
| period | 1 | 0.00420387 | 0.01888838 | 0.30 | 0.8081 |
| trt | 1 | 0.00056004 | 0.00056004 | 0.07 | 0.8081 |
| | _ | | | | |
| subject(sequence | <i>)</i> 4 | 1.36582781 | 0.34145695 | 5.47 | 0.0643 |

Comparison: A vs B

Dependent Variable: V<sub>d</sub>/F (L) Weight Group: 51-62

# The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_VZFO

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.018889 | 0.018889 | 0.06 | 0.8256 |
| Error | 4 | 1.365828 | 0.341457 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| *period | 1 | 0.003649 | 0.003649 | 0.06 | 0.8209 |
| trt | 1 | 0.000560 | 0.000560 | 0.01 | 0.9291 |
| subject(sequence) | 4 | 1.365828 | 0.341457 | 5.47 | 0.0643 |
| Error: MS(Error) 4 0.249704 0.062426 | | | | | |
| * This test assumes one or more other fixed effects are zero. | | | | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.018889 | 0.018889 | 0.06 | 0.8256 |
| Error 4 1.365828 | | | 0.341457 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.004204 | 0.004204 | 0.07 | 0.8081 |
| trt | 1 | 0.000560 | 0.000560 | 0.01 | 0.9291 |
| subject(sequence) | 4 | 1.365828 | 0.341457 | 5.47 | 0.0643 |
| Error: MS(Error) | 4 | 0.249704 | 0.062426 | | |

Comparison: A vs B

Dependent Variable: V<sub>d</sub>/F (L) Weight Group: 51-62

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_VZFO

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.018889 | 0.018889 | 0.06 | 0.8256 |
| Error | 4 | 1.365828 | 0.341457 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 0.004204 | 0.004204 | 0.07 | 0.8081 |
| trt | 1 | 0.000560 | 0.000560 | 0.01 | 0.9291 |
| subject(sequence) | 4 | 1.365828 | 0.341457 | 5.47 | 0.0643 |
| Error: MS(Error) | 4 | 0.249704 | 0.062426 | | - |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.018889 | 0.018889 | 0.06 | 0.8256 |
| Error | 4 | 1.365828 | 0.341457 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.004204 | 0.004204 | 0.07 | 0.8081 |
| trt | 1 | 0.000560 | 0.000560 | 0.01 | 0.9291 |
| subject(sequence) | 4 | 1.365828 | 0.341457 | 5.47 | 0.0643 |
| Error: MS(Error) | 4 | 0.249704 | 0.062426 | | |

Comparison: A vs B

Dependent Variable: V<sub>d</sub>/F (L) Weight Group: 51-62

#### Least Squares Means

| | | H0:LSMean1=LSMean2 | |
|-----|----------------|--------------------|---------|
| trt | LN_VZFO LSMEAN | | Pr > t |
| A | 4.26178039 | | 0.9291 |
| В | 4.24728854 | | |

| trt | LN_VZFO LSMEAN | | 90% Confidence Limits |
|-----|----------------|----------|-----------------------|
| A | 4.261780 | 4.031138 | 4.492423 |
| В | 4.247289 | 4.016646 | 4.477931 |

| Le | Least Squares Means for Effect trt | | | |
|---|---|---|---|---|
| | | Difference Between | | |
| i | j | Means | 90% Confider | nce Limits for LSMean(i)-LSMean(j) |
| 1 | 2 | 0.014492 | -0.311686 | 0.340670 |

| | | Standard | | | |
|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confidence Limits |
| A - B | 0.01449185 | 0.15300260 | 0.09 | 0.9291-0 | 0.31168624 |

Comparison: A vs B

Dependent Variable: T<sub>max</sub> (h) Weight Group: 51-62

#### The GLM Procedure

| Class Level In | formation | | |
|---|---|---|---|
| Class | Levels | Values | |
| subject | 6 | 101 201 302 412 414 503 | |
| sequence | 2 | AB BA | |
| period | 2 | 1 2 | |
| trt | 2 | AΒ | |
| Number of Observations Read 12 | | | |
| Number of Ob | servations Use | d | 12 |

Comparison: A vs B

Dependent Variable: T<sub>max</sub> (h) Weight Group: 51-62

#### The GLM Procedure

| R-Square | Coeff Var | Root | MSE | | TMAX Mean |
|---|---|---|---|---|---|
| 0.730498 | 75.37925 | 0.965 | 3357 | 1.280667 | |
| Source | DF | Type I SS | Mean Square | e F Value | e $Pr > F$ |
| sequence | 1 | 0.25317604 | 0.25317604 | 0.27 | 0.6297 |
| period | 1 | 1.54083333 | 1.54083333 | 1.65 | 0.2679 |
| trt | 1 | 3.84080004 | 3.84080004 | 4.12 | 0.1122 |
| subject(sequence) | 4 | 4.46918363 | 1.11729591 | 1.20 | 0.4323 |
| Source | DF | Type II SS | Mean Square | F Value | e $Pr > F$ |
| sequence | 1 | 0.25317604 | 0.25317604 | 0.27 | 0.6297 |
| period | 1 | 0.26733704 | 0.26733704 | 0.29 | 0.6206 |
| trt | 1 | 3.84080004 | 3.84080004 | 4.12 | 0.1122 |
| subject(sequence) | 4 | 4.46918363 | 1.11729591 | 1.20 | 0.4323 |
| Source | DF | Type III SS | Mean Square | F Value | e $Pr > F$ |
| sequence | 1 | 0.25317604 | 0.25317604 | 0.27 | 0.6297 |
| period | 1 | 0.26733704 | 0.26733704 | 0.29 | 0.6206 |
| trt | 1 | 3.84080004 | 3.84080004 | 4.12 | 0.1122 |
| subject(sequence) | 4 | 4.46918363 | 1.11729591 | 1.20 | 0.4323 |
| Source | DF | Type IV SS | Mean Square | e F Value | e Pr > F |
| sequence | 1 | 0.25317604 | 0.25317604 | 0.27 | 0.6297 |
| period | 1 | 0.26733704 | 0.26733704 | 0.29 | 0.6206 |
| trt | 1 | 3.84080004 | 3.84080004 | 4.12 | 0.1122 |
| subject(sequence) | 4 | 4.46918363 | 1.11729591 | 1.20 | 0.4323 |

Comparison: A vs B

Dependent Variable: T<sub>max</sub> (h) Weight Group: 51-62

# The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: TMAX

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.253176 | 0.253176 | 0.23 | 0.6589 |
| Error | 4 | 4.469184 | 1.117296 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| *period | 1 | 1.540833 | 1.540833 | 1.65 | 0.2679 |
| trt | 1 | 3.840800 | 3.840800 | 4.12 | 0.1122 |
| subject(sequence) | 4 | 4.469184 | 1.117296 | 1.20 | 0.4323 |
| Error: MS(Error) | 4 | 3.727656 | 0.931914 | | |
| * This test assumes one or m | ore oth | ner fixed effects | are zero. | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.253176 | 0.253176 | 0.23 | 0.6589 |
| Error | | | | | |
| Error: MS(s | Error: MS(subject(sequence)) | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.267337 | 0.267337 | 0.29 | 0.6206 |
| trt | 1 | 3.840800 | 3.840800 | 4.12 | 0.1122 |
| subject(sequence) | 4 | 4.469184 | 1.117296 | 1.20 | 0.4323 |
| Error: MS(Error) | 4 | 3.727656 | 0.931914 | | |

Comparison: A vs B

Dependent Variable: T<sub>max</sub> (h) Weight Group: 51-62

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: TMAX

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.253176 | 0.253176 | 0.23 | 0.6589 |
| Error | 4 | 4.469184 | 1.117296 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 0.267337 | 0.267337 | 0.29 | 0.6206 |
| trt | 1 | 3.840800 | 3.840800 | 4.12 | 0.1122 |
| subject(sequence) | 4 | 4.469184 | 1.117296 | 1.20 | 0.4323 |
| Error: MS(Error) | 4 | 3.727656 | 0.931914 | - | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.253176 | 0.253176 | 0.23 | 0.6589 |
| Error | 4 | 4.469184 | 1.117296 | | |
| Error: MS(s | Error: MS(subject(sequence)) | | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.267337 | 0.267337 | 0.29 | 0.6206 |
| trt | 1 | 3.840800 | 3.840800 | 4.12 | 0.1122 |
| subject(sequence) | 4 | 4.469184 | 1.117296 | 1.20 | 0.4323 |
| Error: MS(Error) | 4 | 3.727656 | 0.931914 | | |

Comparison: A vs B

Dependent Variable: T<sub>max</sub> (h) Weight Group: 51-62

#### Least Squares Means

| | | Н | I0:LSMean1=LSMean2 | |
|---|---|---|---|---|
| trt | TMAX LSMEAN | | Pı | r > t |
| A | 1.82937500 | | 0. | 1122 |
| В | 0.62925000 | | | |
| trt | TMAX LSMEAN | | 90% Confidence Limits | |
| A | 1.829375 | 0.93823 | 38 2.720512 | |
| В | 0.629250 | -0.2618 | 1.520387 | |
| Le | ast Squares Means for Effe | ct trt | | |
| | Difference Between | | | |
| i | j Means | 90% Confidence | Limits for LSMean(i)-LSMear | 1(j) |
| 1 | 2 1.200125 | -0.060133 | 2.460383 | |

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confi | dence Limits |
| A - B | 1.20012500 | 0.59115794 | 2.03 | 0.1122-0 | 0.06013316 | 2.46038316 |
Comparison: A vs B

Dependent Variable: K<sub>el</sub> (/h) Weight Group: 51-62

| Class Level In | Class Level Information | | |
|---|---|---|---|
| Class | Levels | Values | |
| subject | 6 | 101 201 302 412 414 503 | |
| sequence | 2 | AB BA | |
| period | 2 | 1 2 | |
| trt | 2 | AΒ | |
| Number of Observations Read 12 | | | |
| Number of Ob | servations Use | d | 12 |

Comparison: A vs B

Dependent Variable:  $K_{el}$  (/h) Weight Group: 51-62

### The GLM Procedure

| R-Square | Coeff Var | Root | MSE | I | LAMZ Mean |
|---|---|---|---|---|---|
| 0.984784 | 11.99520 | 0.002 | 2714 | 0.022627 | |
| | | | | | _ |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.00062156 | 0.00062156 | 84.37 | 0.0008 |
| period | 1 | 0.00002840 | 0.00002840 | 3.86 | 0.1211 |
| trt | 1 | 0.00000016 | 0.00000016 | 0.02 | 0.8885 |
| subject(sequence) | 4 | 0.00125697 | 0.00031424 | 42.66 | 0.0016 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.00062156 | 0.00062156 | 84.37 | 0.0008 |
| period | 1 | 0.00002391 | 0.00002391 | 3.25 | 0.1460 |
| trt | 1 | 0.00000016 | 0.00000016 | 0.02 | 0.8885 |
| subject(sequence) | 4 | 0.00125697 | 0.00031424 | 42.66 | 0.0016 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.00062156 | 0.00062156 | 84.37 | 0.0008 |
| period | 1 | 0.00002391 | 0.00002391 | 3.25 | 0.1460 |
| trt | 1 | 0.00000016 | 0.00000016 | 0.02 | 0.8885 |
| subject(sequence) | 4 | 0.00125697 | 0.00031424 | 42.66 | 0.0016 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.00062156 | 0.00062156 | 84.37 | 0.0008 |
| period | 1 | 0.00002391 | 0.00002391 | 3.25 | 0.1460 |
| trt | 1 | 0.00000016 | 0.00000016 | 0.02 | 0.8885 |
| subject(sequence) | 4 | 0.00125697 | 0.00031424 | 42.66 | 0.0016 |

Comparison: A vs B

Dependent Variable: K<sub>el</sub> (/h) Weight Group: 51-62

## The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LAMZ

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.000622 | 0.000622 | 1.98 | 0.2323 |
| Error | 4 | 0.001257 | 0.000314 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| *period | 1 | 0.000028401 | 0.000028401 | 3.86 | 0.1211 |
| trt | 1 | 0.000000164 | 0.000000164 | 0.02 | 0.8885 |
| subject(sequence) | 4 | 0.001257 | 0.000314 | 42.66 | 0.0016 |
| Error: MS(Error) 4 0.000029467 0.000007367 | | | | | |
| * This test assumes one or more other fixed effects are zero. | | | | | |

### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.000622 | 0.000622 | 1.98 | 0.2323 |
| Error | 4 | 0.001257 | 0.000314 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 0.000023907 | 0.000023907 | 3.25 | 0.1460 |
| trt | 1 | 0.000000164 | 0.000000164 | 0.02 | 0.8885 |
| subject(sequence) | 4 | 0.001257 | 0.000314 | 42.66 | 0.0016 |
| Error: MS(Error) | 4 | 0.000029467 | 0.000007367 | | |

Comparison: A vs B

Dependent Variable: K<sub>el</sub> (/h) Weight Group: 51-62

### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LAMZ

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.000622 | 0.000622 | 1.98 | 0.2323 |
| Error | 4 | 0.001257 | 0.000314 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 0.000023907 | 0.000023907 | 3.25 | 0.1460 |
| trt | 1 | 0.000000164 | 0.000000164 | 0.02 | 0.8885 |
| subject(sequence) | 4 | 0.001257 | 0.000314 | 42.66 | 0.0016 |
| Error: MS(Error) | 4 | 0.000029467 | 0.000007367 | | - |

### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.000622 | 0.000622 | 1.98 | 0.2323 |
| Error | 4 | 0.001257 | 0.000314 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 0.000023907 | 0.000023907 | 3.25 | 0.1460 |
| trt | 1 | 0.000000164 | 0.000000164 | 0.02 | 0.8885 |
| subject(sequence) | 4 | 0.001257 | 0.000314 | 42.66 | 0.0016 |
| Error: MS(Error) | 4 | 0.000029467 | 0.000007367 | | |

Comparison: A vs B

Dependent Variable: K<sub>el</sub> (/h) Weight Group: 51-62

0.000248

### Least Squares Means

| | | H0:LSMean1=LSMean2 | | |
|---|---|---|---|---|
| trt | LAMZ LSMEAN | | | Pr > t |
| A | 0.02020687 | | | 0.8885 |
| В | 0.01995872 | | | |
| trt | LAMZ LSMEAN | 90% ( | Confidence Limits | |
| A | 0.020207 | 0.017701 | 0.022712 | |
| В | 0.019959 | 0.017453 | 0.022464 | |
| _ | A DEC | | | |
| Lea | ast Squares Means for Effec | t trt | | |
| | Difference Between | | | |
| i | j Means | 90% Confidence Limits f | for LSMean(i)-LSM | Iean(j) |

### Dependent Variable: LAMZ

0.003791

-0.003295

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confid | dence Limits |
| A - B | 0.00024814 | 0.00166210 | 0.15 | 0.8885-0 | 0.00329519 | 0.00379148 |

Comparison: A vs B

Dependent Variable: T<sub>1/2 el</sub> (h) Weight Group: 51-62

| Class Level In | nformation | | |
|---|---|---|---|
| Class | Levels | Values | |
| subject | 6 | 101 201 302 412 414 503 | |
| sequence | 2 | AB BA | |
| period | 2 | 1 2 | |
| trt | 2 | AΒ | |
| Number of Ob | oservations Rea | d | 12 |
| Number of Ob | Number of Observations Used 12 | | |

Comparison: A vs B

Dependent Variable: T<sub>1/2 el</sub> (h) Weight Group: 51-62

### The GLM Procedure

| R-Square | Coeff Var | Root MSE | | LAMZ | ZHL Mean |
|---|---|---|---|---|---|
| 0.912041 | 30.75229 | 13.38035 | 43.5101 | 0 | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 2163.641142 | 2163.641142 | 12.09 | 0.0254 |
| period | 1 | 231.387288 | 231.387288 | 1.29 | 0.3191 |
| trt | 1 | 354.611103 | 354.611103 | 1.98 | 0.2321 |
| subject(sequence) | ) 4 | 4675.957475 | 1168.989369 | 6.53 | 0.0482 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 2163.641142 | 2163.641142 | 12.09 | 0.0254 |
| period | 1 | 425.122715 | 425.122715 | 2.37 | 0.1982 |
| trt | 1 | 354.611103 | 354.611103 | 1.98 | 0.2321 |
| subject(sequence) | ) 4 | 4675.957475 | 1168.989369 | 6.53 | 0.0482 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 2163.641142 | 2163.641142 | 12.09 | 0.0254 |
| period | 1 | 425.122715 | 425.122715 | 2.37 | 0.1982 |
| trt | 1 | 354.611103 | 354.611103 | 1.98 | 0.2321 |
| subject(sequence) | ) 4 | 4675.957475 | 1168.989369 | 6.53 | 0.0482 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 2163.641142 | 2163.641142 | 12.09 | 0.0254 |
| period | 1 | 425.122715 | 425.122715 | 2.37 | 0.1982 |
| trt | 1 | 354.611103 | 354.611103 | 1.98 | 0.2321 |
| subject(sequence) | ) 4 | 4675.957475 | 1168.989369 | 6.53 | 0.0482 |

Comparison: A vs B

Dependent Variable: T<sub>1/2 el</sub> (h) Weight Group: 51-62

### The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LAMZHL

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 2163.641142 | 2163.641142 | 1.85 | 0.2453 |
| Error | 4 | 4675.957475 | 1168.989369 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| *period | 1 | 231.387288 | 231.387288 | 1.29 | 0.3191 |
| trt | 1 | 354.611103 | 354.611103 | 1.98 | 0.2321 |
| subject(sequence) | 4 | 4675.957475 | 1168.989369 | 6.53 | 0.0482 |
| Error: MS(Error) | 4 | 716.135395 | 179.033849 | | |
| * This test assumes one or n | nore other | fixed effects a | re zero. | | |

### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 2163.641142 | 2163.641142 | 1.85 | 0.2453 |
| Error | 4 | 4675.957475 | 1168.989369 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 425.122715 | 425.122715 | 2.37 | 0.1982 |
| trt | 1 | 354.611103 | 354.611103 | 1.98 | 0.2321 |
| subject(sequence) | 4 | 4675.957475 | 1168.989369 | 6.53 | 0.0482 |
| Error: MS(Error) | 4 | 716.135395 | 179.033849 | | |

Comparison: A vs B

Dependent Variable: T<sub>1/2 el</sub> (h) Weight Group: 51-62

### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LAMZHL

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 2163.641142 | 2163.641142 | 1.85 | 0.2453 |
| Error | 4 | 4675.957475 | 1168.989369 | | _ |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|-------------|
| period | 1 | 425.122715 | 425.122715 | 2.37 | 0.1982 |
| trt | 1 | 354.611103 | 354.611103 | 1.98 | 0.2321 |
| subject(sequence) | 4 | 4675.957475 | 1168.989369 | 6.53 | 0.0482 |
| Error: MS(Error) | 4 | 716.135395 | 179.033849 | | <del></del> |

### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 2163.641142 | 2163.641142 | 1.85 | 0.2453 |
| Error | 4 | 4675.957475 | 1168.989369 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 425.122715 | 425.122715 | 2.37 | 0.1982 |
| trt | 1 | 354.611103 | 354.611103 | 1.98 | 0.2321 |
| subject(sequence) | 4 | 4675.957475 | 1168.989369 | 6.53 | 0.0482 |
| Error: MS(Error) | 4 | 716.135395 | 179.033849 | | |

Comparison: A vs B

Dependent Variable: T<sub>1/2 el</sub> (h) Weight Group: 51-62

11.531659

### Least Squares Means

| | | | H0:LSMean1=LSMean2 | |
|---|---|---|---|---|
| trt | LAMZHL LSMEAN | | | Pr > t |
| A | 54.0233424 | | | 0.2321 |
| В | 42.4916832 | | | |
| trt | LAMZHL LSMEAN | | 90% Confidence Limits | |
| A | 54.023342 | 41.671714 | 66.374970 | |
| В | 42.491683 | 30.140055 | 54.843311 | |
| Lea | ast Squares Means for Effe | ct trt | | |
| | Difference Between | | | |
| i | j Means | 90% Confide | ence Limits for LSMean(i)-L | SMean(j) |

### Dependent Variable: LAMZHL

28.999499

-5.936180

| | | Standard | | |
|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t 90% Confidence Limits |
| A - B | 11.5316592 | 8.19375941 | 1.41 | 0.2321-5.9361805 28.9994989 |

Comparison: C vs B

Dependent Variable: AUC<sub>0-t</sub> (h\*ng/mL) Weight Group: 51-62

| Class | Levels | Values | |
|-----------------------|----------|---------|---|
| subject | 2 | 101 201 | |
| sequence | 1 | ABC | |
| trt | 2 | ВС | |
| N. 1 001 | | | |
| Number of Observation | ons Read | | 4 |
| Number of Observati | ons Used | | 4 |

Comparison: C vs B

Dependent Variable: AUC<sub>0-t</sub> (h\*ng/mL) Weight Group: 51-62

### The GLM Procedure

Dependent Variable: LN\_AUCLST

| R-Square | Coeff Var | Root MSE | | LN_AUC | LST Mean |
|---|---|---|---|---|---|
| 0.995425 | 0.993048 | 0.089625 | 9.025241 | | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.00000000 | | | |
| trt | 1 | 0.00308741 | 0.00308741 | 0.38 | 0.6467 |
| subject(sequence | ce) 1 | 1.74458843 | 1.74458843 | 217.19 | 0.0431 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.00000000 | | | |
| trt | 1 | 0.00308741 | 0.00308741 | 0.38 | 0.6467 |
| subject(sequence | ce) 1 | 1.74458843 | 1.74458843 | 217.19 | 0.0431 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.00000000 | | | |
| trt | 1 | 0.00308741 | 0.00308741 | 0.38 | 0.6467 |
| subject(sequence | ce) 1 | 1.74458843 | 1.74458843 | 217.19 | 0.0431 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.00000000 | | | |
| trt | 1 | 0.00308741 | 0.00308741 | 0.38 | 0.6467 |
| subject(sequence | ce) 1 | 1.74458843 | 1.74458843 | 217.19 | 0.0431 |

Comparison: C vs B

Dependent Variable: AUC<sub>0-t</sub> (h\*ng/mL) Weight Group: 51-62

### The GLM Procedure Least Squares Means

| | | H0:LSMean1=LSMean2 |
|-----|------------------|--------------------|
| trt | LN_AUCLST LSMEAN | Pr > t |
| В | 9.05302332 | 0.6467 |
| C | 8.99745888 | |

| trt | LN_AUCLST LSMEAN | 90% Confidence Limits | |
|-----|------------------|-----------------------|----------|
| В | 9.053023 | 8.652893 | 9.453154 |
| C | 8.997459 | 8.597329 | 9.397589 |

| Le | Least Squares Means for Effect trt | | | |
|---|---|---|---|---|
| | | Difference Between | | |
| i | j | Means | 90% Confide | ence Limits for LSMean(i)-LSMean(j) |
| 1 | 2 | 0.055564 | -0.510305 | 0.621434 |

### The GLM Procedure

Dependent Variable: LN\_AUCLST

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confide | ence Limits |
| C - B | -0.05556445 | 0.08962497 | -0.62 | 0.6467-0 | 0.62143424 | 0.51030535 |

Comparison: C vs B

Dependent Variable: AUC<sub>0-inf</sub> (h\*ng/mL) Weight Group: 51-62

| Class Level Informatical Class | Levels | Values | |
|--------------------------------|----------|---------|---|
| subject | 2 | 101 201 | |
| sequence | 1 | ABC | |
| trt | 2 | ВС | |
| Number of Observati | ons Read | | 4 |
| Number of Observati | ons Used | | 4 |

Comparison: C vs B

Dependent Variable: AUC<sub>0-inf</sub> (h\*ng/mL) Weight Group: 51-62

### The GLM Procedure

Dependent Variable: LN\_AUCIFO

| R-Square | Coeff Var | Root MSE | | LN_AUC | IFO Mean |
|---|---|---|---|---|---|
| 0.999287 | 0.422185 | 0.038401 | 9.095817 | | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.00000000 | | | |
| trt | 1 | 0.00001005 | 0.00001005 | 0.01 | 0.9476 |
| subject(sequence | ce) 1 | 2.06771611 | 2.06771611 | 1402.17 | 0.0170 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.00000000 | | | |
| trt | 1 | 0.00001005 | 0.00001005 | 0.01 | 0.9476 |
| subject(sequence | ce) 1 | 2.06771611 | 2.06771611 | 1402.17 | 0.0170 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.00000000 | | | |
| trt | 1 | 0.00001005 | 0.00001005 | 0.01 | 0.9476 |
| subject(sequence | ce) 1 | 2.06771611 | 2.06771611 | 1402.17 | 0.0170 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.00000000 | | | |
| trt | 1 | 0.00001005 | 0.00001005 | 0.01 | 0.9476 |
| subject(sequence | ce) 1 | 2.06771611 | 2.06771611 | 1402.17 | 0.0170 |

Comparison: C vs B

Dependent Variable: AUC<sub>0-inf</sub> (h\*ng/mL) Weight Group: 51-62

### The GLM Procedure Least Squares Means

| | | H0:LSMean1=LSMean2 | |
|-----|------------------|--------------------|---------|
| trt | LN_AUCIFO LSMEAN | | Pr > t |
| В | 9.09740260 | | 0.9476 |
| C | 9.09423224 | | |

| trt | LN_AUCIFO LSMEAN | 90% Confidence Limits | |
|-----|------------------|-----------------------|----------|
| В | 9.097403 | 8.925960 | 9.268845 |
| C | 9.094232 | 8.922790 | 9.265674 |

| Le | Least Squares Means for Effect trt | | | |
|---|---|---|---|---|
| | | Difference Between | | |
| i | j | Means | 90% Confid | ence Limits for LSMean(i)-LSMean(j) |
| 1 | 2 | 0.003170 | -0.239285 | 0.245626 |

### The GLM Procedure

Dependent Variable: LN\_AUCIFO

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confid | lence Limits |
| C - B | -0.00317035 | 0.03840122 | -0.08 | 0.9476-0 | 0.24562613 | 0.23928542 |

Comparison: C vs B

Dependent Variable: C<sub>max</sub> (ng/mL) Weight Group: 51-62

| Class Level Informa | | 77.1 | |
|---------------------|----------|---------|---|
| Class | Levels | Values | |
| subject | 2 | 101 201 | |
| sequence | 1 | ABC | |
| trt | 2 | ВС | |
| Number of Observati | ons Read | | 4 |
| Number of Observati | ons Used | | 4 |

Comparison: C vs B

Dependent Variable:  $C_{max}$  (ng/mL) Weight Group: 51-62

### The GLM Procedure

Dependent Variable: LN\_CMAX

| R-Square ( | Coeff Var | Root MSE | | LN_CM | IAX Mean |
|---|---|---|---|---|---|
| 0.996701 | 1.022835 | 0.056591 | 5.532719 | _ | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.00000000 | | | |
| trt | 1 | 0.27556715 | 0.27556715 | 86.05 | 0.0684 |
| subject(sequence) | ) 1 | 0.69186372 | 0.69186372 | 216.04 | 0.0432 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.00000000 | | | |
| trt | 1 | 0.27556715 | 0.27556715 | 86.05 | 0.0684 |
| subject(sequence) | ) 1 | 0.69186372 | 0.69186372 | 216.04 | 0.0432 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.00000000 | | | |
| trt | 1 | 0.27556715 | 0.27556715 | 86.05 | 0.0684 |
| subject(sequence) | ) 1 | 0.69186372 | 0.69186372 | 216.04 | 0.0432 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.00000000 | | | |
| trt | 1 | 0.27556715 | 0.27556715 | 86.05 | 0.0684 |
| subject(sequence) | ) 1 | 0.69186372 | 0.69186372 | 216.04 | 0.0432 |

Comparison: C vs B

Dependent Variable: C<sub>max</sub> (ng/mL) Weight Group: 51-62

### The GLM Procedure Least Squares Means

| | | H0:LSMean1=LSMean2 | |
|-----|----------------|--------------------|---------|
| trt | LN_CMAX LSMEAN | | Pr > t |
| В | 5.79519172 | | 0.0684 |
| C | 5.27024682 | | |

| trt | LN_CMAX LSMEAN | 90% Confidence Limits | |
|-----|----------------|-----------------------|----------|
| В | 5.795192 | 5.542543 | 6.047840 |
| C | 5.270247 | 5.017598 | 5.522895 |

| Le | ast S | Squares Means for Effect | et trt | |
|---|---|---|---|---|
| | | Difference Between | | |
| i | j | Means | 90% Confid | ence Limits for LSMean(i)-LSMean(j) |
| 1 | 2 | 0.524945 | 0.167646 | 0.882244 |

### The GLM Procedure

Dependent Variable: LN\_CMAX

| - | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confi | dence Limits |
| C - B | -0.52494490 | 0.05659061 | -9.28 | 0.0684-0 | .88224396 | -0.16764585 |

Comparison: C vs B

Dependent Variable: Cl/F/kg ((L/h)/kg) Weight Group: 51-62

| Class Level Informatical Class | Levels | Values | |
|--------------------------------|----------|---------|---|
| subject | 2 | 101 201 | |
| sequence | 1 | ABC | |
| trt | 2 | ВС | |
| Number of Observati | ons Read | | 4 |
| Number of Observati | ons Used | | 4 |

Comparison: C vs B

Dependent Variable: Cl/F/kg ((L/h)/kg) Weight Group: 51-62

### The GLM Procedure

Dependent Variable: LN\_CLFOW

| R-Square | Coeff Var | Root MSE | | LN_CLF | OW Mean |
|------------------|-----------|-------------|-------------|---------|---------|
| 0.999296 | -1.025649 | 0.038401 | -3.744090 | | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.00000000 | | | |
| trt | 1 | 0.00001005 | 0.00001005 | 0.01 | 0.9476 |
| subject(sequence | e) 1 | 2.09205676 | 2.09205676 | 1418.68 | 0.0169 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.00000000 | | | |
| trt | 1 | 0.00001005 | 0.00001005 | 0.01 | 0.9476 |
| subject(sequence | e) 1 | 2.09205676 | 2.09205676 | 1418.68 | 0.0169 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.00000000 | | | |
| trt | 1 | 0.00001005 | 0.00001005 | 0.01 | 0.9476 |
| subject(sequence | e) 1 | 2.09205676 | 2.09205676 | 1418.68 | 0.0169 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.00000000 | · | | |
| trt | 1 | 0.00001005 | 0.00001005 | 0.01 | 0.9476 |
| subject(sequence | e) 1 | 2.09205676 | 2.09205676 | 1418.68 | 0.0169 |

Comparison: C vs B

Dependent Variable: Cl/F/kg ((L/h)/kg) Weight Group: 51-62

### The GLM Procedure Least Squares Means

| | | H0:LSMean1=LSMean2 | |
|-----|-----------------|--------------------|---------|
| trt | LN_CLFOW LSMEAN | | Pr > t |
| В | -3.74567555 | | 0.9476 |
| C | -3.74250520 | | |

| trt | LN_CLFOW LSMEAN | 90% Confidence Limits | |
|-----|-----------------|-----------------------|-----------|
| В | -3.745676 | -3.917118 | -3.574233 |
| C | -3.742505 | -3.913947 | -3.571063 |

| Le | Least Squares Means for Effect trt | | | |
|---|---|---|---|---|
| | | Difference Between | | |
| i | j | Means | 90% Confider | ace Limits for LSMean(i)-LSMean(j) |
| 1 | 2 | -0.003170 | -0.245626 | 0.239285 |

### The GLM Procedure

Dependent Variable: LN\_CLFOW

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confi | dence Limits |
| C - B | 0.00317035 | 0.03840122 | 0.08 | 0.9476-0 | 0.23928542 | 0.24562613 |

Comparison: C vs B

Dependent Variable: Cl/F (L/h) Weight Group: 51-62

| Class | Levels | Values | |
|---------------------|-----------|---------|---|
| subject | 2 | 101 201 | |
| sequence | 1 | ABC | |
| trt | 2 | ВС | |
| Number of Observati | ions Read | | 4 |
| Number of Observati | ions Used | | 4 |

Comparison: C vs B

Dependent Variable: Cl/F (L/h) Weight Group: 51-62

### The GLM Procedure

Dependent Variable: LN\_CLFO

| R-Square | Coeff Var | Root MSE | 3 | LN_0 | CLFO Mean |
|---|---|---|---|---|---|
| 0.999287 | 11.37253 | 0.038401 | 0.337667 | | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.00000000 | | | |
| trt | 1 | 0.00001005 | 0.00001005 | 0.01 | 0.9476 |
| subject(sequence | e) 1 | 2.06771611 | 2.06771611 | 1402.17 | 0.0170 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.00000000 | | | |
| trt | 1 | 0.00001005 | 0.00001005 | 0.01 | 0.9476 |
| subject(sequence | e) 1 | 2.06771611 | 2.06771611 | 1402.17 | 0.0170 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.00000000 | | | |
| trt | 1 | 0.00001005 | 0.00001005 | 0.01 | 0.9476 |
| subject(sequence | e) 1 | 2.06771611 | 2.06771611 | 1402.17 | 0.0170 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.00000000 | | | |
| trt | 1 | 0.00001005 | 0.00001005 | 0.01 | 0.9476 |
| subject(sequence | e) 1 | 2.06771611 | 2.06771611 | 1402.17 | 0.0170 |

Comparison: C vs B

Dependent Variable: Cl/F (L/h) Weight Group: 51-62

### The GLM Procedure Least Squares Means

| | | H0:LSMean1=LSMean2 | |
|-----|----------------|--------------------|---------|
| trt | LN_CLFO LSMEAN | | Pr > t |
| В | 0.33608132 | | 0.9476 |
| C | 0.33925168 | | |

| trt | LN_CLFO LSMEAN | 90% Confidence Limits | |
|-----|----------------|-----------------------|----------|
| В | 0.336081 | 0.164639 | 0.507523 |
| C | 0.339252 | 0.167810 | 0.510694 |

| Le | Least Squares Means for Effect trt | | | |
|---|---|---|---|---|
| | | Difference Between | | |
| i | j | Means | 90% Confid | ence Limits for LSMean(i)-LSMean(j) |
| 1 | 2 | -0.003170 | -0.245626 | 0.239285 |

#### The GLM Procedure

Dependent Variable: LN\_CLFO

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confid | dence Limits |
| C - B | 0.00317035 | 0.03840122 | 0.08 | 0.9476-0 | .23928542 | 0.24562613 |

Comparison: C vs B

Dependent Variable: V<sub>d</sub>/F/kg (L/kg) Weight Group: 51-62

| Class Level Informa | | 77.1 | |
|---------------------|----------|---------|---|
| Class | Levels | Values | |
| subject | 2 | 101 201 | |
| sequence | 1 | ABC | |
| trt | 2 | ВС | |
| Number of Observati | ons Read | | 4 |
| Number of Observati | ons Used | | 4 |

Comparison: C vs B

Dependent Variable: V<sub>d</sub>/F/kg (L/kg) Weight Group: 51-62

### The GLM Procedure

Dependent Variable: LN\_VZFOW

| R-Square | Coeff Var | Root MSE | | LN_VZF | OW Mean |
|----------------|-----------|-------------|-------------|---------|---------|
| 0.507929 | 87.10023 | 0.257878 | 0.296071 | | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.00000000 | | | |
| trt | 1 | 0.06357519 | 0.06357519 | 0.96 | 0.5072 |
| subject(sequen | ce) 1 | 0.00506924 | 0.00506924 | 0.08 | 0.8285 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.00000000 | | | |
| trt | 1 | 0.06357519 | 0.06357519 | 0.96 | 0.5072 |
| subject(sequen | ce) 1 | 0.00506924 | 0.00506924 | 0.08 | 0.8285 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.00000000 | - | | |
| trt | 1 | 0.06357519 | 0.06357519 | 0.96 | 0.5072 |
| subject(sequen | ce) 1 | 0.00506924 | 0.00506924 | 0.08 | 0.8285 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.00000000 | | | |
| trt | 1 | 0.06357519 | 0.06357519 | 0.96 | 0.5072 |
| subject(sequen | ce) 1 | 0.00506924 | 0.00506924 | 0.08 | 0.8285 |

Comparison: C vs B

Dependent Variable: V<sub>d</sub>/F/kg (L/kg) Weight Group: 51-62

### The GLM Procedure Least Squares Means

| | | H0:LS | Mean1=LSMean2 | |
|-----|-----------------|-----------|-------------------|---------|
| trt | LN_VZFOW LSMEAN | | | Pr > t |
| В | 0.17000011 | | | 0.5072 |
| C | 0.42214132 | | | |
| trt | LN_VZFOW LSMEAN | 90% | Confidence Limits | |
| В | 0.170000 | -0.981296 | 1.321297 | |
| C | 0.422141 | -0.729155 | 1 573438 | |

| Le | ast | Squares Means for Effec | t trt | |
|---|---|---|---|---|
| | | Difference Between | | |
| i | j | Means | 90% Confide | ence Limits for LSMean(i)-LSMean(j) |
| 1 | 2 | -0.252141 | -1.880320 | 1.376038 |

#### The GLM Procedure

Dependent Variable: LN\_VZFOW

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confi | dence Limits |
| C - B | 0.25214122 | 0.25787826 | 0.98 | 0.5072-1 | .37603804 | 1.88032048 |

Comparison: C vs B

Dependent Variable: V<sub>d</sub>/F (L) Weight Group: 51-62

| Class Level Informa<br>Class | Levels | Values | |
|------------------------------|-----------|---------|---|
| | Levels | | |
| subject | 2 | 101 201 | |
| sequence | 1 | ABC | |
| trt | 2 | ВС | |
| Number of Observation | ions Read | | 4 |
| Number of Observati | ions Used | | 4 |

Comparison: C vs B

Dependent Variable: V<sub>d</sub>/F (L) Weight Group: 51-62

### The GLM Procedure

Dependent Variable: LN\_VZFO

| R-Square | Coeff Var | Root MSE | ·<br>· | LN_ | VZFO Mean |
|---|---|---|---|---|---|
| 0.512521 | 5.890553 | 0.257878 | 4.377828 | | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.00000000 | | | |
| trt | 1 | 0.06357519 | 0.06357519 | 0.96 | 0.5072 |
| subject(sequence) | ) 1 | 0.00634213 | 0.00634213 | 0.10 | 0.8093 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.00000000 | | | |
| trt | 1 | 0.06357519 | 0.06357519 | 0.96 | 0.5072 |
| subject(sequence) | ) 1 | 0.00634213 | 0.00634213 | 0.10 | 0.8093 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.00000000 | | | |
| trt | 1 | 0.06357519 | 0.06357519 | 0.96 | 0.5072 |
| subject(sequence) | ) 1 | 0.00634213 | 0.00634213 | 0.10 | 0.8093 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.00000000 | | | |
| trt | 1 | 0.06357519 | 0.06357519 | 0.96 | 0.5072 |
| subject(sequence) | ) 1 | 0.00634213 | 0.00634213 | 0.10 | 0.8093 |

Comparison: C vs B

Dependent Variable: V<sub>d</sub>/F (L) Weight Group: 51-62

### The GLM Procedure Least Squares Means

| | | H0:LSMean1=LSMean2 |
|-----|----------------|--------------------|
| trt | LN_VZFO LSMEAN | Pr > t |
| В | 4.25175698 | 0.5072 |
| C | 4.50389820 | |

| trt | LN_VZFO LSMEAN | 90% Confidence Limits | |
|-----|----------------|-----------------------|----------|
| В | 4.251757 | 3.100460 | 5.403054 |
| C | 4.503898 | 3.352602 | 5.655195 |

| Le | Least Squares Means for Effect trt | | | |
|---|---|---|---|---|
| | | Difference Between | | |
| i | j | Means | 90% Confid | ence Limits for LSMean(i)-LSMean(j) |
| 1 | 2 | -0.252141 | -1.880320 | 1.376038 |

### The GLM Procedure

Dependent Variable: LN\_VZFO

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confiden | nce Limits |
| C - B | 0.25214122 | 0.25787826 | 0.98 | 0.5072-1 | .37603804 1 | .88032048 |

Comparison: C vs B

Dependent Variable: T<sub>max</sub> (h) Weight Group: 51-62

| Class Level Informa<br>Class | Levels | Values | |
|------------------------------|----------|---------|---|
| | Levels | | |
| subject | 2 | 101 201 | |
| sequence | 1 | ABC | |
| trt | 2 | ВС | |
| Number of Observation | ons Read | | 4 |
| Number of Observation | ons Used | | 4 |

Comparison: C vs B

Dependent Variable: T<sub>max</sub> (h) Weight Group: 51-62

### The GLM Procedure

Dependent Variable: TMAX

| R-Square | Coeff Var | Root | MSE | Т | MAX Mean |
|---|---|---|---|---|---|
| 0.470588 | 120.0000 | 1.500 | 0000 1.2 | 250000 | |
| | D.F. | T. 100 | | | B . E |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.00000000 | | | |
| trt | 1 | 1.00000000 | 1.00000000 | 0.44 | 0.6257 |
| subject(sequence) | 1 | 1.00000000 | 1.00000000 | 0.44 | 0.6257 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| | | 71 | Mean Square | 1 value | 11/1 |
| sequence | 0 | 0.00000000 | 1 0000000 | 0.44 | 0.6257 |
| trt | 1 | 1.00000000 | 1.00000000 | 0.44 | 0.6257 |
| subject(sequence) | l | 1.00000000 | 1.00000000 | 0.44 | 0.6257 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.00000000 | | | |
| trt | 1 | 1.00000000 | 1.00000000 | 0.44 | 0.6257 |
| subject(sequence) | 1 | 1.00000000 | 1.00000000 | 0.44 | 0.6257 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.00000000 | | | |
| trt | 1 | 1.00000000 | 1.00000000 | 0.44 | 0.6257 |
| subject(sequence) | 1 | 1.00000000 | 1.00000000 | 0.44 | 0.6257 |

Comparison: C vs B

Dependent Variable: T<sub>max</sub> (h) Weight Group: 51-62

### The GLM Procedure Least Squares Means

| | | H0:LS | Mean1=LSMean2 | |
|---|---|---|---|---|
| trt | TMAX LSMEAN | | | Pr > t |
| В | 0.75000000 | | | 0.6257 |
| C | 1.75000000 | | | |
| trt | TMAX LSMEAN | 90% | 6 Confidence Limits | |
| В | 0.750000 | -5.946745 | 7.446745 | |
| C | 1.750000 | -4.946745 | 8.446745 | |
| Le | ast Squares Means for Effec | et trt | | |
| | Difference Between | | | |
| i | j Means | 90% Confidence Limit | s for LSMean(i)-LSN | Aean(j) |
| 1 | 2 -1.000000 | -10.470627 | 8.470627 | |

### The GLM Procedure

Dependent Variable: TMAX

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confi | idence Limits |
| C - B | 1.00000000 | 1.50000000 | 0.67 | 0.6257-8 | .47062727 | 10.47062727 |

Comparison: C vs B

Dependent Variable: K<sub>el</sub> (/h) Weight Group: 51-62

| Class | Levels | Values | |
|---------------------|----------|---------|---|
| subject | 2 | 101 201 | |
| sequence | 1 | ABC | |
| trt | 2 | ВС | |
| Number of Observati | ons Read | | 4 |
| Number of Observati | ons Used | | 4 |

Comparison: C vs B

Dependent Variable: K<sub>el</sub> (/h) Weight Group: 51-62

### The GLM Procedure

| R-Square | Coeff Var | Root | MSE | | LAMZ Mean |
|---|---|---|---|---|---|
| 0.997732 | 6.051039 | 0.00 | 1393 | 0.023023 | |
| Source | DF | Type I SS | Mean Square | F Value | e Pr > F |
| sequence | 0 | 0.00000000 | | | |
| trt | 1 | 0.00000626 | 0.00000626 | 3.22 | 0.3235 |
| subject(sequence) | 1 | 0.00084772 | 0.00084772 | 436.78 | 0.0304 |
| Source | DF | Type II SS | Mean Square | F Value | e Pr > F |
| sequence | 0 | 0.00000000 | | | _ |
| trt | 1 | 0.00000626 | 0.00000626 | 3.22 | 0.3235 |
| subject(sequence) | 1 | 0.00084772 | 0.00084772 | 436.78 | 0.0304 |
| Source | DF | Type III SS | Mean Square | F Value | e Pr > F |
| sequence | 0 | 0.00000000 | | | |
| trt | 1 | 0.00000626 | 0.00000626 | 3.22 | 0.3235 |
| subject(sequence) | 1 | 0.00084772 | 0.00084772 | 436.78 | 0.0304 |
| Course | DE | Trme IV/CC | Maan Sayara | F Value | e Pr > F |
| Source | DF | Type IV SS | Mean Square | e r vaiue | 2 PI > F |
| sequence | 0 | 0.00000000 | 0.00000626 | 2 22 | 0.2225 |
| trt | 1 | 0.00000626 | 0.00000626 | 3.22 | 0.3235 |
| subject(sequence) | 1 | 0.00084772 | 0.00084772 | 436.78 | 0.0304 |
## Listing 16.1.9-5 ANOVA for Treatment Comparison of Diazepam for Weight Group $51\text{-}62~\mathrm{kg}$ - PK Population

Comparison: C vs B

Dependent Variable: K<sub>el</sub> (/h) Weight Group: 51-62

#### The GLM Procedure Least Squares Means

| | | H0:LSMe | ean1=LSMean2 |
|-----|-------------|----------|-------------------|
| trt | LAMZ LSMEAN | | Pr > t |
| В | 0.02427392 | | 0.3235 |
| C | 0.02177245 | | |
| trt | LAMZ LSMEAN | 90% ( | Confidence Limits |
| В | 0.024274 | 0.018054 | 0.030494 |
| C | 0.021772 | 0.015553 | 0.027992 |

| Le | Least Squares Means for Effect trt | | | |
|---|---|---|---|---|
| | | Difference Between | | |
| i | j | Means | 90% Confide | nce Limits for LSMean(i)-LSMean(j) |
| 1 | 2 | 0.002501 | -0.006294 | 0.011297 |

#### The GLM Procedure

Dependent Variable: LAMZ

| | | Standard | | | |
|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confidence Limits |
| C - B | -0.00250147 | 0.00139314 | -1.80 | 0.3235-0 | 0.01129742 0.00629448 |

Comparison: C vs B

Dependent Variable: T<sub>1/2 el</sub> (h) Weight Group: 51-62

| Class | Levels | Values | |
|--------------------|-----------|---------|---|
| subject | 2 | 101 201 | |
| sequence | 1 | ABC | |
| trt | 2 | ВС | |
| Number of Observat | ions Read | | 4 |
| Number of Observat | | | 4 |

Comparison: C vs B

Dependent Variable: T<sub>1/2 el</sub> (h) Weight Group: 51-62

#### The GLM Procedure

Dependent Variable: LAMZHL

| R-Square | Coeff Var | Root MSE | | LAMZ | HL Mean |
|---|---|---|---|---|---|
| 0.928959 | 37.39729 | 19.61552 | 52.45171 | | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.000000 | | | |
| trt | 1 | 406.408780 | 406.408780 | 1.06 | 0.4913 |
| subject(sequence | ) 1 | 4624.986296 | 4624.986296 | 12.02 | 0.1788 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| | 0 | 0.000000 | Wican Square | 1 value | 11 > 1 |
| sequence<br>trt | 1 | 406.408780 | 406.408780 | 1.06 | 0.4913 |
| | - | | | | |
| subject(sequence | ) 1 | 4624.986296 | 4624.986296 | 12.02 | 0.1788 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.000000 | | | |
| trt | 1 | 406.408780 | 406.408780 | 1.06 | 0.4913 |
| subject(sequence | ) 1 | 4624.986296 | 4624.986296 | 12.02 | 0.1788 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.000000 | | | |
| trt | 1 | 406.408780 | 406.408780 | 1.06 | 0.4913 |
| subject(sequence | ) 1 | 4624.986296 | 4624.986296 | 12.02 | 0.1788 |

Comparison: C vs B

Dependent Variable: T<sub>1/2 el</sub> (h) Weight Group: 51-62

#### The GLM Procedure Least Squares Means

| | | H0:LSMean1=LSMean2 | |
|-----|---------------|--------------------|---------|
| trt | LAMZHL LSMEAN | | Pr > t |
| В | 42.3719162 | | 0.4913 |
| C | 62.5314991 | | |

| trt | LAMZHL LSMEAN | | 90% Confidence Limits |
|-----|---------------|------------|-----------------------|
| В | 42.371916 | -45.201494 | 129.945327 |
| C | 62.531499 | -25.041912 | 150.104910 |

| Le | Least Squares Means for Effect trt | | | |
|---|---|---|---|---|
| | | Difference Between | | |
| i | j | Means | 90% Confidence | ce Limits for LSMean(i)-LSMean(j) |
| 1 | 2 | -20.159583 | -144.007088 | 103.687922 |

#### The GLM Procedure

Dependent Variable: LAMZHL

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confid | dence Limits |
| C - B | 20.1595828 | 19.6155178 | 1.03 | 0.4913-1 | 03.6879223 | 144.0070879 |

Comparison: A vs B

Dependent Variable: AUC<sub>0-t</sub> (h\*ng/mL) Weight Group: 63-75

| Class Level Info | rmation | | |
|-----------------------------|---------------|-----------------|---|
| Class | Levels | Values | |
| subject | 4 | 202 303 408 413 | |
| sequence | 2 | AB BA | |
| period | 2 | 1 2 | |
| trt | 2 | A B | |
| Number of Observations Read | | | |
| Number of Obse | rvations Used | | 8 |

Comparison: A vs B

Dependent Variable: AUC<sub>0-t</sub> (h\*ng/mL) Weight Group: 63-75

#### The GLM Procedure

Dependent Variable: LN\_AUCLST

| R-Square | Coeff Var | Root MSE | | LN_AUC | LST Mean |
|---|---|---|---|---|---|
| 0.998187 | 0.385829 | 0.032800 | 8.501081 | | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.09031713 | 0.09031713 | 83.95 | 0.0117 |
| period | 1 | 0.02145914 | 0.02145914 | 19.95 | 0.0467 |
| trt | 1 | 0.00001757 | 0.00001757 | 0.02 | 0.9100 |
| subject(sequence | e) 2 | 1.07303798 | 0.53651899 | 498.71 | 0.0020 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.09031713 | 0.09031713 | 83.95 | 0.0117 |
| period | 1 | 0.02145914 | 0.02145914 | 19.95 | 0.0467 |
| trt | 1 | 0.00001757 | 0.00001757 | 0.02 | 0.9100 |
| subject(sequence | e) 2 | 1.07303798 | 0.53651899 | 498.71 | 0.0020 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.09031713 | 0.09031713 | 83.95 | 0.0117 |
| period | 1 | 0.02145914 | 0.02145914 | 19.95 | 0.0467 |
| trt | 1 | 0.00001757 | 0.00001757 | 0.02 | 0.9100 |
| subject(sequence | e) 2 | 1.07303798 | 0.53651899 | 498.71 | 0.0020 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.09031713 | 0.09031713 | 83.95 | 0.0117 |
| period | 1 | 0.02145914 | 0.02145914 | 19.95 | 0.0467 |
| trt | 1 | 0.00001757 | 0.00001757 | 0.02 | 0.9100 |
| subject(sequence | e) 2 | 1.07303798 | 0.53651899 | 498.71 | 0.0020 |

Comparison: A vs B

Dependent Variable: AUC<sub>0-t</sub> (h\*ng/mL) Weight Group: 63-75

## The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_AUCLST

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.090317 | 0.090317 | 0.17 | 0.7214 |
| Error | 2 | 1.073038 | 0.536519 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 0.021459 | 0.021459 | 19.95 | 0.0467 |
| trt | 1 | 0.000017570 | 0.000017570 | 0.02 | 0.9100 |
| subject(sequence) | 2 | 1.073038 | 0.536519 | 498.71 | 0.0020 |
| Error: MS(Error) | 2 | 0.002152 | 0.001076 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN AUCLST

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------|-----------|------------|-------------|---------|--------|
| sequence | 1 | 0.090317 | 0.090317 | 0.17 | 0.7214 |
| Error | 2 | 1.073038 | 0.536519 | | _ |
| Error: MS(s | subject(s | equence)) | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 0.021459 | 0.021459 | 19.95 | 0.0467 |
| trt | 1 | 0.000017570 | 0.000017570 | 0.02 | 0.9100 |
| subject(sequence) | 2 | 1.073038 | 0.536519 | 498.71 | 0.0020 |
| Error: MS(Error) | 2 | 0.002152 | 0.001076 | | |

Comparison: A vs B

Dependent Variable: AUC<sub>0-t</sub> (h\*ng/mL) Weight Group: 63-75

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_AUCLST

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.090317 | 0.090317 | 0.17 | 0.7214 |
| Error | 2 | 1.073038 | 0.536519 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 0.021459 | 0.021459 | 19.95 | 0.0467 |
| trt | 1 | 0.000017570 | 0.000017570 | 0.02 | 0.9100 |
| subject(sequence) | 2 | 1.073038 | 0.536519 | 498.71 | 0.0020 |
| Error: MS(Error) | 2 | 0.002152 | 0.001076 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_AUCLST

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------|-----------|------------|-------------|---------|--------|
| sequence | 1 | 0.090317 | 0.090317 | 0.17 | 0.7214 |
| Error | 2 | 1.073038 | 0.536519 | | |
| Error: MS(s | subject(s | sequence)) | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 0.021459 | 0.021459 | 19.95 | 0.0467 |
| trt | 1 | 0.000017570 | 0.000017570 | 0.02 | 0.9100 |
| subject(sequence) | 2 | 1.073038 | 0.536519 | 498.71 | 0.0020 |
| Error: MS(Error) | 2 | 0.002152 | 0.001076 | | |

Comparison: A vs B

Dependent Variable: AUC<sub>0-t</sub> (h\*ng/mL) Weight Group: 63-75

#### Least Squares Means

| | | H0:LSM | Iean1=LSMean2 | |
|-----|------------------|----------|-------------------|---------|
| trt | LN_AUCLST LSMEAN | | | Pr > t |
| A | 8.50256332 | | | 0.9100 |
| В | 8.49959937 | | | |
| trt | LN_AUCLST LSMEAN | 90% | Confidence Limits | |
| trt | LN AUCLST LSMEAN | 90% | Confidence Limits | |
| A | 8.502563 | 8.454676 | 8.550451 | |
| В | 8.499599 | 8.451712 | 8.547487 | |

Least Squares Means for Effect trt

Difference Between

i j Means 90% Confidence Limits for LSMean(i)-LSMean(j)

1 2 0.002964 -0.064759 0.070687

Dependent Variable: LN\_AUCLST

| • | | Standard | | | | _ |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confi | dence Limits |
| A - B | 0.00296395 | 0.02319284 | 0.13 | 0.9100-0 | 0.06475879 | 0.07068670 |

Comparison: A vs B

Dependent Variable: AUC<sub>0-inf</sub> (h\*ng/mL) Weight Group: 63-75

| Class Level Info | | 37 1 | |
|---|---|---|---|
| Class | Levels | Values | |
| subject | 4 | 202 303 408 413 | |
| sequence | 2 | AB BA | |
| period | 2 | 1 2 | |
| trt | 2 | A B | |
| Number of Obse | rvations Read | | 8 |
| Number of Obse | Number of Observations Used | | |

Comparison: A vs B

Dependent Variable: AUC<sub>0-inf</sub> (h\*ng/mL) Weight Group: 63-75

#### The GLM Procedure

Dependent Variable: LN\_AUCIFO

| R-Square | Coeff Var | Root MSE | | LN_AUC | IFO Mean |
|-----------------|-----------|-------------|-------------|---------|----------|
| 0.998102 | 0.409031 | 0.034910 | 8.534749 | | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.10836268 | 0.10836268 | 88.92 | 0.0111 |
| period | 1 | 0.01560178 | 0.01560178 | 12.80 | 0.0700 |
| trt | 1 | 0.00019420 | 0.00019420 | 0.16 | 0.7283 |
| subject(sequenc | e) 2 | 1.15775241 | 0.57887620 | 475.00 | 0.0021 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.10836268 | 0.10836268 | 88.92 | 0.0111 |
| period | 1 | 0.01560178 | 0.01560178 | 12.80 | 0.0700 |
| trt | 1 | 0.00019420 | 0.00019420 | 0.16 | 0.7283 |
| subject(sequenc | e) 2 | 1.15775241 | 0.57887620 | 475.00 | 0.0021 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.10836268 | 0.10836268 | 88.92 | 0.0111 |
| period | 1 | 0.01560178 | 0.01560178 | 12.80 | 0.0700 |
| trt | 1 | 0.00019420 | 0.00019420 | 0.16 | 0.7283 |
| subject(sequenc | e) 2 | 1.15775241 | 0.57887620 | 475.00 | 0.0021 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.10836268 | 0.10836268 | 88.92 | 0.0111 |
| period | 1 | 0.01560178 | 0.01560178 | 12.80 | 0.0700 |
| trt | 1 | 0.00019420 | 0.00019420 | 0.16 | 0.7283 |
| subject(sequenc | e) 2 | 1.15775241 | 0.57887620 | 475.00 | 0.0021 |

Comparison: A vs B

Dependent Variable: AUC<sub>0-inf</sub> (h\*ng/mL) Weight Group: 63-75

## The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_AUCIFO

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.108363 | 0.108363 | 0.19 | 0.7074 |
| Error | 2 | 1.157752 | 0.578876 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-------------------|----|-----------|-------------|---------|--------|
| period | 1 | 0.015602 | 0.015602 | 12.80 | 0.0700 |
| trt | 1 | 0.000194 | 0.000194 | 0.16 | 0.7283 |
| subject(sequence) | 2 | 1.157752 | 0.578876 | 475.00 | 0.0021 |
| Error: MS(Error) | 2 | 0.002437 | 0.001219 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN AUCIFO

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------|-----------|------------|-------------|---------|--------|
| sequence | 1 | 0.108363 | 0.108363 | 0.19 | 0.7074 |
| Error | 2 | 1.157752 | 0.578876 | | |
| Error: MS(s | subject(s | equence)) | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.015602 | 0.015602 | 12.80 | 0.0700 |
| trt | 1 | 0.000194 | 0.000194 | 0.16 | 0.7283 |
| subject(sequence) | 2 | 1.157752 | 0.578876 | 475.00 | 0.0021 |
| Error: MS(Error) | 2 | 0.002437 | 0.001219 | | |

Comparison: A vs B

Dependent Variable: AUC<sub>0-inf</sub> (h\*ng/mL) Weight Group: 63-75

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_AUCIFO

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------|-----------|-------------|-------------|---------|--------|
| sequence | 1 | 0.108363 | 0.108363 | 0.19 | 0.7074 |
| Error | 2 | 1.157752 | 0.578876 | | |
| Error: MS(s | subject(s | sequence)) | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 0.015602 | 0.015602 | 12.80 | 0.0700 |
| trt | 1 | 0.000194 | 0.000194 | 0.16 | 0.7283 |
| subject(sequence) | 2 | 1.157752 | 0.578876 | 475.00 | 0.0021 |
| Error: MS(Error) | 2 | 0.002437 | 0.001219 | | - |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_AUCIFO

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------|-----------|------------|-------------|---------|--------|
| sequence | 1 | 0.108363 | 0.108363 | 0.19 | 0.7074 |
| Error | 2 | 1.157752 | 0.578876 | | |
| Error: MS(s | subject(s | sequence)) | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.015602 | 0.015602 | 12.80 | 0.0700 |
| trt | 1 | 0.000194 | 0.000194 | 0.16 | 0.7283 |
| subject(sequence) | 2 | 1.157752 | 0.578876 | 475.00 | 0.0021 |
| Error: MS(Error) | 2 | 0.002437 | 0.001219 | | |

Comparison: A vs B

Dependent Variable: AUC<sub>0-inf</sub> (h\*ng/mL) Weight Group: 63-75

Means 0.009854

#### Least Squares Means

| | | H0:LSM | 1ean1=LSMean2 | |
|---|---|---|---|---|
| trt | LN_AUCIFO LSMEAN | | | Pr > t |
| A | 8.53967571 | | | 0.7283 |
| В | 8.52982180 | | | |
| trt | LN AUCIFO LSMEAN | 90% | Confidence Limits | |
| A | 8.539676 | 8.488708 | 8.590644 | |
| В | 8.529822 | 8.478854 | 8.580790 | |
| Lea | ast Squares Means for Effect | trt | | |
| | Difference Between | | | |
| i | j Means | 90% Confidence Limit | its for LSMean(i)-LS | Mean(j) |

Dependent Variable: LN\_AUCIFO

0.081933

-0.062226

| | | Standard | | | |
|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confidence Limits |
| A - B | 0.00985391 | 0.02468491 | 0.40 | 0.7283-0 | 0.06222566 0.08193349 |

Comparison: A vs B

Dependent Variable: C<sub>max</sub> (ng/mL) Weight Group: 63-75

| Class Level Info | Levels | Values | |
|------------------|----------------|-----------------|---|
| subject | 4 | 202 303 408 413 | |
| sequence | 2 | AB BA | |
| period | 2 | 1 2 | |
| trt | 2 | A B | |
| Number of Obse | ervations Read | | 8 |
| Number of Obse | 8 | | |

Comparison: A vs B

Dependent Variable: C<sub>max</sub> (ng/mL) Weight Group: 63-75

#### The GLM Procedure

Dependent Variable: LN\_CMAX

| R-Square | Coeff Var | Root MSE | | LN_CM | IAX Mean |
|-----------------|-----------|-------------|-------------|---------|----------|
| 0.395997 | 10.38897 | 0.572102 | 5.506819 | | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.24870956 | 0.24870956 | 0.76 | 0.4753 |
| period | 1 | 0.00507523 | 0.00507523 | 0.02 | 0.9123 |
| trt | 1 | 0.01964743 | 0.01964743 | 0.06 | 0.8293 |
| subject(sequenc | e) 2 | 0.15573658 | 0.07786829 | 0.24 | 0.8078 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.24870956 | 0.24870956 | 0.76 | 0.4753 |
| period | 1 | 0.00507523 | 0.00507523 | 0.02 | 0.9123 |
| trt | 1 | 0.01964743 | 0.01964743 | 0.06 | 0.8293 |
| subject(sequenc | e) 2 | 0.15573658 | 0.07786829 | 0.24 | 0.8078 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.24870956 | 0.24870956 | 0.76 | 0.4753 |
| period | 1 | 0.00507523 | 0.00507523 | 0.02 | 0.9123 |
| trt | 1 | 0.01964743 | 0.01964743 | 0.06 | 0.8293 |
| subject(sequenc | e) 2 | 0.15573658 | 0.07786829 | 0.24 | 0.8078 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.24870956 | 0.24870956 | 0.76 | 0.4753 |
| period | 1 | 0.00507523 | 0.00507523 | 0.02 | 0.9123 |
| trt | 1 | 0.01964743 | 0.01964743 | 0.06 | 0.8293 |
| subject(sequenc | e) 2 | 0.15573658 | 0.07786829 | 0.24 | 0.8078 |

Comparison: A vs B

Dependent Variable: C<sub>max</sub> (ng/mL) Weight Group: 63-75

## The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_CMAX

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-------------|----------|-----------|-------------|---------|--------|
| sequence | 1 | 0.248710 | 0.248710 | 3.19 | 0.2158 |
| Error | 2 | 0.155737 | 0.077868 | | _ |
| Error: MS(s | ubject(s | equence)) | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-------------------|----|-----------|-------------|---------|--------|
| period | 1 | 0.005075 | 0.005075 | 0.02 | 0.9123 |
| trt | 1 | 0.019647 | 0.019647 | 0.06 | 0.8293 |
| subject(sequence) | 2 | 0.155737 | 0.077868 | 0.24 | 0.8078 |
| Error: MS(Error) | 2 | 0.654600 | 0.327300 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN CMAX

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------|----------|------------|-------------|---------|--------|
| sequence | 1 | 0.248710 | 0.248710 | 3.19 | 0.2158 |
| Error | 2 | 0.155737 | 0.077868 | | _ |
| Error: MS(s | ubject(s | equence)) | | | |

| G | DE | T II 00 | ) f . G | D 17 1 | D . D |
|-------------------|----|------------|-------------|---------|--------|
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| period | 1 | 0.005075 | 0.005075 | 0.02 | 0.9123 |
| trt | 1 | 0.019647 | 0.019647 | 0.06 | 0.8293 |
| subject(sequence) | 2 | 0.155737 | 0.077868 | 0.24 | 0.8078 |
| Error: MS(Error) | 2 | 0.654600 | 0.327300 | | |

Comparison: A vs B

Dependent Variable: C<sub>max</sub> (ng/mL) Weight Group: 63-75

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_CMAX

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.248710 | 0.248710 | 3.19 | 0.2158 |
| Error | 2 | 0.155737 | 0.077868 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 0.005075 | 0.005075 | 0.02 | 0.9123 |
| trt | 1 | 0.019647 | 0.019647 | 0.06 | 0.8293 |
| subject(sequence) | 2 | 0.155737 | 0.077868 | 0.24 | 0.8078 |
| Error: MS(Error) | 2 | 0.654600 | 0.327300 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_CMAX

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------|-----------|------------|-------------|---------|--------|
| sequence | 1 | 0.248710 | 0.248710 | 3.19 | 0.2158 |
| Error | 2 | 0.155737 | 0.077868 | | |
| Error: MS(s | subject(s | sequence)) | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.005075 | 0.005075 | 0.02 | 0.9123 |
| trt | 1 | 0.019647 | 0.019647 | 0.06 | 0.8293 |
| subject(sequence) | 2 | 0.155737 | 0.077868 | 0.24 | 0.8078 |
| Error: MS(Error) | 2 | 0.654600 | 0.327300 | | |

Comparison: A vs B

Dependent Variable: C<sub>max</sub> (ng/mL) Weight Group: 63-75

Means -0.099115

#### Least Squares Means

| | | H0:LSI | | |
|---|---|---|---|---|
| trt | LN_CMAX LSMEAN | | | Pr > t |
| A | 5.45726168 | | | 0.8293 |
| В | 5.55637635 | | | |
| trt | LN_CMAX LSMEAN | 90% | Confidence Limits | |
| A | 5.457262 | 4.621998 | 6.292526 | |
| В | 5.556376 | 4.721112 | 6.391640 | |
| Lea | ast Squares Means for Effect tr | <u> </u> | | |
| LCC | Difference Between | • | | |

Dependent Variable: LN\_CMAX

-1.280356

90% Confidence Limits for LSMean(i)-LSMean(j)

1.082127

| | | Standard | | | |
|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confidence Limits |
| A - B | -0.09911467 | 0.40453685 | -0.25 | 0.8293-1 | .28035645 1.08212712 |

Comparison: A vs B

Dependent Variable: Cl/F/kg ((L/h)/kg) Weight Group: 63-75

| Class Level Info | Levels | Values | |
|------------------|----------------|-----------------|---|
| subject | 4 | 202 303 408 413 | |
| sequence | 2 | AB BA | |
| period | 2 | 1 2 | |
| trt | 2 | A B | |
| Number of Obse | ervations Read | | 8 |
| Number of Obse | 8 | | |

Comparison: A vs B

Dependent Variable: Cl/F/kg ((L/h)/kg) Weight Group: 63-75

#### The GLM Procedure

Dependent Variable: LN\_CLFOW

| R-Square | Coeff Var | Root MSE | | LN_CLF | OW Mean |
|------------------|-----------|-------------|-------------|---------|---------|
| 0.998313 | -1.114725 | 0.034910 | -3.131690 | | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.13920778 | 0.13920778 | 114.23 | 0.0086 |
| period | 1 | 0.01560178 | 0.01560178 | 12.80 | 0.0700 |
| trt | 1 | 0.00019420 | 0.00019420 | 0.16 | 0.7283 |
| subject(sequence | e) 2 | 1.28746738 | 0.64373369 | 528.22 | 0.0019 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.13920778 | 0.13920778 | 114.23 | 0.0086 |
| period | 1 | 0.01560178 | 0.01560178 | 12.80 | 0.0700 |
| trt | 1 | 0.00019420 | 0.00019420 | 0.16 | 0.7283 |
| subject(sequence | e) 2 | 1.28746738 | 0.64373369 | 528.22 | 0.0019 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.13920778 | 0.13920778 | 114.23 | 0.0086 |
| period | 1 | 0.01560178 | 0.01560178 | 12.80 | 0.0700 |
| trt | 1 | 0.00019420 | 0.00019420 | 0.16 | 0.7283 |
| subject(sequence | e) 2 | 1.28746738 | 0.64373369 | 528.22 | 0.0019 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.13920778 | 0.13920778 | 114.23 | 0.0086 |
| period | 1 | 0.01560178 | 0.01560178 | 12.80 | 0.0700 |
| trt | 1 | 0.00019420 | 0.00019420 | 0.16 | 0.7283 |
| subject(sequence | e) 2 | 1.28746738 | 0.64373369 | 528.22 | 0.0019 |

Comparison: A vs B

Dependent Variable: Cl/F/kg ((L/h)/kg) Weight Group: 63-75

## The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_CLFOW

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.139208 | 0.139208 | 0.22 | 0.6876 |
| Error | 2 | 1.287467 | 0.643734 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-------------------|----|-----------|-------------|---------|--------|
| period | 1 | 0.015602 | 0.015602 | 12.80 | 0.0700 |
| trt | 1 | 0.000194 | 0.000194 | 0.16 | 0.7283 |
| subject(sequence) | 2 | 1.287467 | 0.643734 | 528.22 | 0.0019 |
| Error: MS(Error) | 2 | 0.002437 | 0.001219 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN CLFOW

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------|----------|------------|-------------|---------|--------|
| sequence | 1 | 0.139208 | 0.139208 | 0.22 | 0.6876 |
| Error | 2 | 1.287467 | 0.643734 | | |
| Error: MS(s | ubject(s | equence)) | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.015602 | 0.015602 | 12.80 | 0.0700 |
| trt | 1 | 0.000194 | 0.000194 | 0.16 | 0.7283 |
| subject(sequence) | 2 | 1.287467 | 0.643734 | 528.22 | 0.0019 |
| Error: MS(Error) | 2 | 0.002437 | 0.001219 | | |

Comparison: A vs B

Dependent Variable: Cl/F/kg ((L/h)/kg) Weight Group: 63-75

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_CLFOW

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------|-----------|-------------|-------------|---------|--------|
| sequence | 1 | 0.139208 | 0.139208 | 0.22 | 0.6876 |
| Error | 2 | 1.287467 | 0.643734 | | |
| Error: MS(s | subject(s | sequence)) | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 0.015602 | 0.015602 | 12.80 | 0.0700 |
| trt | 1 | 0.000194 | 0.000194 | 0.16 | 0.7283 |
| subject(sequence) | 2 | 1.287467 | 0.643734 | 528.22 | 0.0019 |
| Error: MS(Error) | 2 | 0.002437 | 0.001219 | | - |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_CLFOW

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------|-----------|------------|-------------|---------|--------|
| sequence | 1 | 0.139208 | 0.139208 | 0.22 | 0.6876 |
| Error | 2 | 1.287467 | 0.643734 | | |
| Error: MS(s | subject(s | sequence)) | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.015602 | 0.015602 | 12.80 | 0.0700 |
| trt | 1 | 0.000194 | 0.000194 | 0.16 | 0.7283 |
| subject(sequence) | 2 | 1.287467 | 0.643734 | 528.22 | 0.0019 |
| Error: MS(Error) | 2 | 0.002437 | 0.001219 | | |

Comparison: A vs B

Dependent Variable: Cl/F/kg ((L/h)/kg) Weight Group: 63-75

-0.009854

#### Least Squares Means

| | | H0:LS | Mean1=LSMean2 | |
|---|---|---|---|---|
| trt | LN_CLFOW LSMEAN | | | Pr > t |
| A | -3.13661745 | | | 0.7283 |
| В | -3.12676354 | | | |
| trt | LN CLFOW LSMEAN | 90% | Confidence Limits | |
| A | -3.136617 | -3.187585 | -3.085649 | |
| В | -3.126764 | -3.177731 | -3.075796 | |
| Lea | ast Squares Means for Effect | trt | | |
| | Difference Between | | | |
| i | j Means | 90% Confidence Li | mits for LSMean(i)-LS | SMean(j) |

#### Dependent Variable: LN\_CLFOW

0.062226

-0.081933

| | | Standard | | |
|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t 90% Confidence Limits |
| A - B | -0.00985391 | 0.02468491 | -0.40 | 0.7283-0.08193349 0.06222566 |

Comparison: A vs B

Dependent Variable: Cl/F (L/h) Weight Group: 63-75

| Class Level Info | Levels | Values | |
|------------------|----------------|-----------------|---|
| subject | 4 | 202 303 408 413 | |
| sequence | 2 | AB BA | |
| period | 2 | 1 2 | |
| trt | 2 | A B | |
| Number of Obse | ervations Read | | 8 |
| Number of Obse | 8 | | |

Comparison: A vs B

Dependent Variable: Cl/F (L/h) Weight Group: 63-75

#### The GLM Procedure

Dependent Variable: LN\_CLFO

| R-Square | Coeff Var | Root MSE | <u>, </u> | LN_ | CLFO Mean |
|---|---|---|---|---|---|
| 0.998102 | 3.229223 | 0.034910 | 1.081057 | | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.10836268 | 0.10836268 | 88.92 | 0.0111 |
| period | 1 | 0.01560178 | 0.01560178 | 12.80 | 0.0700 |
| trt | 1 | 0.00019420 | 0.00019420 | 0.16 | 0.7283 |
| subject(sequence | 2 | 1.15775241 | 0.57887620 | 475.00 | 0.0021 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.10836268 | 0.10836268 | 88.92 | 0.0111 |
| period | 1 | 0.01560178 | 0.01560178 | 12.80 | 0.0700 |
| trt | 1 | 0.00019420 | 0.00019420 | 0.16 | 0.7283 |
| subject(sequence | 2 | 1.15775241 | 0.57887620 | 475.00 | 0.0021 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.10836268 | 0.10836268 | 88.92 | 0.0111 |
| period | 1 | 0.01560178 | 0.01560178 | 12.80 | 0.0700 |
| trt | 1 | 0.00019420 | 0.00019420 | 0.16 | 0.7283 |
| subject(sequence | 2 | 1.15775241 | 0.57887620 | 475.00 | 0.0021 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.10836268 | 0.10836268 | 88.92 | 0.0111 |
| period | 1 | 0.01560178 | 0.01560178 | 12.80 | 0.0700 |
| trt | 1 | 0.00019420 | 0.00019420 | 0.16 | 0.7283 |
| subject(sequence | 2 | 1.15775241 | 0.57887620 | 475.00 | 0.0021 |

Comparison: A vs B

Dependent Variable: Cl/F (L/h) Weight Group: 63-75

## The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_CLFO

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-------------|-----------|-----------|-------------|---------|--------|
| sequence | 1 | 0.108363 | 0.108363 | 0.19 | 0.7074 |
| Error | 2 | 1.157752 | 0.578876 | | |
| Error: MS(s | ubject(se | equence)) | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-------------------|----|-----------|-------------|---------|--------|
| period | 1 | 0.015602 | 0.015602 | 12.80 | 0.0700 |
| trt | 1 | 0.000194 | 0.000194 | 0.16 | 0.7283 |
| subject(sequence) | 2 | 1.157752 | 0.578876 | 475.00 | 0.0021 |
| Error: MS(Error) | 2 | 0.002437 | 0.001219 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN CLFO

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------|-----------|------------|-------------|---------|--------|
| sequence | 1 | 0.108363 | 0.108363 | 0.19 | 0.7074 |
| Error | 2 | 1.157752 | 0.578876 | | |
| Error: MS(s | subject(s | equence)) | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.015602 | 0.015602 | 12.80 | 0.0700 |
| trt | 1 | 0.000194 | 0.000194 | 0.16 | 0.7283 |
| subject(sequence) | 2 | 1.157752 | 0.578876 | 475.00 | 0.0021 |
| Error: MS(Error) | 2 | 0.002437 | 0.001219 | · | |

Comparison: A vs B

Dependent Variable: Cl/F (L/h) Weight Group: 63-75

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_CLFO

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------|-----------|-------------|-------------|---------|--------|
| sequence | 1 | 0.108363 | 0.108363 | 0.19 | 0.7074 |
| Error | 2 | 1.157752 | 0.578876 | | |
| Error: MS(s | subject(s | sequence)) | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 0.015602 | 0.015602 | 12.80 | 0.0700 |
| trt | 1 | 0.000194 | 0.000194 | 0.16 | 0.7283 |
| subject(sequence) | 2 | 1.157752 | 0.578876 | 475.00 | 0.0021 |
| Error: MS(Error) | 2 | 0.002437 | 0.001219 | | - |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_CLFO

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------|-----------|------------|-------------|---------|--------|
| sequence | 1 | 0.108363 | 0.108363 | 0.19 | 0.7074 |
| Error | 2 | 1.157752 | 0.578876 | | |
| Error: MS(s | subject(s | sequence)) | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|----------|--------|
| period | 1 | 0.015602 | 0.015602 | 12.80 | 0.0700 |
| trt | 1 | 0.000194 | 0.000194 | 0.16 | 0.7283 |
| subject(sequence) | 2 | 1.157752 | 0.578876 | 475.00 | 0.0021 |
| Error: MS(Error) | 2 | 0.002437 | 0.001219 | <u>'</u> | |

Comparison: A vs B

Dependent Variable: Cl/F (L/h) Weight Group: 63-75

#### Least Squares Means

| | | H0:LS | Mean1=LSMean2 | |
|---|---|---|---|---|
| trt | LN_CLFO LSMEAN | | | Pr > t |
| A | 1.07612977 | | | 0.7283 |
| В | 1.08598368 | | | |
| trt | LN_CLFO LSMEAN | | 6 Confidence Limits | |
| trt<br>A | LN_CLFO LSMEAN<br>1.076130 | 90% | 6 Confidence Limits<br>1.127098 | |

Least Squares Means for Effect trt

Difference Between

i j Means 90% Confidence Limits for LSMean(i)-LSMean(j)
1 2 -0.009854 -0.081933 0.062226

#### Dependent Variable: LN\_CLFO

| | | Standard | | |
|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t 90% Confidence Limits |
| A - B | -0.00985391 | 0.02468491 | -0.40 | 0.7283-0.08193349 |

Comparison: A vs B

Dependent Variable: V<sub>d</sub>/F/kg (L/kg) Weight Group: 63-75

| Class Level Info | rmation | | |
|------------------|---------------|-----------------|---|
| Class | Levels | Values | |
| subject | 4 | 202 303 408 413 | |
| sequence | 2 | AB BA | |
| period | 2 | 1 2 | |
| trt | 2 | A B | |
| Number of Obse | rvations Read | | 8 |
| Number of Obse | rvations Used | | 8 |

Comparison: A vs B

Dependent Variable: V<sub>d</sub>/F/kg (L/kg) Weight Group: 63-75

#### The GLM Procedure

Dependent Variable: LN\_VZFOW

| R-Square | Coeff Var | Root MSE | | LN_VZF | OW Mean |
|------------------|-----------|-------------|-------------|---------|---------|
| 0.943812 | 10.17324 | 0.088331 | 0.868266 | | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.01194838 | 0.01194838 | 1.53 | 0.3415 |
| period | 1 | 0.10103255 | 0.10103255 | 12.95 | 0.0693 |
| trt | 1 | 0.05015616 | 0.05015616 | 6.43 | 0.1267 |
| subject(sequence | ce) 2 | 0.09897914 | 0.04948957 | 6.34 | 0.1362 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.01194838 | 0.01194838 | 1.53 | 0.3415 |
| period | 1 | 0.10103255 | 0.10103255 | 12.95 | 0.0693 |
| trt | 1 | 0.05015616 | 0.05015616 | 6.43 | 0.1267 |
| subject(sequence | ce) 2 | 0.09897914 | 0.04948957 | 6.34 | 0.1362 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.01194838 | 0.01194838 | 1.53 | 0.3415 |
| period | 1 | 0.10103255 | 0.10103255 | 12.95 | 0.0693 |
| trt | 1 | 0.05015616 | 0.05015616 | 6.43 | 0.1267 |
| subject(sequence | ce) 2 | 0.09897914 | 0.04948957 | 6.34 | 0.1362 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.01194838 | 0.01194838 | 1.53 | 0.3415 |
| period | 1 | 0.10103255 | 0.10103255 | 12.95 | 0.0693 |
| trt | 1 | 0.05015616 | 0.05015616 | 6.43 | 0.1267 |
| subject(sequence | ce) 2 | 0.09897914 | 0.04948957 | 6.34 | 0.1362 |

Comparison: A vs B

Dependent Variable: V<sub>d</sub>/F/kg (L/kg) Weight Group: 63-75

## The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_VZFOW

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-------------|----------|-----------|-------------|---------|--------|
| sequence | 1 | 0.011948 | 0.011948 | 0.24 | 0.6718 |
| Error | 2 | 0.098979 | 0.049490 | | |
| Error: MS(s | ubject(s | equence)) | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-------------------|----|-----------|-------------|---------|--------|
| period | 1 | 0.101033 | 0.101033 | 12.95 | 0.0693 |
| trt | 1 | 0.050156 | 0.050156 | 6.43 | 0.1267 |
| subject(sequence) | 2 | 0.098979 | 0.049490 | 6.34 | 0.1362 |
| Error: MS(Error) | 2 | 0.015605 | 0.007802 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN VZFOW

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------|----------|------------|-------------|---------|--------|
| sequence | 1 | 0.011948 | 0.011948 | 0.24 | 0.6718 |
| Error | 2 | 0.098979 | 0.049490 | | _ |
| Error: MS(s | ubject(s | equence)) | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.101033 | 0.101033 | 12.95 | 0.0693 |
| trt | 1 | 0.050156 | 0.050156 | 6.43 | 0.1267 |
| subject(sequence) | 2 | 0.098979 | 0.049490 | 6.34 | 0.1362 |
| Error: MS(Error) | 2 | 0.015605 | 0.007802 | | |

Comparison: A vs B

Dependent Variable: V<sub>d</sub>/F/kg (L/kg) Weight Group: 63-75

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_VZFOW

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------|-----------|-------------|-------------|---------|--------|
| sequence | 1 | 0.011948 | 0.011948 | 0.24 | 0.6718 |
| Error | 2 | 0.098979 | 0.049490 | | |
| Error: MS(s | subject(s | sequence)) | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 0.101033 | 0.101033 | 12.95 | 0.0693 |
| trt | 1 | 0.050156 | 0.050156 | 6.43 | 0.1267 |
| subject(sequence) | 2 | 0.098979 | 0.049490 | 6.34 | 0.1362 |
| Error: MS(Error) | 2 | 0.015605 | 0.007802 | | - |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_VZFOW

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------|-----------|------------|-------------|---------|--------|
| sequence | 1 | 0.011948 | 0.011948 | 0.24 | 0.6718 |
| Error | 2 | 0.098979 | 0.049490 | | |
| Error: MS(s | subject(s | sequence)) | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.101033 | 0.101033 | 12.95 | 0.0693 |
| trt | 1 | 0.050156 | 0.050156 | 6.43 | 0.1267 |
| subject(sequence) | 2 | 0.098979 | 0.049490 | 6.34 | 0.1362 |
| Error: MS(Error) | 2 | 0.015605 | 0.007802 | | |

Comparison: A vs B

Dependent Variable: V<sub>d</sub>/F/kg (L/kg) Weight Group: 63-75

#### Least Squares Means

| | | H0:LSN | Mean1=LSMean2 | |
|---|---|---|---|---|
| trt | LN_VZFOW LSMEAN | | | Pr > t |
| A | 0.78908533 | | | 0.126 |
| В | 0.94744593 | | | |
| trt | LN_VZFOW LSMEAN | | Confidence Limits | |
| trt A | LN_VZFOW LSMEAN<br>0.789085<br>0.947446 | 90%<br>0.660123<br>0.818484 | 0.918048<br>1.076408 | |

Least Squares Means for Effect trtDifference BetweenijMeans90% Confidence Limits for LSMean(i)-LSMean(j)12-0.158361-0.3407410.024020

Dependent Variable: LN\_VZFOW

| | | Standard | | |
|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t 90% Confidence Limits |
| A - B | -0.15836060 | 0.06245926 | -2.54 | 0.1267-0.34074073 |

Comparison: A vs B

Dependent Variable: V<sub>d</sub>/F (L) Weight Group: 63-75

| Class Level Info | Levels | Values | |
|------------------|----------------|-----------------|---|
| subject | 4 | 202 303 408 413 | |
| sequence | 2 | AB BA | |
| period | 2 | 1 2 | |
| trt | 2 | A B | |
| Number of Obse | ervations Read | | 8 |
| Number of Obse | rvations Used | | 8 |
Comparison: A vs B

Dependent Variable: V<sub>d</sub>/F (L) Weight Group: 63-75

#### The GLM Procedure

Dependent Variable: LN\_VZFO

| R-Square | Coeff Var | Root MSF | 3 | LN_V | ZFO Mean |
|---|---|---|---|---|---|
| 0.940999 | 1.738447 | 0.088331 | 5.081013 | | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.02347924 | 0.02347924 | 3.01 | 0.2249 |
| period | 1 | 0.10103255 | 0.10103255 | 12.95 | 0.0693 |
| trt | 1 | 0.05015616 | 0.05015616 | 6.43 | 0.1267 |
| subject(sequence) | 2 | 0.07420835 | 0.03710417 | 4.76 | 0.1737 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.02347924 | 0.02347924 | 3.01 | 0.2249 |
| period | 1 | 0.10103255 | 0.10103255 | 12.95 | 0.0693 |
| trt | 1 | 0.05015616 | 0.05015616 | 6.43 | 0.1267 |
| subject(sequence) | 2 | 0.07420835 | 0.03710417 | 4.76 | 0.1737 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.02347924 | 0.02347924 | 3.01 | 0.2249 |
| period | 1 | 0.10103255 | 0.10103255 | 12.95 | 0.0693 |
| trt | 1 | 0.05015616 | 0.05015616 | 6.43 | 0.1267 |
| subject(sequence) | 2 | 0.07420835 | 0.03710417 | 4.76 | 0.1737 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.02347924 | 0.02347924 | 3.01 | 0.2249 |
| period | 1 | 0.10103255 | 0.10103255 | 12.95 | 0.0693 |
| trt | 1 | 0.05015616 | 0.05015616 | 6.43 | 0.1267 |
| subject(sequence) | 2 | 0.07420835 | 0.03710417 | 4.76 | 0.1737 |

Comparison: A vs B

Dependent Variable: V<sub>d</sub>/F (L) Weight Group: 63-75

# The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_VZFO

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.023479 | 0.023479 | 0.63 | 0.5097 |
| Error 2 0.074208 0.037104 | | | | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-------------------|----|-----------|-------------|---------|--------|
| period | 1 | 0.101033 | 0.101033 | 12.95 | 0.0693 |
| trt | 1 | 0.050156 | 0.050156 | 6.43 | 0.1267 |
| subject(sequence) | 2 | 0.074208 | 0.037104 | 4.76 | 0.1737 |
| Error: MS(Error) | 2 | 0.015605 | 0.007802 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN VZFO

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.023479 | 0.023479 | 0.63 | 0.5097 |
| Error 2 0.074208 0.037104 | | | | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.101033 | 0.101033 | 12.95 | 0.0693 |
| trt | 1 | 0.050156 | 0.050156 | 6.43 | 0.1267 |
| subject(sequence) | 2 | 0.074208 | 0.037104 | 4.76 | 0.1737 |
| Error: MS(Error) | 2 | 0.015605 | 0.007802 | | |

Comparison: A vs B

Dependent Variable: V<sub>d</sub>/F (L) Weight Group: 63-75

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_VZFO

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.023479 | 0.023479 | 0.63 | 0.5097 |
| Error 2 0.074208 0.037104 | | | | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 0.101033 | 0.101033 | 12.95 | 0.0693 |
| trt | 1 | 0.050156 | 0.050156 | 6.43 | 0.1267 |
| subject(sequence) | 2 | 0.074208 | 0.037104 | 4.76 | 0.1737 |
| Error: MS(Error) | 2 | 0.015605 | 0.007802 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_VZFO

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.023479 | 0.023479 | 0.63 | 0.5097 |
| Error | 2 | 0.074208 | 0.037104 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.101033 | 0.101033 | 12.95 | 0.0693 |
| trt | 1 | 0.050156 | 0.050156 | 6.43 | 0.1267 |
| subject(sequence) | 2 | 0.074208 | 0.037104 | 4.76 | 0.1737 |
| Error: MS(Error) | 2 | 0.015605 | 0.007802 | | |

Comparison: A vs B

Dependent Variable: V<sub>d</sub>/F (L) Weight Group: 63-75

#### Least Squares Means

| | | Н | 0:LSMean1=LSMean2 | _ |
|-----|----------------|----------|-----------------------|---------|
| trt | LN_VZFO LSMEAN | | | Pr > t |
| A | 5.00183256 | | | 0.1267 |
| В | 5.16019315 | | | |
| | | | | _ |
| trt | LN_VZFO LSMEAN | | 90% Confidence Limits | - |
| A | 5.001833 | 4.872870 | 5.130795 | - |
| В | 5.160193 | 5.031231 | 5.289155 | |

| Le | Least Squares Means for Effect trt | | | |
|---|---|---|---|---|
| | | Difference Between | | |
| i | j | Means | 90% Confid | ence Limits for LSMean(i)-LSMean(j) |
| 1 | 2 | -0.158361 | -0.340741 | 0.024020 |

#### Dependent Variable: LN\_VZFO

| | | Standard | | |
|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t 90% Confidence Limits |
| A - B | -0.15836060 | 0.06245926 | -2.54 | 0.1267-0.34074073 |

Comparison: A vs B

Dependent Variable: T<sub>max</sub> (h) Weight Group: 63-75

| Class Level Info | | 37 1 | |
|------------------|---------------|-----------------|---|
| Class | Levels | Values | |
| subject | 4 | 202 303 408 413 | |
| sequence | 2 | AB BA | |
| period | 2 | 1 2 | |
| trt | 2 | A B | |
| Number of Obse | rvations Read | | 8 |
| Number of Obse | 8 | | |

Comparison: A vs B

Dependent Variable: T<sub>max</sub> (h) Weight Group: 63-75

#### The GLM Procedure

| R-Square | Coeff Var | Root | MSE | 7 | MAX Mean |
|---|---|---|---|---|---|
| 0.688311 | 116.3511 | 1.243 | 502 | 1.068750 | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 1.51728200 | 1.51728200 | 0.98 | 0.4263 |
| period | 1 | 1.54528200 | 1.54528200 | 1.00 | 0.4228 |
| trt | 1 | 1.48781250 | 1.48781250 | 0.96 | 0.4301 |
| subject(sequence) | 2 | 2.27909450 | 1.13954725 | 0.74 | 0.5757 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 1.51728200 | 1.51728200 | 0.98 | 0.4263 |
| period | 1 | 1.54528200 | 1.54528200 | 1.00 | 0.4228 |
| trt | 1 | 1.48781250 | 1.48781250 | 0.96 | 0.4301 |
| subject(sequence) | 2 | 2.27909450 | 1.13954725 | 0.74 | 0.5757 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 1.51728200 | 1.51728200 | 0.98 | 0.4263 |
| period | 1 | 1.54528200 | 1.54528200 | 1.00 | 0.4228 |
| trt | 1 | 1.48781250 | 1.48781250 | 0.96 | 0.4301 |
| subject(sequence) | 2 | 2.27909450 | 1.13954725 | 0.74 | 0.5757 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 1.51728200 | 1.51728200 | 0.98 | 0.4263 |
| period | 1 | 1.54528200 | 1.54528200 | 1.00 | 0.4228 |
| trt | 1 | 1.48781250 | 1.48781250 | 0.96 | 0.4301 |
| subject(sequence) | 2 | 2.27909450 | 1.13954725 | 0.74 | 0.5757 |

Comparison: A vs B

Dependent Variable: T<sub>max</sub> (h) Weight Group: 63-75

## The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: TMAX

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 1.517282 | 1.517282 | 1.33 | 0.3678 |
| Error 2 2.279094 1.139547 | | | | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-------------------|----|-----------|-------------|---------|--------|
| period | 1 | 1.545282 | 1.545282 | 1.00 | 0.4228 |
| trt | 1 | 1.487813 | 1.487813 | 0.96 | 0.4301 |
| subject(sequence) | 2 | 2.279095 | 1.139547 | 0.74 | 0.5757 |
| Error: MS(Error) | 2 | 3.092595 | 1.546297 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------|----------|------------|-------------|---------|--------|
| sequence | 1 | 1.517282 | 1.517282 | 1.33 | 0.3678 |
| Error | 2 | 2.279094 | 1.139547 | | _ |
| Error: MS(s | ubject(s | equence)) | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 1.545282 | 1.545282 | 1.00 | 0.4228 |
| trt | 1 | 1.487813 | 1.487813 | 0.96 | 0.4301 |
| subject(sequence) | 2 | 2.279095 | 1.139547 | 0.74 | 0.5757 |
| Error: MS(Error) | 2 | 3.092595 | 1.546297 | | |

Comparison: A vs B

Dependent Variable: T<sub>max</sub> (h) Weight Group: 63-75

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: TMAX

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 1.517282 | 1.517282 | 1.33 | 0.3678 |
| Error | 2 | 2.279094 | 1.139547 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 1.545282 | 1.545282 | 1.00 | 0.4228 |
| trt | 1 | 1.487813 | 1.487813 | 0.96 | 0.4301 |
| subject(sequence) | 2 | 2.279095 | 1.139547 | 0.74 | 0.5757 |
| Error: MS(Error) | 2 | 3.092595 | 1.546297 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 1.517282 | 1.517282 | 1.33 | 0.3678 |
| Error | 2 | 2.279094 | 1.139547 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 1.545282 | 1.545282 | 1.00 | 0.4228 |
| trt | 1 | 1.487813 | 1.487813 | 0.96 | 0.4301 |
| subject(sequence) | 2 | 2.279095 | 1.139547 | 0.74 | 0.5757 |
| Error: MS(Error) | 2 | 3.092595 | 1.546297 | | |

Comparison: A vs B

Dependent Variable: T<sub>max</sub> (h) Weight Group: 63-75

#### Least Squares Means

| | | 110.1.6 | | |
|---|---|---|---|---|
| | | H0:LS | SMean1=LSMean2 | |
| trt | TMAX LSMEAN | | | Pr > t |
| A | 1.50000000 | | | 0.4301 |
| В | 0.63750000 | | | |
| trt | TMAX LSMEAN | 909 | % Confidence Limits | |
| A | 1.500000 | -0.315504 | 3.315504 | |
| В | 0.637500 | -1.178004 | 2.453004 | |
| Le | ast Squares Means for Effec | et trt | | |
| | Difference Between | | | |
| i | j Means | 90% Confidence Limi | ts for LSMean(i)-LSM | Iean(j) |
| 1 | 2 0.862500 | -1 705010 | 3.430010 | |

| | | Standard | | | |
|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confidence Limits |
| A - B | 0.86250000 | 0.87928870 | 0.98 | 0.4301-1 | .70501034 3.43001034 |

Comparison: A vs B

Dependent Variable: K<sub>el</sub> (/h) Weight Group: 63-75

| Class Level Info | Levels | Values | |
|------------------|----------------|-----------------|---|
| subject | 4 | 202 303 408 413 | |
| sequence | 2 | AB BA | |
| period | 2 | 1 2 | |
| trt | 2 | A B | |
| Number of Obse | ervations Read | | 8 |
| Number of Obse | rvations Used | | 8 |

Comparison: A vs B

Dependent Variable: K<sub>el</sub> (/h) Weight Group: 63-75

#### The GLM Procedure

| R-Square | Coeff Var | Root | MSE | | LAMZ Mean |
|---|---|---|---|---|---|
| 0.948689 | 21.40862 | 0.00 | 4371 | 0.020416 | _ |
| Source | DF | Type I SS | Mean Square | F Value | $\frac{1}{2}$ $\frac{1}$ |
| sequence | 1 | 0.00009919 | 0.00009919 | 5.19 | 0.1503 |
| period | 1 | 0.00003519 | 0.00002579 | 1.35 | 0.3652 |
| trt | 1 | 0.00003954 | 0.00003954 | 2.07 | 0.2868 |
| subject(sequence) | 2 | 0.00054187 | 0.00027093 | 14.18 | 0.0659 |
| <u>sucject(sequence)</u> | <del>_</del> | 0.0000 1107 | 0.00027092 | 1 1.10 | 0.0005 |
| Source | DF | Type II SS | Mean Square | F Value | e $Pr > F$ |
| sequence | 1 | 0.00009919 | 0.00009919 | 5.19 | 0.1503 |
| period | 1 | 0.00002579 | 0.00002579 | 1.35 | 0.3652 |
| trt | 1 | 0.00003954 | 0.00003954 | 2.07 | 0.2868 |
| subject(sequence) | 2 | 0.00054187 | 0.00027093 | 14.18 | 0.0659 |
| Source | DF | Type III SS | Mean Square | | |
| sequence | 1 | 0.00009919 | 0.00009919 | 5.19 | 0.1503 |
| period | 1 | 0.00002579 | 0.00002579 | 1.35 | 0.3652 |
| trt | 1 | 0.00003954 | 0.00003954 | 2.07 | 0.2868 |
| subject(sequence) | 2 | 0.00054187 | 0.00027093 | 14.18 | 0.0659 |
| <u> </u> | DE | T. W.CC | M C | F 1/ 1 | D v E |
| Source | DF | Type IV SS | Mean Square | | |
| sequence | 1 | 0.00009919 | 0.00009919 | 5.19 | 0.1503 |
| period | 1 | 0.00002579 | 0.00002579 | 1.35 | 0.3652 |
| trt | 1 | 0.00003954 | 0.00003954 | 2.07 | 0.2868 |
| subject(sequence) | 2 | 0.00054187 | 0.00027093 | 14.18 | 0.0659 |

Comparison: A vs B

Dependent Variable: K<sub>el</sub> (/h) Weight Group: 63-75

# The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LAMZ

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.000099193 | 0.000099193 | 0.37 | 0.6066 |
| Error 2 0.000542 0.000271 | | | | | |
| Error: MS(s | subject( | sequence)) | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 0.000025787 | 0.000025787 | 1.35 | 0.3652 |
| trt | 1 | 0.000039543 | 0.000039543 | 2.07 | 0.2868 |
| subject(sequence) | 2 | 0.000542 | 0.000271 | 14.18 | 0.0659 |
| Error: MS(Error) | 2 | 0.000038206 | 0.000019103 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------|----------|-------------|-------------|---------|--------|
| sequence | 1 | 0.000099193 | 0.000099193 | 0.37 | 0.6066 |
| Error | 2 | 0.000542 | 0.000271 | | |
| Error: MS(s | subject( | sequence)) | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 0.000025787 | 0.000025787 | 1.35 | 0.3652 |
| trt | 1 | 0.000039543 | 0.000039543 | 2.07 | 0.2868 |
| subject(sequence) | 2 | 0.000542 | 0.000271 | 14.18 | 0.0659 |
| Error: MS(Error) | 2 | 0.000038206 | 0.000019103 | | |

Comparison: A vs B

Dependent Variable: K<sub>el</sub> (/h) Weight Group: 63-75

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LAMZ

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.000099193 | 0.000099193 | 0.37 | 0.6066 |
| Error | | | | | |
| Error: MS(s | Error: MS(subject(sequence)) | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 0.000025787 | 0.000025787 | 1.35 | 0.3652 |
| trt | 1 | 0.000039543 | 0.000039543 | 2.07 | 0.2868 |
| subject(sequence) | 2 | 0.000542 | 0.000271 | 14.18 | 0.0659 |
| Error: MS(Error) | 2 | 0.000038206 | 0.000019103 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------|----------|-------------|-------------|---------|--------|
| sequence | 1 | 0.000099193 | 0.000099193 | 0.37 | 0.6066 |
| Error | 2 | 0.000542 | 0.000271 | | |
| Error: MS(s | subject( | sequence)) | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 0.000025787 | 0.000025787 | 1.35 | 0.3652 |
| trt | 1 | 0.000039543 | 0.000039543 | 2.07 | 0.2868 |
| subject(sequence) | 2 | 0.000542 | 0.000271 | 14.18 | 0.0659 |
| Error: MS(Error) | 2 | 0.000038206 | 0.000019103 | | |

Comparison: A vs B

Dependent Variable: K<sub>el</sub> (/h) Weight Group: 63-75

#### Least Squares Means

| | | | H0:LSM | ean1=LSMean2 | |
|---|---|---|---|---|---|
| trt | LAMZ LSMEAN | | | | Pr > t |
| A | 0.02263887 | | | | 0.2868 |
| В | 0.01819235 | | | | |
| trt | LAMZ LSMEAN | | 90% | Confidence Limits | |
| A | 0.022639 | 0.01 | 5258 | 0.029020 | |
| В | 0.018192 | 0.01 | 1811 | 0.024574 | |
| Le | ast Squares Means for Effec | et trt | | | |
| | Difference Between | | | | |
| i | j Means | 90% Confidence | e Limits f | for LSMean(i)-LSM | Iean(j) |
| 1 | 2 0.004447 | -0.004578 | | 0.013471 | |

#### Dependent Variable: LAMZ

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confi | dence Limits |
| A - B | 0.00444652 | 0.00309055 | 1.44 | 0.2868-0 | 0.00457784 | 0.01347089 |

Comparison: A vs B

Dependent Variable: T<sub>1/2 el</sub> (h) Weight Group: 63-75

| Class Level Info | rmation | | |
|---|---|---|---|
| Class | Levels | Values | |
| subject | 4 | 202 303 408 413 | |
| sequence | 2 | AB BA | |
| period | 2 | 1 2 | |
| trt | 2 | A B | |
| Number of Obse | Number of Observations Read | | |
| Number of Obse | rvations Used | | 8 |

Comparison: A vs B

Dependent Variable: T<sub>1/2 el</sub> (h) Weight Group: 63-75

#### The GLM Procedure

| R-Square | Coeff Var | Root MSI | Ξ | LAMZ | ZHL Mean |
|---|---|---|---|---|---|
| 0.992313 | 7.735473 | 3.247983 | 41.9881 | 16 | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 402.676341 | 402.676341 | 38.17 | 0.0252 |
| period | 1 | 43.461721 | 43.461721 | 4.12 | 0.1795 |
| trt | 1 | 22.577445 | 22.577445 | 2.14 | 0.2810 |
| subject(sequence) | ) 2 | 2254.889672 | 1127.444836 | 106.87 | 0.0093 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 402.676341 | 402.676341 | 38.17 | 0.0252 |
| period | 1 | 43.461721 | 43.461721 | 4.12 | 0.1795 |
| trt | 1 | 22.577445 | 22.577445 | 2.14 | 0.2810 |
| subject(sequence) | ) 2 | 2254.889672 | 1127.444836 | 106.87 | 0.0093 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 402.676341 | 402.676341 | 38.17 | 0.0252 |
| period | 1 | 43.461721 | 43.461721 | 4.12 | 0.1795 |
| trt | 1 | 22.577445 | 22.577445 | 2.14 | 0.2810 |
| subject(sequence) | ) 2 | 2254.889672 | 1127.444836 | 106.87 | 0.0093 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 402.676341 | 402.676341 | 38.17 | 0.0252 |
| period | 1 | 43.461721 | 43.461721 | 4.12 | 0.1795 |
| trt | 1 | 22.577445 | 22.577445 | 2.14 | 0.2810 |
| subject(sequence) | ) 2 | 2254.889672 | 1127.444836 | 106.87 | 0.0093 |

Comparison: A vs B

Dependent Variable: T<sub>1/2 el</sub> (h) Weight Group: 63-75

## The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LAMZHL

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 402.676341 | 402.676341 | 0.36 | 0.6107 |
| Error | 2 | 2254.889672 | 1127.444836 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 43.461721 | 43.461721 | 4.12 | 0.1795 |
| trt | 1 | 22.577445 | 22.577445 | 2.14 | 0.2810 |
| subject(sequence) | 2 | 2254.889672 | 1127.444836 | 106.87 | 0.0093 |
| Error: MS(Error) | 2 | 21.098782 | 10.549391 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 402.676341 | 402.676341 | 0.36 | 0.6107 |
| Error | 2 | 2254.889672 | 1127.444836 | | |
| Error: MS(s | Error: MS(subject(sequence)) | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 43.461721 | 43.461721 | 4.12 | 0.1795 |
| trt | 1 | 22.577445 | 22.577445 | 2.14 | 0.2810 |
| subject(sequence) | 2 | 2254.889672 | 1127.444836 | 106.87 | 0.0093 |
| Error: MS(Error) | 2 | 21.098782 | 10.549391 | | |

Comparison: A vs B

Dependent Variable: T<sub>1/2 el</sub> (h) Weight Group: 63-75

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LAMZHL

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 402.676341 | 402.676341 | 0.36 | 0.6107 |
| Error | 2 | 2254.889672 | 1127.444836 | | _ |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 43.461721 | 43.461721 | 4.12 | 0.1795 |
| trt | 1 | 22.577445 | 22.577445 | 2.14 | 0.2810 |
| subject(sequence) | 2 | 2254.889672 | 1127.444836 | 106.87 | 0.0093 |
| Error: MS(Error) | 2 | 21.098782 | 10.549391 | | - |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 402.676341 | 402.676341 | 0.36 | 0.6107 |
| Error | 2 | 1127.444836 | | | |
| Error: MS(s | Error: MS(subject(sequence)) | | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 43.461721 | 43.461721 | 4.12 | 0.1795 |
| trt | 1 | 22.577445 | 22.577445 | 2.14 | 0.2810 |
| subject(sequence) | 2 | 2254.889672 | 1127.444836 | 106.87 | 0.0093 |
| Error: MS(Error) | 2 | 21.098782 | 10.549391 | | |

Comparison: A vs B

Dependent Variable: T<sub>1/2 el</sub> (h) Weight Group: 63-75

#### Least Squares Means

| | | | H0:LSMean1=LSMean2 | |
|---|---|---|---|---|
| trt | LAMZHL LSMEAN | | | Pr > t |
| A | 40.3082215 | | | 0.2810 |
| В | 43.6680910 | | | |
| | | | 200/ 5 51 | |
| trt | LAMZHL LSMEAN | | 90% Confidence Limits | |
| Α | 40.308222 | 35.566190 | 45.050253 | |
| В | 43.668091 | 38.926060 | 48.410122 | |
| Lea | ast Squares Means for Effec | et trt | | |
| | Difference Between | | | |
| i | j Means | 90% Confide | ence Limits for LSMean(i)-LSM | Mean(j) |
| 1 | 2 -3.359869 | -10.066114 | 3.346375 | |

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confid | lence Limits |
| A - B | -3.35986944 | 2.29667055 | -1.46 | 0.2810-1 | 0.06611433 | 3.34637545 |

Comparison: C vs B

Dependent Variable: AUC<sub>0-t</sub> (h\*ng/mL) Weight Group: 63-75

| Class | Levels | Values | |
|-----------------------|--------|--------|---|
| subject | 1 | 202 | |
| sequence | 1 | BAC | |
| trt | 2 | ВС | |
| N | D I | | 2 |
| Number of Observation | | 2 | |
| Number of Observation | | 2 | |

Comparison: C vs B

Dependent Variable: AUC<sub>0-t</sub> (h\*ng/mL) Weight Group: 63-75

#### The GLM Procedure

Dependent Variable: LN\_AUCLST

| R-Square | Coeff Var | Root MSE | | LN_AUCI | ST Mean |
|------------------|-----------|-------------|-------------|---------|---------|
| 1.000000 | | | 8.989924 | | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.00000000 | | | |
| trt | 1 | 0.00749245 | 0.00749245 | | |
| subject(sequence | e) 0 | 0.00000000 | | | |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.00000000 | | | |
| trt | 1 | 0.00749245 | 0.00749245 | | |
| subject(sequence | e) 0 | 0.00000000 | | | |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.00000000 | | | |
| trt | 1 | 0.00749245 | 0.00749245 | | |
| subject(sequence | e) 0 | 0.00000000 | | | |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.00000000 | | | • |
| trt | 1 | 0.00749245 | 0.00749245 | | |
| subject(sequence | e) 0 | 0.00000000 | | | |
| | ee) 0 | | 0.00749243 | | |

Comparison: C vs B

Dependent Variable: AUC<sub>0-t</sub> (h\*ng/mL) Weight Group: 63-75

#### The GLM Procedure Least Squares Means

| | | H0:LSMean1=LSMean2 |
|---|---|---|
| trt | LN_AUCLST LSMEAN | Pr > t |
| В | 8.92871712 | |
| C | 9.05112994 | |
| trt | LN_AUCLST LSMEAN | 90% Confidence Limits |
| В | 8.928717 | |
| C | 9.051130 | |
| Lar | est Squares Means for Effect t | ert. |
| Lea | ast Squares Means for Effect t | 11 |
| | Difference Between | |
| <u>i</u> | j Means | 90% Confidence Limits for LSMean(i)-LSMean(j) |
| 1 | 2 -0.122413 | |

#### The GLM Procedure

Dependent Variable: LN\_AUCLST

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Conf | idence Limits |
| C - B | 0.12241283 | | | 0. | .00000000 | 0.00000000 |

Comparison: C vs B

Dependent Variable: AUC<sub>0-inf</sub> (h\*ng/mL) Weight Group: 63-75

| Class Level Informati | ion | | |
|-----------------------|----------|--------|---|
| Class | Levels | Values | |
| subject | 1 | 202 | |
| sequence | 1 | BAC | |
| trt | 2 | ВС | |
| Number of Observation | ons Read | | 2 |
| Number of Observation | 2 | | |

Comparison: C vs B

Dependent Variable: AUC<sub>0-inf</sub> (h\*ng/mL) Weight Group: 63-75

#### The GLM Procedure

Dependent Variable: LN\_AUCIFO

| R-Square | Coeff Var | Root MSE | | LN_AUC | FO Mean |
|-----------------|-----------|-------------|-------------|---------|---------|
| 1.000000 | | | 9.152155 | <u></u> | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.00000000 | | | |
| trt | 1 | 0.05815112 | 0.05815112 | | |
| subject(sequenc | e) 0 | 0.00000000 | | | |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.00000000 | | | |
| trt | 1 | 0.05815112 | 0.05815112 | | |
| subject(sequenc | e) 0 | 0.00000000 | | | |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.00000000 | | | |
| trt | 1 | 0.05815112 | 0.05815112 | | |
| subject(sequenc | e) 0 | 0.00000000 | | | |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.00000000 | | | |
| trt | 1 | 0.05815112 | 0.05815112 | | |
| subject(sequenc | e) 0 | 0.00000000 | | | |

Comparison: C vs B

Dependent Variable: AUC<sub>0-inf</sub> (h\*ng/mL) Weight Group: 63-75

#### The GLM Procedure Least Squares Means

| | | | H0:LSMean1=LSMean2 |
|---|---|---|---|
| trt | L | N_AUCIFO LSMEAN | Pr > t |
| В | 8. | .98163980 | |
| C | 9. | .32267095 | |
| trt | | LN_AUCIFO LSMEAN | 90% Confidence Limits |
| В | | 8.981640 | |
| C | | 9.322671 | |
| Le | ast | Squares Means for Effect | trt |
| | | Difference Between | |
| i | j | Means | 90% Confidence Limits for LSMean(i)-LSMean(j) |
| 1 | 2 | -0.341031 | ., |

#### The GLM Procedure

Dependent Variable: LN\_AUCIFO

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Conf | idence Limits |
| C - B | 0.34103116 | | | 0 | .00000000 | 0.00000000 |

Comparison: C vs B

Dependent Variable: C<sub>max</sub> (ng/mL) Weight Group: 63-75

| Class Level Informati | on | | |
|-----------------------|----------|--------|---|
| Class | Levels | Values | |
| subject | 1 | 202 | |
| sequence | 1 | BAC | |
| trt | 2 | ВС | |
| Number of Observation | ons Read | | 2 |
| Number of Observation | 2 | | |

Comparison: C vs B

Dependent Variable: C<sub>max</sub> (ng/mL) Weight Group: 63-75

#### The GLM Procedure

| R-Square | Coeff Var | Root MSE | | LN_CM | AX Mean |
|------------------|-----------|-------------|-------------|---------|---------|
| 1.000000 | | | 5.618963 | _ | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.00000000 | | | |
| trt | 1 | 0.36116740 | 0.36116740 | | |
| subject(sequence | e) 0 | 0.00000000 | | | |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.00000000 | | | |
| trt | 1 | 0.36116740 | 0.36116740 | | |
| subject(sequence | e) 0 | 0.00000000 | | | |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.00000000 | | | |
| trt | 1 | 0.36116740 | 0.36116740 | | |
| subject(sequence | e) 0 | 0.00000000 | | | |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.00000000 | | | |
| trt | 1 | 0.36116740 | 0.36116740 | | |
| subject(sequence | e) 0 | 0.00000000 | | | |
| subject(sequence | e) 0 | 0.00000000 | | | |

Comparison: C vs B

Dependent Variable: C<sub>max</sub> (ng/mL) Weight Group: 63-75

#### The GLM Procedure Least Squares Means

| | | H0:LSMean1=LSMean2 |
|---|---|---|
| trt | LN_CMAX LSMEAN | Pr > t |
| В | 6.04391467 | |
| C | 5.19401185 | |
| trt | LN_CMAX LSMEAN | 90% Confidence Limits |
| В | 6.043915 | |
| C | 5.194012 | |
| Lea | ast Squares Means for Effect | trt |
| | Difference Between | |
| i | j Means | 90% Confidence Limits for LSMean(i)-LSMean(j) |
| 1 | 2 0.849903 | |

#### The GLM Procedure

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Conf | idence Limits |
| C - B | -0.84990282 | | | 0 | .00000000 | 0.00000000 |

Comparison: C vs B

Dependent Variable: Cl/F/kg ((L/h)/kg) Weight Group: 63-75

| Class Level Informat | | Values | |
|-----------------------------|----------|--------|---|
| Class | Levels | Values | |
| subject | 1 | 202 | |
| sequence | 1 | BAC | |
| trt | 2 | ВС | |
| Number of Observation | ons Read | | 2 |
| Number of Observations Used | | | |

Comparison: C vs B

Dependent Variable: Cl/F/kg ((L/h)/kg) Weight Group: 63-75

#### The GLM Procedure

Dependent Variable: LN\_CLFOW

| R-Square | Coeff Var | Root MSE | | LN_CLF0 | OW Mean |
|-----------------|-----------|-------------|-------------|---------|---------|
| 1.000000 | | | -3.758794 | | |
| | | | | | _ |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.00000000 | | | |
| trt | 1 | 0.05815112 | 0.05815112 | | |
| subject(sequenc | e) 0 | 0.00000000 | | | |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.00000000 | | | |
| trt | 1 | 0.05815112 | 0.05815112 | | |
| subject(sequenc | e) 0 | 0.00000000 | | | |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.00000000 | | | |
| trt | 1 | 0.05815112 | 0.05815112 | | |
| subject(sequenc | e) 0 | 0.00000000 | | | |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.00000000 | • | | |
| trt | 1 | 0.05815112 | 0.05815112 | | |
| subject(sequenc | e) 0 | 0.00000000 | | | |

Comparison: C vs B

Dependent Variable: Cl/F/kg ((L/h)/kg) Weight Group: 63-75

#### The GLM Procedure Least Squares Means

| | | | H0:LSMean1=LSMean2 |
|---|---|---|---|
| trt | L | N_CLFOW LSMEAN | Pr > t |
| В | -3 | 3.58827888 | |
| C | -3 | 3.92931004 | |
| trt | | LN_CLFOW LSMEAN | 90% Confidence Limits |
| В | | -3.588279 | |
| C | | -3.929310 | |
| T . | 4 1 | C M C ECC / A | |
| Lea | ast | Squares Means for Effect tr | Ţ |
| | | Difference Between | |
| i | j | Means | 90% Confidence Limits for LSMean(i)-LSMean(j) |
| 1 | 2 | 0.341031 | |

#### The GLM Procedure

Dependent Variable: LN\_CLFOW

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Conf | idence Limits |
| C - B | -0.34103116 | | | 0 | .00000000 | 0.00000000 |

Comparison: C vs B

Dependent Variable: Cl/F (L/h) Weight Group: 63-75

| Class Level Informati | on | | |
|-----------------------|----------|--------|---|
| Class | Levels | Values | |
| subject | 1 | 202 | |
| sequence | 1 | BAC | |
| trt | 2 | ВС | |
| Number of Observation | ons Read | | 2 |
| Number of Observation | ons Used | | 2 |

Comparison: C vs B

Dependent Variable: Cl/F (L/h) Weight Group: 63-75

#### The GLM Procedure

Dependent Variable: LN\_CLFO

| R-Square | Coeff Var | Root MS | Е | LN_CL | FO Mean |
|------------------|-----------|-------------|-------------|---------|---------|
| 1.000000 | | | 0.46365 | 50 | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.00000000 | | | |
| trt | 1 | 0.05815112 | 0.05815112 | | |
| subject(sequence | e) 0 | 0.00000000 | | | |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.00000000 | | | |
| trt | 1 | 0.05815112 | 0.05815112 | | |
| subject(sequence | e) 0 | 0.00000000 | | | |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.00000000 | | | |
| trt | 1 | 0.05815112 | 0.05815112 | | |
| subject(sequence | e) 0 | 0.00000000 | | | |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.00000000 | | | |
| trt | 1 | 0.05815112 | 0.05815112 | | |
| subject(sequence | e) 0 | 0.00000000 | | | |

Comparison: C vs B

Dependent Variable: Cl/F (L/h) Weight Group: 63-75

#### The GLM Procedure Least Squares Means

| | | | H0:LSMean1=LSMean2 |
|---|---|---|---|
| trt | L | N_CLFO LSMEAN | Pr > t |
| В | 0 | .63416568 | |
| C | 0 | .29313453 | |
| trt | | LN_CLFO LSMEAN | 90% Confidence Limits |
| В | | 0.634166 | |
| C | | 0.293135 | |
| Le | ast | Squares Means for Effect t | art . |
| | | Difference Between | |
| i | j | Means | 90% Confidence Limits for LSMean(i)-LSMean(j) |
| 1 | 2 | 0.341031 | · |

#### The GLM Procedure

Dependent Variable: LN\_CLFO

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confi | idence Limits |
| C - B | -0.34103116 | | | 0. | .00000000 | 0.00000000 |

Comparison: C vs B

Dependent Variable: V<sub>d</sub>/F/kg (L/kg) Weight Group: 63-75

| Class Level Information | on | | |
|-------------------------|---------|--------|---|
| Class | Levels | Values | |
| subject | 1 | 202 | |
| sequence | 1 | BAC | |
| trt | 2 | ВС | |
| Number of Observatio | ns Read | | 2 |
| Number of Observatio | ns Used | | 2 |

Comparison: C vs B

Dependent Variable: V<sub>d</sub>/F/kg (L/kg) Weight Group: 63-75

#### The GLM Procedure

Dependent Variable: LN\_VZFOW

| R-Square | Coeff Var | Root MSE | | LN_VZFC | W Mean |
|------------------|-----------|-------------|-------------|---------|--------|
| 1.000000 | | | 1.259065 | _ | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.00000000 | | | |
| trt | 1 | 0.17042279 | 0.17042279 | | |
| subject(sequence | ce) 0 | 0.00000000 | | | |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.00000000 | | | |
| trt | 1 | 0.17042279 | 0.17042279 | | |
| subject(sequence | ce) 0 | 0.00000000 | | | |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.00000000 | | | |
| trt | 1 | 0.17042279 | 0.17042279 | | |
| subject(sequence | ce) 0 | 0.00000000 | | | |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.00000000 | | | |
| trt | 1 | 0.17042279 | 0.17042279 | | |
| subject(sequence | ce) 0 | 0.00000000 | | | |
Comparison: C vs B

Dependent Variable: V<sub>d</sub>/F/kg (L/kg) Weight Group: 63-75

#### The GLM Procedure Least Squares Means

| | | | H0:LSMean1=LSMean2 |
|---|---|---|---|
| trt | L | N_VZFOW LSMEAN | Pr > t |
| В | 0. | .96715507 | |
| C | 1. | .55097489 | |
| trt | | LN_VZFOW LSMEAN | 90% Confidence Limits |
| В | | 0.967155 | |
| C | | 1.550975 | |
| Les | act ' | Squares Means for Effect tr | t · |
| LCC | ast i | Difference Between | ı |
| i | ; | Means | 90% Confidence Limits for LSMean(i)-LSMean(j) |
| 1 | <u>J</u> | | 30/0 Confidence Limits for Estrican(1)-Estrican(1) |
| I | 2 | -0.583820 | |

#### The GLM Procedure

Dependent Variable: LN\_VZFOW

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Conf | idence Limits |
| C - B | 0.58381983 | | | 0. | .00000000 | 0.00000000 |

Comparison: C vs B

Dependent Variable: V<sub>d</sub>/F (L) Weight Group: 63-75

| Class | Levels | Values | |
|-----------------------|----------|--------|---|
| subject | 1 | 202 | |
| sequence | 1 | BAC | |
| trt | 2 | ВС | |
| N | D I | | 2 |
| Number of Observation | ons Read | | 2 |
| Number of Observation | | | |

Comparison: C vs B

Dependent Variable: V<sub>d</sub>/F (L) Weight Group: 63-75

#### The GLM Procedure

Dependent Variable: LN\_VZFO

| R-Square | Coeff Var | Root MSE | | $LN_VZ$ | FO Mean |
|------------------|-----------|-------------|-------------|---------|---------|
| 1.000000 | | | 5.481510 | | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.00000000 | | | |
| trt | 1 | 0.17042279 | 0.17042279 | | |
| subject(sequence | e) 0 | 0.00000000 | | | |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.00000000 | | | |
| trt | 1 | 0.17042279 | 0.17042279 | | |
| subject(sequence | e) 0 | 0.00000000 | | | |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.00000000 | | | |
| trt | 1 | 0.17042279 | 0.17042279 | | |
| subject(sequence | e) 0 | 0.00000000 | | | |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.00000000 | | | • |
| trt | 1 | 0.17042279 | 0.17042279 | | |
| subject(sequence | e) 0 | 0.00000000 | | | |

Comparison: C vs B

Dependent Variable: V<sub>d</sub>/F (L) Weight Group: 63-75

#### The GLM Procedure Least Squares Means

| | | | H0:LSMean1=LSMean2 |
|---|---|---|---|
| trt | L | N_VZFO LSMEAN | Pr > t |
| В | 5 | .18959963 | |
| C | 5 | .77341946 | |
| trt | | LN_VZFO LSMEAN | 90% Confidence Limits |
| В | | 5.189600 | |
| C | | 5.773419 | |
| Le | ast | Squares Means for Effect | trt |
| | | Difference Between | |
| i | j | Means | 90% Confidence Limits for LSMean(i)-LSMean(j) |
| 1 | 2 | -0.583820 | |

#### The GLM Procedure

Dependent Variable: LN\_VZFO

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Conf | idence Limits |
| C - B | 0.58381983 | | | 0. | .00000000 | 0.00000000 |

Comparison: C vs B

Dependent Variable: T<sub>max</sub> (h) Weight Group: 63-75

| Class Level Informati | ion | | |
|-----------------------|----------|--------|---|
| Class | Levels | Values | |
| subject | 1 | 202 | |
| sequence | 1 | BAC | |
| trt | 2 | ВС | |
| Number of Observation | ons Read | | 2 |
| Number of Observation | ons Used | | 2 |

Comparison: C vs B

Dependent Variable: T<sub>max</sub> (h) Weight Group: 63-75

#### The GLM Procedure

| R-Square | Coeff Var | Root | MSE | TMAX Mean | |
|---|---|---|---|---|---|
| 1.000000 | | | 1.3 | 75000 | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.00000000 | | | |
| trt | 1 | 0.78125000 | 0.78125000 | | |
| subject(sequence) | 0 | 0.00000000 | | | |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.00000000 | | | |
| trt | 1 | 0.78125000 | 0.78125000 | | |
| subject(sequence) | 0 | 0.00000000 | | | |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.00000000 | | | |
| trt | 1 | 0.78125000 | 0.78125000 | | |
| subject(sequence) | 0 | 0.00000000 | | | |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.00000000 | _ | | |
| trt | 1 | 0.78125000 | 0.78125000 | | |
| subject(sequence) | 0 | 0.00000000 | | | |

Comparison: C vs B

Dependent Variable: T<sub>max</sub> (h) Weight Group: 63-75

#### The GLM Procedure Least Squares Means

| _ | | | H0:LSMean1=LSMean2 |
|---|---|---|---|
| trt | TI | MAX LSMEAN | Pr > t |
| В | 0. | 75000000 | |
| C | 2.0 | 00000000 | |
| trt | - | TMAX LSMEAN | 90% Confidence Limits |
| В | | 0.750000 | 7070 Confidence Emilits |
| C | | 2.000000 | |
| _ | | a 7.00 | |
| Le | ast : | Squares Means for Effect t | rt |
| | | Difference Between | |
| i | j | Means | 90% Confidence Limits for LSMean(i)-LSMean(j) |
| 1 | 2 | -1.250000 | |

#### The GLM Procedure

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Conf | idence Limits |
| C - B | 1.25000000 | | | 0 | .00000000 | 0.00000000 |

Comparison: C vs B

Dependent Variable: K<sub>el</sub> (/h) Weight Group: 63-75

| Class | Levels | Values | |
|-----------------------|----------|--------|---|
| subject | 1 | 202 | |
| sequence | 1 | BAC | |
| trt | 2 | ВС | |
| N | D I | | 2 |
| Number of Observation | ons Read | | 2 |
| Number of Observation | | | |

Comparison: C vs B

Dependent Variable: K<sub>el</sub> (/h) Weight Group: 63-75

#### The GLM Procedure

Dependent Variable: LAMZ

| R-Square | Coeff Var | Root | MSE | LAMZ Mean | |
|---|---|---|---|---|---|
| 1.000000 | | | 0.0 | 07339 | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.00000000 | | | |
| trt | 1 | 0.00002011 | 0.00002011 | | |
| subject(sequence) | 0 | 0.00000000 | | | |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.00000000 | | | |
| trt | 1 | 0.00002011 | 0.00002011 | | |
| subject(sequence) | 0 | 0.00000000 | | | |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.00000000 | | | |
| trt | 1 | 0.00002011 | 0.00002011 | | |
| subject(sequence) | 0 | 0.00000000 | | | |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.00000000 | | | |
| trt | 1 | 0.00002011 | 0.00002011 | | |
| subject(sequence) | 0 | 0.00000000 | | | |
| · | | · | · | · | |

Comparison: C vs B

Dependent Variable: K<sub>el</sub> (/h) Weight Group: 63-75

#### The GLM Procedure Least Squares Means

| | | | H0:LSMean1=LSMean2 |
|---|---|---|---|
| trt | L | AMZ LSMEAN | Pr > t |
| В | 0. | 01050994 | |
| C | 0. | 00416814 | |
| trt | | LAMZ LSMEAN | 90% Confidence Limits |
| В | | 0.010510 | |
| C | | 0.004168 | |
| Le | ast | Squares Means for Effect tr | 1 |
| | ast | Difference Between | • |
| i | j | Means | 90% Confidence Limits for LSMean(i)-LSMean(j) |
| 1 | 2 | 0.006342 | · |

#### The GLM Procedure

Dependent Variable: LAMZ

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Conf | idence Limits |
| C - B | -0.00634180 | | | 0 | .00000000 | 0.00000000 |

Comparison: C vs B

Dependent Variable: T<sub>1/2 el</sub> (h) Weight Group: 63-75

| Class | Levels | Values | |
|-----------------------|----------|--------|---|
| subject | 1 | 202 | |
| sequence | 1 | BAC | |
| trt | 2 | ВС | |
| Number of Observation | ons Read | | 2 |
| Number of Observation | ons Used | | 2 |

Comparison: C vs B

Dependent Variable: T<sub>1/2 el</sub> (h) Weight Group: 63-75

#### The GLM Procedure

Dependent Variable: LAMZHL

| R-Square | Coeff Var | Root MSE | | LAMZ | HL Mean |
|------------------|-----------|-------------|-------------|---------|---------|
| 1.000000 | | | 116.1240 | 0 | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.000000 | | | |
| trt | 1 | 5034.544709 | 5034.544709 | | |
| subject(sequence | e) 0 | 0.000000 | | | |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.000000 | | | |
| trt | 1 | 5034.544709 | 5034.544709 | | |
| subject(sequence | e) 0 | 0.000000 | | | |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.000000 | | | |
| trt | 1 | 5034.544709 | 5034.544709 | | |
| subject(sequence | e) 0 | 0.000000 | | | |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 0 | 0.000000 | | | |
| trt | 1 | 5034.544709 | 5034.544709 | | |
| subject(sequence | e) 0 | 0.000000 | | | |

Comparison: C vs B

Dependent Variable: T<sub>1/2 el</sub> (h) Weight Group: 63-75

#### The GLM Procedure Least Squares Means

| | | H0:LSMean1=LSMean2 |
|---|---|---|
| trt | LAMZHL LSMEAN | Pr > t |
| В | 65.951593 | |
| C | 166.296445 | |
| trt | LAMZHL LSMEAN | 90% Confidence Limits |
| В | 65.951593 | |
| C | 166.296445 | |
| Le | ast Squares Means for Effect trt | |
| i | j Difference Between Means 90° | % Confidence Limits for LSMean(i)-LSMean(j) |
| 1 | 2 -100.344852 | |

#### The GLM Procedure

Dependent Variable: LAMZHL

| | | Standard | | | |
|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t 90% Conf | idence Limits |
| C - B | 100.344852 | | | 0.000000 | 0.000000 |

Comparison: A vs B

Dependent Variable: AUC<sub>0-t</sub> (h\*ng/mL) Weight Group: 76-87

| Class Level In | Class Level Information | |
|---|---|---|
| Class | Levels | Values |
| subject | 6 | 205 301 406 410 411 501 |
| sequence | 2 | AB BA |
| period | 2 | 1 2 |
| trt | 2 | AΒ |
| Number of Ob | Number of Observations Read 12 | |
| Number of Ob | Number of Observations Used 12 | |

Comparison: A vs B

Dependent Variable: AUC<sub>0-t</sub> (h\*ng/mL) Weight Group: 76-87

#### The GLM Procedure

Dependent Variable: LN\_AUCLST

| R-Square | Coeff Var | Root MSE | | LN_AUC | LST Mean |
|-----------------|-----------|-------------|-------------|---------|----------|
| 0.964977 | 1.738422 | 0.154632 | 8.894970 | | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 1.12739488 | 1.12739488 | 47.15 | 0.0024 |
| period | 1 | 0.02008228 | 0.02008228 | 0.84 | 0.4113 |
| trt | 1 | 0.02193858 | 0.02193858 | 0.92 | 0.3924 |
| subject(sequenc | e) 4 | 1.46581263 | 0.36645316 | 15.33 | 0.0108 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 1.12739488 | 1.12739488 | 47.15 | 0.0024 |
| period | 1 | 0.02008228 | 0.02008228 | 0.84 | 0.4113 |
| trt | 1 | 0.02193858 | 0.02193858 | 0.92 | 0.3924 |
| subject(sequenc | e) 4 | 1.46581263 | 0.36645316 | 15.33 | 0.0108 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 1.12739488 | 1.12739488 | 47.15 | 0.0024 |
| period | 1 | 0.02008228 | 0.02008228 | 0.84 | 0.4113 |
| trt | 1 | 0.02193858 | 0.02193858 | 0.92 | 0.3924 |
| subject(sequenc | e) 4 | 1.46581263 | 0.36645316 | 15.33 | 0.0108 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 1.12739488 | 1.12739488 | 47.15 | 0.0024 |
| period | 1 | 0.02008228 | 0.02008228 | 0.84 | 0.4113 |
| trt | 1 | 0.02193858 | 0.02193858 | 0.92 | 0.3924 |
| subject(sequenc | e) 4 | 1.46581263 | 0.36645316 | 15.33 | 0.0108 |

Comparison: A vs B

Dependent Variable: AUC<sub>0-t</sub> (h\*ng/mL) Weight Group: 76-87

## The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_AUCLST

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 1.127395 | 1.127395 | 3.08 | 0.1543 |
| Error | 4 | 1.465813 | 0.366453 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-------------------|----|-----------|-------------|---------|--------|
| period | 1 | 0.020082 | 0.020082 | 0.84 | 0.4113 |
| trt | 1 | 0.021939 | 0.021939 | 0.92 | 0.3924 |
| subject(sequence) | 4 | 1.465813 | 0.366453 | 15.33 | 0.0108 |
| Error: MS(Error) | 4 | 0.095644 | 0.023911 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN AUCLST

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 1.127395 | 1.127395 | 3.08 | 0.1543 |
| Error | 4 | 1.465813 | 0.366453 | | _ |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.020082 | 0.020082 | 0.84 | 0.4113 |
| trt | 1 | 0.021939 | 0.021939 | 0.92 | 0.3924 |
| subject(sequence) | 4 | 1.465813 | 0.366453 | 15.33 | 0.0108 |
| Error: MS(Error) | 4 | 0.095644 | 0.023911 | | |

Comparison: A vs B

Dependent Variable: AUC<sub>0-t</sub> (h\*ng/mL) Weight Group: 76-87

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_AUCLST

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 1.127395 | 1.127395 | 3.08 | 0.1543 |
| Error 4 1.465813 0.366453 | | | | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 0.020082 | 0.020082 | 0.84 | 0.4113 |
| trt | 1 | 0.021939 | 0.021939 | 0.92 | 0.3924 |
| subject(sequence) | 4 | 1.465813 | 0.366453 | 15.33 | 0.0108 |
| Error: MS(Error) | 4 | 0.095644 | 0.023911 | | - |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_AUCLST

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 1.127395 | 1.127395 | 3.08 | 0.1543 |
| Error 4 1.465813 0.366453 | | | | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.020082 | 0.020082 | 0.84 | 0.4113 |
| trt | 1 | 0.021939 | 0.021939 | 0.92 | 0.3924 |
| subject(sequence) | 4 | 1.465813 | 0.366453 | 15.33 | 0.0108 |
| Error: MS(Error) | 4 | 0.095644 | 0.023911 | | |

Comparison: A vs B

Dependent Variable: AUC<sub>0-t</sub> (h\*ng/mL) Weight Group: 76-87

#### Least Squares Means

| | | H0:LSMean1=LSMean2 | |
|-----|------------------|--------------------|---------|
| trt | LN_AUCLST LSMEAN | | Pr > t |
| A | 8.85221198 | | 0.3924 |
| В | 8.93772725 | | |

| trt | LN_AUCLST LSMEAN | 90% | Confidence Limits |
|-----|------------------|----------|-------------------|
| A | 8.852212 | 8.717632 | 8.986792 |
| В | 8.937727 | 8.803147 | 9.072307 |

| Le | Least Squares Means for Effect trt | | | |
|---|---|---|---|---|
| | | Difference Between | | |
| i | j | Means | 90% Confiden | ce Limits for LSMean(i)-LSMean(j) |
| 1 | 2 | -0.085515 | -0.275840 | 0.104809 |

Dependent Variable: LN\_AUCLST

| • | | Standard | | | | _ |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confid | dence Limits |
| A - B | -0.08551527 | 0.08927691 | -0.96 | 0.3924-0 | ).27583996 | 0.10480942 |

Comparison: A vs B

Dependent Variable: AUC<sub>0-inf</sub> (h\*ng/mL) Weight Group: 76-87

| Class Level In | nformation | |
|--------------------------------|------------|-------------------------|
| Class | Levels | Values |
| subject | 6 | 205 301 406 410 411 501 |
| sequence | 2 | AB BA |
| period | 2 | 1 2 |
| trt | 2 | AΒ |
| Number of Observations Read 12 | | |
| Number of Observations Used 1 | | |

Comparison: A vs B

Dependent Variable: AUC<sub>0-inf</sub> (h\*ng/mL) Weight Group: 76-87

#### The GLM Procedure

Dependent Variable: LN\_AUCIFO

| R-Square | Coeff Var | Root MSE | | LN_AUC | IFO Mean |
|---|---|---|---|---|---|
| 0.963280 | 2.122888 | 0.192833 | 9.083543 | | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 1.57345243 | 1.57345243 | 42.31 | 0.0029 |
| period | 1 | 0.02783629 | 0.02783629 | 0.75 | 0.4357 |
| trt | 1 | 0.00812175 | 0.00812175 | 0.22 | 0.6646 |
| subject(sequence | ee) 4 | 2.29244990 | 0.57311247 | 15.41 | 0.0107 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 1.57345243 | 1.57345243 | 42.31 | 0.0029 |
| period | 1 | 0.02783629 | 0.02783629 | 0.75 | 0.4357 |
| trt | 1 | 0.00812175 | 0.00812175 | 0.22 | 0.6646 |
| subject(sequence | e) 4 | 2.29244990 | 0.57311247 | 15.41 | 0.0107 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 1.57345243 | 1.57345243 | 42.31 | 0.0029 |
| period | 1 | 0.02783629 | 0.02783629 | 0.75 | 0.4357 |
| trt | 1 | 0.00812175 | 0.00812175 | 0.22 | 0.6646 |
| subject(sequence | e) 4 | 2.29244990 | 0.57311247 | 15.41 | 0.0107 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 1.57345243 | 1.57345243 | 42.31 | 0.0029 |
| period | 1 | 0.02783629 | 0.02783629 | 0.75 | 0.4357 |
| trt | 1 | 0.00812175 | 0.00812175 | 0.22 | 0.6646 |
| subject(sequence | e) 4 | 2.29244990 | 0.57311247 | 15.41 | 0.0107 |

Comparison: A vs B

Dependent Variable: AUC<sub>0-inf</sub> (h\*ng/mL) Weight Group: 76-87

## The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_AUCIFO

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 1.573452 | 1.573452 | 2.75 | 0.1729 |
| Error 4 2.292450 0.573112 | | | | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-------------------|----|-----------|-------------|---------|--------|
| period | 1 | 0.027836 | 0.027836 | 0.75 | 0.4357 |
| trt | 1 | 0.008122 | 0.008122 | 0.22 | 0.6646 |
| subject(sequence) | 4 | 2.292450 | 0.573112 | 15.41 | 0.0107 |
| Error: MS(Error) | 4 | 0.148739 | 0.037185 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN AUCIFO

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 1.573452 | 1.573452 | 2.75 | 0.1729 |
| Error | 4 | 2.292450 | 0.573112 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.027836 | 0.027836 | 0.75 | 0.4357 |
| trt | 1 | 0.008122 | 0.008122 | 0.22 | 0.6646 |
| subject(sequence) | 4 | 2.292450 | 0.573112 | 15.41 | 0.0107 |
| Error: MS(Error) | 4 | 0.148739 | 0.037185 | | |

Comparison: A vs B

Dependent Variable: AUC<sub>0-inf</sub> (h\*ng/mL) Weight Group: 76-87

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_AUCIFO

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 1.573452 | 1.573452 | 2.75 | 0.1729 |
| Error | 4 | 2.292450 | 0.573112 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 0.027836 | 0.027836 | 0.75 | 0.4357 |
| trt | 1 | 0.008122 | 0.008122 | 0.22 | 0.6646 |
| subject(sequence) | 4 | 2.292450 | 0.573112 | 15.41 | 0.0107 |
| Error: MS(Error) | 4 | 0.148739 | 0.037185 | | - |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_AUCIFO

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 1.573452 | 1.573452 | 2.75 | 0.1729 |
| Error | 4 | 2.292450 | 0.573112 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.027836 | 0.027836 | 0.75 | 0.4357 |
| trt | 1 | 0.008122 | 0.008122 | 0.22 | 0.6646 |
| subject(sequence) | 4 | 2.292450 | 0.573112 | 15.41 | 0.0107 |
| Error: MS(Error) | 4 | 0.148739 | 0.037185 | | |

Comparison: A vs B

Dependent Variable: AUC<sub>0-inf</sub> (h\*ng/mL) Weight Group: 76-87

#### Least Squares Means

| | | H0:LSMean1=LSMean2 |
|-----|------------------|--------------------|
| trt | LN_AUCIFO LSMEAN | Pr > t |
| A | 9.10955867 | 0.6646 |
| В | 9.05752745 | |

| trt | LN_AUCIFO LSMEAN | | 90% Confidence Limits |
|-----|------------------|----------|-----------------------|
| A | 9.109559 | 8.941731 | 9.277386 |
| В | 9.057527 | 8.889700 | 9.225355 |

| Le | Least Squares Means for Effect trt | | | |
|---|---|---|---|---|
| | | Difference Between | | |
| i | j | Means | 90% Confiden | nce Limits for LSMean(i)-LSMean(j) |
| 1 | 2 | 0.052031 | -0.185312 | 0.289375 |

Dependent Variable: LN\_AUCIFO

| | | Standard | | | |
|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confidence Limits |
| A - B | 0.05203123 | 0.11133243 | 0.47 | 0.6646-0 | 0.18531246 |

Comparison: A vs B

Dependent Variable: C<sub>max</sub> (ng/mL) Weight Group: 76-87

| Class Level I | nformation | |
|--------------------------------|------------|-----------------------------|
| Class | Levels | Values |
| subject | 7 | 205 301 406 410 411 501 506 |
| sequence | 2 | AB BA |
| period | 2 | 1 2 |
| trt | 2 | A B |
| Number of Observations Read 14 | | |
| Number of Observations Used 14 | | |

Comparison: A vs B

Dependent Variable: C<sub>max</sub> (ng/mL) Weight Group: 76-87

#### The GLM Procedure

| R-Square | Coeff Var | Root MSE | | LN_C | MAX Mean |
|---|---|---|---|---|---|
| 0.663147 | 6.456680 | 0.353705 | 5.478128 | | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.14298687 | 0.14298687 | 1.14 | 0.3339 |
| period | 1 | 0.05353200 | 0.05353200 | 0.43 | 0.5419 |
| trt | 1 | 0.48189892 | 0.48189892 | 3.85 | 0.1069 |
| subject(sequence | ) 5 | 0.55304583 | 0.11060917 | 0.88 | 0.5521 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.14298687 | 0.14298687 | 1.14 | 0.3339 |
| period | 1 | 0.10769335 | 0.10769335 | 0.86 | 0.3961 |
| trt | 1 | 0.48189892 | 0.48189892 | 3.85 | 0.1069 |
| subject(sequence | ) 5 | 0.55304583 | 0.11060917 | 0.88 | 0.5521 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.14298687 | 0.14298687 | 1.14 | 0.3339 |
| period | 1 | 0.10769335 | 0.10769335 | 0.86 | 0.3961 |
| trt | 1 | 0.48189892 | 0.48189892 | 3.85 | 0.1069 |
| subject(sequence | ) 5 | 0.55304583 | 0.11060917 | 0.88 | 0.5521 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.14298687 | 0.14298687 | 1.14 | 0.3339 |
| period | 1 | 0.10769335 | 0.10769335 | 0.86 | 0.3961 |
| trt | 1 | 0.48189892 | 0.48189892 | 3.85 | 0.1069 |
| subject(sequence | 5 | 0.55304583 | 0.11060917 | 0.88 | 0.5521 |

Comparison: A vs B

Dependent Variable: C<sub>max</sub> (ng/mL) Weight Group: 76-87

## The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_CMAX

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.142987 | 0.142987 | 1.29 | 0.3071 |
| Error 5 0.55304 | | 0.553046 | 0.110609 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| *period | 1 | 0.053532 | 0.053532 | 0.43 | 0.5419 |
| trt | 1 | 0.481899 | 0.481899 | 3.85 | 0.1069 |
| subject(sequence) | 5 | 0.553046 | 0.110609 | 0.88 | 0.5521 |
| Error: MS(Error) | 5 | 0.625537 | 0.125107 | | |
| * This test assumes one or more other fixed effects are zero. | | | | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.142987 | 0.142987 | 1.29 | 0.3071 |
| Error 5 | | 0.553046 | 0.110609 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.107693 | 0.107693 | 0.86 | 0.3961 |
| trt | 1 | 0.481899 | 0.481899 | 3.85 | 0.1069 |
| subject(sequence) | 5 | 0.553046 | 0.110609 | 0.88 | 0.5521 |
| Error: MS(Error) | 5 | 0.625537 | 0.125107 | | |

Comparison: A vs B

Dependent Variable: C<sub>max</sub> (ng/mL) Weight Group: 76-87

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_CMAX

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.142987 | 0.142987 | 1.29 | 0.3071 |
| Error | 5 | 0.553046 | 0.110609 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 0.107693 | 0.107693 | 0.86 | 0.3961 |
| trt | 1 | 0.481899 | 0.481899 | 3.85 | 0.1069 |
| subject(sequence) | 5 | 0.553046 | 0.110609 | 0.88 | 0.5521 |
| Error: MS(Error) | 5 | 0.625537 | 0.125107 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.142987 | 0.142987 | 1.29 | 0.3071 |
| Error | 5 | 0.553046 | 0.110609 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.107693 | 0.107693 | 0.86 | 0.3961 |
| trt | 1 | 0.481899 | 0.481899 | 3.85 | 0.1069 |
| subject(sequence) | 5 | 0.553046 | 0.110609 | 0.88 | 0.5521 |
| Error: MS(Error) | 5 | 0.625537 | 0.125107 | | |

Comparison: A vs B

Dependent Variable: C<sub>max</sub> (ng/mL) Weight Group: 76-87

#### Least Squares Means

| | | H0:LSI | Mean1=LSMean2 | |
|-----|----------------|----------|---------------------|---------|
| trt | LN_CMAX LSMEAN | | | Pr > t |
| A | 5.30526255 | | | 0.1069 |
| В | 5.68016767 | | | |
| trt | LN_CMAX LSMEAN | 90% | 6 Confidence Limits | |
| A | 5.305263 | 5.033083 | 5.577442 | |
| D | 5.680168 | 5.407988 | 5.952347 | |
| В | | | | |
| В | | | | |

Least Squares Means for Effect trt
Difference Between

| i | j | Means | 90% Confidence I | Limits for LSMean(i)-LSMean(j) |
|---|---|-----------|------------------|--------------------------------|
| 1 | 2 | -0.374905 | -0.759825 | 0.010015 |

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confi | dence Limits |
| A - B | -0.37490513 | 0.19102264 | -1.96 | 0.1069-0 | 0.75982499 | 0.01001474 |

Comparison: A vs B

Dependent Variable: Cl/F/kg ((L/h)/kg) Weight Group: 76-87

| Class Level I | nformation | | |
|---|---|---|---|
| Class | Levels | Values | |
| subject | 7 | 205 301 406 410 411 501 506 | |
| sequence | 2 | AB BA | |
| period | 2 | 1 2 | |
| trt | 2 | A B | |
| Number of O | bservations R | ead | 13 |
| Number of O | Number of Observations Used 13 | | |

Comparison: A vs B

Dependent Variable: Cl/F/kg ((L/h)/kg) Weight Group: 76-87

#### The GLM Procedure

Dependent Variable: LN\_CLFOW

| R-Square | Coeff Var | Root MSE | | LN_CLF | OW Mean |
|------------------|-----------|-------------|-------------|---------|---------|
| 0.966101 | -4.963592 | 0.192833 | -3.884957 | | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 1.04930375 | 1.04930375 | 28.22 | 0.0060 |
| period | 1 | 0.00397640 | 0.00397640 | 0.11 | 0.7601 |
| trt | 1 | 0.32070448 | 0.32070448 | 8.62 | 0.0425 |
| subject(sequence | e) 5 | 2.86497841 | 0.57299568 | 15.41 | 0.0101 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 1.12723610 | 1.12723610 | 30.31 | 0.0053 |
| period | 1 | 0.02783629 | 0.02783629 | 0.75 | 0.4357 |
| trt | 1 | 0.12753294 | 0.12753294 | 3.43 | 0.1377 |
| subject(sequence | e) 5 | 2.86497841 | 0.57299568 | 15.41 | 0.0101 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.70022141 | 0.70022141 | 18.83 | 0.0123 |
| period | 1 | 0.02783629 | 0.02783629 | 0.75 | 0.4357 |
| trt | 1 | 0.12753294 | 0.12753294 | 3.43 | 0.1377 |
| subject(sequence | e) 5 | 2.86497841 | 0.57299568 | 15.41 | 0.0101 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.70022141 | 0.70022141 | 18.83 | 0.0123 |
| period | 1 | 0.02783629 | 0.02783629 | 0.75 | 0.4357 |
| trt | 1 | 0.12753294 | 0.12753294 | 3.43 | 0.1377 |
| subject(sequence | 2) 5 | 2.86497841 | 0.57299568 | 15.41 | 0.0101 |

Comparison: A vs B

Dependent Variable: Cl/F/kg ((L/h)/kg) Weight Group: 76-87

## The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN CLFOW

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-----------|-------|-----------|-------------|---------|--------|
| *sequence | 1 | 1.049304 | 1.049304 | 1.71 | 0.2481 |
| Error | 4.955 | 3.036931 | 0.612903 | | |

Error: 1.0745\*MS(subject(sequence)) - 0.0745\*MS(Error)

<sup>\*</sup> This test assumes one or more other fixed effects are zero.

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---------|--------|-----------|-------------|---------|--------|
| *period | 1 | 0.003976 | 0.003976 | 0.07 | 0.8029 |
| Error | 8.2446 | 0.493559 | 0.059865 | | |

Error: 0.0423\*MS(subject(sequence)) + 0.9577\*MS(Error)

<sup>\*</sup> This test assumes one or more other fixed effects are zero.

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|------------|------------|-----------|-------------|---------|--------|
| trt | 1 | 0.320704 | 0.320704 | 5.62 | 0.0455 |
| Error | 7.9206 | 0.451711 | 0.057030 | | |
| Error: 0.0 | 37*MS(subj | | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-------------------|----|-----------|-------------|---------|--------|
| subject(sequence) | 5 | 2.864978 | 0.572996 | 15.41 | 0.0101 |
| Error: MS(Error) | 4 | 0.148739 | 0.037185 | | |

Comparison: A vs B

Dependent Variable: Cl/F/kg ((L/h)/kg) Weight Group: 76-87

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_CLFOW

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 1.127236 | 1.127236 | 1.84 | 0.2335 |
| Error | 4.9552 | 3.035991 | 0.612685 | | |
| Error: 1.0741*MS(subject(sequence)) - 0.0741*MS(Error) | | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.027836 | 0.027836 | 0.75 | 0.4357 |
| trt | 1 | 0.127533 | 0.127533 | 3.43 | 0.1377 |
| subject(sequence) | 5 | 2.864978 | 0.572996 | 15.41 | 0.0101 |
| Error: MS(Error) | 4 | 0.148739 | 0.037185 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_CLFOW

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.700221 | 0.700221 | 1.25 | 0.3134 |
| Error | 5.0185 | 2.800906 | 0.558112 | | |
| Error: 0.9722*MS(subject(sequence)) + 0.0278*MS(Error) | | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 0.027836 | 0.027836 | 0.75 | 0.4357 |
| trt | 1 | 0.127533 | 0.127533 | 3.43 | 0.1377 |
| subject(sequence) | 5 | 2.864978 | 0.572996 | 15.41 | 0.0101 |
| Error: MS(Error) | 4 | 0.148739 | 0.037185 | | |

Comparison: A vs B

Dependent Variable: Cl/F/kg ((L/h)/kg) Weight Group: 76-87

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_CLFOW

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.700221 | 0.700221 | 1.25 | 0.3134 |
| Error | 5.0185 | 2.800906 | 0.558112 | | |
| Error: 0.9722*MS(subject(sequence)) + 0.0278*MS(Error) | | | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.027836 | 0.027836 | 0.75 | 0.4357 |
| trt | 1 | 0.127533 | 0.127533 | 3.43 | 0.1377 |
| subject(sequence) | 5 | 2.864978 | 0.572996 | 15.41 | 0.0101 |
| Error: MS(Error) | 4 | 0.148739 | 0.037185 | | _ |

Comparison: A vs B

Dependent Variable: Cl/F/kg ((L/h)/kg) Weight Group: 76-87

Means -0.206182

#### Least Squares Means

| | | H | H0:LSMean1=LSMean2 | |
|---|---|---|---|---|
| trt | LN_CLFOW LSMEAN | | | Pr > t |
| A | -4.05335533 | | | 0.1377 |
| В | -3.84717342 | | | |
| trt | LN_CLFOW LSMEAN | | 90% Confidence Limits | |
| A | -4.053355 | -4.210343 | -3.896367 | |
| В | -3.847173 | -4.025181 | -3.669166 | |
| Lea | ast Squares Means for Effect trt<br>Difference Between | | | |

#### Dependent Variable: LN\_CLFOW

-0.443526

90% Confidence Limits for LSMean(i)-LSMean(j)

0.031162

| | | Standard | | |
|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t 90% Confidence Limits |
| A - B | -0.20618191 | 0.11133243 | -1.85 | 0.1377-0.44352559 |

Comparison: A vs B

Dependent Variable: Cl/F (L/h) Weight Group: 76-87

| Class Level I | | |
|---------------|--------|-----------------------------|
| Class | Levels | Values |
| subject | 7 | 205 301 406 410 411 501 506 |
| sequence | 2 | AB BA |
| period | 2 | 1 2 |
| trt | 2 | AB |
| Number of O | 13 | |
| Number of O | 13 | |
Comparison: A vs B

Dependent Variable: Cl/F (L/h) Weight Group: 76-87

#### The GLM Procedure

| R-Square | Coeff Var | Root MSE | | LN_C | LFO Mean |
|---|---|---|---|---|---|
| 0.967079 | 34.30586 | 0.192833 | 0.562101 | | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 1.10473169 | 1.10473169 | 29.71 | 0.0055 |
| period | 1 | 0.00520841 | 0.00520841 | 0.14 | 0.7272 |
| trt | 1 | 0.33042950 | 0.33042950 | 8.89 | 0.0407 |
| subject(sequence) | ) 5 | 2.92899343 | 0.58579869 | 15.75 | 0.0097 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 1.18703340 | 1.18703340 | 31.92 | 0.0048 |
| period | 1 | 0.02783629 | 0.02783629 | 0.75 | 0.4357 |
| trt | 1 | 0.12753294 | 0.12753294 | 3.43 | 0.1377 |
| subject(sequence) | ) 5 | 2.92899343 | 0.58579869 | 15.75 | 0.0097 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.73180313 | 0.73180313 | 19.68 | 0.0114 |
| period | 1 | 0.02783629 | 0.02783629 | 0.75 | 0.4357 |
| trt | 1 | 0.12753294 | 0.12753294 | 3.43 | 0.1377 |
| subject(sequence) | ) 5 | 2.92899343 | 0.58579869 | 15.75 | 0.0097 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.73180313 | 0.73180313 | 19.68 | 0.0114 |
| period | 1 | 0.02783629 | 0.02783629 | 0.75 | 0.4357 |
| trt | 1 | 0.12753294 | 0.12753294 | 3.43 | 0.1377 |
| subject(sequence) | ) 5 | 2.92899343 | 0.58579869 | 15.75 | 0.0097 |

Comparison: A vs B

Dependent Variable: Cl/F (L/h) Weight Group: 76-87

### The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_CLFO

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| *sequence | 1 | 1.104732 | 1.104732 | 1.76 | 0.2421 |
| Error | 4.956 | 3.105712 | 0.626660 | | |
| Error: 1.0745*MS(su | bject(seq | uence)) - 0.074 | 5*MS(Error) | | |

\* This test assumes one or more other fixed effects are zero.

| Sour | rce DF | Type I SS | Mean Square | F Value | Pr > F |
|-------|----------|-----------|-------------|---------|--------|
| *peri | od 1 | 0.005208 | 0.005208 | 0.09 | 0.7763 |
| Erro | r 8.2931 | 0.500957 | 0.060406 | | |

Error: 0.0423\*MS(subject(sequence)) + 0.9577\*MS(Error)

<sup>\*</sup> This test assumes one or more other fixed effects are zero.

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|------------|------------|-----------|-------------|---------|--------|
| trt | 1 | 0.330430 | 0.330430 | 5.75 | 0.0435 |
| Error | 7.9739 | 0.458527 | 0.057504 | | |
| Error: 0.0 | 37*MS(subj | | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-------------------|----|-----------|-------------|---------|--------|
| subject(sequence) | 5 | 2.928993 | 0.585799 | 15.75 | 0.0097 |
| Error: MS(Error) | 4 | 0 148739 | 0.037185 | | |

Comparison: A vs B

Dependent Variable: Cl/F (L/h) Weight Group: 76-87

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_CLFO

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 1.187033 | 1.187033 | 1.89 | 0.2276 |
| Error | 4.9562 | 3.104746 | 0.626437 | | |
| Error: 1.07 | 41*MS(sub | iect(sequence)) - | 0.0741*MS(Error | ) | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.027836 | 0.027836 | 0.75 | 0.4357 |
| trt | 1 | 0.127533 | 0.127533 | 3.43 | 0.1377 |
| subject(sequence) | 5 | 2.928993 | 0.585799 | 15.75 | 0.0097 |
| Error: MS(Error) | 4 | 0.148739 | 0.037185 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.731803 | 0.731803 | 1.28 | 0.3086 |
| Error | 5.0181 | 2.863142 | 0.570559 | | |
| Error: 0.97 | 22*MS(sub | ject(sequence)) + | 0.0278*MS(Error | ) | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 0.027836 | 0.027836 | 0.75 | 0.4357 |
| trt | 1 | 0.127533 | 0.127533 | 3.43 | 0.1377 |
| subject(sequence) | 5 | 2.928993 | 0.585799 | 15.75 | 0.0097 |
| Error: MS(Error) | 4 | 0.148739 | 0.037185 | | |

Comparison: A vs B

Dependent Variable: Cl/F (L/h) Weight Group: 76-87

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.731803 | 0.731803 | 1.28 | 0.3086 |
| Error | 5.0181 | 2.863142 | 0.570559 | | <del></del> i |
| Error: 0.97 | 22*MS(sub | ject(sequence)) + | 0.0278*MS(Error | ) | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.027836 | 0.027836 | 0.75 | 0.4357 |
| trt | 1 | 0.127533 | 0.127533 | 3.43 | 0.1377 |
| subject(sequence) | 5 | 2.928993 | 0.585799 | 15.75 | 0.0097 |
| Error: MS(Error) | 4 | 0.148739 | 0.037185 | | |

Comparison: A vs B

Dependent Variable: Cl/F (L/h) Weight Group: 76-87

#### Least Squares Means

| D., 8, 141 |
|------------|
| Pr > t |
| 0.1377 |

| trt | LN_CLFO LSMEAN | 90% Confidence Limits | |
|-----|----------------|-----------------------|----------|
| A | 0.391089 | 0.234101 | 0.548077 |
| В | 0.597271 | 0.419263 | 0.775279 |

| Le | Least Squares Means for Effect trt | | | |
|---|---|---|---|---|
| | | Difference Between | | |
| i | j | Means | 90% Confid | ence Limits for LSMean(i)-LSMean(j) |
| 1 | 2 | -0.206182 | -0.443526 | 0.031162 |

| | | Standard | | |
|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t 90% Confidence Limits |
| A - B | -0.20618191 | 0.11133243 | -1.85 | 0.1377-0.44352559 |

Comparison: A vs B

Dependent Variable: V<sub>d</sub>/F/kg (L/kg) Weight Group: 76-87

#### The GLM Procedure

| Class Level I | nformation | |
|---|---|---|
| Class | Levels | Values |
| subject | 7 | 205 301 406 410 411 501 506 |
| sequence | 2 | AB BA |
| period | 2 | 1 2 |
| trt | 2 | A B |
| Number of O | Number of Observations Read 13 | |
| Number of O | Number of Observations Used 13 | |

Comparison: A vs B

Dependent Variable: V<sub>d</sub>/F/kg (L/kg) Weight Group: 76-87

#### The GLM Procedure

| R-Square | Coeff Var | Root MSE | | LN_VZF | OW Mean |
|------------------|-----------|-------------|-------------|---------|---------|
| 0.827623 | 54.35284 | 0.457834 | 0.842336 | | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.55584599 | 0.55584599 | 2.65 | 0.1788 |
| period | 1 | 0.47525416 | 0.47525416 | 2.27 | 0.2066 |
| trt | 1 | 0.01535182 | 0.01535182 | 0.07 | 0.8001 |
| subject(sequence | e) 5 | 2.97913450 | 0.59582690 | 2.84 | 0.1667 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.61287645 | 0.61287645 | 2.92 | 0.1625 |
| period | 1 | 0.22564597 | 0.22564597 | 1.08 | 0.3581 |
| trt | 1 | 0.10173215 | 0.10173215 | 0.49 | 0.5244 |
| subject(sequence | e) 5 | 2.97913450 | 0.59582690 | 2.84 | 0.1667 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.31250150 | 0.31250150 | 1.49 | 0.2891 |
| period | 1 | 0.22564597 | 0.22564597 | 1.08 | 0.3581 |
| trt | 1 | 0.10173215 | 0.10173215 | 0.49 | 0.5244 |
| subject(sequence | e) 5 | 2.97913450 | 0.59582690 | 2.84 | 0.1667 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.31250150 | 0.31250150 | 1.49 | 0.2891 |
| period | 1 | 0.22564597 | 0.22564597 | 1.08 | 0.3581 |
| trt | 1 | 0.10173215 | 0.10173215 | 0.49 | 0.5244 |
| subject(sequence | e) 5 | 2.97913450 | 0.59582690 | 2.84 | 0.1667 |

Comparison: A vs B

Dependent Variable: V<sub>d</sub>/F/kg (L/kg) Weight Group: 76-87

### The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN VZFOW

| <br>Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|------------|--------|-----------|-------------|---------|--------|
| *sequence | 1 | 0.555846 | 0.555846 | 0.89 | 0.3909 |
| Error | 4.7556 | 2.970298 | 0.624593 | | |

Error: 1.0745\*MS(subject(sequence)) - 0.0745\*MS(Error)

<sup>\*</sup> This test assumes one or more other fixed effects are zero.

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---------|-------|-----------|-------------|---------|--------|
| *period | 1 | 0.475254 | 0.475254 | 2.10 | 0.2066 |
| Error | 5.005 | 1.130933 | 0.225959 | | |

Error: 0.0423\*MS(subject(sequence)) + 0.9577\*MS(Error)

<sup>\*</sup> This test assumes one or more other fixed effects are zero.

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|--------|--------|-----------|-------------|---------|--------|
| trt | 1 | 0.015352 | 0.015352 | 0.07 | 0.8041 |
| Error | 4.8758 | 1.091772 | 0.223916 | | |

Error: 0.037\*MS(subject(sequence)) + 0.963\*MS(Error)

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-------------------|----|-----------|-------------|---------|--------|
| subject(sequence) | 5 | 2.979134 | 0.595827 | 2.84 | 0.1667 |
| Error: MS(Error) | 4 | 0.838447 | 0.209612 | | |

Comparison: A vs B

Dependent Variable: V<sub>d</sub>/F/kg (L/kg) Weight Group: 76-87

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_VZFOW

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.612876 | 0.612876 | 0.98 | 0.3695 |
| Error | 4.7568 | 2.970329 | 0.624435 | | _ |
| Error: 1.0741*MS(subject(sequence)) - 0.0741*MS(Error) | | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.225646 | 0.225646 | 1.08 | 0.3581 |
| trt | 1 | 0.101732 | 0.101732 | 0.49 | 0.5244 |
| subject(sequence) | 5 | 2.979134 | 0.595827 | 2.84 | 0.1667 |
| Error: MS(Error) | 4 | 0.838447 | 0.209612 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.312501 | 0.312501 | 0.53 | 0.4971 |
| Error | 5.1004 | 2.984223 | 0.585099 | | |
| Error: 0.9722*MS(subject(sequence)) + 0.0278*MS(Error) | | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 0.225646 | 0.225646 | 1.08 | 0.3581 |
| trt | 1 | 0.101732 | 0.101732 | 0.49 | 0.5244 |
| subject(sequence) | 5 | 2.979134 | 0.595827 | 2.84 | 0.1667 |
| Error: MS(Error) | 4 | 0.838447 | 0.209612 | | |

Comparison: A vs B

Dependent Variable: V<sub>d</sub>/F/kg (L/kg) Weight Group: 76-87

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------|-----------|------------|-------------|---------|--------|
| sequence | 1 | 0.312501 | 0.312501 | 0.53 | 0.4971 |
| Error | 5.1004 | 2.984223 | 0.585099 | | |
| Error: 0.97 | 22*MS(sub | ) | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.225646 | 0.225646 | 1.08 | 0.3581 |
| trt | 1 | 0.101732 | 0.101732 | 0.49 | 0.5244 |
| subject(sequence) | 5 | 2.979134 | 0.595827 | 2.84 | 0.1667 |
| Error: MS(Error) | 4 | 0.838447 | 0.209612 | | |

Comparison: A vs B

Dependent Variable: V<sub>d</sub>/F/kg (L/kg) Weight Group: 76-87

#### Least Squares Means

| | | H0:L | SMean1=LSMean2 | |
|-----|-----------------|----------|----------------------|---------|
| trt | LN_VZFOW LSMEAN | | | Pr > t |
| A | 0.87243886 | | | 0.5244 |
| В | 0.68829023 | | | |
| trt | LN_VZFOW LSMEAN | 9( | 0% Confidence Limits | |
| A | 0.872439 | 0.499711 | 1.245167 | |
| В | 0.688290 | 0.265656 | 1 110924 | |

Least Squares Means for Effect trt

Difference Between

i j Means 90% Confidence Limits for LSMean(i)-LSMean(j)

1 2 0.184149 -0.379363 0.747661

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confi | dence Limits |
| A - B | 0.18414862 | 0.26433041 | 0.70 | 0.5244-0 | 0.37936331 | 0.74766056 |

Comparison: A vs B

Dependent Variable: V<sub>d</sub>/F (L) Weight Group: 76-87

#### The GLM Procedure

| Class Level I | nformation | |
|---|---|---|
| Class | Levels | Values |
| subject | 7 | 205 301 406 410 411 501 506 |
| sequence | 2 | AB BA |
| period | 2 | 1 2 |
| trt | 2 | A B |
| Number of Observations Read 13 | | |
| Number of O | Number of Observations Used | |

Comparison: A vs B

Dependent Variable: V<sub>d</sub>/F (L) Weight Group: 76-87

#### The GLM Procedure

| R-Square | Coeff Var | Root MSF | 3 | LN_ | VZFO Mean |
|---|---|---|---|---|---|
| 0.829814 | 8.655693 | 0.457834 | 5.289394 | | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.59638193 | 0.59638193 | 2.85 | 0.1669 |
| period | 1 | 0.48789867 | 0.48789867 | 2.33 | 0.2018 |
| trt | 1 | 0.01331260 | 0.01331260 | 0.06 | 0.8134 |
| subject(sequence | ) 5 | 2.99060271 | 0.59812054 | 2.85 | 0.1658 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.65717146 | 0.65717146 | 3.14 | 0.1513 |
| period | 1 | 0.22564597 | 0.22564597 | 1.08 | 0.3581 |
| trt | 1 | 0.10173215 | 0.10173215 | 0.49 | 0.5244 |
| subject(sequence | ) 5 | 2.99060271 | 0.59812054 | 2.85 | 0.1658 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.33371526 | 0.33371526 | 1.59 | 0.2756 |
| period | 1 | 0.22564597 | 0.22564597 | 1.08 | 0.3581 |
| trt | 1 | 0.10173215 | 0.10173215 | 0.49 | 0.5244 |
| subject(sequence | ) 5 | 2.99060271 | 0.59812054 | 2.85 | 0.1658 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.33371526 | 0.33371526 | 1.59 | 0.2756 |
| period | 1 | 0.22564597 | 0.22564597 | 1.08 | 0.3581 |
| trt | 1 | 0.10173215 | 0.10173215 | 0.49 | 0.5244 |
| subject(sequence | ) 5 | 2.99060271 | 0.59812054 | 2.85 | 0.1658 |

Comparison: A vs B

Dependent Variable: V<sub>d</sub>/F (L) Weight Group: 76-87

### The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN VZFO

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| *sequence | 1 | 0.596382 | 0.596382 | 0.95 | 0.3764 |
| Error 4.7565 2.982607 0.627057 | | | | | |
| Error: 1.0745*MS(su | bject(sequ | ence)) - 0.074 | 5*MS(Error) | | |

\* This test assumes one or more other fixed effects are zero.

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---------|--------|-----------|-------------|---------|--------|
| *period | 1 | 0.487899 | 0.487899 | 2.16 | 0.2016 |
| Error | 5.0088 | 1.132283 | 0.226057 | | |

Error: 0.0423\*MS(subject(sequence)) + 0.9577\*MS(Error)

<sup>\*</sup> This test assumes one or more other fixed effects are zero.

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| trt | 1 | 0.013313 | 0.013313 | 0.06 | 0.8173 |
| Error | 4.8792 | 1.092935 | 0.224001 | | |
| Error: 0.0 | Error: $0.027*MS(subject(sequence)) + 0.063*MS(Error)$ | | | | |

Error: 0.037\*MS(subject(sequence)) + 0.963\*MS(Error)

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-------------------|----|-----------|-------------|---------|--------|
| subject(sequence) | 5 | 2.990603 | 0.598121 | 2.85 | 0.1658 |
| Error: MS(Error) | 4 | 0.838447 | 0.209612 | | |

Comparison: A vs B

Dependent Variable: V<sub>d</sub>/F (L) Weight Group: 76-87

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_VZFO

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.657171 | 0.657171 | 1.05 | 0.3551 |
| Error | 4.7578 | 2.982633 | 0.626899 | | |
| Error: 1.0741*MS(subject(sequence)) - 0.0741*MS(Error) | | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|-----------|
| period | 1 | 0.225646 | 0.225646 | 1.08 | 0.3581 |
| trt | 1 | 0.101732 | 0.101732 | 0.49 | 0.5244 |
| subject(sequence) | 5 | 2.990603 | 0.598121 | 2.85 | 0.1658 |
| Error: MS(Error) | 4 | 0.838447 | 0.209612 | | <u></u> ; |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.333715 | 0.333715 | 0.57 | 0.4843 |
| Error | 5.1 | 2.995371 | 0.587329 | | |
| Error: 0.9722*MS(subject(sequence)) + 0.0278*MS(Error) | | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 0.225646 | 0.225646 | 1.08 | 0.3581 |
| trt | 1 | 0.101732 | 0.101732 | 0.49 | 0.5244 |
| subject(sequence) | 5 | 2.990603 | 0.598121 | 2.85 | 0.1658 |
| Error: MS(Error) | 4 | 0.838447 | 0.209612 | | |

Comparison: A vs B

Dependent Variable: V<sub>d</sub>/F (L) Weight Group: 76-87

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.333715 | 0.333715 | 0.57 | 0.4843 |
| Error | 5.1 | 2.995371 | 0.587329 | | |
| Error: 0.9722*MS(subject(sequence)) + 0.0278*MS(Error) | | | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.225646 | 0.225646 | 1.08 | 0.3581 |
| trt | 1 | 0.101732 | 0.101732 | 0.49 | 0.5244 |
| subject(sequence) | 5 | 2.990603 | 0.598121 | 2.85 | 0.1658 |
| Error: MS(Error) | 4 | 0.838447 | 0.209612 | | |

Comparison: A vs B

Dependent Variable: V<sub>d</sub>/F (L) Weight Group: 76-87

#### Least Squares Means

| | | H0:LSMean1=LSMean2 | |
|-----|----------------|--------------------|---------|
| trt | LN_VZFO LSMEAN | | Pr > t |
| A | 5.31688317 | | 0.5244 |
| В | 5.13273455 | | |

| trt | LN_VZFO LSMEAN | 90% Confidence Limits | |
|-----|----------------|-----------------------|----------|
| A | 5.316883 | 4.944155 | 5.689611 |
| В | 5.132735 | 4.710101 | 5.555368 |

| Le | Least Squares Means for Effect trt | | | |
|---|---|---|---|---|
| | | Difference Between | | |
| i | j | Means | 90% Confid | ence Limits for LSMean(i)-LSMean(j) |
| 1 | 2 | 0.184149 | -0.379363 | 0.747661 |

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confi | dence Limits |
| A - B | 0.18414862 | 0.26433041 | 0.70 | 0.5244-0 | 0.37936331 | 0.74766056 |

Comparison: A vs B

Dependent Variable: T<sub>max</sub> (h) Weight Group: 76-87

#### The GLM Procedure

| Class Level I | nformation | |
|---------------|------------|-----------------------------|
| Class | Levels | Values |
| subject | 7 | 205 301 406 410 411 501 506 |
| sequence | 2 | AB BA |
| period | 2 | 1 2 |
| trt | 2 | A B |
| Number of O | 14 | |
| Number of O | 14 | |

Comparison: A vs B

Dependent Variable: T<sub>max</sub> (h) Weight Group: 76-87

#### The GLM Procedure

| R-Square | Coeff Var | Root | MSE | | TMAX Mean |
|---|---|---|---|---|---|
| 0.547486 | 51.70082 | 0.529 | 380 | 1.023929 | |
| Source | DF | Type I SS | Mean Square | e F Value | e Pr > F |
| sequence | 1 | 0.04136010 | 0.04136010 | 0.15 | 0.7166 |
| period | 1 | 0.03837779 | 0.03837779 | 0.14 | 0.7265 |
| trt | 1 | 0.58717038 | 0.58717038 | 2.10 | 0.2074 |
| subject(sequence) | 5 | 1.02838533 | 0.20567707 | 0.73 | 0.6287 |
| Source | DF | Type II SS | Mean Square | F Value | e $Pr > F$ |
| sequence | 1 | 0.04136010 | 0.04136010 | 0.15 | 0.7166 |
| period | 1 | 0.09202752 | 0.09202752 | 0.33 | 0.5914 |
| trt | 1 | 0.58717038 | 0.58717038 | 2.10 | 0.2074 |
| subject(sequence) | 5 | 1.02838533 | 0.20567707 | 0.73 | 0.6287 |
| Source | DF | Type III SS | Mean Square | F Value | e $Pr > F$ |
| sequence | 1 | 0.04136010 | 0.04136010 | 0.15 | 0.7166 |
| period | 1 | 0.09202752 | 0.09202752 | 0.33 | 0.5914 |
| trt | 1 | 0.58717038 | 0.58717038 | 2.10 | 0.2074 |
| subject(sequence) | 5 | 1.02838533 | 0.20567707 | 0.73 | 0.6287 |
| Source | DF | Type IV SS | Mean Square | F Value | e $Pr > F$ |
| sequence | 1 | 0.04136010 | 0.04136010 | 0.15 | 0.7166 |
| period | 1 | 0.09202752 | 0.09202752 | 0.33 | 0.5914 |
| trt | 1 | 0.58717038 | 0.58717038 | 2.10 | 0.2074 |
| subject(sequence) | 5 | 1.02838533 | 0.20567707 | 0.73 | 0.6287 |

Comparison: A vs B

Dependent Variable: T<sub>max</sub> (h) Weight Group: 76-87

### The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: TMAX

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.041360 | 0.041360 | 0.20 | 0.6726 |
| Error | 5 | 1.028385 | 0.205677 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| *period | 1 | 0.038378 | 0.038378 | 0.14 | 0.7265 |
| trt | 1 | 0.587170 | 0.587170 | 2.10 | 0.2074 |
| subject(sequence) | 5 | 1.028385 | 0.205677 | 0.73 | 0.6287 |
| Error: MS(Error) 5 1.401213 0.280243 | | | | | |
| * This test assumes one or more other fixed effects are zero. | | | | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.041360 | 0.041360 | 0.20 | 0.6726 |
| Error | 5 | 1.028385 | 0.205677 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.092028 | 0.092028 | 0.33 | 0.5914 |
| trt | 1 | 0.587170 | 0.587170 | 2.10 | 0.2074 |
| subject(sequence) | 5 | 1.028385 | 0.205677 | 0.73 | 0.6287 |
| Error: MS(Error) | 5 | 1.401213 | 0.280243 | | |

Comparison: A vs B

Dependent Variable: T<sub>max</sub> (h) Weight Group: 76-87

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: TMAX

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.041360 | 0.041360 | 0.20 | 0.6726 |
| Error | 5 | 1.028385 | 0.205677 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 0.092028 | 0.092028 | 0.33 | 0.5914 |
| trt | 1 | 0.587170 | 0.587170 | 2.10 | 0.2074 |
| subject(sequence) | 5 | 1.028385 | 0.205677 | 0.73 | 0.6287 |
| Error: MS(Error) | 5 | 1.401213 | 0.280243 | | - |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------|-----------|------------|-------------|---------|--------|
| sequence | 1 | 0.041360 | 0.041360 | 0.20 | 0.6726 |
| Error | 5 | 1.028385 | 0.205677 | | |
| Error: MS(s | subject(s | sequence)) | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.092028 | 0.092028 | 0.33 | 0.5914 |
| trt | 1 | 0.587170 | 0.587170 | 2.10 | 0.2074 |
| subject(sequence) | 5 | 1.028385 | 0.205677 | 0.73 | 0.6287 |
| Error: MS(Error) | 5 | 1.401213 | 0.280243 | | |

Comparison: A vs B

Dependent Variable: T<sub>max</sub> (h) Weight Group: 76-87

#### Least Squares Means

| trt TMAX LSMEAN A 1.22300000 B 0.80916667 trt TMAX LSMEAN A 1.223000 B 0.809167 Least Squares Means for Effect trt Difference Between | | ean2 |
|---|---|---|
| B 0.80916667 trt TMAX LSMEAN A 1.223000 B 0.809167 Least Squares Means for Effect trt | | Pr > t |
| trt TMAX LSMEAN A 1.223000 B 0.809167 Least Squares Means for Effect trt | | 0.2074 |
| A 1.223000 B 0.809167 Least Squares Means for Effect trt | | |
| A 1.223000 B 0.809167 Least Squares Means for Effect trt | | |
| B 0.809167 Least Squares Means for Effect trt | 90% Confidence | Limits |
| Least Squares Means for Effect trt | 0.815638 1.630 | 0362 |
| 1 | 0.401804 1.216 | 6529 |
| 1 | | |
| Difference Between | | |
| i i Means 90% C | Confidence Limits for LSMean | (i) I CMoon(i) |
| 1 2 0.413833 -0.16220 | | (1)-LSIVICALI(J) |

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confi | dence Limits |
| A - B | 0.41383333 | 0.28589761 | 1.45 | 0.2074-0 | 0.16226418 | 0.98993085 |

Comparison: A vs B

Dependent Variable: K<sub>el</sub> (/h) Weight Group: 76-87

#### The GLM Procedure

| Class Level I | nformation | |
|---|---|---|
| Class | Levels | Values |
| subject | 7 | 205 301 406 410 411 501 506 |
| sequence | 2 | AB BA |
| period | 2 | 1 2 |
| trt | 2 | A B |
| | <del></del> | |
| Number of Observations Read | | |
| Number of Observations Used | | |

Comparison: A vs B

Dependent Variable:  $K_{el}$  (/h) Weight Group: 76-87

#### The GLM Procedure

| R-Square | Coeff Var | Root | MSE | I | LAMZ Mean |
|---|---|---|---|---|---|
| 0.873885 | 28.10434 | 0.002 | 2893 | 0.010293 | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.00000004 | 0.00000004 | 0.01 | 0.9469 |
| period | 1 | 0.00000565 | 0.00000565 | 0.67 | 0.4575 |
| trt | 1 | 0.00002119 | 0.00002119 | 2.53 | 0.1868 |
| subject(sequence) | 5 | 0.00020508 | 0.00004102 | 4.90 | 0.0744 |
| Source | DF | Type II SS | Mean Square | e F Value | Pr > F |
| sequence | 1 | 0.00000000 | 0.00000000 | 0.00 | 0.9827 |
| period | 1 | 0.00000681 | 0.00000681 | 0.81 | 0.4181 |
| trt | 1 | 0.00001972 | 0.00001972 | 2.36 | 0.1996 |
| subject(sequence) | 5 | 0.00020508 | 0.00004102 | 4.90 | 0.0744 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.00000001 | 0.00000001 | 0.00 | 0.9790 |
| period | 1 | 0.00000681 | 0.00000681 | 0.81 | 0.4181 |
| trt | 1 | 0.00001972 | 0.00001972 | 2.36 | 0.1996 |
| subject(sequence) | 5 | 0.00020508 | 0.00004102 | 4.90 | 0.0744 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.00000001 | 0.00000001 | 0.00 | 0.9790 |
| period | 1 | 0.00000681 | 0.00000681 | 0.81 | 0.4181 |
| trt | 1 | 0.00001972 | 0.00001972 | 2.36 | 0.1996 |
| subject(sequence) | 5 | 0.00020508 | 0.00004102 | 4.90 | 0.0744 |

Comparison: A vs B

Dependent Variable: K<sub>el</sub> (/h) Weight Group: 76-87

### The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LAMZ

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| *sequence | 1 | 4.2090894E-8 | 4.2090894E-8 | 0.00 | 0.9764 |
| Error | 4.8584 | 0.000211 | 0.000043447 | | |
| Compan 1 0745*MC(collisat(compan)) 0 0745*MC(Compan) | | | | | |

Error: 1.0745\*MS(subject(sequence)) - 0.0745\*MS(Error)

<sup>\*</sup> This test assumes one or more other fixed effects are zero.

| 9 | Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|----|--------|--------|-------------|-------------|---------|--------|
| *1 | period | 1 | 0.000005647 | 0.000005647 | 0.58 | 0.4769 |
| ] | Error | 5.7064 | 0.000055641 | 0.000009751 | | |

Error: 0.0423\*MS(subject(sequence)) + 0.9577\*MS(Error)

<sup>\*</sup> This test assumes one or more other fixed effects are zero.

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| trt | 1 | 0.000021191 | 0.000021191 | 2.21 | 0.1919 |
| Error | 5.494 | 0.000052620 | 0.000009578 | | |
| Error: 0.0 | )37*MS(sul | piect(sequence)) + 0 | ) 963*MS(Error) | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| subject(sequence) | 5 | 0.000205 | 0.000041015 | 4.90 | 0.0744 |
| Error: MS(Error) | 4 | 0.000033475 | 0.000008369 | | |

Comparison: A vs B

Dependent Variable: K<sub>el</sub> (/h) Weight Group: 76-87

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LAMZ

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 4.4420302E-9 | 4.4420302E-9 | 0.00 | 0.9923 |
| Error | 4.8591 | 0.000211 | 0.000043433 | | |
| Error: 1.07 | Error: 1.0741*MS(subject(sequence)) - 0.0741*MS(Error) | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 0.000006809 | 0.000006809 | 0.81 | 0.4181 |
| trt | 1 | 0.000019719 | 0.000019719 | 2.36 | 0.1996 |
| subject(sequence) | 5 | 0.000205 | 0.000041015 | 4.90 | 0.0744 |
| Error: MS(Error) | 4 | 0.000033475 | 0.000008369 | | - |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 6.5762621E-9 | 6.5762621E-9 | 0.00 | 0.9903 |
| Error | 5.0583 | 0.000203 | 0.000040108 | | |
| Error: 0.97 | 722*MS(su | bject(sequence)) + ( | 0.0278*MS(Error) | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 0.000006809 | 0.000006809 | 0.81 | 0.4181 |
| trt | 1 | 0.000019719 | 0.000019719 | 2.36 | 0.1996 |
| subject(sequence) | 5 | 0.000205 | 0.000041015 | 4.90 | 0.0744 |
| Error: MS(Error) | 4 | 0.000033475 | 0.000008369 | | |

Comparison: A vs B

Dependent Variable: K<sub>el</sub> (/h) Weight Group: 76-87

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 6.5762621E-9 | 6.5762621E-9 | 0.00 | 0.9903 |
| Error | 5.0583 | 0.000203 | 0.000040108 | | |
| Error: 0.97 | Error: 0.9722*MS(subject(sequence)) + 0.0278*MS(Error) | | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 0.000006809 | 0.000006809 | 0.81 | 0.4181 |
| trt | 1 | 0.000019719 | 0.000019719 | 2.36 | 0.1996 |
| subject(sequence) | 5 | 0.000205 | 0.000041015 | 4.90 | 0.0744 |
| Error: MS(Error) | 4 | 0.000033475 | 0.000008369 | | |

Comparison: A vs B

Dependent Variable: K<sub>el</sub> (/h) Weight Group: 76-87

#### Least Squares Means

| _ | | | H0:LSM | Mean1=LSMean2 | |
|---|---|---|---|---|---|
| trt | LAMZ LSMEAN | | | | Pr > t |
| A | 0.00904945 | | | | 0.1996 |
| В | 0.01161324 | | | | |
| trt | LAMZ LSMEAN | | 90% | Confidence Limits | |
| A | 0.009049 | 0. | 006694 | 0.011405 | |
| В | 0.011613 | 0. | 008943 | 0.014284 | |
| Le | ast Squares Means for Effect<br>Difference Between | et trt | | | |
| i | i Means | 90% Confid | ence Limits | for LSMean(i)-LSM | Iean(i) |
| 1 | 2 -0.002564 | -0.006124 | | 0.000997 | 0/ |

| | | Standard | | |
|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t 90% Confidence Limits |
| A - B | -0.00256379 | 0.00167020 | -1.54 | 0.1996-0.00612439 |

Comparison: A vs B

Dependent Variable: T<sub>1/2 el</sub> (h) Weight Group: 76-87

#### The GLM Procedure

| Class Level I | nformation | |
|-----------------------------|------------|-----------------------------|
| Class | Levels | Values |
| subject | 7 | 205 301 406 410 411 501 506 |
| sequence | 2 | AB BA |
| period | 2 | 1 2 |
| trt | 2 | AB |
| Number of O | 13 | |
| Number of Observations Used | | |

Comparison: A vs B

Dependent Variable: T<sub>1/2 el</sub> (h) Weight Group: 76-87

#### The GLM Procedure

| R-Square | Coeff Var | Root MSE | | LAMZ | HL Mean |
|---|---|---|---|---|---|
| 0.658688 | 115.2892 | 120.4972 | 104.51 | 73 | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 9566.77716 | 9566.77716 | 0.66 | 0.4625 |
| period | 1 | 17411.68113 | 17411.68113 | 1.20 | 0.3350 |
| trt | 1 | 15198.84251 | 15198.84251 | 1.05 | 0.3641 |
| subject(sequence) | ) 5 | 69906.18556 | 13981.23711 | 0.96 | 0.5294 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 9246.29628 | 9246.29628 | 0.64 | 0.4696 |
| period | 1 | 18021.71774 | 18021.71774 | 1.24 | 0.3277 |
| trt | 1 | 14534.90061 | 14534.90061 | 1.00 | 0.3737 |
| subject(sequence) | ) 5 | 69906.18556 | 13981.23711 | 0.96 | 0.5294 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 8891.77606 | 8891.77606 | 0.61 | 0.4776 |
| period | 1 | 18021.71774 | 18021.71774 | 1.24 | 0.3277 |
| trt | 1 | 14534.90061 | 14534.90061 | 1.00 | 0.3737 |
| subject(sequence) | ) 5 | 69906.18556 | 13981.23711 | 0.96 | 0.5294 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 8891.77606 | 8891.77606 | 0.61 | 0.4776 |
| period | 1 | 18021.71774 | 18021.71774 | 1.24 | 0.3277 |
| trt | 1 | 14534.90061 | 14534.90061 | 1.00 | 0.3737 |
| subject(sequence) | ) 5 | 69906.18556 | 13981.23711 | 0.96 | 0.5294 |

Comparison: A vs B

Dependent Variable: T<sub>1/2 el</sub> (h) Weight Group: 76-87

### The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LAMZHL

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-----------|--------|-------------|-------------|---------|--------|
| *sequence | 1 | 9566.777155 | 9566.777155 | 0.69 | 0.4512 |
| Error | 4.2783 | 59645 | 13941 | | |

Error: 1.0745\*MS(subject(sequence)) - 0.0745\*MS(Error)

<sup>\*</sup> This test assumes one or more other fixed effects are zero.

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---------|--------|-----------|-------------|---------|--------|
| *period | 1 | 17412 | 17412 | 1.20 | 0.3301 |
| Error | 4.3414 | 62937 | 14497 | | |

Error: 0.0423\*MS(subject(sequence)) + 0.9577\*MS(Error)

<sup>\*</sup> This test assumes one or more other fixed effects are zero.

| Source | e DF | Type I S | S Mean Square | e F Value | Pr > F |
|--------|----------------|----------|--------------------|-----------|--------|
| trt | 1 | 15199 | 15199 | 1.05 | 0.3601 |
| Error | 4.2971 | 62306 | 14500 | | |
| | 0.00549.60/ 1: | | )) . 0.0(0.49 f0/F | ` | |

Error: 0.037\*MS(subject(sequence)) + 0.963\*MS(Error)

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-------------------|----|-----------|-------------|---------|--------|
| subject(sequence) | 5 | 69906 | 13981 | 0.96 | 0.5294 |
| Error: MS(Error) | 4 | 58078 | 14520 | | |

Comparison: A vs B

Dependent Variable: T<sub>1/2 el</sub> (h) Weight Group: 76-87

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LAMZHL

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 9246.296277 | 9246.296277 | 0.66 | 0.4583 |
| Error 4.282 59697 13941 | | | | | |
| Error: 1.07 | Error: 1.0741*MS(subject(sequence)) - 0.0741*MS(Error) | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|---------|
| period | 1 | 18022 | 18022 | 1.24 | 0.3277 |
| trt | 1 | 14535 | 14535 | 1.00 | 0.3737 |
| subject(sequence) | 5 | 69906 | 13981 | 0.96 | 0.5294 |
| Error: MS(Error) | 4 | 58078 | 14520 | | <u></u> |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 8891.776063 | 8891.776063 | 0.64 | 0.4597 |
| Error | Error 5.2953 74114 13996 | | | | |
| Error: 0.9722*MS(subject(sequence)) + 0.0278*MS(Error) | | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 18022 | 18022 | 1.24 | 0.3277 |
| trt | 1 | 14535 | 14535 | 1.00 | 0.3737 |
| subject(sequence) | 5 | 69906 | 13981 | 0.96 | 0.5294 |
| Error: MS(Error) | 4 | 58078 | 14520 | | |

Comparison: A vs B

Dependent Variable: T<sub>1/2 el</sub> (h) Weight Group: 76-87

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 8891.776063 | 8891.776063 | 0.64 | 0.4597 |
| Error 5.2953 74114 13996 | | | | | |
| Error: 0.9722*MS(subject(sequence)) + 0.0278*MS(Error) | | | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 18022 | 18022 | 1.24 | 0.3277 |
| trt | 1 | 14535 | 14535 | 1.00 | 0.3737 |
| subject(sequence) | 5 | 69906 | 13981 | 0.96 | 0.5294 |
| Error: MS(Error) | 4 | 58078 | 14520 | | |

Comparison: A vs B

Dependent Variable: T<sub>1/2 el</sub> (h) Weight Group: 76-87

#### Least Squares Means

| | | H0: | LSMean1=LSMean2 |
|---|---|---|---|
| trt | LAMZHL LSMEAN | | Pr > t |
| A | 141.400412 | | 0.3737 |
| В | 71.794615 | | |
| trt | LAMZHL LSMEAN | 90 | % Confidence Limits |
| A | 141.400412 | 43.302149 | 239.498674 |
| В | 71.794615 | -39.438359 | 183.027590 |
| Le | ast Squares Means for Effe | ct trt | |
| | Difference Between | | |
| i | j Means | 90% Confidence | e Limits for LSMean(i)-LSMean(j) |
| 1 | 2 69 605796 | -78 704837 | 217 916429 |

| | | Standard | | | |
|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confidence Limits |
| A - B | 69.6057962 | 69.5690862 | 1.00 | 0.3737-7 | 8.7048366 217.9164290 |

Comparison: C vs B

Dependent Variable: AUC<sub>0-t</sub> (h\*ng/mL) Weight Group: 76-87

#### The GLM Procedure

| subject 2 301 406 sequence 2 ABC BAC trt 2 B C | |
|------------------------------------------------|---|
| trt 2 BC | |
| Number of Observations Read | 4 |

Comparison: C vs B

Dependent Variable: AUC<sub>0-t</sub> (h\*ng/mL) Weight Group: 76-87

#### The GLM Procedure

Dependent Variable: LN\_AUCLST

| R-Square Coeff Va | | r Root MSE | | LN_AUCLST Mean | |
|---|---|---|---|---|---|
| 0.814181 | 2.448131 | 0.222785 | 9.100215 | | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.20699244 | 0.20699244 | 4.17 | 0.2899 |
| trt | 1 | 0.01047938 | 0.01047938 | 0.21 | 0.7258 |
| subject(sequence | e) 0 | 0.00000000 | | | |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.20699244 | 0.20699244 | 4.17 | 0.2899 |
| trt | 1 | 0.01047938 | 0.01047938 | 0.21 | 0.7258 |
| subject(sequence | ee) 0 | 0.00000000 | | | |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.20699244 | 0.20699244 | 4.17 | 0.2899 |
| trt | 1 | 0.01047938 | 0.01047938 | 0.21 | 0.7258 |
| subject(sequence | ee) 0 | 0.00000000 | | | |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.20699244 | 0.20699244 | 4.17 | 0.2899 |
| trt | 1 | 0.01047938 | 0.01047938 | 0.21 | 0.7258 |
| subject(sequence | e) 0 | 0.00000000 | | | |
Comparison: C vs B

Dependent Variable: AUC<sub>0-t</sub> (h\*ng/mL) Weight Group: 76-87

## The GLM Procedure Least Squares Means

| | | H0:LSMean1=LSMean2 | |
|-----|------------------|--------------------|---------|
| trt | LN_AUCLST LSMEAN | | Pr > t |
| В | 9.15139922 | | 0.7258 |
| C | 9.04903038 | | |

| trt | LN_AUCLST LSMEAN | 90% Confidence Limits | |
|-----|------------------|-----------------------|-----------|
| В | 9.151399 | 8.156775 | 10.146023 |
| C | 9.049030 | 8.054407 | 10.043654 |

| Le | Least Squares Means for Effect trt | | | |
|---|---|---|---|---|
| | | Difference Between | | |
| i | j | Means | 90% Confide | nce Limits for LSMean(i)-LSMean(j) |
| 1 | 2 | 0.102369 | -1.304242 | 1.508979 |

#### The GLM Procedure

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confid | dence Limits |
| C - B | -0.10236884 | 0.22278522 | -0.46 | 0.7258-1 | .50897936 | 1.30424169 |

Comparison: C vs B

Dependent Variable: AUC<sub>0-inf</sub> (h\*ng/mL) Weight Group: 76-87

| Class Level Inform | Levels | Values | |
|-----------------------------|-------------|---------|---|
| subject | 2 | 301 406 | |
| sequence | 2 | ABC BAC | |
| trt | 2 | ВС | |
| Number of Observa | ations Read | | 4 |
| lumber of Observations Read | | | |

Comparison: C vs B

Dependent Variable: AUC<sub>0-inf</sub> (h\*ng/mL) Weight Group: 76-87

## The GLM Procedure

Dependent Variable: LN\_AUCIFO

| R-Square | Coeff Var | Root MSE | | LN_AUC | IFO Mean |
|---|---|---|---|---|---|
| 0.932143 | 1.708233 | 0.157513 | 9.220795 | <u>-</u> | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.34080541 | 0.34080541 | 13.74 | 0.1678 |
| trt | 1 | 0.00000719 | 0.00000719 | 0.00 | 0.9892 |
| subject(sequence | ee) 0 | 0.00000000 | | | |
| | | | | | _ |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.34080541 | 0.34080541 | 13.74 | 0.1678 |
| trt | 1 | 0.00000719 | 0.00000719 | 0.00 | 0.9892 |
| subject(sequence | ce) 0 | 0.00000000 | | | |
| <u> </u> | DE | T. HIGG | M. C | F 1/ 1 | D > F |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.34080541 | 0.34080541 | 13.74 | 0.1678 |
| trt | 1 | 0.00000719 | 0.00000719 | 0.00 | 0.9892 |
| subject(sequence | (e) 0 | 0.00000000 | | | |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| | 1 | 0.34080541 | 0.34080541 | 13.74 | 0.1678 |
| sequence<br>trt | 1 | 0.00000719 | 0.00000719 | 0.00 | 0.1678 |
| | | 0.00000719 | 0.00000/19 | 0.00 | 0.9692 |
| subject(sequence | 0 | 0.00000000 | | | |

Comparison: C vs B

Dependent Variable: AUC<sub>0-inf</sub> (h\*ng/mL) Weight Group: 76-87

## The GLM Procedure Least Squares Means

| | | H0:LSMean1=LSMean2 | |
|-----|------------------|--------------------|---------|
| trt | LN_AUCIFO LSMEAN | | Pr > t |
| В | 9.21945385 | | 0.9892 |
| C | 9.22213570 | | |

| trt | LN_AUCIFO LSMEAN | 90% | Confidence Limits |
|-----|------------------|----------|-------------------|
| В | 9.219454 | 8.516239 | 9.922668 |
| C | 9.222136 | 8.518921 | 9.925350 |

| Le | Least Squares Means for Effect trt | | | |
|---|---|---|---|---|
| | | Difference Between | | |
| i | j | Means | 90% Confid | ence Limits for LSMean(i)-LSMean(j) |
| 1 | 2 | -0.002682 | -0.997177 | 0.991814 |

#### The GLM Procedure

Dependent Variable: LN\_AUCIFO

| - | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confi | dence Limits |
| C - B | 0.00268185 | 0.15751262 | 0.02 | 0.9892-0 | 0.99181367 | 0.99717736 |

Comparison: C vs B

Dependent Variable: C<sub>max</sub> (ng/mL) Weight Group: 76-87

| Class Level Inform | Levels | Values | |
|-----------------------------|-------------|---------|---|
| subject | 2 | 301 406 | |
| sequence | 2 | ABC BAC | |
| trt | 2 | ВС | |
| Number of Observa | ations Read | | 4 |
| lumber of Observations Read | | | |

Comparison: C vs B

Dependent Variable: C<sub>max</sub> (ng/mL) Weight Group: 76-87

## The GLM Procedure

Dependent Variable: LN\_CMAX

| R-Square | Coeff Var | Root MSE | | LN_CI | MAX Mean |
|---|---|---|---|---|---|
| 0.263645 | 10.67177 | 0.587305 | 5.503351 | | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.00664457 | 0.00664457 | 0.02 | 0.9122 |
| trt | 1 | 0.11685348 | 0.11685348 | 0.34 | 0.6644 |
| subject(sequence | e) 0 | 0.00000000 | | | |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.00664457 | 0.00664457 | 0.02 | 0.9122 |
| trt | 1 | 0.11685348 | 0.11685348 | 0.34 | 0.6644 |
| subject(sequence | e) 0 | 0.00000000 | | | |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.00664457 | 0.00664457 | 0.02 | 0.9122 |
| trt | 1 | 0.11685348 | 0.11685348 | 0.34 | 0.6644 |
| subject(sequence | e) 0 | 0.00000000 | | | |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.00664457 | 0.00664457 | 0.02 | 0.9122 |
| trt | 1 | 0.11685348 | 0.11685348 | 0.34 | 0.6644 |
| subject(sequence | e) 0 | 0.00000000 | | | |

Comparison: C vs B

Dependent Variable: C<sub>max</sub> (ng/mL) Weight Group: 76-87

## The GLM Procedure Least Squares Means

| | | H0:LSMean1=LSMean2 | |
|-----|----------------|--------------------|---------|
| trt | LN_CMAX LSMEAN | | Pr > t |
| В | 5.67427068 | | 0.6644 |
| C | 5.33243229 | | |

| trt | LN_CMAX LSMEAN | 90% Confidence Limits | |
|-----|----------------|-----------------------|----------|
| В | 5.674271 | 3.052250 | 8.296291 |
| C | 5.332432 | 2.710412 | 7.954453 |

| Le | Least Squares Means for Effect trt | | | |
|---|---|---|---|---|
| | | Difference Between | | |
| i | j | Means | 90% Confid | ence Limits for LSMean(i)-LSMean(j) |
| 1 | 2 | 0.341838 | -3.366259 | 4.049935 |

#### The GLM Procedure

Dependent Variable: LN\_CMAX

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confid | dence Limits |
| C - B | -0.34183838 | 0.58730486 | -0.58 | 0.6644-4 | 1.04993531 | 3.36625855 |

Comparison: C vs B

Dependent Variable: Cl/F/kg ((L/h)/kg) Weight Group: 76-87

| Class | Levels | Values | |
|-------------------|----------------------------|---------|---|
| subject | 2 | 301 406 | |
| sequence | 2 | ABC BAC | |
| trt | 2 | ВС | |
| Number of Observa | ations Read | | 4 |
| Number of Observa | umber of Observations Read | | |

Comparison: C vs B

Dependent Variable: Cl/F/kg ((L/h)/kg) Weight Group: 76-87

## The GLM Procedure

Dependent Variable: LN\_CLFOW

| R-Square | Coeff Var | Root MSE | | LN_CLF | OW Mean |
|------------------|-----------|-------------|-------------|---------|---------|
| 0.930720 | -3.964760 | 0.157513 | -3.972816 | | |
| | | | | | _ |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.30870751 | 0.30870751 | 12.44 | 0.1759 |
| trt | 1 | 0.02459644 | 0.02459644 | 0.99 | 0.5014 |
| subject(sequence | ce) 0 | 0.00000000 | | | |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.30870751 | 0.30870751 | 12.44 | 0.1759 |
| trt | 1 | 0.02459644 | 0.02459644 | 0.99 | 0.5014 |
| subject(sequence | ce) 0 | 0.00000000 | | | |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.30870751 | 0.30870751 | 12.44 | 0.1759 |
| trt | 1 | 0.02459644 | 0.02459644 | 0.99 | 0.5014 |
| subject(sequence | ce) 0 | 0.00000000 | | | |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.30870751 | 0.30870751 | 12.44 | 0.1759 |
| trt | 1 | 0.02459644 | 0.02459644 | 0.99 | 0.5014 |
| subject(sequence | ce) 0 | 0.00000000 | | | |

Comparison: C vs B

Dependent Variable: Cl/F/kg ((L/h)/kg) Weight Group: 76-87

## The GLM Procedure Least Squares Means

| | | H0:LSMean1=LSMean2 | |
|-----|-----------------|--------------------|---------|
| trt | LN_CLFOW LSMEAN | | Pr > t |
| В | -3.89439993 | | 0.5014 |
| C | -4.05123246 | | |

| trt | LN_CLFOW LSMEAN | 90' | % Confidence Limits |
|-----|-----------------|-----------|---------------------|
| В | -3.894400 | -4.597614 | -3.191185 |
| C | -4.051232 | -4.754447 | -3.348018 |

| Le | Least Squares Means for Effect trt | | | |
|---|---|---|---|---|
| | | Difference Between | | |
| i | j | Means | 90% Confide | ence Limits for LSMean(i)-LSMean(j) |
| 1 | 2 | 0.156833 | -0.837663 | 1.151328 |

#### The GLM Procedure

Dependent Variable: LN\_CLFOW

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confidence | ce Limits |
| C - B | -0.15683253 | 0.15751262 | -1.00 | 0.5014-1 | .15132804 0.8 | 33766299 |

Comparison: C vs B

Dependent Variable: Cl/F (L/h) Weight Group: 76-87

| Class | Levels | Values |
|------------------|--------|---------|
| subject | 2 | 301 406 |
| sequence | 2 | ABC BAC |
| trt | 2 | ВС |
| Number of Observ | 4 | |
| T TOTAL OF CODE | | |

Comparison: C vs B

Dependent Variable: Cl/F (L/h) Weight Group: 76-87

## The GLM Procedure

Dependent Variable: LN\_CLFO

| R-Square | Coeff Var | Root MSE | | LN_C | LFO Mean |
|---|---|---|---|---|---|
| 0.936419 | 33.36523 | 0.157513 | 0.472086 | | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.34080541 | 0.34080541 | 13.74 | 0.1678 |
| trt | 1 | 0.02459644 | 0.02459644 | 0.99 | 0.5014 |
| subject(sequence | 9 0 | 0.00000000 | | | |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.34080541 | 0.34080541 | 13.74 | 0.1678 |
| trt | 1 | 0.02459644 | 0.02459644 | 0.99 | 0.5014 |
| subject(sequence | 9 0 | 0.00000000 | | | |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.34080541 | 0.34080541 | 13.74 | 0.1678 |
| trt | 1 | 0.02459644 | 0.02459644 | 0.99 | 0.5014 |
| subject(sequence | ) 0 | 0.00000000 | | | |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.34080541 | 0.34080541 | 13.74 | 0.1678 |
| trt | 1 | 0.02459644 | 0.02459644 | 0.99 | 0.5014 |
| subject(sequence | 9 0 | 0.00000000 | | | |

Comparison: C vs B

Dependent Variable: Cl/F (L/h) Weight Group: 76-87

## The GLM Procedure Least Squares Means

| | | H0:LSMean1=LSMean2 | |
|-----|----------------|--------------------|---------|
| trt | LN_CLFO LSMEAN | | Pr > t |
| В | 0.55050231 | | 0.5014 |
| C | 0.39366978 | | |

| trt | LN_CLFO LSMEAN | 90 | % Confidence Limits |
|-----|----------------|-----------|---------------------|
| В | 0.550502 | -0.152712 | 1.253717 |
| C | 0.393670 | -0.309545 | 1.096884 |

| Le | Least Squares Means for Effect trt | | | |
|---|---|---|---|---|
| | | Difference Between | | |
| i | j | Means | 90% Confi | dence Limits for LSMean(i)-LSMean(j) |
| 1 | 2 | 0.156833 | -0.837663 | 1.151328 |

#### The GLM Procedure

Dependent Variable: LN\_CLFO

| - | | Standard | | | |
|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confidence Limits |
| C - B | -0.15683253 | 0.15751262 | -1.00 | 0.5014-1 | 1.15132804 0.83766299 |

Comparison: C vs B

Dependent Variable: V<sub>d</sub>/F/kg (L/kg) Weight Group: 76-87

| subject 2 301 406 sequence 2 ABC BAC trt 2 B C |
|------------------------------------------------|
| trt 2 B C |
| Number of Observations Read |

Comparison: C vs B

Dependent Variable: V<sub>d</sub>/F/kg (L/kg) Weight Group: 76-87

## The GLM Procedure

Dependent Variable: LN\_VZFOW

| R-Square | Coeff Var | Root MSE | | LN_VZF | OW Mean |
|------------------|-----------|-------------|-------------|---------|---------|
| 0.677827 | 40.68762 | 0.281952 | 0.692967 | | |
| | | | | | _ |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.00005645 | 0.00005645 | 0.00 | 0.9830 |
| trt | 1 | 0.16719912 | 0.16719912 | 2.10 | 0.3843 |
| subject(sequence | ce) 0 | 0.00000000 | | | |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.00005645 | 0.00005645 | 0.00 | 0.9830 |
| trt | 1 | 0.16719912 | 0.16719912 | 2.10 | 0.3843 |
| subject(sequence | ce) 0 | 0.00000000 | | | |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.00005645 | 0.00005645 | 0.00 | 0.9830 |
| trt | 1 | 0.16719912 | 0.16719912 | 2.10 | 0.3843 |
| subject(sequence | ce) 0 | 0.00000000 | | | |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.00005645 | 0.00005645 | 0.00 | 0.9830 |
| trt | 1 | 0.16719912 | 0.16719912 | 2.10 | 0.3843 |
| subject(sequence | ee) 0 | 0.00000000 | | | |

Comparison: C vs B

Dependent Variable: V<sub>d</sub>/F/kg (L/kg) Weight Group: 76-87

## The GLM Procedure Least Squares Means

| | | H0:LSMean1=LSMean2 | |
|-----|-----------------|-----------------------|---------|
| trt | LN_VZFOW LSMEAN | | Pr > t |
| В | 0.48851732 | | 0.3843 |
| C | 0.89741721 | | |
| trt | LN VZFOW LSMEAN | 90% Confidence Limits | |

| В | 0.488517 | -0.770256 | 1.747291 |
|---|----------|-----------|----------|
| C | 0.897417 | -0.361356 | 2.156191 |

| Le | ast S | Squares Means for Effect | et trt | Least Squares Means for Effect trt |
|---|---|---|---|---|
| | | Difference Between | | |
| i | j | Means | 90% Confide | nce Limits for LSMean(i)-LSMean(j) |
| 1 | 2 | -0.408900 | -2.189074 | 1.371274 |

#### The GLM Procedure

Dependent Variable: LN\_VZFOW

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confi | dence Limits |
| C - B | 0.40889990 | 0.28195191 | 1.45 | 0.3843-1 | .37127442 | 2.18907421 |

Comparison: C vs B

Dependent Variable: V<sub>d</sub>/F (L) Weight Group: 76-87

| subject 2 301 406 sequence 2 ABC BAC trt 2 B C |
|------------------------------------------------|
| trt 2 B C |
| Number of Observations Read |

Comparison: C vs B

Dependent Variable: V<sub>d</sub>/F (L) Weight Group: 76-87

## The GLM Procedure

Dependent Variable: LN\_VZFO

| R-Square | Coeff Var | Root MSE | | LN V | ZFO Mean |
|---|---|---|---|---|---|
| 0.678310 | 5.487720 | 0.281952 | 5.137870 | _ | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.00042674 | 0.00042674 | 0.01 | 0.9534 |
| trt | 1 | 0.16719912 | 0.16719912 | 2.10 | 0.3843 |
| subject(sequence | e) 0 | 0.00000000 | | | |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.00042674 | 0.00042674 | 0.01 | 0.9534 |
| trt | 1 | 0.16719912 | 0.16719912 | 2.10 | 0.3843 |
| subject(sequence | e) 0 | 0.00000000 | | | |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.00042674 | 0.00042674 | 0.01 | 0.9534 |
| trt | 1 | 0.16719912 | 0.16719912 | 2.10 | 0.3843 |
| subject(sequence | e) 0 | 0.00000000 | | | |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.00042674 | 0.00042674 | 0.01 | 0.9534 |
| trt | 1 | 0.16719912 | 0.16719912 | 2.10 | 0.3843 |
| subject(sequence | e) 0 | 0.00000000 | | | |

Comparison: C vs B

Dependent Variable: V<sub>d</sub>/F (L) Weight Group: 76-87

## The GLM Procedure Least Squares Means

| | | H0:LSMean1=LSMean2 | |
|-----|----------------|--------------------|---------|
| trt | LN_VZFO LSMEAN | | Pr > t |
| В | 4.93341956 | | 0.3843 |
| C | 5.34231945 | | |

| trt | LN_VZFO LSMEAN | 90% Confidence Limits | |
|-----|----------------|-----------------------|----------|
| В | 4.933420 | 3.674646 | 6.192193 |
| C | 5.342319 | 4.083546 | 6.601093 |

| Le | Least Squares Means for Effect trt | | | |
|---|---|---|---|---|
| | | Difference Between | | |
| i | j | Means | 90% Confide | ence Limits for LSMean(i)-LSMean(j) |
| 1 | 2 | -0.408900 | -2.189074 | 1.371274 |

#### The GLM Procedure

Dependent Variable: LN\_VZFO

| | | Standard | | | |
|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confidence Limits |
| C - B | 0.40889990 | 0.28195191 | 1.45 | 0.3843-1 | .37127442 2.18907421 |

Comparison: C vs B

Dependent Variable: T<sub>max</sub> (h) Weight Group: 76-87

| Class | Levels | Values |
|-----------------------------|--------|---------|
| subject | 2 | 301 406 |
| sequence | 2 | ABC BAC |
| trt | 2 | ВС |
| Number of Observations Read | | |
| Number of Observations Used | | |

Comparison: C vs B

Dependent Variable: T<sub>max</sub> (h) Weight Group: 76-87

## The GLM Procedure

Dependent Variable: TMAX

| R-Square | Coeff Var | Root | MSE | T | MAX Mean |
|---|---|---|---|---|---|
| 0.500070 | 50.63480 | 0.508 | 3500 1 | .004250 | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.00007225 | 0.00007225 | 0.00 | 0.9894 |
| trt | 1 | 0.25857225 | 0.25857225 | 1.00 | 0.5000 |
| subject(sequence) | 0 | 0.00000000 | | | |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.00007225 | 0.00007225 | 0.00 | 0.9894 |
| trt | 1 | 0.25857225 | 0.25857225 | 1.00 | 0.5000 |
| subject(sequence) | 0 | 0.00000000 | | | |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.00007225 | 0.00007225 | 0.00 | 0.9894 |
| trt | 1 | 0.25857225 | 0.25857225 | 1.00 | 0.5000 |
| subject(sequence) | 0 | 0.00000000 | | | |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.00007225 | 0.00007225 | 0.00 | 0.9894 |
| trt | 1 | 0.25857225 | 0.25857225 | 1.00 | 0.5000 |
| subject(sequence) | 0 | 0.00000000 | | | |

Comparison: C vs B

Dependent Variable: T<sub>max</sub> (h) Weight Group: 76-87

## The GLM Procedure Least Squares Means

| | | H0: | LSMean1=LSMean2 | |
|---|---|---|---|---|
| trt | TMAX LSMEAN | | Pr > | > t |
| В | 0.75000000 | | 0.50 | 000 |
| C | 1.25850000 | | | |
| trt | TMAX LSMEAN | 9 | 0% Confidence Limits | |
| В | 0.750000 | -1.520196 | 3.020196 | |
| C | 1.258500 | -1.011696 | 3.528696 | |
| Le | ast Squares Means for Effec | et trt | | — |
| | Difference Between | | | |
| 1 | j Means | 90% Confidence Lir | nits for LSMean(i)-LSMean(j | <u>)</u> |
| 1 | 2 -0.508500 | -3.719043 | 2.702043 | |

#### The GLM Procedure

Dependent Variable: TMAX

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confid | dence Limits |
| C - B | 0.50850000 | 0.50850000 | 1.00 | 0.5000-2 | 2.70204265 | 3.71904265 |

Comparison: C vs B

Dependent Variable: K<sub>el</sub> (/h) Weight Group: 76-87

| Class | Levels | Values | |
|------------------|-------------|---------|---|
| subject | 2 | 301 406 | |
| sequence | 2 | ABC BAC | |
| trt | 2 | ВС | |
| Number of Observ | ations Read | | 4 |

Comparison: C vs B

Dependent Variable: K<sub>el</sub> (/h) Weight Group: 76-87

## The GLM Procedure

Dependent Variable: LAMZ

| R-Square | Coeff Var | Root | MSE | | LAMZ Mean |
|---|---|---|---|---|---|
| 0.998640 | 2.704657 | 0.000 | 0275 | 0.010153 | |
| Source | DF | Type I SS | Mean Square | F Value | e $Pr > F$ |
| sequence | 1 | 0.00002754 | 0.00002754 | 365.23 | 0.0333 |
| trt | 1 | 0.00002782 | 0.00002782 | 368.87 | 0.0331 |
| subject(sequence) | 0 | 0.00000000 | | | |
| Source | DF | Type II SS | Mean Square | F Value | e $Pr > F$ |
| sequence | 1 | 0.00002754 | 0.00002754 | 365.23 | 0.0333 |
| trt | 1 | 0.00002782 | 0.00002782 | 368.87 | 0.0331 |
| <pre>subject(sequence)</pre> | 0 | 0.00000000 | | | |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.00002754 | 0.00002754 | 365.23 | 0.0333 |
| trt | 1 | 0.00002782 | 0.00002782 | 368.87 | 0.0331 |
| <pre>subject(sequence)</pre> | 0 | 0.00000000 | | | |
| Source | DF | Type IV SS | Mean Square | F Value | e $Pr > F$ |
| sequence | 1 | 0.00002754 | 0.00002754 | 365.23 | 0.0333 |
| trt | 1 | 0.00002782 | 0.00002782 | 368.87 | 0.0331 |
| subject(sequence) | 0 | 0.00000000 | | | |

Comparison: C vs B

Dependent Variable: K<sub>el</sub> (/h) Weight Group: 76-87

## The GLM Procedure Least Squares Means

| | | | | H0:LS | Mean1=LSMean2 | |
|---|---|---|---|---|---|---|
| trt | LA | AMZ LSMEAN | | | | Pr > t |
| В | 0.0 | )1279051 | | | | 0.0331 |
| C | 0.0 | 00751627 | | | | |
| trt | L | AMZ LSMEAN | | 90% | % Confidence Limits | |
| В | 0. | 012791 | | 0.011564 | 0.014017 | |
| C | 0. | 007516 | | 0.006290 | 0.008742 | |
| Le | ast S | Squares Means for Effec | et trt | | | |
| | | Difference Between | | | | |
| i | j | Means | 90% Con | fidence Limit | s for LSMean(i)-LSM | Iean(j) |
| 1 | 2 | 0.005274 | 0.003540 | | 0.007008 | |

#### The GLM Procedure

Dependent Variable: LAMZ

| <u>, </u> | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confi | dence Limits |
| C - B | -0.00527424 | 0.00027461 | -19.21 | 0.0331-0 | 0.00700808 | -0.00354039 |

Comparison: C vs B

Dependent Variable: T<sub>1/2 el</sub> (h) Weight Group: 76-87

| subject 2 301 406 sequence 2 ABC BAC trt 2 B C | |
|---|---|
| trt 2 B C | |
| Number of Observations Read | 4 |

Comparison: C vs B

Dependent Variable: T<sub>1/2 el</sub> (h) Weight Group: 76-87

## The GLM Procedure

Dependent Variable: LAMZHL

| R-Square Coeff Var Roo | | Root MSE | | LAM | ZHL Mean |
|---|---|---|---|---|---|
| 0.899909 | 27.41894 | 21.98952 | 80.19828 | | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 2165.315655 | 2165.315655 | 4.48 | 0.2810 |
| trt | 1 | 2182.123274 | 2182.123274 | 4.51 | 0.2801 |
| subject(sequence | - | 0.000000 | 2102.123274 | 4.51 | 0.2001 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | <u>Dr</u><br>1 | 2165.315655 | 2165.315655 | 4.48 | 0.2810 |
| trt | 1 | 2182.123274 | 2182.123274 | 4.51 | 0.2801 |
| subject(sequence | _ | 0.000000 | 2102.123271 | 1.51 | 0.2001 |
| | / | | | | |
| <u>C</u> | DE | T-ma III CC | Maan Canana | E Walna | D <sub>n</sub> × E |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 2165.315655 | 2165.315655 | 4.48 | 0.2810 |
| trt | 1 | 2182.123274 | 2182.123274 | 4.51 | 0.2801 |
| subject(sequence | e) 0 | 0.000000 | | | |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 2165.315655 | 2165.315655 | 4.48 | 0.2810 |
| trt | 1 | 2182.123274 | 2182.123274 | 4.51 | 0.2801 |
| subject(sequence | e) 0 | 0.000000 | | | |

Comparison: C vs B

Dependent Variable: T<sub>1/2 el</sub> (h) Weight Group: 76-87

## The GLM Procedure Least Squares Means

| | | HO | :LSMean1=LSMean2 |
|---|---|---|---|
| trt | LAMZHL LSMEAN | | Pr > |
| В | 56.841678 | | 0.280 |
| C | 103.554880 | | |
| trt | LAMZHL LSMEAN | 9 | 0% Confidence Limits |
| В | 56.841678 | -41.330441 | 155.013796 |
| C | 103.554880 | 5.382761 | 201.726999 |
| Lea | ast Squares Means for Effect | et trt | |
| | Difference Between | | |
| i | j Means | 90% Confidence | ee Limits for LSMean(i)-LSMean(j) |
| 1 | 2 -46.713202 | -185.549544 | 92.123140 |

#### The GLM Procedure

Dependent Variable: LAMZHL

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Conf | idence Limits |
| C - B | 46.7132024 | 21.9895163 | 2.12 | 0.2801-9 | 2.1231396 | 185.5495443 |

Comparison: A vs B

Dependent Variable: AUC<sub>0-t</sub> (h\*ng/mL) Weight Group: 88-111

| Class Leve | l Informa | tion |
|---|---|---|
| Class | Levels | Values |
| subject | 11 | 203 204 304 402 404 407 409 502 505 507 508 |
| sequence | 2 | AB BA |
| period | 2 | 1 2 |
| trt | 2 | A B |
| Number of Observations Read 22 | | |
| Number of | Number of Observations Used 22 | |

Comparison: A vs B

Dependent Variable: AUC<sub>0-t</sub> (h\*ng/mL) Weight Group: 88-111

## The GLM Procedure

| R-Square Coeff Var | | Root MSE | | LN_AUCI | LST Mean |
|---|---|---|---|---|---|
| 0.624540 | 10.97272 | 0.944959 | 8.611893 | | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.34347906 | 0.34347906 | 0.38 | 0.5505 |
| period | 1 | 0.00482396 | 0.00482396 | 0.01 | 0.9430 |
| trt | 1 | 2.32311575 | 2.32311575 | 2.60 | 0.1412 |
| subject(sequence | e) 9 | 10.69654172 | 1.18850464 | 1.33 | 0.3385 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.34347906 | 0.34347906 | 0.38 | 0.5505 |
| period | 1 | 0.04315122 | 0.04315122 | 0.05 | 0.8309 |
| trt | 1 | 2.32311575 | 2.32311575 | 2.60 | 0.1412 |
| subject(sequence | e) 9 | 10.69654172 | 1.18850464 | 1.33 | 0.3385 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.34347906 | 0.34347906 | 0.38 | 0.5505 |
| period | 1 | 0.04315122 | 0.04315122 | 0.05 | 0.8309 |
| trt | 1 | 2.32311575 | 2.32311575 | 2.60 | 0.1412 |
| subject(sequence | e) 9 | 10.69654172 | 1.18850464 | 1.33 | 0.3385 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.34347906 | 0.34347906 | 0.38 | 0.5505 |
| period | 1 | 0.04315122 | 0.04315122 | 0.05 | 0.8309 |
| trt | 1 | 2.32311575 | 2.32311575 | 2.60 | 0.1412 |
| subject(sequence | e) 9 | 10.69654172 | 1.18850464 | 1.33 | 0.3385 |

Comparison: A vs B

Dependent Variable: AUC<sub>0-t</sub> (h\*ng/mL) Weight Group: 88-111

## The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_AUCLST

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.343479 | 0.343479 | 0.29 | 0.6039 |
| Error | 9 | 10.696542 | 1.188505 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| *period | 1 | 0.004824 | 0.004824 | 0.01 | 0.9430 |
| trt | 1 | 2.323116 | 2.323116 | 2.60 | 0.1412 |
| subject(sequence) | 9 | 10.696542 | 1.188505 | 1.33 | 0.3385 |
| Error: MS(Error) | 9 | 8.036520 | 0.892947 | | |
| This test assumes one or more other fixed effects are zero. | | | | | |

## Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.343479 | 0.343479 | 0.29 | 0.6039 |
| Error 9 10.696542 1.188505 | | | | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.043151 | 0.043151 | 0.05 | 0.8309 |
| trt | 1 | 2.323116 | 2.323116 | 2.60 | 0.1412 |
| subject(sequence) | 9 | 10.696542 | 1.188505 | 1.33 | 0.3385 |
| Error: MS(Error) | 9 | 8.036520 | 0.892947 | | |

Comparison: A vs B

Dependent Variable: AUC<sub>0-t</sub> (h\*ng/mL) Weight Group: 88-111

## Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_AUCLST

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.343479 | 0.343479 | 0.29 | 0.6039 |
| Error 9 10.696542 1.188505 | | | | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 0.043151 | 0.043151 | 0.05 | 0.8309 |
| trt | 1 | 2.323116 | 2.323116 | 2.60 | 0.1412 |
| subject(sequence) | 9 | 10.696542 | 1.188505 | 1.33 | 0.3385 |
| Error: MS(Error) | 9 | 8.036520 | 0.892947 | | |

## Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------|-----------|------------|-------------|---------|--------|
| sequence | 1 | 0.343479 | 0.343479 | 0.29 | 0.6039 |
| Error | 9 | 10.696542 | 1.188505 | | |
| Error: MS(s | subject(s | sequence)) | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.043151 | 0.043151 | 0.05 | 0.8309 |
| trt | 1 | 2.323116 | 2.323116 | 2.60 | 0.1412 |
| subject(sequence) | 9 | 10.696542 | 1.188505 | 1.33 | 0.3385 |
| Error: MS(Error) | 9 | 8.036520 | 0.892947 | | |

Comparison: A vs B

Dependent Variable: AUC<sub>0-t</sub> (h\*ng/mL) Weight Group: 88-111

## Least Squares Means

| | | H0:LSM | Iean1=LSMean2 | |
|-----|------------------|----------|-------------------|---------|
| trt | LN_AUCLST LSMEAN | | | Pr > t |
| A | 8.92679321 | | | 0.1412 |
| В | 8.27417958 | | | |
| trt | LN_AUCLST LSMEAN | 90% | Confidence Limits | |
| A | 8.926793 | 8.402339 | 9.451248 | |
| | 8.274180 | 7.749725 | 8.798634 | |

Least Squares Means for Effect trt
Difference Between

| i | j | Means | 90% Confidence L | imits for LSMean(i)-LSMean(j) |
|---|---|----------|------------------|-------------------------------|
| 1 | 2 | 0.652614 | -0.089077 | 1.394304 |

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confi | dence Limits |
| A - B | 0.65261363 | 0.40460708 | 1.61 | 0.1412-0 | 0.08907684 | 1.39430410 |

Comparison: A vs B

Dependent Variable: AUC<sub>0-inf</sub> (h\*ng/mL) Weight Group: 88-111

| Class Leve | l Informa | tion |
|---|---|---|
| Class | Levels | Values |
| subject | 11 | 203 204 304 402 404 407 409 502 505 507 508 |
| sequence | 2 | AB BA |
| period | 2 | 1 2 |
| trt | 2 | A B |
| Number of Observations Read 22 | | |
| Number of | Number of Observations Used 22 | |

Comparison: A vs B

Dependent Variable: AUC<sub>0-inf</sub> (h\*ng/mL) Weight Group: 88-111

## The GLM Procedure

Dependent Variable: LN\_AUCIFO

| R-Square | Coeff Var | Root MSE | | LN_AUC | IFO Mean |
|-----------------|-----------|-------------|-------------|---------|----------|
| 0.810830 | 6.590357 | 0.587678 | 8.917241 | | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.69862990 | 0.69862990 | 2.02 | 0.1887 |
| period | 1 | 0.23085126 | 0.23085126 | 0.67 | 0.4347 |
| trt | 1 | 1.60598632 | 1.60598632 | 4.65 | 0.0594 |
| subject(sequenc | e) 9 | 10.78744135 | 1.19860459 | 3.47 | 0.0389 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.69862990 | 0.69862990 | 2.02 | 0.1887 |
| period | 1 | 0.35246442 | 0.35246442 | 1.02 | 0.3388 |
| trt | 1 | 1.60598632 | 1.60598632 | 4.65 | 0.0594 |
| subject(sequenc | e) 9 | 10.78744135 | 1.19860459 | 3.47 | 0.0389 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.69862990 | 0.69862990 | 2.02 | 0.1887 |
| period | 1 | 0.35246442 | 0.35246442 | 1.02 | 0.3388 |
| trt | 1 | 1.60598632 | 1.60598632 | 4.65 | 0.0594 |
| subject(sequenc | e) 9 | 10.78744135 | 1.19860459 | 3.47 | 0.0389 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.69862990 | 0.69862990 | 2.02 | 0.1887 |
| period | 1 | 0.35246442 | 0.35246442 | 1.02 | 0.3388 |
| trt | 1 | 1.60598632 | 1.60598632 | 4.65 | 0.0594 |
| subject(sequenc | e) 9 | 10.78744135 | 1.19860459 | 3.47 | 0.0389 |
Comparison: A vs B

Dependent Variable: AUC<sub>0-inf</sub> (h\*ng/mL) Weight Group: 88-111

### The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN AUCIFO

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.698630 | 0.698630 | 0.58 | 0.4647 |
| Error | 9 | 10.787441 | 1.198605 | | _ |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| *period | 1 | 0.230851 | 0.230851 | 0.67 | 0.4347 |
| trt | 1 | 1.605986 | 1.605986 | 4.65 | 0.0594 |
| subject(sequence) | 9 | 10.787441 | 1.198605 | 3.47 | 0.0389 |
| Error: MS(Error) | 9 | 3.108289 | 0.345365 | | |
| * This test assumes one or m | ore oth | er fixed effects | are zero. | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.698630 | 0.698630 | 0.58 | 0.4647 |
| Error | 9 | 10.787441 | 1.198605 | | |
| Error: MS(s | Error: MS(subject(sequence)) | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.352464 | 0.352464 | 1.02 | 0.3388 |
| trt | 1 | 1.605986 | 1.605986 | 4.65 | 0.0594 |
| subject(sequence) | 9 | 10.787441 | 1.198605 | 3.47 | 0.0389 |
| Error: MS(Error) | 9 | 3.108289 | 0.345365 | | |

Comparison: A vs B

Dependent Variable: AUC<sub>0-inf</sub> (h\*ng/mL) Weight Group: 88-111

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_AUCIFO

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.698630 | 0.698630 | 0.58 | 0.4647 |
| Error | 9 | 10.787441 | 1.198605 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 0.352464 | 0.352464 | 1.02 | 0.3388 |
| trt | 1 | 1.605986 | 1.605986 | 4.65 | 0.0594 |
| subject(sequence) | 9 | 10.787441 | 1.198605 | 3.47 | 0.0389 |
| Error: MS(Error) | 9 | 3.108289 | 0.345365 | | - |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.698630 | 0.698630 | 0.58 | 0.4647 |
| Error | 9 | 10.787441 | 1.198605 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.352464 | 0.352464 | 1.02 | 0.3388 |
| trt | 1 | 1.605986 | 1.605986 | 4.65 | 0.0594 |
| subject(sequence) | 9 | 10.787441 | 1.198605 | 3.47 | 0.0389 |
| Error: MS(Error) | 9 | 3.108289 | 0.345365 | | |

Comparison: A vs B

Dependent Variable: AUC<sub>0-inf</sub> (h\*ng/mL) Weight Group: 88-111

#### Least Squares Means

| | | H0:LSM | Iean1=LSMean2 | |
|---|---|---|---|---|
| trt | LN_AUCIFO LSMEAN | | | Pr > t |
| A | 9.17228121 | | | 0.0594 |
| В | 8.62966640 | | | |
| trt | LN AUCIFO LSMEAN | 90% | Confidence Limits | |
| trt<br>A | LN_AUCIFO LSMEAN<br>9.172281 | 90%<br>8.846118 | Confidence Limits<br>9.498444 | |

Least Squares Means for Effect trtDifference BetweenijMeans90% Confidence Limits for LSMean(i)-LSMean(j)120.5426150.0813511.003879

| | | Standard | | |
|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t 90% Confidence Limits |
| A - B | 0.54261480 | 0.25162870 | 2.16 | 0.05940.08135098 1.00387863 |

Comparison: A vs B

Dependent Variable: C<sub>max</sub> (ng/mL) Weight Group: 88-111

#### The GLM Procedure

| Class Leve | el Informa | tion |
|---|---|---|
| Class | Levels | Values |
| subject | 11 | 203 204 304 402 404 407 409 502 505 507 508 |
| sequence | 2 | AB BA |
| period | 2 | 1 2 |
| trt | 2 | A B |
| Number of | Number of Observations Read 22 | |
| Number of | Number of Observations Used 22 | |

Comparison: A vs B

Dependent Variable: C<sub>max</sub> (ng/mL) Weight Group: 88-111

#### The GLM Procedure

| R-Square | Coeff Var | Root MSE | | LN_CM | IAX Mean |
|---|---|---|---|---|---|
| 0.462659 | 19.25038 | 0.955689 | 4.964517 | | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.05327995 | 0.05327995 | 0.06 | 0.8146 |
| period | 1 | 0.73440347 | 0.73440347 | 0.80 | 0.3932 |
| trt | 1 | 0.94378043 | 0.94378043 | 1.03 | 0.3359 |
| subject(sequence | e) 9 | 5.34614197 | 0.59401577 | 0.65 | 0.7341 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.05327995 | 0.05327995 | 0.06 | 0.8146 |
| period | 1 | 0.88687719 | 0.88687719 | 0.97 | 0.3502 |
| trt | 1 | 0.94378043 | 0.94378043 | 1.03 | 0.3359 |
| subject(sequence | e) 9 | 5.34614197 | 0.59401577 | 0.65 | 0.7341 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.05327995 | 0.05327995 | 0.06 | 0.8146 |
| period | 1 | 0.88687719 | 0.88687719 | 0.97 | 0.3502 |
| trt | 1 | 0.94378043 | 0.94378043 | 1.03 | 0.3359 |
| subject(sequence | e) 9 | 5.34614197 | 0.59401577 | 0.65 | 0.7341 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.05327995 | 0.05327995 | 0.06 | 0.8146 |
| period | 1 | 0.88687719 | 0.88687719 | 0.97 | 0.3502 |
| trt | 1 | 0.94378043 | 0.94378043 | 1.03 | 0.3359 |
| subject(sequence | e) 9 | 5.34614197 | 0.59401577 | 0.65 | 0.7341 |

Comparison: A vs B

Dependent Variable: C<sub>max</sub> (ng/mL) Weight Group: 88-111

### The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_CMAX

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.053280 | 0.053280 | 0.09 | 0.7714 |
| Error 9 5.346142 0.594016 | | | | | |
| Error: MS(s | Error: MS(subject(sequence)) | | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| *period | 1 | 0.734403 | 0.734403 | 0.80 | 0.3932 |
| trt | 1 | 0.943780 | 0.943780 | 1.03 | 0.3359 |
| subject(sequence) | 9 | 5.346142 | 0.594016 | 0.65 | 0.7341 |
| Error: MS(Error) | 9 | 8.220065 | 0.913341 | | |
| * This test assumes one or m | ore oth | ner fixed effects | are zero. | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------|----------|------------|-------------|---------|--------|
| sequence | 1 | 0.053280 | 0.053280 | 0.09 | 0.7714 |
| Error | 9 | 5.346142 | 0.594016 | | |
| Error: MS(s | ubiect(s | equence)) | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.886877 | 0.886877 | 0.97 | 0.3502 |
| trt | 1 | 0.943780 | 0.943780 | 1.03 | 0.3359 |
| subject(sequence) | 9 | 5.346142 | 0.594016 | 0.65 | 0.7341 |
| Error: MS(Error) | 9 | 8.220065 | 0.913341 | | |

Comparison: A vs B

Dependent Variable: C<sub>max</sub> (ng/mL) Weight Group: 88-111

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_CMAX

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.053280 | 0.053280 | 0.09 | 0.7714 |
| Error | 9 | 5.346142 | 0.594016 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 0.886877 | 0.886877 | 0.97 | 0.3502 |
| trt | 1 | 0.943780 | 0.943780 | 1.03 | 0.3359 |
| subject(sequence) | 9 | 5.346142 | 0.594016 | 0.65 | 0.7341 |
| Error: MS(Error) | 9 | 8.220065 | 0.913341 | | - |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.053280 | 0.053280 | 0.09 | 0.7714 |
| Error | 9 | 5.346142 | 0.594016 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.886877 | 0.886877 | 0.97 | 0.3502 |
| trt | 1 | 0.943780 | 0.943780 | 1.03 | 0.3359 |
| subject(sequence) | 9 | 5.346142 | 0.594016 | 0.65 | 0.7341 |
| Error: MS(Error) | 9 | 8.220065 | 0.913341 | | |

Comparison: A vs B

Dependent Variable: C<sub>max</sub> (ng/mL) Weight Group: 88-111

#### Least Squares Means

| | | H0:LS | SMean1=LSMean2 | |
|-----|----------------|----------|---------------------|---------|
| trt | LN_CMAX LSMEAN | | | Pr > t |
| A | 5.16800682 | | | 0.3359 |
| В | 4.75204239 | | | |
| trt | LN_CMAX LSMEAN | 909 | % Confidence Limits | |
| A | 5.168007 | 4.637597 | 5.698416 | |
| B | 4.752042 | 4.221633 | 5.282452 | |

Least Squares Means for Effect trt
Difference Between
i j Means 90% Confidence Limits for LSMean(i)-LSMean(j)
1 2 0.415964 -0.334148 1.166077

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confi | dence Limits |
| A - B | 0.41596444 | 0.40920138 | 1.02 | 0.3359-0 | 0.33414790 | 1.16607677 |

Comparison: A vs B

Dependent Variable: Cl/F/kg ((L/h)/kg) Weight Group: 88-111

#### The GLM Procedure

| Class Leve | el Informa | tion | |
|---|---|---|---|
| Class | Levels | Values | |
| subject | 11 | 203 204 304 402 404 407 409 502 505 507 508 | |
| sequence | 2 | AB BA | |
| period | 2 | 1 2 | |
| trt | 2 | A B | |
| Number of | f Observat | tions Read | 22 |
| Number of | Number of Observations Used 2 | | |

Comparison: A vs B

Dependent Variable: Cl/F/kg ((L/h)/kg) Weight Group: 88-111

#### The GLM Procedure

| R-Square | Coeff Var | Root MSE | | LN_CLF | OW Mean |
|------------------|-----------|-------------|-------------|---------|---------|
| 0.840724 | -15.77847 | 0.587678 | -3.724556 | | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.95042330 | 0.95042330 | 2.75 | 0.1315 |
| period | 1 | 0.20430477 | 0.20430477 | 0.59 | 0.4615 |
| trt | 1 | 2.49367461 | 2.49367461 | 7.22 | 0.0249 |
| subject(sequence | e) 9 | 12.75844172 | 1.41760464 | 4.10 | 0.0236 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.95042330 | 0.95042330 | 2.75 | 0.1315 |
| period | 1 | 0.35246442 | 0.35246442 | 1.02 | 0.3388 |
| trt | 1 | 2.49367461 | 2.49367461 | 7.22 | 0.0249 |
| subject(sequence | e) 9 | 12.75844172 | 1.41760464 | 4.10 | 0.0236 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.95042330 | 0.95042330 | 2.75 | 0.1315 |
| period | 1 | 0.35246442 | 0.35246442 | 1.02 | 0.3388 |
| trt | 1 | 2.49367461 | 2.49367461 | 7.22 | 0.0249 |
| subject(sequence | e) 9 | 12.75844172 | 1.41760464 | 4.10 | 0.0236 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.95042330 | 0.95042330 | 2.75 | 0.1315 |
| period | 1 | 0.35246442 | 0.35246442 | 1.02 | 0.3388 |
| trt | 1 | 2.49367461 | 2.49367461 | 7.22 | 0.0249 |
| subject(sequence | e) 9 | 12.75844172 | 1.41760464 | 4.10 | 0.0236 |

Comparison: A vs B

Dependent Variable: Cl/F/kg ((L/h)/kg) Weight Group: 88-111

### The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_CLFOW

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.950423 | 0.950423 | 0.67 | 0.4340 |
| Error | 9 | 12.758442 | 1.417605 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| *period | 1 | 0.204305 | 0.204305 | 0.59 | 0.4615 |
| trt | 1 | 2.493675 | 2.493675 | 7.22 | 0.0249 |
| subject(sequence) | 9 | 12.758442 | 1.417605 | 4.10 | 0.0236 |
| Error: MS(Error) 9 3.108289 0.345365 | | | | | |
| * This test assumes one or more other fixed effects are zero. | | | | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------|----------|------------|-------------|---------|--------|
| sequence | 1 | 0.950423 | 0.950423 | 0.67 | 0.4340 |
| Error | 9 | 12.758442 | 1.417605 | | |
| Error: MS(s | ubject(s | equence)) | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.352464 | 0.352464 | 1.02 | 0.3388 |
| trt | 1 | 2.493675 | 2.493675 | 7.22 | 0.0249 |
| subject(sequence) | 9 | 12.758442 | 1.417605 | 4.10 | 0.0236 |
| Error: MS(Error) | 9 | 3.108289 | 0.345365 | | |

Comparison: A vs B

Dependent Variable: Cl/F/kg ((L/h)/kg) Weight Group: 88-111

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_CLFOW

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.950423 | 0.950423 | 0.67 | 0.4340 |
| Error | 9 | 12.758442 | 1.417605 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 0.352464 | 0.352464 | 1.02 | 0.3388 |
| trt | 1 | 2.493675 | 2.493675 | 7.22 | 0.0249 |
| subject(sequence) | 9 | 12.758442 | 1.417605 | 4.10 | 0.0236 |
| Error: MS(Error) | 9 | 3.108289 | 0.345365 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.950423 | 0.950423 | 0.67 | 0.4340 |
| Error | 9 | 12.758442 | 1.417605 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.352464 | 0.352464 | 1.02 | 0.3388 |
| trt | 1 | 2.493675 | 2.493675 | 7.22 | 0.0249 |
| subject(sequence) | 9 | 12.758442 | 1.417605 | 4.10 | 0.0236 |
| Error: MS(Error) | 9 | 3.108289 | 0.345365 | | |

Comparison: A vs B

Dependent Variable: Cl/F/kg ((L/h)/kg) Weight Group: 88-111

-0.676146

#### Least Squares Means

| | | H0:LSMean1=LSMean2 | | |
|---|---|---|---|---|
| trt | LN_CLFOW LSMEAN | | | Pr > t |
| A | -4.04365537 | | | 0.0249 |
| В | -3.36750918 | | | |
| trt | LN_CLFOW LSMEAN | 90 | % Confidence Limits | |
| A | -4.043655 | -4.369818 | -3.717493 | |
| В | -3.367509 | -3.693672 | -3.041346 | |
| Lea | ast Squares Means for Effect | trt | | |
| | Difference Between | | | |
| i j Means 90% Confidence Limits for LSMean(i)-LSMe | | | | |

#### Dependent Variable: LN\_CLFOW

-0.214882

-1.137410

| | | Standard | | | |
|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confidence Limits |
| A - B | -0.67614620 | 0.25162870 | -2.69 | 0.0249-1 | .13741002 -0.21488237 |

Dependent Variable: Cl/F (L/h) Weight Group: 88-111

#### The GLM Procedure

| Class Leve | l Informa | tion |
|---|---|---|
| Class | Levels | Values |
| subject | 11 | 203 204 304 402 404 407 409 502 505 507 508 |
| sequence | 2 | AB BA |
| period | 2 | 1 2 |
| trt | 2 | A B |
| Number of | Number of Observations Read 22 | |
| Number of | Number of Observations Used | |

Comparison: A vs B

Dependent Variable: Cl/F (L/h) Weight Group: 88-111

#### The GLM Procedure

| R-Square | Coeff Var | Root MSE | | LN_CI | LFO Mean |
|---|---|---|---|---|---|
| 0.820251 | 63.91414 | 0.587678 | 0.919481 | | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > I |
| sequence | 1 | 0.69862990 | 0.69862990 | 2.02 | 0.1887 |
| period | 1 | 0.20430477 | 0.20430477 | 0.59 | 0.4615 |
| trt | 1 | 2.49367461 | 2.49367461 | 7.22 | 0.0249 |
| subject(sequence) | 9 | 10.78744135 | 1.19860459 | 3.47 | 0.0389 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.69862990 | 0.69862990 | 2.02 | 0.1887 |
| period | 1 | 0.35246442 | 0.35246442 | 1.02 | 0.3388 |
| trt | 1 | 2.49367461 | 2.49367461 | 7.22 | 0.0249 |
| subject(sequence) | 9 | 10.78744135 | 1.19860459 | 3.47 | 0.0389 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.69862990 | 0.69862990 | 2.02 | 0.1887 |
| period | 1 | 0.35246442 | 0.35246442 | 1.02 | 0.3388 |
| trt | 1 | 2.49367461 | 2.49367461 | 7.22 | 0.0249 |
| subject(sequence) | 9 | 10.78744135 | 1.19860459 | 3.47 | 0.0389 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.69862990 | 0.69862990 | 2.02 | 0.1887 |
| period | 1 | 0.35246442 | 0.35246442 | 1.02 | 0.3388 |
| trt | 1 | 2.49367461 | 2.49367461 | 7.22 | 0.0249 |
| subject(sequence) | 9 | 10.78744135 | 1.19860459 | 3.47 | 0.0389 |

Comparison: A vs B

Dependent Variable: Cl/F (L/h) Weight Group: 88-111

### The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_CLFO

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.698630 | 0.698630 | 0.58 | 0.4647 |
| Error | 9 | 10.787441 | 1.198605 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| *period | 1 | 0.204305 | 0.204305 | 0.59 | 0.4615 |
| trt | 1 | 2.493675 | 2.493675 | 7.22 | 0.0249 |
| subject(sequence) | 9 | 10.787441 | 1.198605 | 3.47 | 0.0389 |
| Error: MS(Error) 9 3.108289 0.345365 | | | | | |
| * This test assumes one or more other fixed effects are zero. | | | | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.698630 | 0.698630 | 0.58 | 0.4647 |
| Error | 9 | 10.787441 | 1.198605 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.352464 | 0.352464 | 1.02 | 0.3388 |
| trt | 1 | 2.493675 | 2.493675 | 7.22 | 0.0249 |
| subject(sequence) | 9 | 10.787441 | 1.198605 | 3.47 | 0.0389 |
| Error: MS(Error) | 9 | 3.108289 | 0.345365 | | |

Comparison: A vs B

Dependent Variable: Cl/F (L/h) Weight Group: 88-111

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_CLFO

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.698630 | 0.698630 | 0.58 | 0.4647 |
| Error | 9 | 10.787441 | 1.198605 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 0.352464 | 0.352464 | 1.02 | 0.3388 |
| trt | 1 | 2.493675 | 2.493675 | 7.22 | 0.0249 |
| subject(sequence) | 9 | 10.787441 | 1.198605 | 3.47 | 0.0389 |
| Error: MS(Error) | 9 | 3.108289 | 0.345365 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.698630 | 0.698630 | 0.58 | 0.4647 |
| Error | 9 | 10.787441 | 1.198605 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.352464 | 0.352464 | 1.02 | 0.3388 |
| trt | 1 | 2.493675 | 2.493675 | 7.22 | 0.0249 |
| subject(sequence) | 9 | 10.787441 | 1.198605 | 3.47 | 0.0389 |
| Error: MS(Error) | 9 | 3.108289 | 0.345365 | | |

Comparison: A vs B

Dependent Variable: Cl/F (L/h) Weight Group: 88-111

#### Least Squares Means

| | | H0:LSMean1=LSMean2 | |
|-----|----------------|-----------------------|---------|
| trt | LN_CLFO LSMEAN | | Pr > t |
| A | 0.59767495 | | 0.0249 |
| В | 1.27382115 | | |
| trt | LN CLFO LSMEAN | 90% Confidence Limits | |

| trt | LN_CLFO LSMEAN | 9 | 0% Confidence Limits |
|-----|----------------|----------|----------------------|
| A | 0.597675 | 0.271512 | 0.923838 |
| В | 1.273821 | 0.947658 | 1.599984 |

| Le | Least Squares Means for Effect trt | | | |
|---|---|---|---|---|
| | | Difference Between | | |
| i | j | Means | 90% Confide | nce Limits for LSMean(i)-LSMean(j) |
| 1 | 2 | -0.676146 | -1.137410 | -0.214882 |

| | | Standard | | | |
|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confidence Limits |
| A - B | -0.67614620 | 0.25162870 | -2.69 | 0.0249-1 | .13741002 -0.21488237 |

Comparison: A vs B

Dependent Variable: V<sub>d</sub>/F/kg (L/kg) Weight Group: 88-111

#### The GLM Procedure

| Class | Levels | Values | |
|---|---|---|---|
| subject | 11 | 203 204 304 402 404 407 409 502 505 507 508 | |
| sequence | 2 | AB BA | |
| period | 2 | 1 2 | |
| trt | 2 | A B | |
| Number of | f Observat | tions Read | 22 |
| Number of Observations Used | | | 22 |

Comparison: A vs B

Dependent Variable: V<sub>d</sub>/F/kg (L/kg) Weight Group: 88-111

#### The GLM Procedure

| R-Square | Coeff Var | Root MSE | | LN_VZF | OW Mean |
|------------------|-----------|-------------|-------------|---------|---------|
| 0.530952 | 83.84526 | 1.109423 | 1.323179 | | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.27195823 | 0.27195823 | 0.22 | 0.6495 |
| period | 1 | 0.01551644 | 0.01551644 | 0.01 | 0.9131 |
| trt | 1 | 3.73511476 | 3.73511476 | 3.03 | 0.1155 |
| subject(sequence | e) 9 | 8.51675186 | 0.94630576 | 0.77 | 0.6491 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.27195823 | 0.27195823 | 0.22 | 0.6495 |
| period | 1 | 0.00266729 | 0.00266729 | 0.00 | 0.9639 |
| trt | 1 | 3.73511476 | 3.73511476 | 3.03 | 0.1155 |
| subject(sequence | e) 9 | 8.51675186 | 0.94630576 | 0.77 | 0.6491 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.27195823 | 0.27195823 | 0.22 | 0.6495 |
| period | 1 | 0.00266729 | 0.00266729 | 0.00 | 0.9639 |
| trt | 1 | 3.73511476 | 3.73511476 | 3.03 | 0.1155 |
| subject(sequence | e) 9 | 8.51675186 | 0.94630576 | 0.77 | 0.6491 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.27195823 | 0.27195823 | 0.22 | 0.6495 |
| period | 1 | 0.00266729 | 0.00266729 | 0.00 | 0.9639 |
| trt | 1 | 3.73511476 | 3.73511476 | 3.03 | 0.1155 |
| subject(sequence | e) 9 | 8.51675186 | 0.94630576 | 0.77 | 0.6491 |

Comparison: A vs B

Dependent Variable: V<sub>d</sub>/F/kg (L/kg) Weight Group: 88-111

### The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_VZFOW

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.271958 | 0.271958 | 0.29 | 0.6049 |
| Error | 9 | 8.516752 | 0.946306 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| *period | 1 | 0.015516 | 0.015516 | 0.01 | 0.9131 |
| trt | 1 | 3.735115 | 3.735115 | 3.03 | 0.1155 |
| subject(sequence) | 9 | 8.516752 | 0.946306 | 0.77 | 0.6491 |
| Error: MS(Error) 9 11.077366 1.230818 | | | | | |
| * This test assumes one or more other fixed effects are zero. | | | | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.271958 | 0.271958 | 0.29 | 0.6049 |
| Error | 9 | 8.516752 | 0.946306 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.002667 | 0.002667 | 0.00 | 0.9639 |
| trt | 1 | 3.735115 | 3.735115 | 3.03 | 0.1155 |
| subject(sequence) | 9 | 8.516752 | 0.946306 | 0.77 | 0.6491 |
| Error: MS(Error) | 9 | 11.077366 | 1.230818 | | |

Comparison: A vs B

Dependent Variable: V<sub>d</sub>/F/kg (L/kg) Weight Group: 88-111

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_VZFOW

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.271958 | 0.271958 | 0.29 | 0.6049 |
| Error | 9 | 8.516752 | 0.946306 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|-------------|
| period | 1 | 0.002667 | 0.002667 | 0.00 | 0.9639 |
| trt | 1 | 3.735115 | 3.735115 | 3.03 | 0.1155 |
| subject(sequence) | 9 | 8.516752 | 0.946306 | 0.77 | 0.6491 |
| Error: MS(Error) | 9 | 11.077366 | 1.230818 | · | <del></del> |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.271958 | 0.271958 | 0.29 | 0.6049 |
| Error | 9 | 8.516752 | 0.946306 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.002667 | 0.002667 | 0.00 | 0.9639 |
| trt | 1 | 3.735115 | 3.735115 | 3.03 | 0.1155 |
| subject(sequence) | 9 | 8.516752 | 0.946306 | 0.77 | 0.6491 |
| Error: MS(Error) | 9 | 11.077366 | 1.230818 | | |

Comparison: A vs B

Dependent Variable: V<sub>d</sub>/F/kg (L/kg) Weight Group: 88-111

#### Least Squares Means

| | | H0: | LSMean1=LSMean2 | |
|-----|-----------------|----------|-----------------------|---------|
| trt | LN_VZFOW LSMEAN | | | Pr > t |
| A | 0.91957377 | | | 0.1155 |
| В | 1.74708271 | | | |
| trt | LN_VZFOW LSMEAN | ! | 90% Confidence Limits | |
| A | 0.919574 | 0.303841 | 1.535306 | |
| В | 1.747083 | 1.131350 | 2.362815 | |

Least Squares Means for Effect trt

Difference Between

i j Means 90% Confidence Limits for LSMean(i)-LSMean(j)

1 2 -0.827509 -1.698286 0.043268

| | | Standard | | |
|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t 90% Confidence Limits |
| A - B | -0.82750894 | 0.47502636 | -1.74 | 0.1155-1.69828590 0.04326803 |

Comparison: A vs B

Dependent Variable: V<sub>d</sub>/F (L) Weight Group: 88-111

#### The GLM Procedure

| Class | Levels | Values | |
|-----------|------------|---------------------------------------------|----|
| subject | 11 | 203 204 304 402 404 407 409 502 505 507 508 | |
| sequence | 2 | AB BA | |
| period | 2 | 1 2 | |
| trt | 2 | A B | |
| Number of | f Observat | tions Read | 22 |
| 3.7 1 | 0.01 | tions Used | 22 |

Comparison: A vs B

Dependent Variable: V<sub>d</sub>/F (L) Weight Group: 88-111

#### The GLM Procedure

| R-Square | Coeff Var | Root MSE | <u>C</u> | LN_ | VZFO Mean |
|---|---|---|---|---|---|
| 0.511939 | 18.59196 | 1.109423 | 5.967215 | | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.14626067 | 0.14626067 | 0.12 | 0.7382 |
| period | 1 | 0.01551644 | 0.01551644 | 0.01 | 0.9131 |
| trt | 1 | 3.73511476 | 3.73511476 | 3.03 | 0.1155 |
| subject(sequence | ) 9 | 7.72241356 | 0.85804595 | 0.70 | 0.7002 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.14626067 | 0.14626067 | 0.12 | 0.7382 |
| period | 1 | 0.00266729 | 0.00266729 | 0.00 | 0.9639 |
| trt | 1 | 3.73511476 | 3.73511476 | 3.03 | 0.1155 |
| subject(sequence | ) 9 | 7.72241356 | 0.85804595 | 0.70 | 0.7002 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.14626067 | 0.14626067 | 0.12 | 0.7382 |
| period | 1 | 0.00266729 | 0.00266729 | 0.00 | 0.9639 |
| trt | 1 | 3.73511476 | 3.73511476 | 3.03 | 0.1155 |
| subject(sequence | ) 9 | 7.72241356 | 0.85804595 | 0.70 | 0.7002 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.14626067 | 0.14626067 | 0.12 | 0.7382 |
| period | 1 | 0.00266729 | 0.00266729 | 0.00 | 0.9639 |
| trt | 1 | 3.73511476 | 3.73511476 | 3.03 | 0.1155 |
| subject(sequence | ) 9 | 7.72241356 | 0.85804595 | 0.70 | 0.7002 |

Comparison: A vs B

Dependent Variable: V<sub>d</sub>/F (L) Weight Group: 88-111

### The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_VZFO

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.146261 | 0.146261 | 0.17 | 0.6894 |
| Error | 9 | 7.722414 | 0.858046 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| *period | 1 | 0.015516 | 0.015516 | 0.01 | 0.9131 |
| trt | 1 | 3.735115 | 3.735115 | 3.03 | 0.1155 |
| subject(sequence) | 9 | 7.722414 | 0.858046 | 0.70 | 0.7002 |
| Error: MS(Error) | 9 | 11.077366 | 1.230818 | | |
| * This test assumes one or m | ore othe | er fixed effects | are zero. | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.146261 | 0.146261 | 0.17 | 0.6894 |
| Error | 9 | 7.722414 | 0.858046 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.002667 | 0.002667 | 0.00 | 0.9639 |
| trt | 1 | 3.735115 | 3.735115 | 3.03 | 0.1155 |
| subject(sequence) | 9 | 7.722414 | 0.858046 | 0.70 | 0.7002 |
| Error: MS(Error) | 9 | 11.077366 | 1.230818 | | |

Comparison: A vs B

Dependent Variable: V<sub>d</sub>/F (L) Weight Group: 88-111

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_VZFO

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.146261 | 0.146261 | 0.17 | 0.6894 |
| Error | 9 | 7.722414 | 0.858046 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 0.002667 | 0.002667 | 0.00 | 0.9639 |
| trt | 1 | 3.735115 | 3.735115 | 3.03 | 0.1155 |
| subject(sequence) | 9 | 7.722414 | 0.858046 | 0.70 | 0.7002 |
| Error: MS(Error) | 9 | 11.077366 | 1.230818 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.146261 | 0.146261 | 0.17 | 0.6894 |
| Error | 9 | 7.722414 | 0.858046 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 0.002667 | 0.002667 | 0.00 | 0.9639 |
| trt | 1 | 3.735115 | 3.735115 | 3.03 | 0.1155 |
| subject(sequence) | 9 | 7.722414 | 0.858046 | 0.70 | 0.7002 |
| Error: MS(Error) | 9 | 11.077366 | 1.230818 | | |

Comparison: A vs B

Dependent Variable: V<sub>d</sub>/F (L) Weight Group: 88-111

#### Least Squares Means

| | | Н | 0:LSMean1=LSMean2 | |
|-----|----------------|----------|-----------------------|---------|
| trt | LN_VZFO LSMEAN | | | Pr > t |
| A | 5.56090410 | | | 0.1155 |
| В | 6.38841304 | | | |
| trt | LN_VZFO LSMEAN | | 90% Confidence Limits | |
| A | 5.560904 | 4.945172 | 6.176636 | |
| В | 6.388413 | 5.772681 | 7.004145 | |

Least Squares Means for Effect trt

Difference Between

i j Means 90% Confidence Limits for LSMean(i)-LSMean(j)

1 2 -0.827509 -1.698286 0.043268

| - | | Standard | | | |
|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confidence Limits |
| A - B | -0.82750894 | 0.47502636 | -1.74 | 0.1155-1 | .69828590 0.04326803 |

Comparison: A vs B

Dependent Variable: T<sub>max</sub> (h) Weight Group: 88-111

#### The GLM Procedure

| Class Leve | el Informa | tion |
|---|---|---|
| Class | Levels | Values |
| subject | 11 | 203 204 304 402 404 407 409 502 505 507 508 |
| sequence | 2 | AB BA |
| period | 2 | 1 2 |
| trt | 2 | A B |
| Number of | Number of Observations Read 22 | |
| Number of | Number of Observations Used 22 | |

Comparison: A vs B

Dependent Variable: T<sub>max</sub> (h) Weight Group: 88-111

#### The GLM Procedure

| R-Square | Coeff Var | Root | MSE | - | ГМАХ Mean |
|---|---|---|---|---|---|
| 0.669722 | 79.33433 | 0.875 | 5058 | 1.103000 | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.59202165 | 0.59202165 | 0.77 | 0.4021 |
| period | 1 | 6.15015564 | 6.15015564 | 8.03 | 0.0196 |
| trt | 1 | 1.22817855 | 1.22817855 | 1.60 | 0.2371 |
| subject(sequence) | 9 | 6.00394735 | 0.66710526 | 0.87 | 0.5797 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.59202165 | 0.59202165 | 0.77 | 0.4021 |
| period | 1 | 5.61184527 | 5.61184527 | 7.33 | 0.0241 |
| trt | 1 | 1.22817855 | 1.22817855 | 1.60 | 0.2371 |
| subject(sequence) | 9 | 6.00394735 | 0.66710526 | 0.87 | 0.5797 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.59202165 | 0.59202165 | 0.77 | 0.4021 |
| period | 1 | 5.61184527 | 5.61184527 | 7.33 | 0.0241 |
| trt | 1 | 1.22817855 | 1.22817855 | 1.60 | 0.2371 |
| subject(sequence) | 9 | 6.00394735 | 0.66710526 | 0.87 | 0.5797 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.59202165 | 0.59202165 | 0.77 | 0.4021 |
| period | 1 | 5.61184527 | 5.61184527 | 7.33 | 0.0241 |
| trt | 1 | 1.22817855 | 1.22817855 | 1.60 | 0.2371 |
| subject(sequence) | 9 | 6.00394735 | 0.66710526 | 0.87 | 0.5797 |

Comparison: A vs B

Dependent Variable: T<sub>max</sub> (h) Weight Group: 88-111

### The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: TMAX

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.592022 | 0.592022 | 0.89 | 0.3708 |
| Error 9 6.003947 0.667105 | | | | | |
| Error: MS(s | Error: MS(subject(sequence)) | | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| *period | 1 | 6.150156 | 6.150156 | 8.03 | 0.0196 |
| trt | 1 | 1.228179 | 1.228179 | 1.60 | 0.2371 |
| subject(sequence) | 9 | 6.003947 | 0.667105 | 0.87 | 0.5797 |
| Error: MS(Error) | 9 | 6.891533 | 0.765726 | | |
| * This test assumes one or m | ore oth | ner fixed effects | are zero. | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.592022 | 0.592022 | 0.89 | 0.3708 |
| Error | 9 | 6.003947 | 0.667105 | | _ |
| Error: MS(s | Error: MS(subject(sequence)) | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 5.611845 | 5.611845 | 7.33 | 0.0241 |
| trt | 1 | 1.228179 | 1.228179 | 1.60 | 0.2371 |
| subject(sequence) | 9 | 6.003947 | 0.667105 | 0.87 | 0.5797 |
| Error: MS(Error) | 9 | 6.891533 | 0.765726 | | |

Comparison: A vs B

Dependent Variable: T<sub>max</sub> (h) Weight Group: 88-111

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: TMAX

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.592022 | 0.592022 | 0.89 | 0.3708 |
| Error | 9 | 0.667105 | | <u></u> ; | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 5.611845 | 5.611845 | 7.33 | 0.0241 |
| trt | 1 | 1.228179 | 1.228179 | 1.60 | 0.2371 |
| subject(sequence) | 9 | 6.003947 | 0.667105 | 0.87 | 0.5797 |
| Error: MS(Error) | 9 | 6.891533 | 0.765726 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------|-----------|------------|-------------|---------|--------|
| sequence | 1 | 0.592022 | 0.592022 | 0.89 | 0.3708 |
| Error | 9 | 6.003947 | 0.667105 | | |
| Error: MS(s | subject(s | sequence)) | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| period | 1 | 5.611845 | 5.611845 | 7.33 | 0.0241 |
| trt | 1 | 1.228179 | 1.228179 | 1.60 | 0.2371 |
| subject(sequence) | 9 | 6.003947 | 0.667105 | 0.87 | 0.5797 |
| Error: MS(Error) | 9 | 6.891533 | 0.765726 | | |

Comparison: A vs B

Dependent Variable: T<sub>max</sub> (h) Weight Group: 88-111

#### Least Squares Means

| | | | H0:LSN | Mean1=LSMean2 | |
|---|---|---|---|---|---|
| trt | TMAX LSMEAN | | | | Pr > t |
| A | 1.32528333 | | | | 0.2371 |
| В | 0.85076667 | | | | |
| trt | TMAX LSMEAN | | 90% | 6 Confidence Limits | |
| A | 1.325283 | 0. | 839624 | 1.810943 | |
| В | 0.850767 | 0. | 365107 | 1.336426 | |
| Le | ast Squares Means for Effec | et trt | | | |
| | Difference Between | | | | |
| i | j Means | 90% Confide | ence Limits | for LSMean(i)-LSM | 1ean(j) |
| 1 | 2 0.474517 | -0.212309 | • | 1.161342 | |

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confi | dence Limits |
| A - B | 0.47451667 | 0.37467730 | 1.27 | 0.2371-0 | 0.21230913 | 1.16134246 |

Comparison: A vs B

Dependent Variable: K<sub>el</sub> (/h) Weight Group: 88-111

#### The GLM Procedure

| Class Level Information | | |
|---|---|---|
| Class | Levels | Values |
| subject | 11 | 203 204 304 402 404 407 409 502 505 507 508 |
| sequence | 2 | AB BA |
| period | 2 | 1 2 |
| trt | 2 | A B |
| • | | |
| Number of Observations Read 22 | | |
| Number of Observations Used 22 | | |

Comparison: A vs B

Dependent Variable: K<sub>el</sub> (/h) Weight Group: 88-111

#### The GLM Procedure

Dependent Variable: LAMZ

| R-Square | Coeff Var | Root MSE | | | LAMZ Mean |
|---|---|---|---|---|---|
| 0.660697 | 38.44030 | 0.002 | 853 0.007423 | | |
| Source | DF | Type I SS | Mean Square | e F Value | e Pr > F |
| sequence | 1 | 0.00000972 | 0.00000972 | 1.19 | 0.3028 |
| period | 1 | 0.00000474 | 0.00000474 | 0.58 | 0.4649 |
| trt | 1 | 0.00000587 | 0.00000587 | 0.72 | 0.4177 |
| subject(sequence) | 9 | 0.00012234 | 0.00001359 | 1.67 | 0.2285 |
| Source | DF | Type II SS | Mean Square | F Value | e $Pr > F$ |
| sequence | 1 | 0.00000972 | 0.00000972 | 1.19 | 0.3028 |
| period | 1 | 0.00000380 | 0.00000380 | 0.47 | 0.5119 |
| trt | 1 | 0.00000587 | 0.00000587 | 0.72 | 0.4177 |
| subject(sequence) | 9 | 0.00012234 | 0.00001359 | 1.67 | 0.2285 |
| Source | DF | Type III SS | Mean Square | F Value | e $Pr > F$ |
| sequence | 1 | 0.00000972 | 0.00000972 | 1.19 | 0.3028 |
| period | 1 | 0.00000380 | 0.00000380 | 0.47 | 0.5119 |
| trt | 1 | 0.00000587 | 0.00000587 | 0.72 | 0.4177 |
| subject(sequence) | 9 | 0.00012234 | 0.00001359 | 1.67 | 0.2285 |
| Source | DF | Type IV SS | Mean Square | F Value | e $Pr > F$ |
| sequence | 1 | 0.00000972 | 0.00000972 | 1.19 | 0.3028 |
| period | 1 | 0.00000380 | 0.00000380 | 0.47 | 0.5119 |
| trt | 1 | 0.00000587 | 0.00000587 | 0.72 | 0.4177 |
| subject(sequence) | 9 | 0.00012234 | 0.00001359 | 1.67 | 0.2285 |

Comparison: A vs B

Dependent Variable: K<sub>el</sub> (/h) Weight Group: 88-111

### The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LAMZ

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.000009724 | 0.000009724 | 0.72 | 0.4196 |
| Error | 9 | 0.000122 | 0.000013594 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| *period | 1 | 0.000004743 | 0.000004743 | 0.58 | 0.4649 |
| trt | 1 | 0.000005875 | 0.000005875 | 0.72 | 0.4177 |
| subject(sequence) | 9 | 0.000122 | 0.000013594 | 1.67 | 0.2285 |
| Error: MS(Error) | 9 | 0.000073276 | 0.000008142 | | |
| * This test assumes one or more other fixed effects are zero. | | | | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LAMZ

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------|----------|-------------|-------------|---------|--------|
| sequence | 1 | 0.000009724 | 0.000009724 | 0.72 | 0.4196 |
| Error | 9 | 0.000122 | 0.000013594 | | |
| Error: MS(s | subject( | sequence)) | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 0.000003796 | 0.000003796 | 0.47 | 0.5119 |
| trt | 1 | 0.000005875 | 0.000005875 | 0.72 | 0.4177 |
| subject(sequence) | 9 | 0.000122 | 0.000013594 | 1.67 | 0.2285 |
| Error: MS(Error) | 9 | 0.000073276 | 0.000008142 | | |
Comparison: A vs B

Dependent Variable: K<sub>el</sub> (/h) Weight Group: 88-111

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LAMZ

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.000009724 | 0.000009724 | 0.72 | 0.4196 |
| Error | 9 | 0.000122 | 0.000013594 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| period | 1 | 0.000003796 | 0.000003796 | 0.47 | 0.5119 |
| trt | 1 | 0.000005875 | 0.000005875 | 0.72 | 0.4177 |
| subject(sequence) | 9 | 0.000122 | 0.000013594 | 1.67 | 0.2285 |
| Error: MS(Error) | 9 | 0.000073276 | 0.000008142 | <del></del> | <del></del> |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.000009724 | 0.000009724 | 0.72 | 0.4196 |
| Error | 9 | 0.000122 | 0.000013594 | | |
| Error: MS(subject(sequence)) | | | | | |

| Carras | DE | T-ma IV/CC | Maan Canana | E Malara | D E |
|-------------------|----|-------------|-------------|----------|--------|
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| period | 1 | 0.000003796 | 0.000003796 | 0.47 | 0.5119 |
| trt | 1 | 0.000005875 | 0.000005875 | 0.72 | 0.4177 |
| subject(sequence) | 9 | 0.000122 | 0.000013594 | 1.67 | 0.2285 |
| Error: MS(Error) | 9 | 0.000073276 | 0.000008142 | | |

Comparison: A vs B

Dependent Variable: K<sub>el</sub> (/h) Weight Group: 88-111

#### Least Squares Means

| | | H0:LSN | Mean1=LSMean2 |
|---|---|---|---|
| trt | LAMZ LSMEAN | | Pr > t |
| A | 0.00800245 | | 0.4177 |
| В | 0.00696467 | | |
| trt | LAMZ LSMEAN | 90% | Confidence Limits |
| A | 0.008002 | 0.006419 | 0.009586 |
| В | 0.006965 | 0.005381 | 0.008548 |
| Le | ast Squares Means for Effec | et trt | |
| | Difference Between | | |
| i | j Means | 90% Confidence Limits | for LSMean(i)-LSMean(j) |
| 1 | 2 0.001038 | -0.001202 | 0.003277 |

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confid | dence Limits |
| A - B | 0.00103779 | 0.00122174 | 0.85 | 0.4177-0 | 0.00120180 | 0.00327738 |

Comparison: A vs B

Dependent Variable: T<sub>1/2 el</sub> (h) Weight Group: 88-111

#### The GLM Procedure

| Class Leve | el Informa | tion |
|---|---|---|
| Class | Levels | Values |
| subject | 11 | 203 204 304 402 404 407 409 502 505 507 508 |
| sequence | 2 | AB BA |
| period | 2 | 1 2 |
| trt | 2 | A B |
| Number of Observations Read 22 | | |
| Number of Observations Used 22 | | |

Comparison: A vs B

Dependent Variable: T<sub>1/2 el</sub> (h) Weight Group: 88-111

#### The GLM Procedure

| R-Square | Coeff Var | Root MSE | , | LAMZ | ZHL Mean |
|---|---|---|---|---|---|
| 0.574882 | 99.33196 | 138.5731 | 139.505 | 51 | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 5649.2726 | 5649.2726 | 0.29 | 0.6007 |
| period | 1 | 25232.1129 | 25232.1129 | 1.31 | 0.2812 |
| trt | 1 | 3972.7356 | 3972.7356 | 0.21 | 0.6600 |
| subject(sequence) | ) 9 | 198852.1366 | 22094.6818 | 1.15 | 0.4189 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 5649.2726 | 5649.2726 | 0.29 | 0.6007 |
| period | 1 | 23243.5863 | 23243.5863 | 1.21 | 0.2998 |
| trt | 1 | 3972.7356 | 3972.7356 | 0.21 | 0.6600 |
| subject(sequence) | _ | 198852.1366 | 22094.6818 | 1.15 | 0.4189 |
| <u> </u> | , | | | | |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 5649.2726 | 5649.2726 | 0.29 | 0.6007 |
| period | 1 | 23243.5863 | 23243.5863 | 1.21 | 0.2998 |
| trt | 1 | 3972.7356 | 3972.7356 | 0.21 | 0.6600 |
| subject(sequence) | ) 9 | 198852.1366 | 22094.6818 | 1.15 | 0.4189 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 5649.2726 | 5649.2726 | 0.29 | 0.6007 |
| period | 1 | 23243.5863 | 23243.5863 | 1.21 | 0.2998 |
| trt | 1 | 3972.7356 | 3972.7356 | 0.21 | 0.6600 |
| subject(sequence) | ) 9 | 198852.1366 | 22094.6818 | 1.15 | 0.4189 |

Comparison: A vs B

Dependent Variable: T<sub>1/2 el</sub> (h) Weight Group: 88-111

## The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LAMZHL

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 5649.272565 | 5649.272565 | 0.26 | 0.6253 |
| Error | 9 | 198852 | 22095 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| *period | 1 | 25232 | 25232 | 1.31 | 0.2812 |
| trt | 1 | 3972.735582 | 3972.735582 | 0.21 | 0.6600 |
| subject(sequence) | 9 | 198852 | 22095 | 1.15 | 0.4189 |
| Error: MS(Error) | 9 | 172823 | 19203 | | |
| * This test assumes one or more other fixed effects are zero. | | | | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 5649.272565 | 5649.272565 | 0.26 | 0.6253 |
| Error | 9 | 198852 | 22095 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 23244 | 23244 | 1.21 | 0.2998 |
| trt | 1 | 3972.735582 | 3972.735582 | 0.21 | 0.6600 |
| subject(sequence) | 9 | 198852 | 22095 | 1.15 | 0.4189 |
| Error: MS(Error) | 9 | 172823 | 19203 | | |

Comparison: A vs B

Dependent Variable: T<sub>1/2 el</sub> (h) Weight Group: 88-111

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LAMZHL

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 5649.272565 | 5649.272565 | 0.26 | 0.6253 |
| Error | 9 | 198852 | 22095 | | _ |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 23244 | 23244 | 1.21 | 0.2998 |
| trt | 1 | 3972.735582 | 3972.735582 | 0.21 | 0.6600 |
| subject(sequence) | 9 | 198852 | 22095 | 1.15 | 0.4189 |
| Error: MS(Error) | 9 | 172823 | 19203 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 5649.272565 | 5649.272565 | 0.26 | 0.6253 |
| Error | 9 | 198852 | 22095 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| period | 1 | 23244 | 23244 | 1.21 | 0.2998 |
| trt | 1 | 3972.735582 | 3972.735582 | 0.21 | 0.6600 |
| subject(sequence) | 9 | 198852 | 22095 | 1.15 | 0.4189 |
| Error: MS(Error) | 9 | 172823 | 19203 | | |

Comparison: A vs B

Dependent Variable: T<sub>1/2 el</sub> (h) Weight Group: 88-111

#### Least Squares Means

| | | ] | H0:LSMean1=LSMean2 | |
|---|---|---|---|---|
| trt | LAMZHL LSMEAN | | | Pr > t |
| A | 124.548382 | | | 0.6600 |
| В | 151.536062 | | | |
| _ | | | | |
| trt | LAMZHL LSMEAN | | 90% Confidence Limits | |
| A | 124.548382 | 47.639963 | 201.456802 | |
| В | 151.536062 | 74.627643 | 228.444482 | |
| Le | ast Squares Means for Effe | et trt | | |
| | Difference Between | | | |
| i | j Means | 90% Confide | ence Limits for LSMean(i)-LS | Mean(j) |
| 1 | 2 -26.987680 | -135.752610 | 81.777250 | |

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confid | ence Limits |
| A - B | -26.9876797 | 59.3334584 | -0.45 | 0.6600-1 | 35.7526097 | 81.7772502 |

Dependent Variable: AUC<sub>0-t</sub> (h\*ng/mL) Weight Group: 88-111

#### The GLM Procedure

| Class | Levels | Values | |
|----------------------------------|----------------|-----------------|---|
| subject | 4 | 203 204 402 404 | |
| sequence | 2 | ABC BAC | |
| trt | 2 | ВС | |
| Number of Obse | ervations Read | | 8 |
| Number of Obse<br>Number of Obse | | | |
| Number of Obse | ervations Used | | |

Comparison: C vs B

Dependent Variable: AUC<sub>0-t</sub> (h\*ng/mL) Weight Group: 88-111

#### The GLM Procedure

Dependent Variable: LN\_AUCLST

| R-Square | Coeff Var | Root MSE | | LN_AUC | LST Mean |
|---|---|---|---|---|---|
| 0.443329 | 5.254932 | 0.467887 | 8.903767 | | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.36557536 | 0.36557536 | 1.67 | 0.2868 |
| trt | 1 | 0.10103184 | 0.10103184 | 0.46 | 0.5456 |
| subject(sequence | ce) 2 | 0.05642733 | 0.02821366 | 0.13 | 0.8837 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.36557536 | 0.36557536 | 1.67 | 0.2868 |
| trt | 1 | 0.10103184 | 0.10103184 | 0.46 | 0.5456 |
| subject(sequence | ce) 2 | 0.05642733 | 0.02821366 | 0.13 | 0.8837 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.36557536 | 0.36557536 | 1.67 | 0.2868 |
| trt | 1 | 0.10103184 | 0.10103184 | 0.46 | 0.5456 |
| subject(sequence | ce) 2 | 0.05642733 | 0.02821366 | 0.13 | 0.8837 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.36557536 | 0.36557536 | 1.67 | 0.2868 |
| trt | 1 | 0.10103184 | 0.10103184 | 0.46 | 0.5456 |
| subject(sequence | ce) 2 | 0.05642733 | 0.02821366 | 0.13 | 0.8837 |

Comparison: C vs B

Dependent Variable: AUC<sub>0-t</sub> (h\*ng/mL) Weight Group: 88-111

## The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_AUCLST

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.365575 | 0.365575 | 12.96 | 0.0693 |
| Error 2 0.056427 0.028214 | | | | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-------------------|----|-----------|-------------|---------|--------|
| trt | 1 | 0.101032 | 0.101032 | 0.46 | 0.5456 |
| subject(sequence) | 2 | 0.056427 | 0.028214 | 0.13 | 0.8837 |
| Error: MS(Error) | 3 | 0.656755 | 0.218918 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_AUCLST

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.365575 | 0.365575 | 12.96 | 0.0693 |
| Error | 2 | 0.056427 | 0.028214 | | _ |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| trt | 1 | 0.101032 | 0.101032 | 0.46 | 0.5456 |
| subject(sequence) | 2 | 0.056427 | 0.028214 | 0.13 | 0.8837 |
| Error: MS(Error) | 3 | 0.656755 | 0.218918 | | |

Comparison: C vs B

Dependent Variable: AUC<sub>0-t</sub> (h\*ng/mL) Weight Group: 88-111

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_AUCLST

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.365575 | 0.365575 | 12.96 | 0.0693 |
| Error | 2 | 0.056427 | 0.028214 | | <u></u> ; |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| trt | 1 | 0.101032 | 0.101032 | 0.46 | 0.5456 |
| subject(sequence) | 2 | 0.056427 | 0.028214 | 0.13 | 0.8837 |
| Error: MS(Error) | 3 | 0.656755 | 0.218918 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN AUCLST

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.365575 | 0.365575 | 12.96 | 0.0693 |
| Error | 2 | 0.056427 | 0.028214 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| trt | 1 | 0.101032 | 0.101032 | 0.46 | 0.5456 |
| subject(sequence) | 2 | 0.056427 | 0.028214 | 0.13 | 0.8837 |
| Error: MS(Error) | 3 | 0.656755 | 0.218918 | | |

Comparison: C vs B

Dependent Variable: AUC<sub>0-t</sub> (h\*ng/mL) Weight Group: 88-111

#### Least Squares Means

| - | | H0:LSMean1=LSMean2 | |
|-----|------------------|-----------------------|---------|
| trt | LN_AUCLST LSMEAN | | Pr > t |
| В | 8.66796917 | ( | ).5456 |
| C | 8.89272663 | | |
| trt | LN_AUCLST LSMEAN | 90% Confidence Limits | |
| D | 0.667060 | 0.072202 0.262625 | |

| В | 8.66/969 | 8.0/3303 | 9.262635 |
|---|----------|----------|----------|
| C | 8.892727 | 8.298060 | 9.487393 |

| Le | Least Squares Means for Effect trt | | | |
|---|---|---|---|---|
| | | Difference Between | | |
| i | j | Means | 90% Confid | ence Limits for LSMean(i)-LSMean(j) |
| 1 | 2 | -0.224757 | -1.003358 | 0.553843 |

Dependent Variable: LN\_AUCLST

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confid | dence Limits |
| C - B | 0.22475747 | 0.33084602 | 0.68 | 0.5456-0 | 0.55384345 | 1.00335839 |

Comparison: C vs B

Dependent Variable: AUC<sub>0-inf</sub> (h\*ng/mL) Weight Group: 88-111

#### The GLM Procedure

| Class Level Info | rmation | |
|-----------------------------|---------|-----------------|
| Class | Levels | Values |
| subject | 4 | 203 204 402 404 |
| sequence | 2 | ABC BAC |
| trt | 2 | ВС |
| Number of Observations Read | | |
| Number of Observations Used | | |

Comparison: C vs B

Dependent Variable: AUC<sub>0-inf</sub> (h\*ng/mL) Weight Group: 88-111

#### The GLM Procedure

Dependent Variable: LN\_AUCIFO

| R-Square | Coeff Var | Root MSE | | LN AUC | IFO Mean |
|----------------|-----------|-------------|-------------|---------|----------|
| 0.498012 | 5.187536 | 0.468583 | 9.032871 | _ | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.50748249 | 0.50748249 | 2.31 | 0.2258 |
| trt | 1 | 0.06707153 | 0.06707153 | 0.31 | 0.6190 |
| subject(sequen | ce) 2 | 0.07893896 | 0.03946948 | 0.18 | 0.8439 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.50748249 | 0.50748249 | 2.31 | 0.2258 |
| trt | 1 | 0.06707153 | 0.06707153 | 0.31 | 0.6190 |
| subject(sequen | ce) 2 | 0.07893896 | 0.03946948 | 0.18 | 0.8439 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.50748249 | 0.50748249 | 2.31 | 0.2258 |
| trt | 1 | 0.06707153 | 0.06707153 | 0.31 | 0.6190 |
| subject(sequen | ce) 2 | 0.07893896 | 0.03946948 | 0.18 | 0.8439 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.50748249 | 0.50748249 | 2.31 | 0.2258 |
| trt | 1 | 0.06707153 | 0.06707153 | 0.31 | 0.6190 |
| subject(sequen | ce) 2 | 0.07893896 | 0.03946948 | 0.18 | 0.8439 |
| | • | - | | | |

Comparison: C vs B

Dependent Variable: AUC<sub>0-inf</sub> (h\*ng/mL) Weight Group: 88-111

## The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_AUCIFO

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.507482 | 0.507482 | 12.86 | 0.0697 |
| Error | 2 | 0.078939 | 0.039469 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-------------------|----|-----------|-------------|---------|--------|
| trt | 1 | 0.067072 | 0.067072 | 0.31 | 0.6190 |
| subject(sequence) | 2 | 0.078939 | 0.039469 | 0.18 | 0.8439 |
| Error: MS(Error) | 3 | 0.658711 | 0.219570 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_AUCIFO

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.507482 | 0.507482 | 12.86 | 0.0697 |
| Error | 2 | 0.078939 | 0.039469 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|-------------|
| trt | 1 | 0.067072 | 0.067072 | 0.31 | 0.6190 |
| subject(sequence) | 2 | 0.078939 | 0.039469 | 0.18 | 0.8439 |
| Error: MS(Error) | 3 | 0.658711 | 0.219570 | | <del></del> |

Comparison: C vs B

Dependent Variable: AUC<sub>0-inf</sub> (h\*ng/mL) Weight Group: 88-111

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_AUCIFO

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.507482 | 0.507482 | 12.86 | 0.0697 |
| Error | 2 | 0.078939 | 0.039469 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| trt | 1 | 0.067072 | 0.067072 | 0.31 | 0.6190 |
| subject(sequence) | 2 | 0.078939 | 0.039469 | 0.18 | 0.8439 |
| Error: MS(Error) | 3 | 0.658711 | 0.219570 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN AUCIFO

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.507482 | 0.507482 | 12.86 | 0.0697 |
| Error | 2 | 0.078939 | 0.039469 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| trt | 1 | 0.067072 | 0.067072 | 0.31 | 0.6190 |
| subject(sequence) | 2 | 0.078939 | 0.039469 | 0.18 | 0.8439 |
| Error: MS(Error) | 3 | 0.658711 | 0.219570 | | |

Comparison: C vs B

Dependent Variable: AUC<sub>0-inf</sub> (h\*ng/mL) Weight Group: 88-111

#### Least Squares Means

| | H0:LSMean1=LSMean2 | | |
|---------|--------------------|------------------|----------|
| Pr > t | | LN_AUCIFO LSMEAN | trt |
| 0.6190 | | 8.79589362 | В |
| | | 8.97902135 | C |
| | | ********* | <u>C</u> |

| trt | LN_AUCIFO LSMEAN | | 90% Confidence Limits |
|-----|------------------|----------|-----------------------|
| В | 8.795894 | 8.200342 | 9.391445 |
| C | 8.979021 | 8.383470 | 9.574573 |

| Le | Least Squares Means for Effect trt | | | |
|---|---|---|---|---|
| | | Difference Between | | |
| i | j | Means | 90% Confider | nce Limits for LSMean(i)-LSMean(j) |
| 1 | 2 | -0.183128 | -0.962888 | 0.596632 |

Dependent Variable: LN\_AUCIFO

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confi | dence Limits |
| C - B | 0.18312773 | 0.33133856 | 0.55 | 0.6190-0 | 0.59663231 | 0.96288777 |

Dependent Variable: C<sub>max</sub> (ng/mL) Weight Group: 88-111

#### The GLM Procedure

| Class Level Info | Levels | Values | |
|------------------|---------------|-----------------|---|
| subject | 4 | 203 204 402 404 | |
| sequence | 2 | ABC BAC | |
| trt | 2 | ВС | |
| Number of Obse | rvations Read | | 8 |
| Number of Obse | 8 | | |

Comparison: C vs B

Dependent Variable: C<sub>max</sub> (ng/mL) Weight Group: 88-111

#### The GLM Procedure

| R-Square C | Coeff Var | Root MSE | | LN_CN | MAX Mean |
|---|---|---|---|---|---|
| 0.422220 8 | 3.993728 | 0.448513 | 4.986958 | _ | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.09754320 | 0.09754320 | 0.48 | 0.5363 |
| trt | 1 | 0.09487043 | 0.09487043 | 0.47 | 0.5416 |
| subject(sequence) | 2 | 0.24859694 | 0.12429847 | 0.62 | 0.5960 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.09754320 | 0.09754320 | 0.48 | 0.5363 |
| trt | 1 | 0.09487043 | 0.09487043 | 0.47 | 0.5416 |
| subject(sequence) | 2 | 0.24859694 | 0.12429847 | 0.62 | 0.5960 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.09754320 | 0.09754320 | 0.48 | 0.5363 |
| trt | 1 | 0.09487043 | 0.09487043 | 0.47 | 0.5416 |
| subject(sequence) | 2 | 0.24859694 | 0.12429847 | 0.62 | 0.5960 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.09754320 | 0.09754320 | 0.48 | 0.5363 |
| trt | 1 | 0.09487043 | 0.09487043 | 0.47 | 0.5416 |
| subject(sequence) | 2 | 0.24859694 | 0.12429847 | 0.62 | 0.5960 |

Comparison: C vs B

Dependent Variable: C<sub>max</sub> (ng/mL) Weight Group: 88-111

## The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_CMAX

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.097543 | 0.097543 | 0.78 | 0.4691 |
| Error 2 0.248597 | | | 0.124298 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-------------------|----|-----------|-------------|---------|--------|
| trt | 1 | 0.094870 | 0.094870 | 0.47 | 0.5416 |
| subject(sequence) | 2 | 0.248597 | 0.124298 | 0.62 | 0.5960 |
| Error: MS(Error) | 3 | 0.603493 | 0.201164 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.097543 | 0.097543 | 0.78 | 0.4691 |
| Error | 2 | 0.248597 | 0.124298 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| trt | 1 | 0.094870 | 0.094870 | 0.47 | 0.5416 |
| subject(sequence) | 2 | 0.248597 | 0.124298 | 0.62 | 0.5960 |
| Error: MS(Error) | 3 | 0.603493 | 0.201164 | | |

Comparison: C vs B

Dependent Variable: C<sub>max</sub> (ng/mL) Weight Group: 88-111

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_CMAX

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.097543 | 0.097543 | 0.78 | 0.4691 |
| Error | 2 | 0.248597 | 0.124298 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| trt | 1 | 0.094870 | 0.094870 | 0.47 | 0.5416 |
| subject(sequence) | 2 | 0.248597 | 0.124298 | 0.62 | 0.5960 |
| Error: MS(Error) | 3 | 0.603493 | 0.201164 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.097543 | 0.097543 | 0.78 | 0.4691 |
| Error | 2 | 0.248597 | 0.124298 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| trt | 1 | 0.094870 | 0.094870 | 0.47 | 0.5416 |
| subject(sequence) | 2 | 0.248597 | 0.124298 | 0.62 | 0.5960 |
| Error: MS(Error) | 3 | 0.603493 | 0.201164 | | |

Comparison: C vs B

Dependent Variable: C<sub>max</sub> (ng/mL) Weight Group: 88-111

5.032104

-0.217796

#### Least Squares Means

| | | H0:LSN | Mean1=LSMean2 | |
|-----|----------------|----------|-------------------|----------|
| trt | LN_CMAX LSMEAN | | | Pr > t |
| В | 4.81430790 | | ( | 0.5416 |
| C | 5.03210417 | | | |
| trt | LN_CMAX LSMEAN | 90% | Confidence Limits | <u> </u> |
| В | 4.814308 | 4.244265 | 5.384351 | |

| Leas | t Squares Means for Effect | trt |
|---|---|---|
| | Difference Between | |
| i j | Means | 90% Confidence Limits for LSMean(i)-LSMean(j) |

-0.964158

4.462061

5.602147

0.528566

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confi | dence Limits |
| C - B | 0.21779627 | 0.31714689 | 0.69 | 0.5416-0 | ).52856563 | 0.96415818 |

Dependent Variable: Cl/F/kg ((L/h)/kg) Weight Group: 88-111

#### The GLM Procedure

| Class Level Info | Levels | Values | |
|------------------|---------------|-----------------|---|
| subject | 4 | 203 204 402 404 | |
| sequence | 2 | ABC BAC | |
| trt | 2 | ВС | |
| Number of Obse | rvations Read | | 8 |
| Number of Obse | 8 | | |

Comparison: C vs B

Dependent Variable: Cl/F/kg ((L/h)/kg) Weight Group: 88-111

#### The GLM Procedure

Dependent Variable: LN\_CLFOW

| R-Square | Coeff Var | Root MSE | | LN_CLF | OW Mean |
|------------------|-----------|-------------|-------------|---------|---------|
| 0.651142 | -12.11538 | 0.468583 | -3.867674 | | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.77546793 | 0.77546793 | 3.53 | 0.1568 |
| trt | 1 | 0.20054600 | 0.20054600 | 0.91 | 0.4097 |
| subject(sequence | 2 | 0.25347050 | 0.12673525 | 0.58 | 0.6136 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.77546793 | 0.77546793 | 3.53 | 0.1568 |
| trt | 1 | 0.20054600 | 0.20054600 | 0.91 | 0.4097 |
| subject(sequence | 2 | 0.25347050 | 0.12673525 | 0.58 | 0.6136 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.77546793 | 0.77546793 | 3.53 | 0.1568 |
| trt | 1 | 0.20054600 | 0.20054600 | 0.91 | 0.4097 |
| subject(sequence | 2 | 0.25347050 | 0.12673525 | 0.58 | 0.6136 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.77546793 | 0.77546793 | 3.53 | 0.1568 |
| trt | 1 | 0.20054600 | 0.20054600 | 0.91 | 0.4097 |
| subject(sequence | 2 | 0.25347050 | 0.12673525 | 0.58 | 0.6136 |

Comparison: C vs B

Dependent Variable: Cl/F/kg ((L/h)/kg) Weight Group: 88-111

## The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_CLFOW

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.775468 | 0.775468 | 6.12 | 0.1319 |
| Error | 2 | 0.253471 | 0.126735 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-------------------|----|-----------|-------------|---------|--------|
| trt | 1 | 0.200546 | 0.200546 | 0.91 | 0.4097 |
| subject(sequence) | 2 | 0.253471 | 0.126735 | 0.58 | 0.6136 |
| Error: MS(Error) | 3 | 0.658711 | 0.219570 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_CLFOW

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.775468 | 0.775468 | 6.12 | 0.1319 |
| Error | 2 | 0.253471 | 0.126735 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| trt | 1 | 0.200546 | 0.200546 | 0.91 | 0.4097 |
| subject(sequence) | 2 | 0.253471 | 0.126735 | 0.58 | 0.6136 |
| Error: MS(Error) | 3 | 0.658711 | 0.219570 | | |

Comparison: C vs B

Dependent Variable: Cl/F/kg ((L/h)/kg) Weight Group: 88-111

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_CLFOW

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.775468 | 0.775468 | 6.12 | 0.1319 |
| Error 2 0.253471 0.126735 | | | | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| trt | 1 | 0.200546 | 0.200546 | 0.91 | 0.4097 |
| subject(sequence) | 2 | 0.253471 | 0.126735 | 0.58 | 0.6136 |
| Error: MS(Error) | 3 | 0.658711 | 0.219570 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN CLFOW

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.775468 | 0.775468 | 6.12 | 0.1319 |
| Error | 2 | 0.253471 | 0.126735 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| trt | 1 | 0.200546 | 0.200546 | 0.91 | 0.4097 |
| subject(sequence) | 2 | 0.253471 | 0.126735 | 0.58 | 0.6136 |
| Error: MS(Error) | 3 | 0.658711 | 0.219570 | | |

Comparison: C vs B

Dependent Variable: Cl/F/kg ((L/h)/kg) Weight Group: 88-111

Means 0.316659

#### Least Squares Means

| | | Н | I0:LSMean1=LSMean2 | |
|---|---|---|---|---|
| trt | LN_CLFOW LSMEAN | | | Pr > t |
| В | -3.52959127 | | | 0.4097 |
| C | -3.84625040 | | | |
| trt | LN_CLFOW LSMEAN | | 90% Confidence Limits | |
| В | -3.529591 | -4.125143 | -2.934040 | |
| C | -3.846250 | -4.441802 | -3.250699 | |
| Lea | ast Squares Means for Effect trt | | | |
| | Difference Between | | | |

#### Dependent Variable: LN\_CLFOW

-0.463101

90% Confidence Limits for LSMean(i)-LSMean(j)

1.096419

| | | Standard | | |
|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t 90% Confidence Limits |
| C - B | -0.31665913 | 0.33133856 | -0.96 | 0.4097-1.09641917 |

Dependent Variable: Cl/F (L/h) Weight Group: 88-111

#### The GLM Procedure

| Class Level Infor | mation | | _ |
|-------------------|--------|-----------------|---|
| Class | Levels | Values | |
| subject | 4 | 203 204 402 404 | _ |
| sequence | 2 | ABC BAC | |
| trt | 2 | ВС | |
| Number of Obser | 8 | | |
| Number of Obser | 8 | | |

Dependent Variable: Cl/F (L/h) Weight Group: 88-111

#### The GLM Procedure

Dependent Variable: LN\_CLFO

| R-Square | Coeff Var | Root MSE | | LN_0 | CLFO Mean |
|---|---|---|---|---|---|
| 0.544358 | 58.29234 | 0.468583 | 0.803851 | _ | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.50748249 | 0.50748249 | 2.31 | 0.2258 |
| trt | 1 | 0.20054600 | 0.20054600 | 0.91 | 0.4097 |
| subject(sequence | 2 | 0.07893896 | 0.03946948 | 0.18 | 0.8439 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.50748249 | 0.50748249 | 2.31 | 0.2258 |
| trt | 1 | 0.20054600 | 0.20054600 | 0.91 | 0.4097 |
| subject(sequence | 2 | 0.07893896 | 0.03946948 | 0.18 | 0.8439 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.50748249 | 0.50748249 | 2.31 | 0.2258 |
| trt | 1 | 0.20054600 | 0.20054600 | 0.91 | 0.4097 |
| subject(sequence | 2 | 0.07893896 | 0.03946948 | 0.18 | 0.8439 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.50748249 | 0.50748249 | 2.31 | 0.2258 |
| trt | 1 | 0.20054600 | 0.20054600 | 0.91 | 0.4097 |
| subject(sequence | 2 | 0.07893896 | 0.03946948 | 0.18 | 0.8439 |

Comparison: C vs B

Dependent Variable: Cl/F (L/h) Weight Group: 88-111

## The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_CLFO

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.507482 | 0.507482 | 12.86 | 0.0697 |
| Error | 2 | 0.078939 | 0.039469 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-------------------|----|-----------|-------------|---------|--------|
| trt | 1 | 0.200546 | 0.200546 | 0.91 | 0.4097 |
| subject(sequence) | 2 | 0.078939 | 0.039469 | 0.18 | 0.8439 |
| Error: MS(Error) | 3 | 0.658711 | 0.219570 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_CLFO

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.507482 | 0.507482 | 12.86 | 0.0697 |
| Error | 2 | 0.078939 | 0.039469 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| trt | 1 | 0.200546 | 0.200546 | 0.91 | 0.4097 |
| subject(sequence) | 2 | 0.078939 | 0.039469 | 0.18 | 0.8439 |
| Error: MS(Error) | 3 | 0.658711 | 0.219570 | | |

Comparison: C vs B

Dependent Variable: Cl/F (L/h) Weight Group: 88-111

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_CLFO

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.507482 | 0.507482 | 12.86 | 0.0697 |
| Error | 2 | 0.078939 | 0.039469 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| trt | 1 | 0.200546 | 0.200546 | 0.91 | 0.4097 |
| subject(sequence) | 2 | 0.078939 | 0.039469 | 0.18 | 0.8439 |
| Error: MS(Error) | 3 | 0.658711 | 0.219570 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN CLFO

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.507482 | 0.507482 | 12.86 | 0.0697 |
| Error | 2 | 0.078939 | 0.039469 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| trt | 1 | 0.200546 | 0.200546 | 0.91 | 0.4097 |
| subject(sequence) | 2 | 0.078939 | 0.039469 | 0.18 | 0.8439 |
| Error: MS(Error) | 3 | 0.658711 | 0.219570 | | |

Comparison: C vs B

Dependent Variable: Cl/F (L/h) Weight Group: 88-111

#### Least Squares Means

| | | H0:LSMean1=LSMean2 | |
|-----|----------------|--------------------|---------|
| trt | LN_CLFO LSMEAN | | Pr > t |
| В | 1.10759394 | | 0.4097 |
| C | 0.79093481 | | |

| trt | LN_CLFO LSMEAN | | 90% Confidence Limits |
|-----|----------------|----------|-----------------------|
| В | 1.107594 | 0.512042 | 1.703146 |
| C | 0.790935 | 0.195383 | 1.386486 |

| Le | Least Squares Means for Effect trt | | | |
|---|---|---|---|---|
| | | Difference Between | | |
| i | j | Means | 90% Confider | nce Limits for LSMean(i)-LSMean(j) |
| 1 | 2 | 0.316659 | -0.463101 | 1.096419 |

#### Dependent Variable: LN\_CLFO

| | | Standard | | |
|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t 90% Confidence Limits |
| C - B | -0.31665913 | 0.33133856 | -0.96 | 0.4097-1.09641917 |

Dependent Variable: V<sub>d</sub>/F/kg (L/kg) Weight Group: 88-111

#### The GLM Procedure

| Class Level Info | Levels | Values | |
|------------------|---------------|-----------------|---|
| subject | 4 | 203 204 402 404 | |
| sequence | 2 | ABC BAC | |
| trt | 2 | ВС | |
| Number of Obse | rvations Read | | 8 |
| Number of Obse | 8 | | |

Comparison: C vs B

Dependent Variable: V<sub>d</sub>/F/kg (L/kg) Weight Group: 88-111

#### The GLM Procedure

Dependent Variable: LN\_VZFOW

| R-Square | Coeff Var | Root MSE | | LN_VZF | OW Mean |
|------------------|-----------|-------------|-------------|---------|---------|
| 0.449575 | 63.64188 | 0.548837 | 0.862384 | _ | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.16265602 | 0.16265602 | 0.54 | 0.5157 |
| trt | 1 | 0.45894271 | 0.45894271 | 1.52 | 0.3049 |
| subject(sequence | ce) 2 | 0.11649724 | 0.05824862 | 0.19 | 0.8337 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.16265602 | 0.16265602 | 0.54 | 0.5157 |
| trt | 1 | 0.45894271 | 0.45894271 | 1.52 | 0.3049 |
| subject(sequence | ce) 2 | 0.11649724 | 0.05824862 | 0.19 | 0.8337 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.16265602 | 0.16265602 | 0.54 | 0.5157 |
| trt | 1 | 0.45894271 | 0.45894271 | 1.52 | 0.3049 |
| subject(sequence | ce) 2 | 0.11649724 | 0.05824862 | 0.19 | 0.8337 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.16265602 | 0.16265602 | 0.54 | 0.5157 |
| trt | 1 | 0.45894271 | 0.45894271 | 1.52 | 0.3049 |
| subject(sequence | ce) 2 | 0.11649724 | 0.05824862 | 0.19 | 0.8337 |

Comparison: C vs B

Dependent Variable: V<sub>d</sub>/F/kg (L/kg) Weight Group: 88-111

## The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_VZFOW

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.162656 | 0.162656 | 2.79 | 0.2367 |
| Error | 2 | 0.116497 | 0.058249 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-------------------|----|-----------|-------------|---------|--------|
| trt | 1 | 0.458943 | 0.458943 | 1.52 | 0.3049 |
| subject(sequence) | 2 | 0.116497 | 0.058249 | 0.19 | 0.8337 |
| Error: MS(Error) | 3 | 0.903667 | 0.301222 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_VZFOW

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.162656 | 0.162656 | 2.79 | 0.2367 |
| Error | 2 | 0.116497 | 0.058249 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| trt | 1 | 0.458943 | 0.458943 | 1.52 | 0.3049 |
| subject(sequence) | 2 | 0.116497 | 0.058249 | 0.19 | 0.8337 |
| Error: MS(Error) | 3 | 0.903667 | 0.301222 | | |

Comparison: C vs B

Dependent Variable: V<sub>d</sub>/F/kg (L/kg) Weight Group: 88-111

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_VZFOW

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.162656 | 0.162656 | 2.79 | 0.2367 |
| Error | 2 | 0.116497 | 0.058249 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| trt | 1 | 0.458943 | 0.458943 | 1.52 | 0.3049 |
| subject(sequence) | 2 | 0.116497 | 0.058249 | 0.19 | 0.8337 |
| Error: MS(Error) | 3 | 0.903667 | 0.301222 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN VZFOW

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.162656 | 0.162656 | 2.79 | 0.2367 |
| Error | 2 | 0.116497 | 0.058249 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| trt | 1 | 0.458943 | 0.458943 | 1.52 | 0.3049 |
| subject(sequence) | 2 | 0.116497 | 0.058249 | 0.19 | 0.8337 |
| Error: MS(Error) | 3 | 0.903667 | 0.301222 | | |
Comparison: C vs B

Dependent Variable: V<sub>d</sub>/F/kg (L/kg) Weight Group: 88-111

#### Least Squares Means

| | | H0:LSMean1=LSMean2 | |
|-----|-----------------|--------------------|---------|
| trt | LN_VZFOW LSMEAN | | Pr > t |
| В | 1.18422404 | | 0.3049 |
| C | 0.70519235 | | |

| trt | LN_VZFOW LSMEAN | 90% Confidence Limits | |
|-----|-----------------|-----------------------|----------|
| В | 1.184224 | 0.486673 | 1.881775 |
| C | 0.705192 | 0.007642 | 1.402743 |

| Le | Least Squares Means for Effect trt | | | |
|---|---|---|---|---|
| | Difference Between | | | |
| i | j | Means | 90% Confide | ence Limits for LSMean(i)-LSMean(j) |
| 1 | 2 | 0.479032 | -0.434277 | 1.392340 |

#### Dependent Variable: LN\_VZFOW

| | | Standard | | | |
|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confidence Limits |
| C - B | -0.47903169 | 0.38808644 | -1.23 | 0.3049- | 1.39234013 0.43427676 |

Dependent Variable: V<sub>d</sub>/F (L) Weight Group: 88-111

#### The GLM Procedure

| Class Level Info | Levels | Values | |
|-----------------------------|---------------|-----------------|---|
| subject | 4 | 203 204 402 404 | |
| sequence | 2 | ABC BAC | |
| trt | 2 | ВС | |
| Number of Obse | rvations Read | | 8 |
| Number of Observations Used | | | |

Comparison: C vs B

Dependent Variable: V<sub>d</sub>/F (L) Weight Group: 88-111

#### The GLM Procedure

Dependent Variable: LN\_VZFO

| R-Square | Coeff Var Root MSI | | 1 | LN | VZFO Mean |
|---|---|---|---|---|---|
| 0.393998 | 9.917712 | 0.548837 | 5.533908 | | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.05526159 | 0.05526159 | 0.18 | 0.6973 |
| trt | 1 | 0.45894271 | 0.45894271 | 1.52 | 0.3049 |
| subject(sequence | ) 2 | 0.07332197 | 0.03666098 | 0.12 | 0.8896 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.05526159 | 0.05526159 | 0.18 | 0.6973 |
| trt | 1 | 0.45894271 | 0.45894271 | 1.52 | 0.3049 |
| subject(sequence | ) 2 | 0.07332197 | 0.03666098 | 0.12 | 0.8896 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.05526159 | 0.05526159 | 0.18 | 0.6973 |
| trt | 1 | 0.45894271 | 0.45894271 | 1.52 | 0.3049 |
| subject(sequence | ) 2 | 0.07332197 | 0.03666098 | 0.12 | 0.8896 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 0.05526159 | 0.05526159 | 0.18 | 0.6973 |
| trt | 1 | 0.45894271 | 0.45894271 | 1.52 | 0.3049 |
| subject(sequence | ) 2 | 0.07332197 | 0.03666098 | 0.12 | 0.8896 |

Comparison: C vs B

Dependent Variable: V<sub>d</sub>/F (L) Weight Group: 88-111

## The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_VZFO

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.055262 | 0.055262 | 1.51 | 0.3444 |
| Error | 2 | 0.073322 | 0.036661 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-------------------|----|-----------|-------------|---------|--------|
| trt | 1 | 0.458943 | 0.458943 | 1.52 | 0.3049 |
| subject(sequence) | 2 | 0.073322 | 0.036661 | 0.12 | 0.8896 |
| Error: MS(Error) | 3 | 0.903667 | 0.301222 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_VZFO

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.055262 | 0.055262 | 1.51 | 0.3444 |
| Error | 2 | 0.073322 | 0.036661 | | _ |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| trt | 1 | 0.458943 | 0.458943 | 1.52 | 0.3049 |
| subject(sequence) | 2 | 0.073322 | 0.036661 | 0.12 | 0.8896 |
| Error: MS(Error) | 3 | 0.903667 | 0.301222 | | |

Comparison: C vs B

Dependent Variable: V<sub>d</sub>/F (L) Weight Group: 88-111

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN\_VZFO

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.055262 | 0.055262 | 1.51 | 0.3444 |
| Error | 2 | 0.073322 | 0.036661 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| trt | 1 | 0.458943 | 0.458943 | 1.52 | 0.3049 |
| subject(sequence) | 2 | 0.073322 | 0.036661 | 0.12 | 0.8896 |
| Error: MS(Error) | 3 | 0.903667 | 0.301222 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LN VZFO

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.055262 | 0.055262 | 1.51 | 0.3444 |
| Error | 2 | 0.073322 | 0.036661 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| trt | 1 | 0.458943 | 0.458943 | 1.52 | 0.3049 |
| subject(sequence) | 2 | 0.073322 | 0.036661 | 0.12 | 0.8896 |
| Error: MS(Error) | 3 | 0.903667 | 0.301222 | | |

Comparison: C vs B

Dependent Variable: V<sub>d</sub>/F (L) Weight Group: 88-111

#### Least Squares Means

| | | H0:LSMean1=LSMean2 | |
|-----|----------------|--------------------|---------|
| trt | LN_VZFO LSMEAN | | Pr > t |
| В | 5.82140924 | | 0.3049 |
| C | 5.34237756 | | |

| trt | LN_VZFO LSMEAN | 90% Confidence Limits | |
|-----|----------------|-----------------------|----------|
| В | 5.821409 | 5.123858 | 6.518960 |
| C | 5.342378 | 4.644827 | 6.039928 |

| Le | Least Squares Means for Effect trt | | | |
|---|---|---|---|---|
| | | Difference Between | | |
| i | j | Means | 90% Confidence | ee Limits for LSMean(i)-LSMean(j) |
| 1 | 2 | 0.479032 | -0.434277 | 1.392340 |

#### Dependent Variable: LN\_VZFO

| | | Standard | | | |
|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t 90% Confidence Li | mits |
| C - B | -0.47903169 | 0.38808644 | -1.23 | 0.3049-1.39234013 0.4342 | 7676 |

Comparison: C vs B

Dependent Variable: T<sub>max</sub> (h) Weight Group: 88-111

#### The GLM Procedure

| Class Level Info | rmation | |
|---|---|---|
| Class | Levels | Values |
| subject | 4 | 203 204 402 404 |
| sequence | 2 | ABC BAC |
| trt | 2 | ВС |
| Number of Observations Read | | |
| Number of Obse | Number of Observations Used | |

Comparison: C vs B

Dependent Variable: T<sub>max</sub> (h) Weight Group: 88-111

#### The GLM Procedure

| R-Square | Coeff Var | Root | MSE | | TMAX Mean |
|---|---|---|---|---|---|
| 0.749116 | 73.44244 | 1.038 | 8935 | 1.414625 | |
| Source | DF | Type I SS | Mean Square | F Value | e Pr > F |
| sequence | 1 | 1.86093704 | 1.86093704 | 1.72 | 0.2806 |
| trt | 1 | 6.51063613 | 6.51063613 | 6.03 | 0.0912 |
| subject(sequence) | 2 | 1.29724633 | 0.64862317 | 0.60 | 0.6033 |
| Source | DF | Type II SS | Mean Square | F Value | e Pr > F |
| sequence | 1 | 1.86093704 | 1.86093704 | 1.72 | 0.2806 |
| trt | 1 | 6.51063613 | 6.51063613 | 6.03 | 0.0912 |
| subject(sequence) | 2 | 1.29724633 | 0.64862317 | 0.60 | 0.6033 |
| Source | DF | Type III SS | Mean Square | F Value | e $Pr > F$ |
| sequence | 1 | 1.86093704 | 1.86093704 | 1.72 | 0.2806 |
| trt | 1 | 6.51063613 | 6.51063613 | 6.03 | 0.0912 |
| subject(sequence) | 2 | 1.29724633 | 0.64862317 | 0.60 | 0.6033 |
| Source | DF | Type IV SS | Mean Square | F Value | e $Pr > F$ |
| sequence | 1 | 1.86093704 | 1.86093704 | 1.72 | 0.2806 |
| trt | 1 | 6.51063613 | 6.51063613 | 6.03 | 0.0912 |
| subject(sequence) | 2 | 1.29724633 | 0.64862317 | 0.60 | 0.6033 |

Comparison: C vs B

Dependent Variable: T<sub>max</sub> (h) Weight Group: 88-111

## The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: TMAX

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 1.860937 | 1.860937 | 2.87 | 0.2324 |
| Error | 2 | 1.297246 | 0.648623 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-------------------|----|-----------|-------------|---------|--------|
| trt | 1 | 6.510636 | 6.510636 | 6.03 | 0.0912 |
| subject(sequence) | 2 | 1.297246 | 0.648623 | 0.60 | 0.6033 |
| Error: MS(Error) | 3 | 3.238158 | 1.079386 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 1.860937 | 1.860937 | 2.87 | 0.2324 |
| Error | 2 | 1.297246 | 0.648623 | | _ |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| trt | 1 | 6.510636 | 6.510636 | 6.03 | 0.0912 |
| subject(sequence) | 2 | 1.297246 | 0.648623 | 0.60 | 0.6033 |
| Error: MS(Error) | 3 | 3.238158 | 1.079386 | | |

Comparison: C vs B

Dependent Variable:  $T_{max}$  (h) Weight Group: 88-111

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: TMAX

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 1.860937 | 1.860937 | 2.87 | 0.2324 |
| Error | 2 | 1.297246 | 0.648623 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| trt | 1 | 6.510636 | 6.510636 | 6.03 | 0.0912 |
| subject(sequence) | 2 | 1.297246 | 0.648623 | 0.60 | 0.6033 |
| Error: MS(Error) | 3 | 3.238158 | 1.079386 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------|-----------|------------|-------------|---------|--------|
| sequence | 1 | 1.860937 | 1.860937 | 2.87 | 0.2324 |
| Error | 2 | 1.297246 | 0.648623 | | |
| Error: MS(s | subject(s | sequence)) | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| trt | 1 | 6.510636 | 6.510636 | 6.03 | 0.0912 |
| subject(sequence) | 2 | 1.297246 | 0.648623 | 0.60 | 0.6033 |
| Error: MS(Error) | 3 | 3.238158 | 1.079386 | | |

Comparison: C vs B

Dependent Variable: T<sub>max</sub> (h) Weight Group: 88-111

#### Least Squares Means

| | | | H0:LSMean1: | =LSMean2 | |
|---|---|---|---|---|---|
| trt | TMAX LSMEAN | | | | Pr > t |
| В | 0.79095833 | | | | 0.0912 |
| C | 2.59520833 | | | | |
| trt | TMAX LSMEAN | | 90% Confi | dence Limits | |
| В | 0.790958 | -0.529 | 9488 | 2.111405 | |
| C | 2.595208 | 1.274 | 762 | 3.915655 | |
| Le | ast Squares Means for Effec | t trt | | | |
| | Difference Between | 000/ G | T | 31.6 (2) 1.61 | |
| 1 | j Means | 90% Confidenc | e Limits for LS | SMean(1)-LSN | Aean(j) |
| 1 | 2 -1.804250 | -3.533120 | -0.07 | 75380 | |

| | | Standard | | |
|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t 90% Confidence Limits |
| C - B | 1.80425000 | 0.73463805 | 2.46 | 0.09120.07537968 3.53312032 |

Dependent Variable: K<sub>el</sub> (/h) Weight Group: 88-111

#### The GLM Procedure

| Class Level Infor | mation | | _ |
|-------------------|--------|-----------------|---|
| Class | Levels | Values | |
| subject | 4 | 203 204 402 404 | _ |
| sequence | 2 | ABC BAC | |
| trt | 2 | ВС | |
| Number of Obser | 8 | | |
| Number of Obser | 8 | | |

Comparison: C vs B

Dependent Variable: K<sub>el</sub> (/h) Weight Group: 88-111

#### The GLM Procedure

| R-Square | Coeff Var | Root MSE | | | LAMZ Mean |
|---|---|---|---|---|---|
| 0.779248 | 18.43795 | 0.001 | 672 | 0.009066 | |
| Source | DF | Type I SS | Mean Square | F Value | e Pr > F |
| sequence | 1 | 0.00002132 | 0.00002132 | 7.63 | 0.0700 |
| trt | 1 | 0.00000528 | 0.00000528 | 1.89 | 0.2629 |
| subject(sequence) | 2 | 0.00000299 | 0.00000150 | 0.54 | 0.6325 |
| Source | DF | Type II SS | Mean Square | F Value | e Pr > F |
| sequence | 1 | 0.00002132 | 0.00002132 | 7.63 | 0.0700 |
| trt | 1 | 0.00000528 | 0.00000528 | 1.89 | 0.2629 |
| subject(sequence) | 2 | 0.00000299 | 0.00000150 | 0.54 | 0.6325 |
| <u> </u> | DE | Toma III CC | Maan Carrage | E Valer | |
| Source | DF | Type III SS | Mean Square | | |
| sequence | 1 | 0.00002132 | 0.00002132 | 7.63 | 0.0700 |
| trt | 1 | 0.00000528 | 0.00000528 | 1.89 | 0.2629 |
| subject(sequence) | 2 | 0.00000299 | 0.00000150 | 0.54 | 0.6325 |
| Source | DF | Type IV SS | Mean Square | F Value | e Pr > F |
| sequence | 1 | 0.00002132 | 0.00002132 | 7.63 | 0.0700 |
| trt | 1 | 0.00000528 | 0.00000528 | 1.89 | 0.2629 |
| subject(sequence) | 2 | 0.00000299 | 0.00000150 | 0.54 | 0.6325 |

Comparison: C vs B

Dependent Variable: K<sub>el</sub> (/h) Weight Group: 88-111

## The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LAMZ

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.000021316 | 0.000021316 | 14.24 | 0.0636 |
| Error | 2 | 0.000002993 | 0.000001497 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| trt | 1 | 0.000005281 | 0.000005281 | 1.89 | 0.2629 |
| subject(sequence) | 2 | 0.000002993 | 0.000001497 | 0.54 | 0.6325 |
| Error: MS(Error) | 3 | 0.000008382 | 0.000002794 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.000021316 | 0.000021316 | 14.24 | 0.0636 |
| Error | 2 | 0.000002993 | 0.000001497 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| trt | 1 | 0.000005281 | 0.000005281 | 1.89 | 0.2629 |
| subject(sequence) | 2 | 0.000002993 | 0.000001497 | 0.54 | 0.6325 |
| Error: MS(Error) | 3 | 0.000008382 | 0.000002794 | | |

Comparison: C vs B

Dependent Variable: K<sub>el</sub> (/h) Weight Group: 88-111

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LAMZ

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.000021316 | 0.000021316 | 14.24 | 0.0636 |
| Error 2 0.000002993 0.000001497 | | | | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| trt | 1 | 0.000005281 | 0.000005281 | 1.89 | 0.2629 |
| subject(sequence) | 2 | 0.000002993 | 0.000001497 | 0.54 | 0.6325 |
| Error: MS(Error) | 3 | 0.000008382 | 0.000002794 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 0.000021316 | 0.000021316 | 14.24 | 0.0636 |
| Error | 2 | 0.000002993 | 0.000001497 | | |
| Error: MS(s | Error: MS(subject(sequence)) | | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| trt | 1 | 0.000005281 | 0.000005281 | 1.89 | 0.2629 |
| subject(sequence) | 2 | 0.000002993 | 0.000001497 | 0.54 | 0.6325 |
| Error: MS(Error) | 3 | 0.000008382 | 0.000002794 | | |

Comparison: C vs B

Dependent Variable: K<sub>el</sub> (/h) Weight Group: 88-111

#### Least Squares Means

| | | | H0:LSN | Mean1=LSMean2 | |
|---|---|---|---|---|---|
| trt | LAMZ LSMEAN | | | | Pr > t |
| В | 0.00919589 | | | | 0.2629 |
| C | 0.01082078 | | | | |
| trt | LAMZ LSMEAN | | 90% | Confidence Limits | |
| В | 0.009196 | ( | 0.007071 | 0.011320 | |
| C | 0.010821 | ( | 0.008696 | 0.012945 | |
| Le | ast Squares Means for Effec | t trt | | | |
| | Difference Between | | | | |
| i | j Means | 90% Confi | dence Limits | for LSMean(i)-LSM | Iean(j) |
| 1 | 2 -0.001625 | -0.004407 | | 0.001157 | |

| | | Standard | | | | |
|---|---|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t | 90% Confi | dence Limits |
| C - B | 0.00162489 | 0.00118198 | 1.37 | 0.2629-0 | 0.00115673 | 0.00440651 |

Comparison: C vs B

Dependent Variable: T<sub>1/2 el</sub> (h) Weight Group: 88-111

#### The GLM Procedure

| Class Level Infor | mation | | _ |
|---|---|---|---|
| Class | Levels | Values | |
| subject | 4 | 203 204 402 404 | |
| sequence | 2 | ABC BAC | |
| trt | 2 | ВС | |
| Number of Observations Read | | | |
| Number of Observations Read Number of Observations Used | | | |

Comparison: C vs B

Dependent Variable: T<sub>1/2 el</sub> (h) Weight Group: 88-111

#### The GLM Procedure

| R-Square | Coeff Var | Root MSE | | LAMZ | ZHL Mean |
|---|---|---|---|---|---|
| 0.717423 | 18.29114 | 14.72222 | 80.48823 | | |
| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 1233.320675 | 1233.320675 | 5.69 | 0.0971 |
| trt | 1 | 270.127861 | 270.127861 | 1.25 | 0.3456 |
| subject(sequence | ) 2 | 147.396875 | 73.698437 | 0.34 | 0.7360 |
| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 1233.320675 | 1233.320675 | 5.69 | 0.0971 |
| trt | 1 | 270.127861 | 270.127861 | 1.25 | 0.3456 |
| subject(sequence | ) 2 | 147.396875 | 73.698437 | 0.34 | 0.7360 |
| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 1233.320675 | 1233.320675 | 5.69 | 0.0971 |
| trt | 1 | 270.127861 | 270.127861 | 1.25 | 0.3456 |
| subject(sequence | ) 2 | 147.396875 | 73.698437 | 0.34 | 0.7360 |
| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
| sequence | 1 | 1233.320675 | 1233.320675 | 5.69 | 0.0971 |
| trt | 1 | 270.127861 | 270.127861 | 1.25 | 0.3456 |
| subject(sequence | ) 2 | 147.396875 | 73.698437 | 0.34 | 0.7360 |

Comparison: C vs B

Dependent Variable: T<sub>1/2 el</sub> (h) Weight Group: 88-111

## The GLM Procedure Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LAMZHL

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 1233.320675 | 1233.320675 | 16.73 | 0.0549 |
| Error | 2 | 147.396875 | 73.698437 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type I SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| trt | 1 | 270.127861 | 270.127861 | 1.25 | 0.3456 |
| subject(sequence) | 2 | 147.396875 | 73.698437 | 0.34 | 0.7360 |
| Error: MS(Error) | 3 | 650.230939 | 216.743646 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 1233.320675 | 1233.320675 | 16.73 | 0.0549 |
| Error | 2 | 147.396875 | 73.698437 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type II SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| trt | 1 | 270.127861 | 270.127861 | 1.25 | 0.3456 |
| subject(sequence) | 2 | 147.396875 | 73.698437 | 0.34 | 0.7360 |
| Error: MS(Error) | 3 | 650.230939 | 216.743646 | | |

Comparison: C vs B

Dependent Variable: T<sub>1/2 el</sub> (h) Weight Group: 88-111

#### Tests of Hypotheses for Mixed Model Analysis of Variance

Dependent Variable: LAMZHL

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 1233.320675 | 1233.320675 | 16.73 | 0.0549 |
| Error | 2 | 147.396875 | 73.698437 | | |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type III SS | Mean Square | F Value | Pr > F |
|-------------------|----|-------------|-------------|---------|--------|
| trt | 1 | 270.127861 | 270.127861 | 1.25 | 0.3456 |
| subject(sequence) | 2 | 147.396875 | 73.698437 | 0.34 | 0.7360 |
| Error: MS(Error) | 3 | 650.230939 | 216.743646 | | |

#### Tests of Hypotheses for Mixed Model Analysis of Variance

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|---|---|---|---|---|---|
| sequence | 1 | 1233.320675 | 1233.320675 | 16.73 | 0.0549 |
| Error | 2 | 147.396875 | 73.698437 | | _ |
| Error: MS(subject(sequence)) | | | | | |

| Source | DF | Type IV SS | Mean Square | F Value | Pr > F |
|-------------------|----|------------|-------------|---------|--------|
| trt | 1 | 270.127861 | 270.127861 | 1.25 | 0.3456 |
| subject(sequence) | 2 | 147.396875 | 73.698437 | 0.34 | 0.7360 |
| Error: MS(Error) | 3 | 650.230939 | 216.743646 | | |

Comparison: C vs B

Dependent Variable: T<sub>1/2 el</sub> (h) Weight Group: 88-111

#### Least Squares Means

| | | Н | 0:LSMean1=LSMean2 |
|---|---|---|---|
| trt | LAMZHL LSMEAN | | Pr > t |
| В | 79.1305102 | | 0.3456 |
| C | 67.5088094 | | |
| trt | LAMZHL LSMEAN | 9 | 00% Confidence Limits |
| В | 79.130510 | 60.419140 | 97.841880 |
| C | 67.508809 | 48.797439 | 86.220179 |
| Lea | ast Squares Means for Effec | et trt | |
| | Difference Between | | |
| i | j Means | 90% Confiden | ce Limits for LSMean(i)-LSMean(j) |
| 1 | 2 11.621701 | -12.877233 | 36.120635 |

#### Dependent Variable: LAMZHL

| | | Standard | | |
|---|---|---|---|---|
| Parameter | Estimate | Error | t Value | Pr > t 90% Confidence Limits |
| C - B | -11.6217008 | 10.4101788 | -1.12 | 0.3456-36.1206350 12.8772334 |